**Statistical Analysis Plan** 

**Study ID: 217710** 

Official Title of Study: A Phase 4, randomized, open-label, two-arm study evaluating

implementation strategies for the delivery of Cabotegravir in low and high-volume pre-

exposure prophylaxis (PrEP) sites in the U.S. for HIV uninfected MSM and transgender

 $men \ge 18$ 

NCT number: NCT05374525

**Date of Document:** 04 Oct 2024

A Phase 4, Randomized, Open-label, Two-arm Study **Evaluating Implementation Strategies for the** Delivery of Cabotegravir in Low- and High-volume Pre-exposure Prophylaxis (PrEP) Sites in the US for HIV Uninfected MSM and Transgender Men ≥18: **217710 PILLAR** 

**Statistical Analysis Plan: Patient Study Participants Questionnaires** 

### EVA-32399 | October 4, 2024 | Version 2.0

#### Prepared For:

Study Delivery Lead—Respiratory & Specialty, GSK , PhD, MPH | PPD , Global Implementation Science, ViiV Healthcare



#### Prepared By:

| PPD | , MA Senior Research Scientist, Patient Centered Research PPD |
|-----|-------------------------------------------------------------------|
| PPD | , MPH Research Scientist, Patient Centered Research PPD |
| PPD | , MSc Lead Data Analyst, Patient Centered Research PPD |
| PPD | , MPH Research Associate III, Patient Centered Research PPD |

#### Project Contact:

, MS, PMP | Tel: PPD







## **Table of Contents**

| 1 | INT | RODUCTION | 1 |
|---|---|---|---|
| 2 | PILL | AR STUDY DESIGN | 1 |
| | 2.1 | Feasibility of Intervention Measure | 3 |
| | 2.2 | Acceptability of Intervention Measure | 3 |
| | 2.3 | Analysis Population | 4 |
| | 2.4 | Missing Data Handling Scheme | 4 |
| | 2.5 | Significance Levels and Multiplicity | 4 |
| 3 | STA | TISTICAL METHODS | 4 |
| | 3.1 | Cross-sectional Distributional Characteristics of Study Variables and Features of Score Distributions | 5 |
| | | 3.1.1 PSP Demographics, Behavioral History, and Attitudes/Knowledge about PrEP and APRETUDE | 5 |
| | 3.2 | Feasibility and Acceptability of APRETUDE and Telehealth | 5 |
| | | 3.2.1 Cross sectional Descriptive Statistics by Visits | 5 |
| | | 3.2.2 Assessment of Variability Within vs. Between Clusters Error! Bookmark not defi | ned. |
| | | 3.2.3 Mixed-effects Models at M6/7 and M12/13 | 5 |
| | | 3.2.4 Change from Baseline Mixed Models | 6 |
| | 3.3 | PSP Perception of Facilitators and Barriers to Feasibility and Acceptability of APRETUDE | 7 |
| | 3.4 | Acceptability and Utility of DI Compared to RI for APRETUDE Administration | 7 |
| | 3.5 | PSP Perceptions of Sexual Health Assessment | 7 |
| | 3.6 | Experience of Implementation | 7 |
| | 3.7 | HIV Knowledge, Stigma, and Quality of Care | 7 |
| | 3.8 | Differences by Implementation Arm and Site Volume, FIM APRETUDE and FIM Telehealth | 8 |
| 4 | REF | ERENCES | 9 |
| TAB | LE SH | HELLS FOR BASELINE ANALYSIS | 10 |
| TAB | LE SH | HELLS FOR MONTH 6/7 ANALYSIS | . 205 |
| TAB | LE SH | HELLS FOR MONTH 12/13 ANALYSIS | . 420 |



## **List of Abbreviations**

| Abbreviation | Definition |
|--------------|---------------------------------------|
| AIM | Acceptability of Intervention Measure |
| BL | Baseline |
| CAB | Cabotegravir |
| DI | Dynamic implementation |
| DTI | Direct to injection |
| FIM | Feasibility of Intervention Measure |
| HIV | Human immunodeficiency virus |
| ISQ | Implementation Science Questionnaire |
| LA | Long-acting |
| MSM | Men who have sex with men |
| OLI | Oral lead-in |
| PrEP | Pre-exposure prophylaxis |
| PSP | Patient Study Participant |
| REML | Residual maximum likelihood |
| RI | Routine implementation |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SSP | Staff study participant |
| TGM | Transgender men |
| US | United States |



### 1 Introduction

This study is being conducted following the Food and Drug Administration approval and commercial availability of cabotegravir (CAB) long-acting (LA) for pre-exposure prophylaxis (PrEP, also known as of APRETUDE) in the United States (US). This is an open-label, phase IV, two-arm (dynamic implementation and routine implementation) study of the delivery of APRETUDE in low- and high-volume sites in the US for men who have sex with men (MSM) and transgender men (TGM) ≥18 years of age, referred to herein as patient study participants (PSPs). Eighteen clinics (~9 high and ~9 low volume) were randomized 2:1 to dynamic implementation (DI) or routine implementation (RI) (protocol # 217710/ Amendment 2.0), and one site was lost in the DI arm.

This statistical analysis plan (SAP) describes the analysis of the PSP questionnaires, which includes the analyses assessing PSP responses to questions regarding the acceptability and feasibility of receiving cabotegravir (GKS1265744) long-acting (APRETUDE).

### 2 Pillar Study Design

The phase 4 study is designed to evaluate DI versus RI strategies on the feasibility of delivering APRETUDE at high- and low-volume PrEP centers over 12 months. The patient population includes approximately 220 human immunodeficiency virus (HIV)-negative PSPs across sites who will be prescribed CAB PrEP and enrolled in the study. At least 50% of the PSPs will be Black or Latino. While the primary objective and associated endpoints are aimed at assessing the feasibility of the administration of APRETUDE from the site perspective, secondary and tertiary objectives/endpoints will address the perspective of PSPs, including the feasibility and acceptability for APRETUDE and telehealth. The comparison of DI vs. RI at the site level with PSPs nested within the randomization (i.e., cluster-randomized) will also be performed in the same way as has been described for the staff study participants (SSPs) SAP. As was stated in the SSP SAP, this design may affect the interpretation of certain outcomes as the independence of responses of PSPs within the same site may not hold.

Objectives/endpoints relevant to the current SAP are listed in Table A.



### Table A. Study Objectives for PSP Data

| Objective<br>Type | Objectives | Endpoints |
|---|---|---|
| Secondary | To evaluate feasibility and acceptability of APRETUDE | PSPs mean FIM and AIM scores as well as ISQ responses at BL, M7(OLI)/M6(DTI) and M13(OLI)/M12(DTI). |
| | for MSM and TGM. | Change from baseline in PSPs' AIM and FIM scores as well as ISQ responses FIN score at M7(OLI)/M6(DTI) and M13(OLI)/M12(DTI) |
| | | PSPs perception of facilitators and barriers to feasibility and acceptability of APRETUDE through M13(OLI)/M12(DTI). |
| | To evaluate feasibility and acceptability of telehealth | PSPs' mean FIM and AIM scores as well as ISQ responses for telehealth delivery at BL, M7(OLI)/M6(DTI) and M13(OLI)/M12(DTI) |
| | delivery for APRETUDE administration by clinical staff. | Change from baseline in PSPs' FIM and AIM scores as well as ISQ responses for telehealth delivery at M7(OLI)/M6(DTI) and M13(OLI)/M12(DTI). |
| | stan. | PSPs perception of facilitators and barriers to feasibility and acceptability of telehealth use through M13(OLI)/M12(DTI) |
| | To evaluate acceptability and utility of DI compared | PSPs' mean AIM score and ISQ responses by implementation strategy at BL, M7(OLI)/M6(DTI). and M13(OLI)/M12(DTI) |
| | to RI for APRETUDE administration | Change from baseline in PSPs' mean AIM score and ISQ responses by implementation strategy at M7(OLI)/M6(DTI) and M13(OLI)/M12(DTI) |
| | | Proportion of PSPs who respond in agreement on relevant items on the ISQ that each implementation strategy is fit for use through M13(OLI)/M12(DTI) |
| | To evaluate fidelity to injection and dosing window | PSPs perception of barriers and facilitators to fidelity to injections through M13 |
| | To evaluate fidelity and<br>reach of client Sexual<br>Health Assessment | Proportion of eligible PSPs for which Sexual Health Assessment are administered through M13 and by clinic characteristics, patient subgroups, and service delivery method (e.g., telehealth vs. face-to-face in clinic) |
| | | Proportion of MSM and TGM who take the Sexual Health Assessment through M13 |
| | | Proportion of MSM and TGM who expressed interest in PrEP or never heard of PrEP out of those who report having had sex in the last 6 months through M13 |
| | | Proportion of PSPs who initiate APRETUDE after taking the Sexual Health<br>Assessment through M13 |
| | | PSPs perceptions of Sexual Health Assessment through M13 |
| | To evaluate switch from oral PrEP to APRETUDE | Proportion of PSPs with history of PrEP use that complete the Sexual Health<br>Assessment and ISQ and start APRETUDE through M13 |
| | | PSPs reasons for choosing APRETUDE, including switching, as assessed by SSIs and ISQ |
| | To evaluate perceptions,<br>barriers, and facilitators<br>with PSPs | PSPs perception of barriers and facilitators through M13. |
| Tertiary | CCI | |





### 2.1 Feasibility of Intervention Measure

The Feasibility of Intervention Measure (FIM) is employed to evaluate the extent to which an intervention can be carried out. This four-item measure assesses perceived intervention feasibility by employing a standard item stem to various aspects of feasibility. The items are measured on a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The FIM has been validated with other implementation outcome measures. Higher scores for FIM indicate greater feasibility and there are no reverse-scored items on the FIM. The FIM has been adapted to measure PSPs' assessments of implementation of APRETUDE and telehealth. Mean scores for the FIM are derived by averaging the four items at each administration where at least two of four item responses are available. This mechanism for handling scoring in the presence of missing item-level responses has been used widely in patient- and clinician-reported outcomes.<sup>2</sup>

### 2.2 Acceptability of Intervention Measure

The Acceptability of Intervention Measure (AIM) is employed to evaluate the perception that a given intervention or treatment is satisfactory. It is similar to the FIM as it is a four-item measure, but it assesses perceived intervention acceptability instead of feasibility. The items are measured on a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The AIM was validated with a suite of implementation outcome measures. Higher scores for AIM indicate greater acceptability. As with the FIM, there are no reverse-scored items on the AIM, and the mean score for acceptability of the intervention is calculated by averaging the responses from four items, provided at least two of the four items have viable responses. The AIM has been



adapted to measure PSPs' assessments of the implementation of: APRETUDE, implementation support, and telehealth.

### 2.3 Analysis Population

The study population in this analysis will be all respondents who complete any item on the PSP questionnaire at any timepoint.

### 2.4 Missing Data Handling Scheme

Missing data at the item level are anticipated to be rare. However, in some cases, the PSP may terminate before completing the survey in its entirety. The scoring algorithm and handling of missing values for FIM and AIM are described in Sections 2.1, 2.2, and 3.2.1. If a participant decides to withdraw from the study, the data will be handled according to the protocol: "If the PSP withdraws consent for disclosure of future information, the sponsor may retain and continue to use any data collected before such a withdrawal of consent." PSPs will be analyzed according to the data as given, and no data imputation will be implemented.

### 2.5 Significance Levels and Multiplicity

Any statistical significance tests will be two-tailed and will be conducted with type I error probability fixed at 0.05. Statistical significance, then, will be determined if the p-value is less than 0.05. No multiplicity adjustment will be performed. The general null and alternative hypotheses for statistical tests will be for a given parameter  $(\theta)$ —e.g., mean:

 $H_0: \theta = 0$ 

Versus

 $H_A: \theta \neq 0$ 

### 3 Statistical Methods

Continuous and interval-like variables will be summarized using descriptive statistics (e.g., n, mean, standard deviation [SD], minimum, first quartile, median, third quartile, and maximum). Means and quartiles will be summarized to one decimal place beyond the data values, SD will be reported to two decimal places more than the source data, and minima and maxima will be reported to the same precision level as the source data. Categorical variables will be reported as frequency counts: the percentage of PSPs in corresponding categories, expressed as whole numbers and percentages with one decimal (e.g., 10.1%). Continuous outcomes will be evaluated depending on the number of group comparisons being made. Grouping variables with two levels will be compared with t-tests. Grouping variables with three or more categories, or which have more than one independent variable (see sections 3.2.3 or 3.2.4 below), or analyses which include a stratification factor, will be evaluated with F-tests and pairwise comparisons will be calculated to aid in interpretation of main effects. Categorical variables will be analyzed with Cochran-Mantel-Haenszel test or Fisher's Exact Test depending on data availability per



category, i.e., if any cell of a given contingency table has a cell with incidence of five or less the Fisher test will be used.

# 3.1 Cross-sectional Distributional Characteristics of Study Variables and Features of Score Distributions

For questions with ordinal responses, a univariate distribution of every item will be tabulated. Standard distributional statistics will be tabulated for interval-like (ordinal) variables, including mean, SD, median, percentage missing, minimum, and maximum of responses, percentage of the sample at the ceiling and floor, first and third quartiles, and 95% confidence intervals around means. For questions with categorical responses, a frequency distribution of all responses will be presented with the number and percentage of a given response.



### 3.2 Feasibility and Acceptability of APRETUDE and Telehealth

### 3.2.1 Cross sectional Descriptive Statistics by Visits

PSP mean FIM and AIM scores focusing on APRETUDE and Telehealth at baseline, M6/M7, and M12/M13 will be evaluated by the study arms using descriptive statistics and mixed-effects modeling approaches described below. Descriptive statistics of scores and coded item response will include those listed in Section 3.1 for continuous variables. Additionally, item response frequencies and percentages will be produced for individual items to further assess the distribution of responses.

### 3.2.2 Mixed-effects Models at M6/7 and M12/13

Cross-sectional mixed-effects models will be fit to the FIM and AIM mean scores at M6/7 and M12/13. These mixed-effects models will be fit using residual maximum likelihood (REML) and will assume data are missing at random. All data will be included regardless of early cessation from the implementation arm. The dependent variables will be the FIM and AIM mean scores. In the model, implementation arm (DI vs. RI), site volume (high vs. low), and the implementation arm by site volume interaction will be fitted as fixed terms, with separate random intercepts fitted to allow for clustering within sites, and for variability within the sites. Site volume was categorized as high versus low according to the reported estimate of PrEP patient seen monthly. These data were split at the median of 50; values above 50 were considered high and those below 50 were considered low. The baseline scores centered around their site mean will be fitted as fixed and random covariates. An unstructured covariance structure will be fitted to account



for the dependence of the residuals within the patient. Should the unstructured covariance structure cause model fitting problems (e.g., nonconvergence), heterogenous compound symmetry will be considered followed by homogenous compound symmetry. Should model fitting problems persist, the random effect on centered mean baseline score will be removed and models will be fit according to the same order of covariance structures (unstructured, then heterogenous compound symmetry, then homogenous compound symmetry).

The corresponding multilevel model for the FIM and AIM scores,  $Y_{ij}$ , for the  $i^{th}$  individual at the  $j^{th}$  site is expressed as:

$$\begin{split} Y_{ij} &= \beta_{00} + \beta_{01}I_j + \beta_{02}V_j + \beta_{03}I_jV_j + \beta_{10}\big(B_{ij} - \bar{B}_j\big) + u_{0j} + u_{1j}\big(B_{ij} - \bar{B}_j\big) + e_{ij} \\ & e_{ij} \sim N(0, \sigma^2) \\ \binom{u_{0j}}{u_{1j}} \sim N\left[\binom{0}{0}, \binom{\tau_{00} & \tau_{01}}{\tau_{10} & \tau_{11}}\right] \end{split}$$

With fixed effects for baseline score  $(B_{ij} - \bar{B}_j)$ , implementation arm  $(I_j)$ , site volume  $(V_j)$ , and the arm by volume interaction. The parameter  $\beta_{00}$  is the fixed mean for the RI arm with low volume. The parameters  $\beta_{01}$ ,  $\beta_{02}$ ,  $\beta_{03}$ , and  $\beta_{10}$  are regression weights for the fixed effects of DI arm, high volume, arm by volume, and baseline score, respectively. Random effects for sites  $(u_{0j})$ , baseline scores across sites  $(u_{1j})$ , and the residual error  $(e_{ij})$  are also included. All random effects and the error term are assumed to be independent. Coding of the mixed-effects models will be done as suggested by Singer (1998).<sup>3</sup> It is worth noting that there is likely a range restriction on FIM and AIM endpoints given that the measures are fairly discrete (i.e., on a 1–5 scale with 0.25 increments) and adjustment of the mixed-effects models may be necessary if the model fits are determined to be affected by this range restriction. The study implementation arms and specific timepoint contrasts will be calculated within the mixed-effects modeling framework.

#### 3.2.3 Change from Baseline Mixed Models

Change from baseline in PSPs' AIM and FIM scores at M6/7, and M12/M13 will be modeled similarly to those described in Section  The dependent variables in this case, however, will be the change from baseline in FIM and AIM mean scores.

The corresponding multilevel model for the changes from baseline in FIM and AIM scores,  $(Y_{ij} - B_{ij})$ , for the  $i^{th}$  individual at the  $j^{th}$  site is expressed as:

$$(Y_{ij} - B_{ij}) = \beta_{00} + \beta_{01}I_j + \beta_{02}V_j + \beta_{03}I_jV_j + \beta_{10}(B_{ij} - \bar{B}_j) + u_{0j} + u_{1j}(B_{ij} - \bar{B}_j) + e_{ij}$$

$$e_{ij} \sim N(0, \sigma^2)$$

$$\binom{u_{0j}}{u_{1j}} \sim N\left[\binom{0}{0}, \binom{\tau_{00}}{\tau_{10}}, \frac{\tau_{01}}{\tau_{11}}\right]$$

Similar to the model in Section , we include the same fixed and random effects. All random effects and the error term are assumed to be independent and random effects will be fit with an unstructured covariance matrix. Model fitting will be attempted until an adequately fitting model is found according to the hierarchy of covariance structures and model specifications described in section 3.2.2. REML will be used to estimate the model's parameters.



# 3.3 PSP Perception of Facilitators and Barriers to Feasibility and Acceptability of APRETUDE

The PSP perception of facilitators and barriers to feasibility and acceptability of APRETUDE will be tabulated by gender (MSM, TGM), implementation arm (RI, DI), and site volume (high, low). For select items tabulation will also be performed by race, ethnicity, as well as race and ethnicity by implementation arm (RI, DI). Descriptive analyses of the facilitators and barriers will be conducted at all timepoints.

## 3.4 Acceptability and Utility of DI Compared to RI for APRETUDE Administration

The proportion of PSPs responding in agreement on relevant items that the respective implementation strategy that they experienced is fit for use at M12/M13 will be estimated.

### 3.5 PSP Perceptions of Sexual Health Assessment

PSP perceptions of the Sexual Health Assessment through M6/7 and M12/M13 will be tabulated by subgroup (MSM, TGM), implementation arm, and site volume. For select items tabulation will also be performed by race, ethnicity, as well as race and ethnicity by implementation arm (RI, DI). All analyses will be conducted at each timepoint.

### 3.6 Experience of Implementation

Attitudes regarding aspects of the experience of implementation, including regarding oral lead-in vs. direct-to-injection, missed doses and following steps, injections and injection reactions, scheduling/appointments, clinics, and quality of care will be tabulated by gender timepoint, implementation arm, and site volume. For select items tabulation will also be performed by race, ethnicity, as well as race and ethnicity by implementation arm (RI, DI). All analyses will be conducted at each timepoint.

### 3.7 HIV Knowledge, Stigma, and Quality of Care

Three subscales regarding HIV Knowledge,<sup>4</sup> Stigma,<sup>5</sup> and Quality of Care<sup>6</sup> are included at all three timepoints. The items of these scales will be tabulated by gender (MSM, TGM), implementation arm (RI, DI), and site volume (high, low); tabulation by race, ethnicity, as well as race and ethnicity by implementation arm will, will be conducted for select items.

For scale scores, distributional characteristics will be summarized by subgroup (MSM, TGM), implementation arm (RI, DI), site volume (high, low), race, ethnicity, as well as race and ethnicity by implementation arm. Cronbach's alpha will also be calculated for items comprising scale scores across the available sample. All analyses will be conducted at each timepoint.



# 3.8 Differences by Implementation Arm and Site Volume, FIM/AIM APRETUDE, and FIM/AIM Telehealth

Difference for FIM/AIM means scores in PSP by implementation arm (RI, DI), site volume (high, low), and the interaction of these variables will be tested using a 2 x 2 between-subjects analysis of variance. The FIM/AIM for APRETUDE and telehealth will be tested, separately, in all analyses all factors will be fixed. Significant interactions will be followed up with appropriate simple effects.



### 4 References

- 1. Weiner BJ, Lewis CC, Stanick C, et al. Psychometric assessment of three newly developed implementation outcome measures. *Implement Sci.* 2017;12(1):108. doi:10.1186/s13012-017-0635-3
- 2. Cella D. Manual of the Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System—Version 4. Center on Outcomes, Research & Education (CORE), Evanston Northwestern Healthcare and Northwestern University; 1997.
- 3. Singer JD. Using SAS PROC MIXED to fit multilevel models, hierarchical models, and individual growth models. *J Educational Behavioral Stat*. 1998;24(4):323-355.
- 4. Janulis P, Newcomb ME, Sullivan P, Mustanski B. Evaluating HIV Knowledge Questionnaires Among Men Who Have Sex with Men: A Multi-Study Item Response Theory Analysis. *Arch Sex Behav*. 2018;47(1):107-119. doi:10.1007/s10508-016-0910-4
- 5. Siegler AJ, Wiatrek S, Mouhanna F, et al. Validation of the HIV Pre-exposure Prophylaxis Stigma Scale: Performance of Likert and Semantic Differential Scale Versions. *AIDS Behav*. 2020;24(9):2637-2649. doi:10.1007/s10461-020-02820-6
- 6. Pilgrim N, Jani N, Mathur S, et al. Provider perspectives on PrEP for adolescent girls and young women in Tanzania: The role of provider biases and quality of care. *PLoS One*. 2018;13(4):e0196280. doi:10.1371/journal.pone.0196280



## **Table Shells for Baseline Analysis**

| Table 5.001. | Demographic Characteristics of New Patient Study Participants (Baseline), N=XX | 15 |
|---|---|---|
| Table 5.003. | Summary of Behaviors of Patient Study Participants (Baseline), N=XX | 18 |
| Table 5.004. | Summary of Patient Study Participants' Sexual History and Behaviors (Baseline), N=XX, Study Arms | 20 |
| Table 5.005. | Summary of Patient Study Participants' Sexual History and Behaviors (Baseline), N=XX, Race, Dynamic Implementation | 23 |
| Table 5.006. | Summary of Patient Study Participants' Sexual History and Behaviors (Baseline), N=XX, Race, Routine Implementation | 26 |
| Table 5.007. | Summary of Patient Study Participants' Sexual History and Behaviors (Baseline), N=XX, Race, Total | 29 |
| Table 5.008. | Summary of Patient Study Participants' Sexual History and Behaviors (Baseline), N=XX, Ethnicity, Study Arms | 32 |
| Table 5.009. | Summary of Patient Study Participants' Sexual History and Behaviors (Baseline), N=XX, Ethnicity, Total | 35 |
| Table 5.0010 | ). Summary of Patient Study Participants' Sexual History and Behaviors (Baseline),<br>N=XX, Gender, Total | 38 |
| Table 5.101. | Summary of Patient Study Participants' HIV and PrEP Knowledge (Baseline), N=XX | 41 |
| Table 5.102. | Summary of Patient Study Participants' HIV and PrEP Knowledge (Baseline), N=XX, Scale Questions, Study Arms | 42 |
| Table 5.103. | Distributional Characteristics of Patient Study Participants' HIV and PrEP Knowledge (Baseline), N=XX, Scale Questions, Overall Score | 44 |
| Table 5.104. | Summary of Patient Study Participants' Perception of Stigma Associated with PrEP Usage (Baseline), N=XX, Stigma, Study Arms | 46 |
| Table 5.105. | Distributional Characteristics of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Stigma, Overall Score | 50 |
| Table 5.106. | Summary of Patient Study Participants' Choice of APRETUDE (Baseline), N=XX | 52 |
| Table 5.107 | Summary of Knowledge of APRETUDE and Utility of Implementation Strategies (Baseline), N=XX | 56 |
| Table 5.108. | Attitude Regarding APRETUDE and Utility of Implementation Strategies (Baseline), N=XX | 60 |
| Table 5.109. | Summary of Patient Study Participant Acquisition Process (Baseline), N=XX | 62 |
| Table 5.110. | Summary of Patient Study Participant Acquisition Process, Insurance (Baseline), N=XX | 63 |
| Table 5.111. | Summary of Patient Study Participants' Perception of Stigma Associated with PrEP Usage (Baseline), N=XX | 67 |
| Table 5.112. | Summary of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Study Arms | 70 |
| Table 5.113. | Summary of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Race, Dynamic Implementation | 71 |
| Table 5.114. | Summary of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX. Race. Routine Implementation | |



| Table 5.115. | Summary of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Race, Total | 75 |
|---|---|---|
| Table 5.116. | Summary of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Ethnicity, Study Arms | 77 |
| Table 5.117. | Summary of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Ethnicity, Total | 79 |
| Table 5.118. | Summary of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Gender, Total | 81 |
| Table 5.201. | Distributional Characteristics of Acceptability of Intervention (AIM) (APRETUDE) (PSP) (Baseline), N=XX | 82 |
| Table 5.202. | Distributional Characteristics of Feasibility of Intervention (FIM) (APRETUDE) (PSP) (Baseline), N=XX | 84 |
| Table 5.203. | Distributional Characteristics of Accessibility of Intervention (AIM) (Telehealth) (PSP) (Baseline), N=XX | 86 |
| Table 5.204. | Distributional Characteristics of Feasibility of Intervention (FIM) (Telehealth) (PSP) (Baseline), N=XX | 88 |
| Table 5.205. | Summary of Acceptability of Intervention (AIM) (APRETUDE) (PSP) (Baseline), N=XX | 90 |
| Table 5.206. | Summary of Feasibility of Intervention (FIM) (APRETUDE) (PSP) (Baseline), N=XX | 92 |
| Table 5.207. | Summary of Acceptability of Intervention (AIM) (Telehealth) (PSP) (Baseline), N=XX | 94 |
| Table 5.208. | Summary of Feasibility of Intervention (FIM) (Telehealth) (PSP) (Baseline), N=XX | 96 |
| Table 5.301. | Summary of Feasibility and Acceptability of Telehealth (Baseline), N=XX | 98 |
| Table 5.302. | Summary of Quality of Care for Patient Study Participants (Baseline), N=XX | 102 |
| Table 5.303. | Summary of Quality of Care for Patient Study Participants (Baseline), N=XX, Non-Score Questions | 106 |
| Table 5.304. | Summary of Quality of Care for Patient Study Participants (Baseline), N=XX, Score Questions | 121 |
| Table 5.305. | Distributional Characteristics of Quality of Care for Patient Study Participants (Baseline), N=XX, Score Questions, Overall Score | 138 |
| Table 5.306. | Summary of Utility of Proposed Implementation Strategies (Baseline), N=XX | 141 |
| Table 5.307. | Summary of Patient Study Participants' Preferences/Acceptability of APRETUDE Information, Appointment Reminders, and Locations (Baseline), N=XX | 146 |
| Table 5.401. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Baseline), N=XX, Study Arms | 149 |
| Table 5.402. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Baseline), N=XX, Race, Dynamic Implementation | 152 |
| Table 5.403. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Baseline), N=XX, Race, Routine Implementation | 155 |
| Table 5.404. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Baseline), N=XX, Race, Total | 158 |
| Table 5.405. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Baseline), N=XX, Ethnicity, Study Arms | 161 |



| Table 5.406. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Baseline), N=XX, Ethnicity, Total | 164 |
|---|---|---|
| Table 5.407. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Baseline), N=XX, Gender, Total | 167 |
| Table 5.408. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Study Arms | 170 |
| Table 5.409. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Race, Dynamic Implementation | 174 |
| Table 5.410. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Race, Routine Implementation | 178 |
| Table 5.411. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Race, Total | 182 |
| Table 5.412. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Ethnicity, Study Arms. | 186 |
| Table 5.413. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Ethnicity, Total | 190 |
| Table 5.414. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Gender | 194 |
| Table 5.415. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Site Volume | 198 |
| Table 5.416. | Distributional Characteristics of Estimated Amount of Money Spent on Transportation for Each Injection Visit (Baseline), N=XX | 202 |
| Table 5.417 | Summary of Optional Oral Lead-In vs. Direct to Injection (Baseline), N=XX | |



Table 5.000. Demographic Characteristics of New Patient Study Participants (Baseline), N=XX

| | | | Total | Dynamic<br>Implementation | Routine<br>Implementation |
|---|---|---|---|---|---|
| Question<br>Number | Question | Response | (N=XX)<br>n (%) | (N=XX)<br>n (%) | (N=XX)<br>n (%) |
| DM1 | Age (years) | N | XX | XX | XX |
| | | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| DM2 | Age (years), High Volume | N | XX | XX | XX |
| | <i>S</i> (, , , , , <i>S</i> | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| DM3 | Age (years), Low Volume | N | XX | XX | XX |
| | <i>C</i> ,, ,, | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| DM4 | Age | | | | |
| | | 18-25 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 26-35 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 36-49 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 50+ | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| DM5 | Study Arm | | | | |
| | | Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| DM6 | Site Volume | | | | |
| | | High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| DM7 | Gender | | | | |
| | | Men who have sex with men | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Transgender men | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| DM8 | Race | | | | |
| | | Asian | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Black or African American | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | White | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Missing/Unknown | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | | uestion | Response | Total<br>(N=XX)<br>n (%) | Dynamic<br>Implementation<br>(N=XX)<br>n (%) | Routine<br>Implementation<br>(N=XX)<br>n (%) |
|---|---|---|---|---|---|---|
| DM9 | Ethnicity | | | | | |
| | | | Hispanic or Latino | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | | Not Hispanic or Latino | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | | Missing/Unknown | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 5.001. Demographic Characteristics of New Patient Study Participants (Baseline), N=XX

| | <u> </u> | | | | ** |
|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
| 1 | How would you describe your current sexual orientation? | Heterosexual or straight | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Gay or lesbian | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bisexual | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Asexual | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Pansexual and/or questioning | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Same gender loving | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Queer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other gender | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 2 | Which of the following best describes your <u>current</u> relationship status? | Single, never married | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Single, widowed | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Single, separated or divorced | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dating, but not living with a partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dating and living with a partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Domestic partnership/civil union | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Married | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 3 | How would you describe your current living situation? | I live in my own house or apartment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I live in my parent's house or apartment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | I live in a family member's house or apartment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I live in a friend's house or apartment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I sleep on various friends'<br>or relatives' couches | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am homeless or am living in a shelter | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I live in motel(s)/hotel(s) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 4 | What is the highest level of education you have completed? | Never attended school | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Less than high school | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some high school; no diploma | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Regular high school<br>diploma/GED or<br>alternative | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some college; no degree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Associate's or technical degree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | College degree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Postgraduate or professional degree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 5 | What <u>best</u> describes your current employment status? | Employed for wages full-<br>time (1 employer) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Employed for wages full-<br>time (2 or more<br>employers) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Employed for wages part-<br>time (1 employer) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Employed for wages part-<br>time (2 or more<br>employers) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Self-employed | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A homemaker | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Student | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Retired | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not employed | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unable to work (disabled) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 6 | What type of medical insurance do you currently have? | My parents' insurance | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | My partner's/spouse's insurance | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Private insurance provided by my workplace | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Private insurance I<br>purchased through an<br>exchange (e.g.,<br>Obamacare, Affordable<br>Care Act) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Federal Insurance (e.g., VA, TRICARE) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Medicare or Medicaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some other health care plan | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't have any health insurance currently | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.002. Summary of Behaviors of Patient Study Participants (Baseline), N=XX

| Question | | | Total<br>(N = XX) | Dynamic<br>Implementation<br>(N = XX) | Routine<br>Implementation<br>(N = XX) |
|---|---|---|---|---|---|
| Number | Question | Response | n (%) | n (%) | n (%) |
| 76 | How often do you have a drink co | ntaining aiconoi? | | 207 | \n, |
| | | Never | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Monthly or less | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 2 to 4 times a month | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 2 to 3 times a week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 4 or more times a week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 77 | On days when you drink alcohol, bottle/ can of beer, 1 glass of win | | | | |
| | | 1 or 2 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 3 to 4 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 5 to 6 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 7 to 9 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 10 or more | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 78 | In the last 6 months, have you she<br>provider, such as speedball, hero<br>a needle, either by mainlining, ski | in, or crack? By shooting up, v | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 79 | In the last 6 months, have you use substances), <u>that</u> were not prescr<br>cocaine? | | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | I prefer not to answer | XX | XX | XX |



Table 5.003. Summary of Patient Study Participants' Sexual History and Behaviors (Baseline), N=XX, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 14 | Have you h<br>oral sex. | nad sex in the last 6 months? This could be vaginal sex | x (penis in va | gina) OR anal sex (p | enis in butt) OR |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | How would | d you describe your sexual behaviors in the last 6 mor | nths? | | |
| | | I have had vaginal sex (penis in vagina) with only<br>1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex (penis in vagina) with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a bottom (penis in butt as a bottom) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a bottom (penis in butt as a bottom) with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top (penis in butt as a top) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top (penis in butt as a top) with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth, tongue, or lips on a vagina, penis, or butt) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth, tongue, or lips on a vagina, penis, or butt) with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 16 | How often | did you use a condom when you had sex in the last 6 | months? | | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 17 | In the last | 6 months, how would you describe the HIV status of | your sexual p | partner(s)? | I |
| | | I know that none of my sexual partners from the last 6 months have HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one sexual partner from the last 6 months is living with HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 18 | | ou know, were any of your sexual partner(s) from the<br>PrEP is a medication that prevents HIV. | last 6 montl | ns taking PrEP to pre | event HIV |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 19 | | oned that you had a least one partner in the last 6 m<br>e any of your partners taking HIV medications (antire | | | |
| | | Yes, my partner(s) was/were taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s) was/were taking HIV medications and was/were undetectable, meaning HIV tests were not finding the virus | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, my partner(s) was/were not taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether my partner(s) was/were taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 20 | Have you h | nad sex in the last 12 months? <i>This could be vaginal s</i> | ex (penis in v | agina) OR anal sex ( | penis in butt) OR |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 21 | | 12 months, have you experienced any incidents of se<br>m a partner? | exual violence | e, physical abuse, or | any other type of |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 22 | In the last | 12 months, have you exchanged things like money or | drugs for se | x with a sexual partr | ner? |
| | | Yes, I have a sexual partner things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave me things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.004. Summary of Patient Study Participants' Sexual History and Behaviors (Baseline), N=XX, Race, Dynamic Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 14 | Have you h<br>OR oral sex | ad sex in the last 6 months? <i>Th</i> | is could be vagin | al sex (penis in vag | gina) OR anal sex | (penis in butt) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | How would | l you describe your sexual beha | viors in the last 6 | 5 months? | | |
| | | I have had vaginal sex<br>(penis in vagina) with only<br>1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex<br>(penis in vagina) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a top)<br>with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a top)<br>with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips on<br>a vagina, penis, or butt)<br>with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips on<br>a vagina, penis, or butt)<br>with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 17 | In the last ( | 6 months, how would you desc | ribe the HIV stati | us of your sexual p | artner(s)? | |
| | | I know that none of my<br>sexual partners from the<br>last 6 months have<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one<br>sexual partner from the<br>last 6 months is living with<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 18 | As far as you know, were any of your sexual partner(s) from the last 6 months taking PrEP to prevent HIV infection? PrEP is a medication that prevents HIV. | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 19 | | oned that you had a least one p<br>e any of your partners taking H | | | | |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s) was/were taking HIV medications and was/were undetectable, | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | meaning HIV tests were not finding the virus | | | | |
| | | No, my partner(s)<br>was/were not taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether my<br>partner(s) was/were<br>taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 20 | Have you h<br>OR oral sex | and sex in the last 12 months? $7$ | his could be vagi | inal sex (penis in vo | agina) OR anal se: | x (penis in butt) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 21 | In the last 12 months, have you experienced any incidents of sexual violence, physical abuse, or any other type of trauma form a partner? | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 22 | In the last 12 months, have you exchanged things like money or drugs for sex with a sexual partner? | | | | | |
| | | Yes, I have a sexual partner things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave<br>me things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.005. Summary of Patient Study Participants' Sexual History and Behaviors (Baseline), N=XX, Race, Routine Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 14 | Have you h<br>OR oral sex | ad sex in the last 6 months? T | This could be vagin | al sex (penis in vag | gina) OR anal sex | (penis in butt) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | How would | l you describe your sexual bel | haviors in the last 6 | 5 months? | | |
| | | I have had vaginal sex<br>(penis in vagina) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex<br>(penis in vagina) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as<br>a bottom) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as<br>a bottom) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a<br>top) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a<br>top) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips<br>on a vagina, penis, or<br>butt) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips<br>on a vagina, penis, or<br>butt) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 16 | How often | did you use a condom when y | ou had sex in the | last 6 months? | | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 17 | In the last ( | 6 months, how would you des | cribe the HIV stat | us of your sexual p | artner(s)? | |
| | | I know that none of my<br>sexual partners from the<br>last 6 months have<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one<br>sexual partner from the<br>last 6 months is living<br>with HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 18 | | ou know, were any of your sex<br>PrEP is a medication that prev | | n the last 6 month | s taking PrEP to p | revent HIV |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 19 | | oned that you had a least one<br>e any of your partners taking H | | | | |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications and | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | was/were undetectable,<br>meaning HIV tests were<br>not finding the virus | | | | |
| | | No, my partner(s)<br>was/were not taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether<br>my partner(s) was/were<br>taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 20 | Have you h<br>OR oral sex | rad sex in the last 12 months? | This could be vag | inal sex (penis in vo | agina) OR anal se: | x (penis in butt) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 21 | In the last 12 months, have you experienced any incidents of sexual violence, physical abuse, or any other type of trauma form a partner? | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 22 | In the last : | 12 months, have you exchange | ed things like mor | ney or drugs for sex | with a sexual pa | rtner? |
| | | Yes, I have a sexual partner things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner<br>gave me things like drugs<br>or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.006. Summary of Patient Study Participants' Sexual History and Behaviors (Baseline), N=XX, Race, Total

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 14 | Have you h<br>OR oral sex | ad sex in the last 6 months? T | This could be vagin | al sex (penis in vag | gina) OR anal sex | (penis in butt) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | How would | l you describe your sexual bel | haviors in the last 6 | 5 months? | | |
| | | I have had vaginal sex<br>(penis in vagina) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex<br>(penis in vagina) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as<br>a bottom) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as<br>a bottom) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a<br>top) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a<br>top) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips<br>on a vagina, penis, or<br>butt) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips<br>on a vagina, penis, or<br>butt) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 16 | How often did you use a condom when you had sex in the last 6 months? | | | | | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 17 | In the last 6 months, how would you describe the HIV status of your sexual partner(s)? | | | | | |
| | | I know that none of my<br>sexual partners from the<br>last 6 months have<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one<br>sexual partner from the<br>last 6 months is living<br>with HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual<br>partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 18 | As far as you know, were any of your sexual partner(s) from the last 6 months taking PrEP to prevent HIV infection? PrEP is a medication that prevents HIV. | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 19 | You mentioned that you had a least one partner in the last 6 months who is living with HIV/AIDS. As far as you know, were any of your partners taking HIV medications (antiretrovirals) to treat their HIV infection? | | | | | |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s) was/were taking HIV medications and | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | was/were undetectable,<br>meaning HIV tests were<br>not finding the virus | | | | |
| | | No, my partner(s)<br>was/were not taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether<br>my partner(s) was/were<br>taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 20 | Have you had sex in the last 12 months? This could be vaginal sex (penis in vagina) OR anal sex (penis in butt) OR oral sex. | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 21 | In the last 12 months, have you experienced any incidents of sexual violence, physical abuse, or any other type of trauma form a partner? | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 22 | In the last 12 months, have you exchanged things like money or drugs for sex with a sexual partner? | | | | | |
| | | Yes, I have a sexual partner things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner<br>gave me things like drugs<br>or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged<br>things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.007. Summary of Patient Study Participants' Sexual History and Behaviors (Baseline), N=XX, Ethnicity, Study Arms

| | | | Dynamic Implementation | | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) |
| 14 | Have you had sex in the last 6 months? This could be vaginal sex (penis in vagina) OR anal sex (penis in butt) OR oral sex. | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | How would you describe your sexual behaviors in the last 6 months? | | | | | |
| | | I have had vaginal sex (penis<br>in vagina) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex (penis<br>in vagina) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 16 | How often | did you use a condom when you | had sex in the last | 6 months? | | |


| | | | Dynamic Imp | olementation | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 17 | In the last ( | 6 months, how would you describ | e the HIV status o | of your sexual partr | ner(s)? | |
| | | I know that none of my<br>sexual partners from the last<br>6 months have HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one<br>sexual partner from the last<br>6 months is living with<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual<br>partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 18 | | ou know, were any of your sexual<br>PrEP is a medication that prevent. | | ne last 6 months ta | aking PrEP to prevent HIV | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 19 | | oned that you had a least one par<br>e any of your partners taking HIV | | | | |
| | | Yes, my partner(s) was/were taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s) was/were taking HIV medications and was/were undetectable, meaning HIV tests were not finding the virus | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic Imp | plementation | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) |
| | | No, my partner(s) was/were not taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether my<br>partner(s) was/were taking<br>HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 20 | Have you h | nad sex in the last 12 months? <i>Thi</i> s | s could be vagina | l sex (penis in vagin | na) OR anal sex (p | enis in butt) OR |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 21 | | 12 months, have you experienced<br>m a partner? | any incidents of | sexual violence, ph | ysical abuse, or a | any other type o |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 22 | In the last 12 months, have you exchanged things like money or drugs for sex with a sexual partner? | | | | | |
| | | Yes, I have a sexual partner<br>things like drugs or money<br>for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave<br>me things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | | _ | | A CONTRACTOR OF THE PARTY OF TH |



Table 5.008. Summary of Patient Study Participants' Sexual History and Behaviors (Baseline), N=XX, Ethnicity, Total

| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 14 | Have you h | ad sex in the last 6 months? <i>This</i> | could be vaginal sex (penis in vagina) | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | How would | l you describe your sexual behavi | ors in the last 6 months? | |
| | | I have had vaginal sex (penis<br>in vagina) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex (penis<br>in vagina) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I have had oral sex (mouth, tongue, or lips on a vagina, penis, or butt) with more than 1 partner | | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 16 | How often | did you use a condom when you | had sex in the last 6 months? | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | · · · · · · | · · · |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | · · · · · · | |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | XX | XX |
| | | None of the time | (XX.X%) | (XX.X%) |
| | | | XX | XX |
| | | I prefer not to answer | (XX.X%) | (XX.X%) |
| .7 | In the last ( | 6 months, how would you describe t | | <u> </u> |
| .7 | III tile last t | | ne niv status oi your sexual par | tilei(s): |
| | | I know that none of my sexual partners from the last | XX | XX |
| | | 6 months have HIV/AIDS | (XX.X%) | (XX.X%) |
| | | I know that at least one | | |
| | | sexual partner from the last | XX | XX |
| | | 6 months is living with | (XX.X%) | (XX.X%) |
| | | HIV/AIDS | , , | , , |
| | | I do not know my sexual | XX | XX |
| | | partners' HIV status | (XX.X%) | (XX.X%) |
| | | | XX | XX |
| | | I prefer not to answer | (XX.X%) | (XX.X%) |
| 18 | | ou know, were any of your sexual par<br>PrEP is a medication that prevents H | | taking PrEP to prevent HIV |
| | | | XX | XX |
| | | No | (XX.X%) | (XX.X%) |
| | | | XX | XX |
| | | Yes | (XX.X%) | (XX.X%) |
| | | | XX | XX |
| | | I don't know | (XX.X%) | (XX.X%) |
| | | | XX | XX |
| | | I prefer not to answer | (XX.X%) | (XX.X%) |
| 19 | | oned that you had a least one partne<br>e any of your partners taking HIV me | | |
| | | Yes, my partner(s) was/were | XX | XX |
| | | taking HIV medications | (XX.X%) | (XX.X%) |
| | | Yes, my partner(s) was/were | | |
| | | taking HIV medications and | XX | XX |
| | | was/were undetectable, | (XX.X%) | (XX.X%) |
| | | meaning HIV tests were not finding the virus | | |
| | | | WW | V07 |
| | | No, my partner(s) was/were | XX<br>(YX Y%) | XX<br>(XX X%) |
| | | not taking HIV medications | (XX.X%) | (XX.X%) |
| | | I do not know whether my partner(s) was/were taking | XX | XX |
| | | HIV medications | (XX.X%) | (XX.X%) |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 20 | Have you h | ad sex in the last 12 months? <i>Thi</i> | is could be vaginal sex (penis in vagin | na) OR anal sex (penis in butt) OR |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 21 | | 12 months, have you experienced<br>m a partner? | d any incidents of sexual violence, ph | ysical abuse, or any other type of |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 22 | In the last 12 months, have you exchanged things like money or drugs for sex with a sexual partner? | | | |
| | | Yes, I have a sexual partner things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave<br>me things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.09. Summary of Patient Study Participants' Sexual History and Behaviors (Baseline), N=XX, Gender, Total

| Question<br>Number | Question | Response | Men who have sex with men<br>(N = XX)<br>n (%) | Transgender Men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 14 | Have you h | ad sex in the last 6 months? <i>This</i> | could be vaginal sex (penis in vagina) ( | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | How would | l you describe your sexual behavi | ors in the last 6 months? | |
| | | I have had vaginal sex (penis<br>in vagina) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex (penis<br>in vagina) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 16 | How often | did you use a condom when you | had sex in the last 6 months? | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Men who have sex with men (N = XX) | Transgender Men (N = XX) |
|---|---|---|---|---|
| | | | n (%) | n (%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | · · · | <u> </u> |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | XX | XX |
| | | A little of the time | (XX.X%) | (XX.X%) |
| | | | XX | XX |
| | | None of the time | (XX.X%) | (XX.X%) |
| | | | XX | XX |
| | | I prefer not to answer | (XX.X%) | (XX.X%) |
| <br>17 | In the last 6 | 6 months, how would you describ | e the HIV status of your sexual partne | |
| | III the last ( | I know that none of my | e the fire status of your sexual partite | . (3). |
| | | sexual partners from the last | XX | XX |
| | | 6 months have HIV/AIDS | (XX.X%) | (XX.X%) |
| | | I know that at least one | | |
| | | sexual partner from the last | XX | XX |
| | | 6 months is living with | (XX.X%) | (XX.X%) |
| | | HIV/AIDS | | |
| | | I do not know my sexual | XX | XX |
| | | partners' HIV status | (XX.X%) | (XX.X%) |
| | | I prefer not to answer | XX | XX |
| | | | (XX.X%) | (XX.X%) |
| 18 | | ou know, were any of your sexual<br>PrEP is a medication that prevents | partner(s) from the last 6 months taki<br>s HIV. | ng PrEP to prevent HIV |
| | | No | XX | XX |
| | | NO | (XX.X%) | (XX.X%) |
| | | Yes | XX | XX |
| | | 165 | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX |
| | | T don't know | (XX.X%) | (XX.X%) |
| | | I prefer not to answer | XX | XX |
| | | i prefer flot to answer | (XX.X%) | (XX.X%) |
| 19 | | | tner in the last 6 months who is living medications (antiretrovirals) to treat t | |
| | | Yes, my partner(s) was/were | XX | XX |
| | | taking HIV medications | (XX.X%) | (XX.X%) |
| | | Yes, my partner(s) was/were | | |
| | | taking HIV medications and | XX | XX |
| | | was/were undetectable, | (XX.X%) | (XX.X%) |
| | | meaning HIV tests were not finding the virus | | . , |
| | | | XX | XX |
| | | No, my partner(s) was/were not taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether my | (700070) | (////////////////////////////////////// |
| | | partner(s) was/were taking | XX | XX |
| | 1 | HIV medications | (XX.X%) | (XX.X%) |



| Question<br>Number | Question | Response | Men who have sex with men<br>(N = XX)<br>n (%) | Transgender Men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 20 | Have you h | and sex in the last 12 months? <i>Thi</i> | is could be vaginal sex (penis in vagina) | OR anal sex (penis in butt) OR |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 21 | | 12 months, have you experienced<br>m a partner? | d any incidents of sexual violence, phys | ical abuse, or any other type of |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 22 | In the last 12 months, have you exchanged things like money or drugs for sex with a sexual partner? | | | |
| | | Yes, I have a sexual partner things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave<br>me things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.101. Summary of Patient Study Participants' HIV and PrEP Knowledge (Baseline), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 7 | Do you personally know of someone living with HIV? | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 9 | Before enrolling in this study, had you ever heard of people who do not have HIV taking oral PrEP pills (the medicine taken every day to reduce the risk of getting HIV)? | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 10 | Do you personally <b>know</b> of a person or people who have ever taken oral PrEP? | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.102. Summary of Patient Study Participants' HIV and PrEP Knowledge (Baseline), N=XX, Scale Questions, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 8 | Please answer true or false to the following s | tatements abo | out HIV. | | |
| А | A person who has HIV can look healthy. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | There is a vaccine that can stop you from getting HIV. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | l don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | A person will NOT get HIV if they are taking antibiotics. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | If you only have sex once with a partner, you cannot get HIV from them. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | People living with HIV on HIV medications cannot spread HIV. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Everybody who has HIV knows that they have HIV. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | A natural (lamb skin) condom works better against HIV than a latex condom. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | When using condoms during sex, it is safer to use water-based lubricants than oilbased lubricants. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.103. Distributional Characteristics of Patient Study Participants' HIV and PrEP Knowledge (Baseline), N=XX, Scale Questions, Overall Score

| 8. Please answer<br>true or false to the<br>following statements<br>about HIV. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | 0.xx |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Gender | | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Not Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| | | | Dyna | amic Implement | ation | | | |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Gender | | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |



| 8. Please answer<br>true or false to the<br>following statements<br>about HIV. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Not Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| | | | Rou | tine Implementa | ation | | | |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Gender | | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Not Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |

Mean score = mean of responses to all of the items under 8 save for A and E; "Don't know" responses coded as false.



Table 5.104. Summary of Patient Study Participants' Perception of Stigma Associated with PrEP Usage (Baseline), N=XX, Stigma, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 13 | To what extent do you agree with each | h of the following : | statements about | PrEP? | |
| А | My <i>friends</i> would be supportive of me taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | People experience problems when they tell their sexual partner(s) they are taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | People experience negative judgement because they take PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | My <i>family</i> would be supportive of me taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Completely<br>agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | People taking PrEP receive praise for being responsible. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | I would feel ashamed to take PrEP in front of others. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | Someone taking PrEP would be seen by others as having sex with a lot of different people. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | People on PrEP are taking care of their health. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| I | People talking PrEP experience verbal harassment. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| J | I would not want others to know if I was taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| K | Someone taking PrEP should keep their pills hidden. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| L | I would feel proud to take PrEP every day. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| M | I would have sex with someone who is taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.105. Distributional Characteristics of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Stigma, Overall Score

| 13. To what extent do you agree with each of the following statements about PrEP? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | X.XX |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Gender | | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Dynamic Implementation | | | | | | | | |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Gender | | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |



| 13. To what extent do you agree with each of the following statements about PrEP? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Routine Implementation | | | | | | | | |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Gender | | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Not Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |

Mean score = mean of responses to all of the items under 13 save for J with the following items are reverse scored: A,D,E,H,L, & M. Higher total score indicates higher stigma.



Table 5.106. Summary of Patient Study Participants' Choice of APRETUDE (Baseline), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 11 | Before enrolling in this study, had<br>you heard of APRETUDE, the long<br>acting injectable (shot) form of<br>PrEP? | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 12 | Where did you first learn about APR | ETUDE? | | | |
| | | Healthcare provider<br>(e.g., doctor, nurse) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Community organization | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Friend | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Family Member | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Internet (website) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Internet (social<br>media) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Advertisement (radio, magazine, television) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 29 | Why have you chosen to take (or sw | vitch to) APRETUDE? | | | |
| | | I never tried PrEP<br>before, but I want to<br>protect myself from<br>HIV | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I think APRETUDE is<br>the most effective<br>HIV prevention<br>method available | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will not have to<br>worry about HIV<br>every day | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will be able to have sex at any moment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | and I know I am<br>protected | | | |
| | | I want to keep taking<br>PrEP a secret | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I want a prevention<br>option that is more<br>convenient for my life | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | My sexual partner<br>will not know I am<br>taking PrEP | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | My doctor suggested I take APRETUDE | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I won't have to<br>remember to take<br>PrEP everyday | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I often forget to take pills | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I want to try a new<br>approach and see if it<br>fits into my life | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer an injection<br>to PrEP because I<br>have difficulty<br>swallowing pills | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned<br>about the long-term<br>side effects of my<br>oral PrEP | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not have to<br>worry or stress about<br>missing a dose like<br>oral PrEP | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I would feel more<br>comfortable not<br>taking pills with me<br>when going out with<br>people/friends | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I would feel more<br>comfortable not<br>taking pills with me<br>when travelling | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I hope that injections<br>will be easier on my<br>stomach/digestive<br>system | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 30 | Do you have any concerns about A | PRETUDE? | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 31 | What concerns do you have about APRETUDE? | | | | |
| | | Pain or soreness from the injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other side effects<br>from APRETUDE | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Fear of needles | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Being approved by<br>my insurance to take<br>it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Having to take oral<br>PrEP first before I<br>take APRETUDE<br>injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Possible long-term<br>effects of the<br>injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | How it affects other medications I take | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Scheduling or<br>rescheduling<br>injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Forgetting my appointment for the injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Missing an injection<br>visit and then getting<br>HIV | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Missing work for the injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Making time to go to the clinic/practice for the injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Travelling to the clinic/practice for the injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Limited<br>clinic/practice hours<br>for injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Childcare/caregiver<br>responsibilities<br>during injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Lack of privacy at injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | My dignity not being<br>respected during<br>injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | People asking why I<br>go to the<br>clinic/doctor every 2<br>months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | My hectic lifestyle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | My travel or holiday schedules | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Taking medication<br>during times when I<br>am not having sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The medication not<br>being effective at<br>preventing HIV | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Worrying people<br>would think I have<br>HIV | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Worrying that people<br>would think I have a<br>lot of sexual partners<br>because I am on CAB<br>LA for PrEP | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Worrying about my<br>privacy because I live<br>with someone | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.107 Summary of Knowledge of APRETUDE and Utility of Implementation Strategies (Baseline), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 67 | Overall, how much do you kno | ow about APRETUDE? | | | |
| | | A lot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Nothing | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 68 | How confident are you with yo | How confident are you with your current level of knowledge about APRETUDE? | | | |
| | | Extremely confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 69 | How helpful was the information, if any, shared by the medical staff about APRETUDE? | | | | |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not receive any<br>information from medical staff | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 70 | How helpful has each of the fo | ollowing materials been in learning | about APRE | ETUDE? | |
| А | Getting Started Brochure –<br>the brochure that gives you<br>an overview of how to get<br>started with APRETUDE | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Patient Brochure – this<br>brochure helps you<br>understand the process of<br>receiving APRETUDE<br>injections, including side<br>effects and insurance<br>information | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | Let's talk about HIV & PrEP<br>video – the video giving key<br>facts about HIV and PrEP<br>options (DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| D | The APRETUDE Myths and Facts video – the game show video addressing common myths about APRETUDE (DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| E | The What to Expect video which shows you what to expect during the APRETUDE process (DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| F | The ViiV Connect Video,<br>which tells you about the<br>ViiV Connect program and<br>frequently asked questions<br>(DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| G | The study website where you access APRETDUE information (RI) | Very helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| Н | The study app where you access APRETUDE information (DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |



Table 5.108. Attitude Regarding APRETUDE and Utility of Implementation Strategies (Baseline), N=XX

| Question | | | | | | |
|---|---|---|---|---|---|---|
| 75. Overall, ho | w are you feeling about<br>DE? | Very positive | Somewhat positive | Neither<br>positive nor<br>negative | Somewhat<br>negative | Very<br>negative |
| Study Arms | | | | | | |
| | Total<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Routine<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynamic | Implementation | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routine I | mplementation | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | | | Response | | |
|---|---|---|---|---|---|---|
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Dyna | amic Implementation | | | | | |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Rout | ine Implementation | | | | | |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Total | I | | | | | |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Total | 1 | | | | | |
| | Men who have sex<br>with men<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Transgender men<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.109. Summary of Patient Study Participant Acquisition Process (Baseline), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 71 | Have you e | ever heard of ViiV Connect? | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 72 | Where did | you learn about ViiV Connect? | | | |
| | | My healthcare provider/healthcare clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The ViiV Connect video on the study app<br>(DI arm only) | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | ViiV Connect brochure | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A friend/family member told me | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The ViiV Connect website | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.110. Summary of Patient Study Participant Acquisition Process, Insurance (Baseline), N=XX

| Question | | | | Response | | |
|---|---|---|---|---|---|---|
| | extent do you agree with following statements? | Completely Agree | Agree | Neither<br>agree nor<br>disagree | Disagree | Completely<br>disagree |
| A. The sta | ff at the clinic helped me un | derstand the insurance a | pproval proces | S | | |
| Study Arms | | | | | | |
| | Total<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Routine<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynan | nic Implementation | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routir | ne Implementation | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | | | Response | | |
|---|---|---|---|---|---|---|
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Dy | namic Implementation | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Ro | utine Implementation | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Tot | | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Tota | al | | | | | |
| | Men who have sex<br>with men<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Transgender men | | | | | |



| Question | | | | Response | | |
|---|---|---|---|---|---|---|
| | Total<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Routine<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynami | ic Implementation | | -1 | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routine | Implementation | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Total | | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | | | Response | | |
|---|---|---|---|---|---|---|
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Dynam | nic Implementation | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Routin | e Implementation | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Total | | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Total | | | | | | |
| | Men who have sex<br>with men<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Transgender men<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.111. Summary of Patient Study Participants' Perception of Stigma Associated with PrEP Usage (Baseline), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 27 | Before deciding to take or switch to AF<br>PrEP? <i>Do not count oral Cabotegravir</i> µ | | | | while taking oral |
| А | Side effects | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Experienced Insurance issues | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | The cost being too high | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | Problems remembering to take oral PrEP | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | Concerns about running out of oral PrEP | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Feeling you had to hide oral PrEP from others | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | Thinking oral PrEP is not convenient for you | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | Difficulty paying for oral PrEP | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| I | Difficulty swallowing oral PrEP | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| J | Worried about potential interaction with other medicines | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| К | Not liking to take oral PrEP so frequently | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| L | Worrying that people may find out you are taking oral PrEP | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| М | Worrying that people will think you have HIV if they see you taking oral PrEP | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| N | Worrying that people would think you have a lot of sexual partners because you take oral PrEP | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 0 | Worrying about your privacy because you live with someone | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Р | Worrying about your privacy<br>because you're on you parent's<br>health insurance plan | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Q | Other concerns (please specify) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 28 | What side effects have you experience | ed on oral PrEP? | | | |
| | | Headache | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Diarrhea | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Nausea | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Vomiting | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Rash | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |


| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Loss of appetite | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Weight loss | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Stomach pain | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | New or worse<br>kidney<br>problems | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bone<br>problems | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Gas or<br>bloating | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.112. Summary of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 23 | Have you take<br>receiving APR | en oral PrEP in the last 6 months? <i>Do not count ETUDE</i> | oral cabotegravi | r pills you might be | taking before |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 24 | How would yo | ou describe your oral PrEP use in the last 6 mon | ths? | | |
| | | I take oral PrEP consistently (at least 5 or<br>more days a week,) each week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP consistently (at least 5 or<br>more days a week) off and on when I need<br>to, but not every week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP for <u>less than</u> 5 days a week<br>each week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP on demand/when I need it;<br>this is also called PrEP 2-1-1 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 25 | How many m | onths in a row have you been taking oral PrEP? | | | |
| | | Less than 2 month | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 2 to 6 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 7 to 12 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 12 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | l don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 26 | Have you eve | r taken oral PrEP? | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.113. Summary of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Race, Dynamic Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 23 | Have you taken oral PrE receiving APRETUDE | P in the last 6 months? <i>Do not c</i> | ount oral cabo | otegravir pills yc | ou might be tal | king before |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 24 | How would you describe | e your oral PrEP use in the last 6 | months? | | | |
| | | I take oral PrEP<br>consistently (at least 5<br>or more days a week,)<br>each week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP<br>consistently (at least 5<br>or more days a week)<br>off and on when I need<br>to, but not every week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP for <u>less</u><br><u>than</u> 5 days a week each<br>week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP on<br>demand/when I need it;<br>this is also called PrEP 2-<br>1-1 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 25 | How many months in a r | row have you been taking oral P | rEP? | | | |
| | | Less than 2 month | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 2 to 6 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 7 to 12 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 12 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 26 | Have you ever taken ora | ll PrEP? | | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.114. Summary of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Race, Routine Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 23 | Have you taken oral Pr receiving APRETUDE | EP in the last 6 months? <i>Do not c</i> | ount oral cabo | tegravir pills yc | ou might be tal | king before |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 24 | How would you describ | pe your oral PrEP use in the last 6 | months? | | | |
| | | I take oral PrEP<br>consistently (at least 5<br>or more days a week,)<br>each week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP<br>consistently (at least 5<br>or more days a week)<br>off and on when I need<br>to, but not every week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP for <u>less</u><br><u>than</u> 5 days a week<br>each week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP on<br>demand/when I need it;<br>this is also called PrEP<br>2-1-1 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 25 | How many months in a | row have you been taking oral P | rEP? | | | |
| | | Less than 2 month | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 2 to 6 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 7 to 12 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 12 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 26 | Have you ever taken o | ral PrEP? | | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.115. Summary of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Race, Total

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 23 | Have you taken oral F receiving APRETUDE | PrEP in the last 6 months? <i>Do not c</i> | ount oral cabo | tegravir pills yc | ou might be tak | king before |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 24 | How would you descr | ibe your oral PrEP use in the last 6 | months? | | | |
| | | I take oral PrEP<br>consistently (at least 5 or<br>more days a week,) each<br>week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP<br>consistently (at least 5 or<br>more days a week) off<br>and on when I need to,<br>but not every week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP for <u>less</u><br><u>than</u> 5 days a week each<br>week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP on<br>demand/when I need it;<br>this is also called PrEP 2-<br>1-1 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 25 | How many months in | a row have you been taking oral P | rEP? | | | |
| | | Less than 2 month | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 2 to 6 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 7 to 12 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 12 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 26 | Have you ever taken | oral PrEP? | | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.116. Summary of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Ethnicity, Study Arms

| | | | Dynamic Im | olementation | Routine Im | plementation |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| 23 | Have you taken ora<br>receiving APRETUDI | l PrEP in the last 6 mon <sup>.</sup><br>E | ths? Do not count | t oral cabotegravir | pills you might i | be taking before |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 24 | How would you des | cribe your oral PrEP use | e in the last 6 mo | nths? | | |
| | | I take oral PrEP consistently (at least 5 or more days a week,) each week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP consistently (at least 5 or more days a week) off and on when I need to, but not every week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral<br>PrEP for <u>less</u><br><u>than</u> 5 days a<br>week each<br>week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral<br>PrEP on<br>demand/when<br>I need it; this<br>is also called<br>PrEP 2-1-1 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 25 | How many months | in a row have you been | taking oral PrEP? | ) | I | |
| | | Less than 2<br>month | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 2 to 6 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic Im | plementation | Routine Im | plementation |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| | | 7 to 12<br>months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 12<br>months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 26 | Have you ever taken ora | al PrEP? | | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.117. Summary of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Ethnicity, Total

| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 23 | Have you taken oral PrEP receiving APRETUDE | in the last 6 months | ? Do not count oral cabotegravir p | oills you might be taking before |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to<br>answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 24 | How would you describe | your oral PrEP use in | the last 6 months? | |
| | | I take oral PrEP<br>consistently (at<br>least 5 or more<br>days a week,)<br>each week | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP<br>consistently (at<br>least 5 or more<br>days a week) off<br>and on when I<br>need to, but not<br>every week | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP<br>for <u>less than</u> 5<br>days a week<br>each week | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP<br>on<br>demand/when I<br>need it; this is<br>also called PrEP<br>2-1-1 | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 25 | How many months in a ro | ow have you been ta | king oral PrEP? | |
| | | Less than 2<br>month | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 2 to 6 months | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 7 to 12 months | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 12<br>months | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 26 | Have you ever taken oral | PrEP? | | |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to<br>answer | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.118. Summary of Patient Study Participants' History and Perception of PrEP Usage (Baseline), N=XX, Gender, Total

| Question<br>Number | Question | Response | Men who have sex with men<br>(N = XX)<br>n (%) | Transgender Men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 23 | Have you ta<br>receiving AP | | s? Do not count oral cabotegravir pil | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 24 | How would | you describe your oral PrEP use | in the last 6 months? | |
| | | I take oral PrEP consistently<br>(at least 5 or more days a<br>week,) each week | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | r | I take oral PrEP consistently<br>(at least 5 or more days a<br>week) off and on when I<br>need to, but not every week | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP for <u>less than</u><br>5 days a week each week | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I take oral PrEP on<br>demand/when I need it; this<br>is also called PrEP 2-1-1 | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 25 | How many r | months in a row have you been t | aking oral PrEP? | |
| | | Less than 2 month | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 2 to 6 months | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 7 to 12 months | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 12 months | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 26 | Have you ev | er taken oral PrEP? | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.201. Distributional Characteristics of Acceptability of Intervention (AIM) (APRETUDE) (PSP) (Baseline), N=XX

| 32. AIM APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Dynamic Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 32. AIM APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



Table 5.202. Distributional Characteristics of Feasibility of Intervention (FIM) (APRETUDE) (PSP) (Baseline), N=XX

| 33. FIM APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Dynamic Implementation | | | | | | | |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 33. FIM APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | | | | | | | |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



Table 5.203. Distributional Characteristics of Accessibility of Intervention (AIM) (Telehealth) (PSP) (Baseline), N=XX

| 34. AIM Telehealth. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | · · · |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Dynamic Implementation | | | | | | | |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 34. AIM Telehealth. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | | | | | | | |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



Table 5.204. Distributional Characteristics of Feasibility of Intervention (FIM) (Telehealth) (PSP) (Baseline), N=XX

| 35. FIM Telehealth. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Dynamic Implementation | | | | | | | |
| Study Arm | | | | | | | |
| Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 35. FIM Telehealth. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | | | | | | | |
| Study Arm | | | | | | | |
| Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



Table 5.205. Summary of Acceptability of Intervention (AIM) (APRETUDE) (PSP) (Baseline), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 32 | Please indicate how much y | ou agree with each sta | atement based | on your current expecta | ations of APRETUDE. |
| | I believe APRETUDE will meet my approval for preventing HIV. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | APRETUDE for the prevention of HIV is appealing to me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I think I will <b>like</b> APRETUDE for the prevention of HIV. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I welcome APRETUDE for the prevention of HIV | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.206. Summary of Feasibility of Intervention (FIM) (APRETUDE) (PSP) (Baseline), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 33 | Please indicate how much y | ou agree with each sta | atement based | on your current expecta | itions of APRETUDE. |
| | Receiving APRETUDE injection every 2-months seems workable in my life | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Receiving APRETUDE injection every 2-months seems possible in my life | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Receiving APRETUDE injection every 2-months seems doable in my life | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Receiving APRETUDE injection every 2-months seems easy in my life | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.207. Summary of Acceptability of Intervention (AIM) (Telehealth) (PSP) (Baseline), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 34 | Please indicate how much you agree with each statement based on your current perceptions and experience with telehealth. | | | | |
| | Using telehealth for APRETUDE services <b>meets my approval</b> . | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Using telehealth for APRETUDE services is appealing to me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I think I will <b>like</b> using<br>telehealth for APRETUDE<br>services. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I welcome using telehealth for APRETUDE services. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.208. Summary of Feasibility of Intervention (FIM) (Telehealth) (PSP) (Baseline), N=XX

| | | • | | | |
|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
| 35 | Please indicate how much you agree with each statement based on your current perceptions and exp<br>with telehealth. | | | | |
| | Using telehealth for APRETUDE services <b>seems</b> workable in my life. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Using telehealth for APRETUDE services <b>seems possible</b> in my life. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Using telehealth for APRETUDE services <b>seems doable</b> in my life. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Using telehealth for APRETUDE services <b>seems easy</b> in my life. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.301. Summary of Feasibility and Acceptability of Telehealth (Baseline), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 36 | | viders offer any type of telehea<br>a portal to check documents? | Ith care, such as | video or phone cor | nsultation, online |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | Have you ever used any of the | telehealth care options that yo | our healthcare p | rovider or clinic offe | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | | convenient do you think it woul<br>well with your life activities and | | | or APRETUDE? <i>By</i> |
| А | Completing relevant clinic visit forms online | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Your doctor ordering an HIV test kit and sending it to your home for you to test yourself | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| С | Your doctor ordering an HIV test at a lab near your home where you can go to take the test | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | Video chatting with your doctor | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | Receiving reminders (e.g.,<br>text, email) about your<br>scheduled injection<br>appointment | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Scheduling your injection appointment online to go to your clinic/doctor's office for the injection | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | Scheduling your injection appointment online for a nurse to come to your home and to give you the injection | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | Scheduling your injection appointment online to go to a pharmacy for the injection | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| I | Sending messages to your doctor online | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| J | Reviewing your health documents, such as test results, online | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Neither convenient nor | XX | XX | XX |
| | | inconvenient | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat inconvenient | XX | XX | XX |
| | | Somewhat inconvenient | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Very inconvenient | XX | XX | XX |
| | | very inconvenient | (XX.X%) | (XX.X%) | (XX.X%) |
| 39 | How comfortable are you or w | ould you be using telehealth to | receive APRETU | JDE services? | |
| | | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | XX | XX | XX |
| | | Somewhat comfortable | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Neither comfortable nor | XX | XX | XX |
| | | uncomfortable | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat uncomfortable | XX | XX | XX |
| | Somewna | Somewhat uncomfortable | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Manus and anti-late | XX | XX | XX |
| | | Very uncomfortable | (XX.X%) | (XX.X%) | (XX.X%) |



Table 5.302. Summary of Quality of Care for Patient Study Participants (Baseline), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 74 | To what extent do you agree v<br>clinic/provider? | vith each of the following sta | tements regarding | g your experience w | ith your |
| А | My provider explained<br>medical words that were<br>used so that I could<br>understand them. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | My provider encouraged me to ask questions. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | My provider really respected me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | My provider gave me<br>enough time to say what I<br>though was important. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | My provider listened carefully to what I had to say. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | Disagree | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | Completely disagree | (XX.X%) | (XX.X%) | (XX.X%) |
| F | My provider explained why tests were being done. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | My provider made me feel comfortable talking about personal things. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | My privacy was respected. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| I | My provider does not judge<br>me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| J | The provider had a respectful attitude towards my sexual orientation. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| K | The staff at the clinic does not judge me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| L | The staff at this clinic is kind and respectful to me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| M | I sometimes felt insulted<br>when the clinic staff spoke<br>to me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| N | I felt judged by the clinic staff for being on PrEP. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 0 | I felt judged by my provider for being on PrEP. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |


| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.303. Summary of Quality of Care for Patient Study Participants (Baseline), N=XX, Non-Score Questions

| Question | Response | | | |
|---|---|---|---|---|
| 74. To what extent do you agree with each of the following statements regarding your experience with your clinical/provider? | Completely Agree | Agree | Neither agree nor<br>disagree | Disagree |
| I. My provider does not judge me. | | | | |
| Study Arms | | | | |
| Total | XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Dynamic<br>Implementation | XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Routine<br>Implementation | XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Race, Dynamic Implementation | | | | |
| Asian | XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Black or African<br>American | XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| White | XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Other | XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Race, Routine Implementation | | | | |
| Asian | XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Black or African<br>American | XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | tal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | estion Response | | | | |
|---|---|---|---|---|---|
| n (%) | | | | | |
| Gender, Total | | | | | |
| Men v | who have sex<br>nen | XX | XX | XX | XX |
| N = XX | ( | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Trans | gender men | XX | XX | XX | XX |
| N = XX | < | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| J. The provider had a | respectful attitude | towards my sexual or | ientation. | | |
| Study Arms | | | | | |
| Total | | XX | XX | XX | XX |
| N = XX | < | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Dynar<br>Imple | mic<br>mentation | XX | XX | XX | XX |
| N = XX | < | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Routi<br>Imple | ne<br>mentation | XX | XX | XX | XX |
| N = XX | < | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Race, Dynamic Imple | mentation | | | | |
| Asian | | XX | XX | XX | XX |
| N = XX | ( | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Black<br>Amer | or African<br>can | XX | XX | XX | XX |
| N = XX | < | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| White | 2 | XX | XX | XX | XX |
| N = X | < | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Other | | XX | XX | XX | XX |
| N = X | < | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Race, Routine Implen | nentation | | | | |
| Asian | | XX | XX | XX | XX |
| N = X | < | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | k or African<br>erican | XX | XX | XX | XX |
| N = | XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | 5) | | | | |
| Whi | te | XX | XX | XX | XX |
| N = | XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | 5) | | | | |
| Oth | er | XX | XX | XX | XX |
| N = | XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | 5) | | | | |
| Race, Total | | | | | |
| Asia | n | XX | XX | XX | XX |
| N = | XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | 5) | | | | |
| | k or African<br>erican | XX | XX | XX | XX |
| N = | XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | 5) | | | | |
| Whi | te | XX | XX | XX | XX |
| N = | XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | 5) | | | | |
| Oth | er | XX | XX | XX | XX |
| N = | XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | 5) | | | | |
| Ethnicity, Dynamic | Implementation | | | | |
| Hisp | oanic or Latino | XX | XX | XX | XX |
| N = | XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | 5) | | | | |
| Not | Hispanic or Latino | XX | XX | XX | XX |
| N = | XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | 5) | | | | |
| Ethnicity, Routine Ir | mplementation | | | | |
| Hisp | anic or Latino | XX | XX | XX | XX |
| N = | XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | 5) | | | | |
| Not | Hispanic or Latino | XX | XX | XX | XX |
| N = | XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | 5) | | | | |
| Ethnicity, Total | | | | | |
| Hisr | oanic or Latino | XX | XX | XX | XX |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tot | al | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| K. The staff | at the clinic does not judge me | ). | | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynar | mic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | · |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | . , | , | , | ` ' |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African | XX | XX | XX | XX |
| | American | ^^ | ^^ | ^^ | ^^ |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dyna | amic Implementation | | | | I |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | <u> </u> | | | · · · · · |
| Ethnicity, Rout | ine Implementation | | 1 | 1 | I |
| • | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | . , | , , | , , | , , |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| Ethnicity, T | otal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, To | otal | | | | |
| | Men who have sex<br>with men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| L. The staff | f at this clinic is kind and respect | ful to me. | | | |
| Study Arms | S | | | | |
| | Total | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dyna | nmic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |



| Question | Response Response | | | | |
|---|---|---|---|---|---|
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routine | Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | ' | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dyn | amic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Rou | tine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | otal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, To | tal | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| M. I someti | mes felt insulted when the clini | c staff spoke to me. | | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynai | mic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | xx |
| | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | N = XX | (^^.^/0) | (///.///// | (,,,,,,,,,, | (, -) |
| | N = XX<br>n (%) | (^^.^/0) | (///.//0) | (70.07.75) | (* * |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routi | ne Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, D | ynamic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | Response | | | | |
|---|---|---|---|---|---|
| Ethnicity, Routine Implementation | | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, | Total | | | | ı |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | , | , , | . , | , , |
| Gender, T | | | I. | I | I |
| , | Men who have sex with men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| N. I felt ju | udged by the clinic staff for being | on PrEP. | I | I | |
| Study Arn | | | | | |
| | Total | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | , | , , | , | , , |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | - | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | * | | | · |
| Race, Dyr | namic Implementation | | 1 | 1 | I |
| . , | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | , , | , , | , , | , |
| | Black or African<br>American | XX | XX | XX | XX |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routir | ne Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | otal | | | | ı |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tot | al | | | | I |
| | Men who have sex with men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| O. I felt judg | ged by my provider for being or | n PrEP. | | | ı |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | - | - | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | · |
| Race, Dynar | mic Implementation | | 1 | 1 | I |
| . , | Asian | XX | XX | XX | XX |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Rou | ıtine Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Tot | al | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | on Response | | | |
|---|---|---|---|---|
| Ethnicity, Dynamic Implementation | | | | |
| Hispanic or La | tino XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Not Hispanic o | or Latino XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Ethnicity, Routine Implement | ation | | | |
| Hispanic or La | tino XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Not Hispanic o | or Latino XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Ethnicity, Total | | | | |
| Hispanic or La | tino XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Not Hispanic o | or Latino XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Gender, Total | | | | |
| Men who have with men | e sex XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Transgender r | nen XX | XX | XX | XX |
| N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |



Table 5.304. Summary of Quality of Care for Patient Study Participants (Baseline), N=XX, Score Questions

| Question | | | Re | esponse | |
|---|---|---|---|---|---|
| each of th | nat extent do you agree with<br>ne following statements<br>your experience with your<br>vider? | Completely Agree | Agree | Neither agree nor<br>disagree | Disagree |
| A. My pro | vider explained medical words | s that were used so that I | could understan | d them. | |
| Study Arm | ns | | | | |
| | Total | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dyn | namic Implementation | , | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Rou | itine Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | tal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | | | Response | | |
|---|---|---|---|---|---|
| n (%) | | | | | |
| Gender, Total | | | | | |
| Men who | have sex | XX | XX | XX | XX |
| N = XX | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Transgen | der men | XX | XX | XX | XX |
| N = XX | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| B. My provider encourag | ed me to ask que | estions. | | | |
| Study Arms | | | | | |
| Total | | XX | XX | XX | XX |
| N = XX | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Dynamic<br>Impleme | ntation | XX | XX | XX | XX |
| N = XX | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Routine<br>Impleme | ntation | XX | XX | XX | XX |
| N = XX | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Race, Dynamic Implemer | ntation | | | | |
| Asian | | XX | XX | XX | XX |
| N = XX | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Black or Americar | | XX | XX | XX | XX |
| N = XX | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| White | | XX | XX | XX | XX |
| N = XX | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Other | | XX | XX | XX | XX |
| N = XX | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Race, Routine Implemen | tation | | | | |
| Asian | | XX | XX | XX | XX |
| N = XX | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | I | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dyr | namic Implementation | | | | ı |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Rou | utine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Tot | al | | 1 | 1 | 1 |
| | Hispanic or Latino | XX | XX | XX | XX |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tot | al | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| C. My provi | der really respected me. | | | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynar | nic Implementation | | | | I |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | <u> </u> | | | · |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | <u> </u> | | | · |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | . , | . , | . , | , |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African | XX | XX | XX | XX |
| | American | ^^ | ^^ | ^^ | ^^ |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dyna | amic Implementation | | | | I |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | <u> </u> | | | · · · · · |
| Ethnicity, Rout | ine Implementation | | 1 | 1 | I |
| • | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | . , | , , | , , | , , |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| Ethnicity, T | otal | | I. | <u> </u> | ı |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, To | tal | | | | |
| | Men who have sex<br>with men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| D. My prov | rider gave me enough time to sa | y what I though was | s important. | | |
| Study Arms | S | | | | |
| | Total | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dyna | mic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routi | ne Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, D | ynamic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, R | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, T | Total | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, To | otal | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| E. My prov | vider listened carefully to what I | had to say. | | | |
| Study Arms | S | | | | |
| | Total | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dyna | amic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | (0() | | | | |
| | n (%) | | + | | |
| | Black or African American | XX | XX | XX | XX |
| | Black or African | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | (XX.X%) |
| | Black or African<br>American | | | | |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routin | e Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| Ethnicity, | Routine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, | Total | | | | ı |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | , | , , | . , | , , |
| Gender, T | | | I. | I | I |
| | Men who have sex with men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| F. My pro | vider explained why tests were b | eing done. | I | I | |
| Study Arn | | | | | |
| | Total | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | , | , , | , | , , |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | * | | | · |
| Race, Dyn | namic Implementation | | 1 | 1 | I |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | , , | , , | , , | , |
| | Black or African<br>American | XX | XX | XX | XX |



| Question | | | Response | | |
|---|---|---|---|---|---|
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routir | ne Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, D | ynamic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | otal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tot | al | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| G. My provi | der made me feel comfortable | talking about perso | nal things. | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | · |
| Race, Dynar | mic Implementation | | 1 | 1 | I |
| · • | Asian | XX | XX | XX | XX |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Rout | ine Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | | Resp | Response | | |
|---|---|---|---|---|---|
| Ethnicity, Dy | namic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | tal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tot | al | | | | |
| | Men who have sex<br>with men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| H. My privad | cy was respected. | | | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynan | nic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routir | ne Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, | Dynamic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, | Routine Implementation | | 1 | 1 | 1 |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, | Total | | | 1 | I |
| | Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, T | otal | | 1 | 1 | 1 |
| | Men who have sex<br>with men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | N = XX | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | , |



Table 5.305. Distributional Characteristics of Quality of Care for Patient Study Participants (Baseline), N=XX, Score Questions, Overall Score

| 74. To what extent do you agree with each of the following statements regarding your experience with your clinic/provider? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | 0.xx |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | - |
| Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | - |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | - |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | - |
| Gender | | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Transgender<br>Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Not Hispanic<br>or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Dynamic Implementat | ion | | | | | | | |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | - |



| 74. To what extent do you agree with each of the following statements regarding your experience with your clinic/provider? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | - |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | - |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | - |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Black or<br>African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Not Hispanic<br>or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | - |
| Routine Implementati | on | | | | | | | |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | - |
| Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | - |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | - |
| Black or<br>African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |



| 74. To what extent do you agree with each of the following statements regarding your experience with your clinic/provider? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |
| Not Hispanic<br>or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) | _ |

Mean score = mean of responses of items A-H. Responses were scored on a scale of 1-4 with higher scores indicating higher quality of care.


Table 5.306. Summary of Utility of Proposed Implementation Strategies (Baseline), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 56 | How useful do you think each | of the following will be in sup | porting you while | e taking APRETUDE? | |
| А | Brochures and other print materials to educate you on APRETUDE. | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Videos to educate you on HIV, PrEP, APRETUDE | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | A digital calendar specifically<br>made for APRETUDE to help<br>you plan your injections | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | Text reminders about your injections | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Fotomorphism follows | XX | XX | XX |
| | | Extremely useful | (XX.X%) | (XX.X%) | (XX.X%) |
| E | Email reminders about your injections | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Phone call reminders about your injections | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | Postal mail reminders about your injection | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | Having video or telephone appointments with your doctor | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Fortuna de la Contraction de l | XX | XX | XX |
| | | Extremely useful | (XX.X%) | (XX.X%) | (XX.X%) |
| | Doing IIIV/tasts at hama | Not at all useful | XX | XX | XX |
| I | Doing HIV tests at home | Not at all userul | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Not very useful | XX | XX | XX |
| | | Not very userui | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat useful | XX | XX | XX |
| | | Somewhat userui | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Useful | XX | XX | XX |
| | | Userui | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Extremely useful | XX | XX | XX |
| | | Extremely useful | (XX.X%) | (XX.X%) | (XX.X%) |
| | Doing HIV tests at a local lab | Nick challacter | XX | XX | XX |
| J | near you | Not at all useful | (XX.X%) | (XX.X%) | (XX.X%) |
| | | N | XX | XX | XX |
| | | Not very useful | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | Somewhat useful | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | Useful | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | Extremely useful | (XX.X%) | (XX.X%) | (XX.X%) |
| 1/ | Having a nurse come to your | Net et ell weeful | XX | XX | XX |
| K | home to conduct your HIV tests | Not at all useful | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Not very useful | XX | XX | XX |
| | | NOT VELY USEIUI | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat useful | XX | XX | XX |
| | | Joinewhat useful | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Useful | XX | XX | XX |
| | | OSCIUI | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Extremely useful | XX | XX | XX |
| | | Extremely useful | (XX.X%) | (XX.X%) | (XX.X%) |
| | Having a nurse come to your | Not at all useful | XX | XX | XX |
| L | home to give your injection | INOL AL AII USEIUI | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Nation | XX | XX | XX |
| | | Not very useful | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Camanula ak ful | XX | XX | XX |
| | | Somewhat useful | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Useful | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| М | Receiving transportation to the clinic/doctor's office for your injection | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| N | Knowing that your clinic/doctor's office offers injections on specific days of the week | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 0 | Ability to show up for your injection without an appointment | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Р | Appointments where you only get your injection and leave | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Q | Ability to schedule your injection appointments on weekends or after-hours | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| R | An app where you access<br>APRETUDE information | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| S | You and your doctor discussing the pros and cons (e.g., side effects, switching) of different PrEP options and together deciding which one is right for you | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.307. Summary of Patient Study Participants' Preferences/Acceptability of APRETUDE Information, Appointment Reminders, and Locations (Baseline), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 57 | If you had questions about APRETUDE <b>before enrolling in the study</b> , where did you find answers? | | | | |
| | | I didn't find answers to my questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Product website | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Written materials such as the study handbook | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Speaking to a healthcare provider | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Social Media | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Internet search | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Friends | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Family | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not had any<br>questions so far | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 58 | How did you receive reminder(s) about your first injection appointment? | | | | |
| | | Phone calls | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Texts/SMS messages | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Existing clinic app reminders | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Emails | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Reminder in the postal mail | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Face-to-face reminder from a healthcare provider | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Written<br>reminder/appointment card<br>with date and time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The study app (DI) | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | I did not receive any reminders | XX | xx | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| 59 | Which type of appointment | reminder(s) would you prefer? | | | |
| | | Phone calls | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Texts/SMS messages | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Existing clinic app reminders | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Emails | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Reminder in the postal mail | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Face-to-face reminder from a healthcare provider | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Written reminder/appointment card with date and time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Another type of reminder (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not wish to receive any reminders | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 60 | Where else would you consi | der receiving your injections? | | | |
| | | Retail pharmacy clinic (e.g.,<br>Minute Clinic, CVS) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other pharmacy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Hospital outpatient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Infusion center | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Community-based organization | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | STD/STI clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Department of Health clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | PrEP clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Community health center | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Mobile van | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Nurse coming to your home | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.401. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Baseline), N=XX, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 46 | How long are you willing you leave? | g to spend in the clinic/practice for your | injection visi | t from arrival at the | clinic to when |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How acceptable is comi | ng to the clinic every 2 months for an inj | jection? | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | How convenient are you with little trouble. | ur clinic's hours? By convenient, we mea | n fitting well | with your life activit | ies and plans, |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 49 | How easy or difficult do | you think it will be getting to the clinic e | | <u> </u> | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Easy | XX | XX | XX |
| | | , | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 50 | Approximately how lor | ng will it take you to get to the clinic/pract | ice from you | r home to receive y | our injection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 51 | How will you most like | ow will you most likely get to the clinic/practice to get your injections? | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drive a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 53 | Do you think you will n<br>your injection visits. | eed to seek additional childcare/eldercar | e/other care | to come to the clini | c/practice for |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 54 | How much time do you | think you will need to take off work to re | eceive injecti | ons? | |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will not need to take time off work for injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a whole day off for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a whole day off for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a partial day off for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a partial day off for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 55 | Do you think your time | off work for injections will be paid or unp | paid? | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.402. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Baseline), N=XX, Race, Dynamic Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 46 | How long are you willing to spend in the clinic/practice for your injection visit from arrival at the clinic to when you leave? | | | | | |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How accept | How acceptable is coming to the clinic every 2 months for an injection? | | | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | How convenient are your clinic's hours? By convenient, we mean fitting well with your life activities and plans, with little trouble. | | | | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 49 | How easy o | or difficult do you think it will be getting to the | clinic every 2 n | nonths for your | injection? | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 50 | Approxima | tely how long will it take you to get to the clinic | c/practice from | your home to | receive your i | njection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 51 | How will yo | ou most likely get to the clinic/practice to get y | our injections? | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drive a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 53 | Do you thii<br>your inject | nk you will need to seek additional childcare/el<br>ion visits. | dercare/other | care to come to | o the clinic/pra | actice for |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 54 | How much time do you think you will need to take off work to receive injections? | | | | | |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will not need to take time off work for injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a whole day off for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a whole day off for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a partial day off<br>for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a partial day off<br>for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 55 | Do you think your time off work for injections will be paid or unpaid? | | | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.403. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Baseline), N=XX, Race, Routine Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 46 | How long a you leave? | re you willing to spend in the clinic/practice fo | r your injectior | ı visit from arri | val at the clinio | to when |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How accep | table is coming to the clinic every 2 months fo | r an injection? | | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | How convenient are your clinic's hours? By convenient, we mean fitting well with your life activities and plans, with little trouble. | | | | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 49 | How easy c | or difficult do you think it will be getting to the | clinic every 2 m | nonths for your | injection? | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 50 | Approxima | tely how long will it take you to get to the clinic | c/practice from | your home to | receive your i | njection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 51 | How will yo | ou most likely get to the clinic/practice to get y | our injections? | I | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drive a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 53 | Do you thii<br>your inject | nk you will need to seek additional childcare/el<br>ion visits. | dercare/other | care to come to | o the clinic/pra | actice for |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 54 | How much | time do you think you will need to take off wo | rk to receive in | jections? | | |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will not need to take time off work for injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a whole day off<br>for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a whole day off for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a partial day off<br>for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a partial day off<br>for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 55 | Do you thi | nk your time off work for injections will be paid | or unpaid? | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.404. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Baseline), N=XX, Race, Total

| | <u> </u> | • | | | | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
| 46 | How long a you leave? | are you willing to spend in the clinic/practice fo | r your injectior | n visit from arri | val at the clinio | to when |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How accep | table is coming to the clinic every 2 months fo | r an injection? | | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | How convenient are your clinic's hours? By convenient, we mean fitting well with your life activities and plans, with little trouble. | | | | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 49 | How easy o | or difficult do you think it will be getting to the | clinic every 2 n | nonths for your | injection? | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 50 | Approxima | tely how long will it take you to get to the clini | c/practice from | your home to | receive your i | njection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 51 | How will yo | ou most likely get to the clinic/practice to get y | our injections? | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drive a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 53 | Do you thii<br>your inject | nk you will need to seek additional childcare/el<br>ion visits. | dercare/other | care to come to | o the clinic/pra | ictice for |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 54 | How much time do you think you will need to take off work to receive injections? | | | | | |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will not need to take time off work for injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a whole day off for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a whole day off for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a partial day off<br>for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a partial day off<br>for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 55 | Do you think your time off work for injections will be paid or unpaid? | | | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.405. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Baseline), N=XX, Ethnicity, Study Arms

| | | | Dynamic Im | plementation | Routine Im | olementation |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) |
| 46 | How long a you leave? | re you willing to spend in the clinic/pra | actice for your in | njection visit from | n arrival at the cl | inic to when |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How accep | table is coming to the clinic every 2 mo | onths for an inje | ction? | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | How conve<br>with little to | nient are your clinic's hours? <i>By conve.</i><br>rouble. | nient, we mean | fitting well with y | our life activitie. | s and plans, |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 49 | How easy o | or difficult do you think it will be getting | g to the clinic ev | ery 2 months for | your injection? | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic Im | plementation | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanio<br>or Latino<br>(N = XX)<br>n (%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 50 | Approxima | stely how long will it take you to get to t | he clinic/practi | ce from your hon | ne to receive yo | ur injection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 51 | How will y | ou most likely get to the clinic/practice | to get your inje | ctions? | ı | ı |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drive a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 53 | Do you thi<br>your inject | nk you will need to seek additional chilo<br>ion visits. | lcare/eldercare | other care to co | me to the clinic/ | practice for |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic Im | plementation | tion Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) |
| 54 | How much | n time do you think you will need to take | e off work to red | ceive injections? | | |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will not need to take time off work for injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a whole day off for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a whole day off for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a partial<br>day off for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a partial day off for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 55 | Do you think your time off work for injections will be paid or unpaid? | | | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.406. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Baseline), N=XX, Ethnicity, Total

| | | | Hispanic or Latino Not Hispanic or Latin | |
|---|---|---|---|---|
| Question | Question | Response | Hispanic or Latino<br>(N = XX) | Not Hispanic or Latino<br>(N = XX) |
| Number | Question | пезропае | n (%) | n (%) |
| 46 | How long a | are you willing to spend in the clinic/pract | | |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How accep | otable is coming to the clinic every 2 mont | ths for an injection? | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | How convenient are your clinic's hours? By convenient, we mean fitting well with your life activities and plans, with little trouble. | | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 49 | How easy | or difficult do you think it will be getting to | o the clinic every 2 months fo | r your injection? |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 50 | Approxima | ately how long will it take you to get to the | e clinic/practice from your ho | me to receive your injection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 51 | How will y | ou most likely get to the clinic/practice to | get your injections? | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drive a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 53 | Do you thi<br>your inject | nk you will need to seek additional childca<br>ion visits. | are/eldercare/other care to co | ome to the clinic/practice for |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 54 | How much | time do you think you will need to take o | off work to receive injections? | |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | I will not need to take time off work for injections | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a whole day off for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a whole day off for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a partial<br>day off for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a partial day off for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 55 | Do you think your time off work for injections will be paid or unpaid? | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.407. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Baseline), N=XX, Gender, Total

| Question<br>Number | Question | Response | Men who have sex with men<br>(N = XX)<br>n (%) | Transgender Men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 46 | How long a<br>you leave? | re you willing to spend in the clinic/pr | | |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 17 | How accep | table is coming to the clinic every 2 mo | onths for an injection? | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | How convenient are your clinic's hours? By convenient, we mean fitting well with your life activities and plans with little trouble. | | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 19 | How easy o | or difficult do you think it will be getting | g to the clinic every 2 months for yo | our injection? |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Men who have sex with men (N = XX) n (%) | Transgender Men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 50 | Approxima | ately how long will it take you to get to t | | <u> </u> |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 51 | How will y | ou most likely get to the clinic/practice | to get your injections? | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drive a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 53 | Do you thi<br>your inject | nk you will need to seek additional chilo<br>ion visits. | dcare/eldercare/other care to come | e to the clinic/practice for |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 54 | How much | time do you think you will need to take | e off work to receive injections? | |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Men who have sex with men<br>(N = XX)<br>n (%) | Transgender Men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | I will not need to take time off work for injections | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a whole day off for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a whole day off for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a partial day off for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I will probably need to take a partial day off for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 55 | Do you thi | nk your time off work for injections will | be paid or unpaid? | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.408. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 40 | Did you complete a S<br>study? | Sexual Health Assessment from your p | provider or clir | nic/practice before be | eing told about this |
| | | Vos | XX | XX | XX |
| | | Yes | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX |
| | | NO | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX |
| | | 1 don't know | (XX.X%) | (XX.X%) | (XX.X%) |
| 41 | Did your provider or | another person at the clinic/practice | discuss the re | sults of the assessme | nt with you? |
| | | Yes | XX | XX | XX |
| | | 163 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| 42 | Who discussed the re | esults of the assessment with you? | | | |
| | | My healthcare | XX | XX | XX |
| | | provider/doctor | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A nurse | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A social worker | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A peer educator | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Other (please specify) | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(YY Y%) | XX<br>(XX X%) |
| 42 | How boles in | nuccing the recults with wave and dis- | | (XX.X%) | (XX.X%) |
| 43 | now neiptul was disc | cussing the results with your provider | | | |
| | | Very helpful | XX<br>(VV VV) | XX<br>(VV VV) | XX<br>(VV V9/) |
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | | (^^.^%)<br>XX | (\lambda \lambda \lamb |
| | | Not at all helpful | XX<br>(XX.X%) | (XX.X%) | (XX.X%) |
| 44 | Please rate vour evo | erience with the Sexual Health Assess | | (70.070) | (70.000) |
| 44 | i lease rate your expi | chence with the Sexual Health ASSESS | JIIICIII | | |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | It was easy to take the<br>Sexual Health Assessment<br>on my digital device | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor sent<br>the assessment before my<br>appointment | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor was<br>assessing my sexual<br>health | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Why did you not complete t | he assessment? | | | |
| | | I did not receive a Sexual<br>Health Assessment from<br>my provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made me feel uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned about the privacy of my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share<br>sexual health information<br>with my doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand why<br>my doctor or clinic was<br>asking me to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.409. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Race, Dynamic Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 40 | Did you complete a Sexual Health Assessment from your provider or clinic/practice before being told about this study? | | | | | |
| | | Yes | XX | XX | XX | XX |
| | | res | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX | XX |
| | | NO | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX | XX |
| | | T don't know | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 41 | Did your provider or a | nother person at the clinic/ | practice dis | cuss the results of t | he assessment wi | th you? |
| | | Yes | XX | XX | XX | XX |
| | | 1 C3 | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX | XX |
| | | 140 | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX | XX |
| | | 1 don't know | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 42 | Who discussed the res | sults of the assessment with | n you? | | | |
| | | My healthcare | XX | XX | XX | XX |
| | | provider/doctor | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A nurse | XX | XX | XX | XX |
| | | 7 ( Turise | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A social worker | XX | XX | XX | XX |
| | | 7 ( Se siai Werker | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A peer educator | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Other (please specify | XX | XX | XX | XX |
| | | ) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 43 | How helpful was discu | issing the results with your | 1 | | · | I |
| | | Very helpful | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat helpful | XX | XX | XX | XX |
| | | <u> </u> | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A little helpful | XX | XX | XX (V/V V/O/) | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Not at all helpful | XX<br>(VV V%) | XX (XX XX XX | XX (VV V0/) | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 44 | Please rate your expe | rience with the Sexual Heal | th Assessme | ent | | |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | It was easy to take<br>the Sexual Health<br>Assessment on my<br>digital device | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor<br>sent the assessment<br>before my<br>appointment | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned<br>about the privacy of<br>my answers | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor<br>was assessing my<br>sexual health | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made<br>me feel<br>uncomfortable | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Why did you not compl | ete the assessment? | | | | |
| | | I did not receive a<br>Sexual Health<br>Assessment from my<br>provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |


| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made<br>me feel<br>uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned about<br>the privacy of my<br>answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share<br>sexual health<br>information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand<br>why my doctor or<br>clinic was asking me to<br>complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.410. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Race, Routine Implementation

| 40 stud | Yes No I do your provider or another Yes No I do o discussed the results of My l | n't know person at the clinic/ n't know the assessment with healthcare vider/doctor | xx (xx.x%) | XX (XX.X%) XX (XX.X%) XX (XX.X%) cuss the results of the second secon | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%) | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%) |
|---|---|---|---|---|---|---|
| | your provider or another Yes No I do I do O discussed the results of My I prov | person at the clinic/<br>n't know<br>the assessment with<br>healthcare<br>vider/doctor | (XX.X%) XX (XX.X%) XX (XX.X%) /practice disc XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) | (XX.X%) XX (XX.X%) XX (XX.X%) cuss the results of ti XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) | (XX.X%) XX (XX.X%) XX (XX.X%) he assessment w XX (XX.X%) XX (XX.X%) XX (XX.X%) XX XX XX XXXX%) | (XX.X%) XX (XX.X%) XX (XX.X%) ith you? XX (XX.X%) XX (XX.X%) XX (XX.X%) XX XX XX XXXXX%) |
| | your provider or another Yes No I do I do O discussed the results of My I prov | person at the clinic/<br>n't know<br>the assessment with<br>healthcare<br>vider/doctor | xx (xx.x%) xx (xx.x%) /practice dis- xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) | XX (XX.X%) XX (XX.X%) cuss the results of the second sec | XX (XX.X%) XX (XX.X%) he assessment w XX (XX.X%) XX (XX.X%) XX (XX.X%) XX X | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>ith you?<br>XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%) |
| | your provider or another Yes No I do o discussed the results of My I | person at the clinic/<br>n't know<br>the assessment with<br>healthcare<br>vider/doctor | (XX.X%) XX (XX.X%) /practice disc XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) | (XX.X%) XX (XX.X%) cuss the results of t XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) | (XX.X%) XX (XX.X%) he assessment w XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) | (XX.X%) XX (XX.X%) ith you? XX (XX.X%) XX (XX.X%) XX (XX.X%) XX X |
| | your provider or another Yes No I do o discussed the results of My I | person at the clinic/<br>n't know<br>the assessment with<br>healthcare<br>vider/doctor | XX (XX.X%) /practice disc XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) | XX (XX.X%) cuss the results of the second o | XX (XX.X%) he assessment w XX (XX.X%) XX (XX.X%) XX (XX.X%) XX XX XX XXXX%) | XX<br>(XX.X%)<br>ith you?<br>XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%) |
| | your provider or another Yes No I do o discussed the results of My l prov | person at the clinic/<br>n't know<br>the assessment with<br>healthcare<br>vider/doctor | (XX.X%) /practice disc XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) | (XX.X%) cuss the results of the second of t | (XX.X%) he assessment w XX (XX.X%) XX (XX.X%) XX (XX.X%) XX XX XX | (XX.X%) ith you? XX (XX.X%) XX (XX.X%) XX (XX.X%) XX XX XX XX |
| | your provider or another Yes No I do o discussed the results of My l prov | person at the clinic/<br>n't know<br>the assessment with<br>healthcare<br>vider/doctor | /practice dist | xX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%) | he assessment w XX (XX.X%) XX (XX.X%) XX (XX.X%) XX XX XX | xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%)<br>xx<br>(xx.x%) |
| | Yes No I do o discussed the results of My l prov | n't know<br>the assessment with<br>healthcare<br>vider/doctor | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>xyou?<br>XX<br>(XX.X%) | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%) | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%) | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%) |
| 42 Who | No I do o discussed the results of My l prov | the assessment with<br>healthcare<br>vider/doctor | (XX.X%) XX (XX.X%) XX (XX.X%) 7 you? XX (XX.X%) | (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) | (XX.X%) XX (XX.X%) XX (XX.X%) | (XX.X%) XX (XX.X%) XX (XX.X%) |
| 42 Who | No I do o discussed the results of My l prov | the assessment with<br>healthcare<br>vider/doctor | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>1 you?<br>XX<br>(XX.X%) | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%) | XX<br>(XX.X%)<br>XX<br>(XX.X%) | XX<br>(XX.X%)<br>XX<br>(XX.X%) |
| 42 Who | o discussed the results of My l | the assessment with<br>healthcare<br>vider/doctor | (XX.X%) XX (XX.X%) 1 you? XX (XX.X%) | (XX.X%) XX (XX.X%) XX (XX.X%) | (XX.X%)<br>XX<br>(XX.X%) | (XX.X%)<br>XX<br>(XX.X%) |
| 42 Who | o discussed the results of My l | the assessment with<br>healthcare<br>vider/doctor | XX<br>(XX.X%)<br>n you?<br>XX<br>(XX.X%) | XX<br>(XX.X%)<br>XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 42 Who | o discussed the results of My l | the assessment with<br>healthcare<br>vider/doctor | (XX.X%) n you? XX (XX.X%) | (XX.X%) XX (XX.X%) | (XX.X%) | (XX.X%) |
| 42 Who | My l | healthcare<br>vider/doctor | xx<br>(XX.X%) | XX<br>(XX.X%) | XX | XX |
| 42 Who | My l | healthcare<br>vider/doctor | XX<br>(XX.X%) | (XX.X%) | | |
| | prov | vider/doctor | (XX.X%) | (XX.X%) | | |
| | | | | ` ' | (XX.X%) | (XX.X%) |
| | A nu | ırse | XX | | | |
| | | | | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | A so | cial worker | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | A pe | eer educator | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | Othe | er (please specify | XX | XX | XX (VV V0/) | XX (XX X0() |
| | / | 1 | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | I do | n't know | XX<br>(VV V0/) | XX<br>(VV V0/) | XX<br>(VV V0/) | XX<br>(VV V0/) |
| 43 11 | المام الم | o rooulto with were | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 43 How | v helpful was discussing th | ie results with your | | | • | |
| | Very | / helpful | XX<br>(VV V0/) | XX<br>(VV V0/) | XX<br>(VV V0/) | XX<br>(VV V0/) |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | Som | newhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | A lit | tle helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not | at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 Plea | | | (^^.^/0) | | | |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | It was easy to take<br>the Sexual Health<br>Assessment on my<br>digital device | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor<br>sent the assessment<br>before my<br>appointment | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned<br>about the privacy of<br>my answers | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor<br>was assessing my<br>sexual health | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made<br>me feel<br>uncomfortable | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Why did you not compl | ete the assessment? | | | | |
| | | I did not receive a<br>Sexual Health<br>Assessment from my<br>provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made me feel uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned about<br>the privacy of my<br>answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share<br>sexual health<br>information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand<br>why my doctor or<br>clinic was asking me to<br>complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.411. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Race, Total

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 40 | Did you complete a Se study? | xual Health Assessment fro | om your pro | vider or clinic/pract | ice before being t | old about this |
| | | Yes | XX | XX | XX | XX |
| | | 163 | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX | XX |
| | | 140 | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX | XX |
| | | T doll t know | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 41 | Did your provider or a | nother person at the clinic | practice dis | cuss the results of t | he assessment wi | th you? |
| | | Yes | XX | XX | XX | XX |
| | | 103 | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX | XX |
| | | 110 | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 42 | Who discussed the res | sults of the assessment with | n you? | | | |
| | | My healthcare | XX | XX | XX | XX |
| | | provider/doctor | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A nurse | XX | XX | XX | XX |
| | | 7110130 | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A social worker | XX | XX | XX | XX |
| | | 7 ( SS SIGN WS) NO. | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A peer educator | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Other (please specify | XX | XX | XX | XX |
| | | ) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 43 | How helpful was discu | ssing the results with your | | | · | I |
| | | Very helpful | XX | XX | XX | XX |
| | | , ' | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat helpful | XX | XX | XX | XX |
| | | · · | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A little helpful | XX | XX | XX | XX |
| | | · · | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Not at all helpful | XX<br>(XX X0/) | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 44 | Please rate your exper | ience with the Sexual Heal | th Assessme | nt | | |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | It was easy to take<br>the Sexual Health<br>Assessment on my<br>digital device | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor<br>sent the assessment<br>before my<br>appointment | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned<br>about the privacy of<br>my answers | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor<br>was assessing my<br>sexual health | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made<br>me feel<br>uncomfortable | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Why did you not compl | ete the assessment? | | | | |
| | | I did not receive a<br>Sexual Health<br>Assessment from my<br>provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made<br>me feel<br>uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned about<br>the privacy of my<br>answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share<br>sexual health<br>information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand<br>why my doctor or<br>clinic was asking me to<br>complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.412. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Ethnicity, Study Arms

| | | | Dynamic Imp | plementation | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) |
| 40 | Did you comple<br>study? | ete a Sexual Health Assess | ment from your pr | ovider or clinic/pr | actice before bein | g told about this |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | Did your provid | ler or another person at t | he clinic/practice c | liscuss the results | of the assessment | with you? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 42 | Who discussed | the results of the assessr | nent with you? | | | |
| | | My healthcare provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 43 | How helpful wa | as discussing the results w | vith your provider o | or another person | at the clinic/practi | ce? |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX (XX.X%) | XX | XX | XX |



| | | | | (XX.X%) | (XX.X%) | (XX.X%) |
|---|---|---|---|---|---|---|
| 44 | Please rate your experience with the Sexual Health Assessment | | | | | |
| | It was easy to<br>take the Sexual<br>Health<br>Assessment on<br>my digital device | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my<br>doctor sent the<br>assessment<br>before my<br>appointment | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned<br>about the<br>privacy of my<br>answers | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my<br>doctor was<br>assessing my<br>sexual health | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
|---|---|---|---|---|---|---|
| | | Agree | XX | XX | XX | XX |
| | | Completely agree | (XX.X%)<br>XX<br>(XX.X%) | (XX.X%)<br>XX<br>(XX.X%) | (XX.X%)<br>XX<br>(XX.X%) | (XX.X%)<br>XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Why did you not complete the assessment? | | | | | |
| | | I did not receive a<br>Sexual Health<br>Assessment from<br>my provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | l forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know<br>how to complete<br>it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| The assessment<br>took too long to<br>complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
|---|---|---|---|---|
| The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| The assessment<br>made me feel<br>uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| I was concerned<br>about the privacy<br>of my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| I did not want to<br>share sexual<br>health<br>information with<br>my doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| I did not<br>understand why<br>my doctor or clinic<br>was asking me to<br>complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.413. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Ethnicity, Total

| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 40 | Did you complete a Sex<br>this study? | xual Health Assessment from your provide | r or clinic/practice befo | re being told about |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | Did your provider or an | nother person at the clinic/practice discuss | s the results of the asse | ssment with you? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 42 | Who discussed the results of the assessment with you? | | | |
| | | My healthcare provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 43 | How helpful was discus | How helpful was discussing the results with your provider or another person at the clinic/practice? | | |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX (XX.X%) | XX<br>(XX.X%) |
| 44 | Please rate your experi | ence with the Sexual Health Assessment | | |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | It was easy to take the Sexual<br>Health Assessment on my<br>digital device | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor sent the assessment before my appointment | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor was assessing my sexual health | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX | XX |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Why did you not complete the assessment? | | | |
| | | I did not receive a Sexual<br>Health Assessment from my<br>provider or clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made me feel uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | I was concerned about the privacy of my answers | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share sexual<br>health information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand why my<br>doctor or clinic was asking<br>me to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.414. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Gender

| Question<br>Number | Question | Response | Men who have<br>sex with men<br>(N = XX)<br>n (%) | Transgender men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 40 | Did you complete a Seath | xual Health Assessment from your provider | r or clinic/practice bef | ore being told about |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | Did your provider or ar | nother person at the clinic/practice discuss | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 42 | Who discussed the res | ults of the assessment with you? | | |
| | | My healthcare provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 43 | How helpful was discussing the results with your provider or another person at the clinic/practice? | | | |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX (XX.X%) | XX<br>(XX.X%) |
| 44 | Please rate your exper | ience with the Sexual Health Assessment | | |



| Question<br>Number | Question | Response | Men who have<br>sex with men<br>(N = XX)<br>n (%) | Transgender men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | It was easy to take the Sexual<br>Health Assessment on my<br>digital device | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor sent the assessment before my appointment | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor was assessing my sexual health | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX | XX |



| Question<br>Number | Question | Response | Men who have<br>sex with men<br>(N = XX)<br>n (%) | Transgender men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Why did you not complete the assessment? | | | |
| | | I did not receive a Sexual<br>Health Assessment from my<br>provider or clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | l forgot | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made me feel uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Men who have<br>sex with men<br>(N = XX)<br>n (%) | Transgender men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | I was concerned about the privacy of my answers | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share sexual<br>health information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand why my<br>doctor or clinic was asking<br>me to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.415. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Baseline), N=XX, Site Volume

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | High Volume<br>(N = XX)<br>n (%) | Low Volume<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 40 | Did you complete a Sexual study? | Did you complete a Sexual Health Assessment from your provider or clinic/practice before being told about this | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | Did your provider or anoth | er person at the clinic/practice | discuss the res | ults of the assessmer | nt with you? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 42 | Who discussed the results of the assessment with you? | | | | |
| | | My healthcare<br>provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 43 | How helpful was discussing the results with your provider or another person at the clinic/practice? | | | | |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please rate your experience | e with the Sexual Health Assess | ment | | |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | High Volume<br>(N = XX)<br>n (%) | Low Volume<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | It was easy to take the<br>Sexual Health Assessment<br>on my digital device | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor sent<br>the assessment before my<br>appointment | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor was<br>assessing my sexual<br>health | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | High Volume<br>(N = XX)<br>n (%) | Low Volume<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Why did you not complete the assessment? | | | | |
| | | I did not receive a Sexual<br>Health Assessment from<br>my provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | High Volume<br>(N = XX)<br>n (%) | Low Volume<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | The assessment made me feel uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned about the privacy of my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share<br>sexual health information<br>with my doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand why<br>my doctor or clinic was<br>asking me to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 5.416. Distributional Characteristics of Estimated Amount of Money Spent on Transportation for Each Injection Visit (Baseline), N=XX

| 52. On average, how much do you think transportation will cost round trip for each injection visit? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



Table 5.417 Summary of Optional Oral Lead-In vs. Direct to Injection (Baseline), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 61 | | Are you currently taking or did you take oral cabotegravir pills in preparation for your first APRETUDE injection? <i>This might have been called oral lead-in.</i> | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 62 | Whose ded | cision was it to use oral cabote | gravir pills in | preparation for your first inj | ection? |
| | | It was primarily my decision | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | It was a joint decision<br>between me and my<br>provider | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | It was primarily my provider's decision | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 63 | 63 What were the main reasons to use oral cabotegravir pills in preparation for your first i | | | | first injection? |
| | | The doctor just started me on them | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The doctor wanted to see<br>how I would react to<br>APRETUDE | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have a history of allergy<br>and reactions to<br>medications and the<br>doctor wanted to assess<br>if I would react to<br>APRETUDE | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The doctor wanted to be cautious with a new medication | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I wanted to make sure<br>the medication was safe | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I wanted to have<br>protection until the<br>injection arrived after it<br>was ordered | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The doctor wanted me to have protection until the injection arrived after it was ordered | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Other (please specify | XX<br>(xx x0/) | XX | XX |
| 64 | | rned would you have been if botegravir pills? | (XX.X%)<br>you had starte | (XX.X%) ed directly with the APRETUI | (XX.X%)<br>DE injections and not |
| | | Very concerned | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Concerned | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat concerned | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very concerned | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all concerned | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 65 | Whose decision was it to start directly with the injections and not use the pills/oral lead-in? | | | | |
| | | It was primarily my<br>decision | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | It was a joint decision<br>between me and my<br>provider | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | It was primarily my provider's decision | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 66 | What were the main reasons that you started directly with the injection and did not use the pill/oral lead-in? | | | | |
| | | I did not know that I<br>could start with the pills | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The doctor just started me with the injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was already on PrEP and<br>wanted to switch<br>immediately | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I believed the medication<br>is effective and didn't<br>want to wait | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | My doctor recommended that start with the injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not think I would<br>have any side effects | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



## **Table Shells for Month 6/7 Analysis**

| Table 6.000. | Demographic Characteristics of Patient Study Participants Completing Surveys (Month 6/7), N=XX | . 208 |
|---|---|---|
| Table 6.001. | Demographic Characteristics of Patient Study Participants (Month 6/7), N=XX | . 210 |
| Table 6.002. | Summary of Behaviors of Patient Study Participants (Month 6/7), N=XX | . 213 |
| Table 6.003. | Summary of Patient Study Participants' Sexual History and Behaviors (Month 6/7), N=XX, Study Arms | . 214 |
| Table 6.004. | Summary of Patient Study Participants' Sexual History and Behaviors (Month 6/7), N=XX, Race, Dynamic Implementation | . 217 |
| Table 6.005. | Summary of Patient Study Participants' Sexual History and Behaviors (Month 6/7), N=XX, Race, Routine Implementation | . 220 |
| Table 6.006. | Summary of Patient Study Participants' Sexual History and Behaviors (Month 6/7), N=XX, Race, Total | . 223 |
| Table 6.007. | Summary of Patient Study Participants' Sexual History and Behaviors (Month 6/7), N=XX, Ethnicity, Study Arms | . 226 |
| Table 6.008. | Summary of Patient Study Participants' Sexual History and Behaviors (Month 6/7), N=XX, Ethnicity, Total | . 229 |
| Table 6.009. | Summary of Patient Study Participants' Sexual History and Behaviors (Month 6/7), N=XX, Gender, Total | . 232 |
| Table 6.101. | Summary of Patient Study Participants' HIV and PrEP Knowledge (Month 6/7), N=XX | . 235 |
| Table 6.102. | Summary of Patient Study Participants' HIV and PrEP Knowledge (Month 6/7), N=XX, Scale Questions, Study Arms | . 236 |
| Table 6.103. | Distributional Characteristics of Patient Study Participants' HIV and PrEP Knowledge (Month 6/7), N=XX, Scale Questions, Overall Score | . 238 |
| Table 6.104. | Summary of Patient Study Participants' Perception of Stigma Associated with PrEP Usage (Month 6/7), N=XX, Stigma, Study Arms | . 240 |
| Table 6.105. | Distributional Characteristics of Patient Study Participants' Perception of Stigma<br>Associated with PrEP Usage (Month 6/7), N=XX, Stigma, Overall Score | . 244 |
| Table 6.106. | Summary of Patient Study Participants' Choice of APRETUDE (Month 6/7), N=XX | . 246 |
| Table 6.107. | Summary of Knowledge of APRETUDE and Utility of Implementation Strategies (Month 6/7), N=XX | . 249 |
| Table 6.108. | Attitude Regarding APRETUDE and Utility of Implementation Strategies (Month 6/7), N=XX | . 254 |
| Table 6.109. | Summary of Patient Study Participant Acquisition Process (Month 6/7), N=XX | . 256 |
| Table 6.110. | Summary of Patient Study Participant Acquisition Process, Insurance (Month 6/7), N=XX | . 257 |
| Table 6.201. | Distributional Characteristics of Acceptability of Intervention (AIM) (APRETUDE) (PSP) (Month 6/7), N=XX | . 267 |
| Table 6.202. | Distributional Characteristics of Feasibility of Intervention (FIM) (APRETUDE) (PSP) (Month 6/7) N=XX | 270 |



| Table 6.203. | Distributional Characteristics of Accessibility of Intervention (AIM) (Telehealth) (PSP) (Month 6/7), N=XX | 273 |
|---|---|---|
| Table 6.204. | Distributional Characteristics of Feasibility of Intervention (FIM) (Telehealth) (PSP) (Month 6/7), N=XX | 276 |
| Table 6.205. | Summary of Acceptability of Intervention (AIM) (APRETUDE) (PSP) (Month 6/7), N=XX | 279 |
| Table 6.206. | Summary of Feasibility of Intervention (FIM) (APRETUDE) (PSP) (Month 6/7), N=XX | 280 |
| Table 6.207. | Summary of Acceptability of Intervention (AIM) (Telehealth) (PSP) (Month 6/7), N=XX | 282 |
| Table 6.208. | Summary of Feasibility of Intervention (FIM) (Telehealth) (PSP) (Month 6/7), N=XX | 284 |
| Table 6.209. | Changes from Baseline to Acceptability of Intervention Measure (AIM - APRETUDE) and Feasibility of Intervention Measure (FIM - APRETUDE) (Month 6/7), N=XX | 286 |
| Table 6.210. | Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – APRETUDE) (Month 6/7), N= XX | 287 |
| Table 6.211. | Mixed-effects Modeling of the Changes from Baseline to Month 6/7 in Acceptability of Intervention Measure (AIM – APRETUDE), N=XX | 288 |
| Table 6.212. | Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – APRETUDE) (Month 6/7), N=XX | 289 |
| Table 6.213. | Mixed-effects Modeling of the Changes from Baseline to Month 6/7 in Feasibility of Intervention Measure (FIM – APRETUDE), N=XX | 290 |
| Table 6.214. | Changes from Baseline for Acceptability of Intervention Measure (AIM - Telehealth) and Feasibility of Intervention Measure (FIM - Telehealth) (Month 6/7), N=XX | 291 |
| Table 6.215. | Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – Telehealth) (Month 6/7), N=XX | 292 |
| Table 6.216. | Mixed-effects Modeling of the Changes from Baseline to Month 6/7 in Acceptability of Intervention Measure (AIM – Telehealth), N=XX | 293 |
| Table 6.217. | Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – Telehealth) (Month 6/7), N=XX | 294 |
| Table 6.218. | Mixed-effects Modeling of the Changes from Baseline to Month 6/7 in Feasibility of Intervention Measure (FIM – Telehealth), N=XX | 295 |
| Table 6.219. | Summary of Pain/Activities After Injection (Month 6/7), N=XX | 296 |
| Table 6.220. | Summary of Patient Study Participants' Labs and Missed Doses (Month 6/7), N=XX | 299 |
| Table 6.301. | Summary of Feasibility and Acceptability of Telehealth (Month 6/7), N=XX | 301 |
| Table 6.302. | Summary of Quality of Care for Patient Study Participants (Month 6/7), N=XX | 309 |
| Table 6.303. | Summary of Quality of Care for Patient Study Participants (Month 6/7), N=XX, Non-Score Questions | 313 |
| Table 6.304. | Summary of Quality of Care for Patient Study Participants (Month 6/7), N=XX, Score Questions | 328 |
| Table 6.305. | Summary of Utility of Proposed Implementation Strategies (Month 6/7), N=XX | 345 |
| Table 6.306. | Summary of Patient Study Participants' Preferences/Acceptability of APRETUDE Information, Appointment Reminders, and Locations (Month 6/7), N=XX | 353 |
| Table 6.307. | Summary of Appointment Scheduling (Month 6/7), N=XX | |



| Table 6.401. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Study Arms | . 358 |
|---|---|---|
| Table 6.402. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Race, Dynamic Implementation | . 362 |
| Table 6.403. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Race, Routine Implementation | .366 |
| Table 6.404. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Race, Total | .370 |
| Table 6.405. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Ethnicity, Study Arms | .374 |
| Table 6.406. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Ethnicity, Total | . 378 |
| Table 6.407. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Gender, Total | . 382 |
| Table 6.408. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Study Arms | .386 |
| Table 6.409. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Race, Dynamic Implementation | . 390 |
| Table 6.410. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Race, Routine Implementation | .394 |
| Table 6.411. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Race, Total | . 398 |
| Table 6.412. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Ethnicity, Study Arms | . 402 |
| Table 6.413. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Ethnicity, Total | . 406 |
| Table 6.414. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Gender | .410 |
| Table 6.415. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Site Volume | . 414 |
| Table 6.416. | Distributional Characteristics of Estimated Amount of Money Spent on Transportation for Each Injection Visit (Month 6/7), N=XX | .418 |



Table 6.000. Demographic Characteristics of Patient Study Participants Completing Surveys (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N=XX)<br>n (%) | Dynamic<br>Implementation<br>(N=XX)<br>n (%) | Routine<br>Implementation<br>(N=XX)<br>n (%) |
|---|---|---|---|---|---|
| DM1 | Age (years) | N | XX | XX | XX |
| | | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| DM2 | Age (years), High Volume | N | XX | XX | XX |
| | | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| DM3 | Age (years), Low Volume | N | XX | XX | XX |
| | | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| DM4 | Age | | | | |
| | | 18-25 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 26-35 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 36-49 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 50+ | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| DM5 | Study Arm | | | | |
| | | Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| DM6 | Site Volume | | | | |
| | | High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| DM7 | Gender | | | | |
| | | Men who have sex with men | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Transgender men | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| DM8 | Race | | | | |
| | | Asian | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Black or African American | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | White | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Missing/Unknown | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | | Question | Response | Total<br>(N=XX)<br>n (%) | Dynamic<br>Implementation<br>(N=XX)<br>n (%) | Routine<br>Implementation<br>(N=XX)<br>n (%) |
|---|---|---|---|---|---|---|
| DM9 | Ethnicity | | | | | |
| | | | Hispanic or Latino | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | | Not Hispanic or Latino | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | | Missing/Unknown | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 6.001. Demographic Characteristics of Patient Study Participants (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 1 | Which of the following best descri | bes your <u>current</u> relationship | status? | | |
| | | Single, never married | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Single, widowed | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Single, separated or divorced | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dating, but not living with a partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dating and living with a partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Domestic partnership/civil union | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Married | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 2 | How would you describe your <u>curr</u> | <u>ent</u> living situation? | ı | | |
| | | I live in my own house or apartment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I live in my parent's<br>house or apartment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I live in a family<br>member's house or<br>apartment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I live in a friend's house or apartment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I sleep on various<br>friends' or relatives'<br>couches | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am homeless or am living in a shelter | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I live in motel(s)/hotel(s) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 3 | What <u>best</u> describes your current | employment status? | | | |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Employed for wages full-<br>time (1 employer) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Employed for wages full-<br>time (2 or more<br>employers) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Employed for wages part-time (1 employer) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Employed for wages<br>part-time (2 or more<br>employers) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Self-employed | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A homemaker | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Student | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Retired | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not employed | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unable to work<br>(disabled) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 4 | What type of medical insurance do | you currently have? | | | |
| | | My parents' insurance | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | My partner's/spouse's insurance | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Private insurance<br>provided by my<br>workplace | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Private insurance I<br>purchased through an<br>exchange (e.g.,<br>Obamacare, Affordable<br>Care Act) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Federal insurance (e.g., VA, TRICARE) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Medicare or Medicaid | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Some other health care plan | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't have any health insurance currently | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |


Table 6.002. Summary of Behaviors of Patient Study Participants (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 84 | How often do you have a drink | containing alcohol? | | | |
| | | Never | XX | XX | XX |
| | | ivevei | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Monthly or less | XX | XX | XX |
| | | Worthing of less | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 2 to 4 times a month | XX | XX | XX |
| | | 2 to 4 times a month | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 2 to 3 times a week | XX | XX | XX |
| | | 2 to 3 times a week | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A or more times a week | XX | XX | XX |
| | | 4 or more times a week | (XX.X%) | (XX.X%) | (XX.X%) |
| 85 | On days when you drink alcoho<br>bottle/ can of beer, 1 glass of w | | | u typically have? (1 o | drink=1 standard |
| | | 1 or 2 | XX | XX | XX |
| | | 1012 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 3 to 4 | XX | XX | XX |
| | | 5 10 4 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 5 to 6 | XX | XX | XX |
| | | 3 10 6 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 7+- 0 | XX | XX | XX |
| | | 7 to 9 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 10 or more | XX | XX | XX |
| | | 10 or more | (XX.X%) | (XX.X%) | (XX.X%) |
| 86 | In the last 6 months, have you s<br>provider, such as speedball, her<br>needle, either by mainlining, ski | oin, or crack? By shooting up, w | | | |
| | | Yes | XX | XX | XX |
| | | Tes | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX |
| | | No | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Lunafan nat ta an an | XX | XX | XX |
| | | I prefer not to answer | (XX.X%) | (XX.X%) | (XX.X%) |
| 87 | In the last 6 months, have you usubstances), that were not prescocaine? | | | | |
| | | V | XX | XX | XX |
| | | Yes | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | | 207 | 107 |
| | | | XX | XX | XX |
| | | No | (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No I prefer not to answer | | | |



Table 6.003. Summary of Patient Study Participants' Sexual History and Behaviors (Month 6/7), N=XX, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 8 | Have you h<br>oral sex. | and sex in the last 6 months? This could be vaginal sex | κ (penis in va | gina) OR anal sex (p | enis in butt) OR |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 9 | How would | you describe your sexual behaviors in the last 6 mor | nths? | | |
| | | I have had vaginal sex (penis in vagina) with only<br>1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex (penis in vagina) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a bottom (penis in butt as<br>a bottom) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a bottom (penis in butt as a bottom) with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top (penis in butt as a<br>top) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top (penis in butt as a<br>top) with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth, tongue, or lips on a vagina, penis, or butt) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth, tongue, or lips on a vagina, penis, or butt) with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 10 | How often | did you use a condom when you had sex in the last 6 | months? | | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 11 | In the last ( | 5 months, how would you describe the HIV status of | your sexual p | partner(s)? | |
| | | I know that none of my sexual partners from the last 6 months have HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one sexual partner from the last 6 months is living with HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 12 | | ou know, were any of your sexual partner(s) from the<br>PrEP is a medication that prevents HIV. | | , , | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | l don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 13 | You mentioned that you had a least one partner in the last 6 months who is living with HIV/AIDS. As far as you know, were any of your partners taking HIV medications (antiretrovirals) to treat their HIV infection? | | | | |
| | | Yes, my partner(s) was/were taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s) was/were taking HIV medications and was/were undetectable, meaning HIV tests were not finding the virus | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, my partner(s) was/were not taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether my partner(s) was/were<br>taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 14 | | 6 months, have you experienced any incidents of sex<br>m a partner? | ual violence, | physical abuse, or a | ny other type of |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 16 | In the last ( | 5 months, have you exchanged things like money or | drugs for sex | with a sexual partne | er? |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Yes, I have a sexual partner things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave me things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.004. Summary of Patient Study Participants' Sexual History and Behaviors (Month 6/7), N=XX, Race, Dynamic Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 8 | Have you ha<br>OR oral sex. | d sex in the last 6 months? <i>Thi</i> | is could be vagin | al sex (penis in vag | nina) OR anal sex | (penis in butt) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| ) | How would | you describe your sexual beha | viors in the last 6 | months? | | |
| | | I have had vaginal sex<br>(penis in vagina) with only<br>1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex<br>(penis in vagina) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a top)<br>with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a top)<br>with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips on<br>a vagina, penis, or butt)<br>with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips on<br>a vagina, penis, or butt)<br>with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify<br>) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 11 | In the last 6 | months, how would you descr | ribe the HIV state | us of your sexual p | artner(s)? | |
| | | I know that none of my<br>sexual partners from the<br>last 6 months have<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one<br>sexual partner from the<br>last 6 months is living with<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual<br>partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 12 | As far as you know, were any of your sexual partner(s) from the last 6 months taking PrEP to prevent HIV infection? PrEP is a medication that prevents HIV. | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 13 | You mentioned that you had a least one partner in the last 6 months who is living with HIV/AIDS. As far as you know, were any of your partners taking HIV medications (antiretrovirals) to treat their HIV infection? | | | | | |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications and<br>was/were undetectable, | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | meaning HIV tests were not finding the virus | | | | |
| | | No, my partner(s)<br>was/were not taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether my<br>partner(s) was/were<br>taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 14 | In the last 6 months, have you experienced any incidents of sexual violence, physical abuse, or any other type of trauma from a partner? | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | In the last 6 | months, have you exchanged | things like mone | y or drugs for sex | with a sexual part | ner? |
| | | Yes, I have a sexual<br>partner things like drugs<br>or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave<br>me things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.005. Summary of Patient Study Participants' Sexual History and Behaviors (Month 6/7), N=XX, Race, Routine Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 8 | Have you ha<br>OR oral sex. | nd sex in the last 6 months? T | his could be vagin | al sex (penis in vag | gina) OR anal sex | (penis in butt) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 9 | How would | you describe your sexual beh | aviors in the last 6 | 5 months? | | |
| | | I have had vaginal sex<br>(penis in vagina) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex<br>(penis in vagina) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as<br>a bottom) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as<br>a bottom) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a<br>top) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a<br>top) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips<br>on a vagina, penis, or<br>butt) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips<br>on a vagina, penis, or<br>butt) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 10 | How often | did you use a condom when y | ou had sex in the | last 6 months? | | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 11 | In the last 6 | months, how would you des | cribe the HIV stat | us of your sexual p | artner(s)? | |
| | | I know that none of my<br>sexual partners from the<br>last 6 months have<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one<br>sexual partner from the<br>last 6 months is living<br>with HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual<br>partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 12 | | u know, were any of your sex<br>PrEP is a medication that preve | | m the last 6 month | is taking PrEP to p | prevent HIV |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 13 | | ned that you had a least one any of your partners taking H | | | | |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications and | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | was/were undetectable,<br>meaning HIV tests were<br>not finding the virus | | | | |
| | | No, my partner(s)<br>was/were not taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether<br>my partner(s) was/were<br>taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 14 | In the last 6 months, have you experienced any incidents of sexual violence, physical abuse, or any other type of trauma form a partner? | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | In the last 6 months, have you exchanged things like money or drugs for sex with a sexual partner? | | | | | |
| | | Yes, I have a sexual partner things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner<br>gave me things like drugs<br>or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged<br>things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.006. Summary of Patient Study Participants' Sexual History and Behaviors (Month 6/7), N=XX, Race, Total

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 8 | Have you ha<br>OR oral sex. | nd sex in the last 6 months? <i>Ti</i> | his could be vagin | al sex (penis in vag | gina) OR anal sex | (penis in butt) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| ) | How would | you describe your sexual beh | aviors in the last 6 | 5 months? | | |
| | | I have had vaginal sex<br>(penis in vagina) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex<br>(penis in vagina) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as<br>a bottom) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as<br>a bottom) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a<br>top) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a<br>top) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips<br>on a vagina, penis, or<br>butt) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips<br>on a vagina, penis, or<br>butt) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | | Black or | | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
| 10 | How often | did you use a condom when y | ou had sex in the | last 6 months? | | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 11 | In the last 6 | 5 months, how would you desc | cribe the HIV stat | us of your sexual p | artner(s)? | |
| | | I know that none of my<br>sexual partners from the<br>last 6 months have<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one<br>sexual partner from the<br>last 6 months is living<br>with HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual<br>partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 12 | As far as you know, were any of your sexual partner(s) from the last 6 months taking PrEP to prevent HIV infection? PrEP is a medication that prevents HIV. | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 13 | | oned that you had a least one pe<br>any of your partners taking H | | | | |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications and | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | was/were undetectable,<br>meaning HIV tests were<br>not finding the virus | | | | |
| | | No, my partner(s)<br>was/were not taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether<br>my partner(s) was/were<br>taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 14 | | 5 months, have you experience form a partner? | ed any incidents c | of sexual violence, | physical abuse, or | any other type |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | In the last 6 months, have you exchanged things like money or drugs for sex with a sexual partner? | | | | | |
| | | Yes, I have a sexual<br>partner things like drugs<br>or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner<br>gave me things like drugs<br>or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged<br>things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.007. Summary of Patient Study Participants' Sexual History and Behaviors (Month 6/7), N=XX, Ethnicity, Study Arms

| | | | Dynamic Implementation | | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) |
| 8 | Have you h oral sex. | ad sex in the last 6 months? <i>This</i> o | could be vaginal s | sex (penis in vagina | ) OR anal sex (pe | nis in butt) OR |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 9 | How would | you describe your sexual behavio | ors in the last 6 m | onths? | | |
| | | I have had vaginal sex (penis<br>in vagina) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex (penis<br>in vagina) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | Question | Response | Dynamic Implementation | | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | | | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanio<br>or Latino<br>(N = XX)<br>n (%) |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 11 | In the last 6 | months, how would you describ | e the HIV status o | of your sexual partr | ner(s)? | |
| | | I know that none of my<br>sexual partners from the last<br>6 months have HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one<br>sexual partner from the last<br>6 months is living with<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual<br>partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 12 | As far as you know, were any of your sexual partner(s) from the last 6 months taking PrEP to prevent HIV infection? PrEP is a medication that prevents HIV. | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 13 | | oned that you had a least one part<br>e any of your partners taking HIV r | | | | |
| | | Yes, my partner(s) was/were taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s) was/were taking HIV medications and was/were undetectable, meaning HIV tests were not finding the virus | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | Question | | Dynamic Implementation | | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) |
| | | No, my partner(s) was/were not taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether my<br>partner(s) was/were taking<br>HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 14 | In the last 6 months, have you experienced any incidents of sexual violence, physical abuse, or any of trauma form a partner? | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | In the last 6 months, have you exchanged things like money or drugs for sex with a sexual partner? | | | | | |
| | | Yes, I have a sexual partner<br>things like drugs or money<br>for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave<br>me things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged<br>things like drugs or money<br>for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.008. Summary of Patient Study Participants' Sexual History and Behaviors (Month 6/7), N=XX, Ethnicity, Total

| Question | | | Hispanic or Latino | Not Hispanic or Latino |
|---|---|---|---|---|
| Number | Question | Response | (N = XX)<br>n (%) | (N = XX)<br>n (%) |
| 8 | Have you h | ad sex in the last 6 months? <i>This co</i> | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 9 | How would you describe your sexual behaviors in the last 6 months? | | | |
| | | I have had vaginal sex (penis<br>in vagina) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex (penis<br>in vagina) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 10 | How often | did you use a condom when you ha | d sex in the last 6 months? | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) |



| 11 | In the last 6 | Most of the time Some of the time A little of the time None of the time I prefer not to answer months, how would you describe to the time of my sexual partners from the last 6 months have HIV/AIDS | XX | n (%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) |
|---|---|---|---|---|
| 11 | In the last 6 | Some of the time A little of the time None of the time I prefer not to answer months, how would you describe to the time the second | (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) AXX (XX.X%) he HIV status of your sexual par | (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) |
| 11 | In the last 6 | A little of the time None of the time I prefer not to answer months, how would you describe to the last of the time. | XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) AX (XX.X%) AX (XX.X%) AX XX XX XX XX XX XX | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%) |
| 11 | In the last 6 | A little of the time None of the time I prefer not to answer months, how would you describe to the last of the time. | XX (XX.X%) XX (XX.X%) XX (XX.X%) he HIV status of your sexual par | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%) |
| 11 | In the last 6 | None of the time I prefer not to answer months, how would you describe t I know that none of my sexual partners from the last | (XX.X%) XX (XX.X%) XX (XX.X%) he HIV status of your sexual par | (XX.X%) XX (XX.X%) XX (XX.X%) tner(s)? |
| 11 | In the last 6 | None of the time I prefer not to answer months, how would you describe t I know that none of my sexual partners from the last | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>he HIV status of your sexual par | XX<br>(XX.X%)<br>XX<br>(XX.X%) |
| 11 | In the last 6 | I prefer not to answer months, how would you describe t I know that none of my sexual partners from the last | (XX.X%) XX (XX.X%) he HIV status of your sexual par XX | (XX.X%) XX (XX.X%) ther(s)? |
| 11 | In the last 6 | months, how would you describe t I know that none of my sexual partners from the last | XX<br>(XX.X%)<br>he HIV status of your sexual par<br>XX | XX<br>(XX.X%)<br>tner(s)? |
| 11 | In the last 6 | months, how would you describe t I know that none of my sexual partners from the last | (XX.X%)<br>he HIV status of your sexual par<br>XX | (XX.X%) |
| 11 | In the last 6 | I know that none of my<br>sexual partners from the last | he HIV status of your sexual par | tner(s)? |
| | | I know that none of my<br>sexual partners from the last | XX | |
| | | sexual partners from the last | | XX |
| | | 6 months have HIV/AIDS | /VV V0/\ | /VV V0/\ |
| | | | (XX.X%) | (XX.X%) |
| | | I know that at least one | | |
| | | sexual partner from the last | XX | XX |
| | | 6 months is living with<br>HIV/AIDS | (XX.X%) | (XX.X%) |
| | | I do not know my sexual | XX | XX |
| | | partners' HIV status | (XX.X%) | (XX.X%) |
| | | I profer not to answer | XX | XX |
| | | I prefer not to answer | (XX.X%) | (XX.X%) |
| | As far as you know, were any of your sexual partner(s) from the last 6 months taking PrEP to prevent HIV infection? PrEP is a medication that prevents HIV. | | | |
| | | No | XX | XX |
| | | INO | (XX.X%) | (XX.X%) |
| | | Yes | XX | XX |
| | | | (XX.X%) | (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | · · · · · · | · · · |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 1 4 | | ned that you had a least one partne<br>any of your partners taking HIV me | er in the last 6 months who is liv | ing with HIV/AIDS. As far as you |
| | | Yes, my partner(s) was/were | XX | XX |
| | | taking HIV medications | (XX.X%) | (XX.X%) |
| | | Yes, my partner(s) was/were | | |
| | | taking HIV medications and | XX | XX |
| | | was/were undetectable,<br>meaning HIV tests were not | (XX.X%) | (XX.X%) |
| | | finding the virus | | |
| | | No, my partner(s) was/were | XX | XX |
| | | not taking HIV medications | (XX.X%) | (XX.X%) |
| | | I do not know whether my | XX | XX |
| | | partner(s) was/were taking<br>HIV medications | (XX.X%) | (XX.X%) |



| Question Number Question | | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 14 | In the last 6 months, have you experienced any incidents of sexual violence, physical abuse, or any oth trauma form a partner? | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | In the last 6 months, have you exchanged things like money or drugs for sex with a sexual partner? | | | |
| | | Yes, I have a sexual partner<br>things like drugs or money<br>for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave<br>me things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged<br>things like drugs or money<br>for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.009. Summary of Patient Study Participants' Sexual History and Behaviors (Month 6/7), N=XX, Gender, Total

| Ougation | | | Men who have sex with men | Transgender Men |
|---|---|---|---|---|
| Question<br>Number | Question | Response | (N = XX)<br>n (%) | (N = XX)<br>n (%) |
| 8 | Have you h | ad sex in the last 6 months? <i>This</i> o | could be vaginal sex (penis in vagina) OR anal sex (penis in butt) OR | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 9 | How would you describe your sexual behaviors in the last 6 months? | | | |
| | | I have had vaginal sex (penis<br>in vagina) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex (penis<br>in vagina) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 10 | How often | did you use a condom when you l | nad sex in the last 6 months? | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Men who have sex with men (N = XX) | Transgender Men<br>(N = XX) |
|---|---|---|---|---|
| Nullibel | | | n (%) | n (%) |
| | | Most of the time | XX | XX |
| | | Most of the time | (XX.X%) | (XX.X%) |
| | | Some of the time | XX | XX |
| | | Some of the time | (XX.X%) | (XX.X%) |
| | | A little of the time | XX | XX |
| | | A little of the time | (XX.X%) | (XX.X%) |
| | | None of the time | XX | XX |
| | | None of the time | (XX.X%) | (XX.X%) |
| | | I prefer not to answer | XX | XX |
| | | r prefer flot to unswer | (XX.X%) | (XX.X%) |
| 11 | In the last 6 months, how would you describe the HIV status of your sexual partner(s)? | | | |
| | | I know that none of my | XX | XX |
| | | sexual partners from the last | (XX.X%) | ^^<br>(XX.X%) |
| | | 6 months have HIV/AIDS | (, , | (, 0,, 1, 0) |
| | | I know that at least one | | |
| | | sexual partner from the last | XX | XX |
| | | 6 months is living with<br>HIV/AIDS | (XX.X%) | (XX.X%) |
| | | | V0/ | <b>NO</b> 4 |
| | | I do not know my sexual<br>partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | partifers filly status | | |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | | , , |
| 12 | As far as you know, were any of your sexual partner(s) from the last 6 months taking PrEP to prevent HIV infection? PrEP is a medication that prevents HIV. | | | |
| | | No | XX | XX |
| | | INO | (XX.X%) | (XX.X%) |
| | | Vos | XX | XX |
| | | Yes | (XX.X%) | (XX.X%) |
| | | L -1 /4- 1 | XX | XX |
| | | I don't know | (XX.X%) | (XX.X%) |
| | | | XX | XX |
| | | I prefer not to answer | (XX.X%) | (XX.X%) |
| 13 | | • | ner in the last 6 months who is living medications (antiretrovirals) to treat t | |
| | | Yes, my partner(s) was/were | XX | XX |
| | | taking HIV medications | (XX.X%) | (XX.X%) |
| | | Yes, my partner(s) was/were | | |
| | | taking HIV medications and | VV | W |
| | | was/were undetectable, | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | meaning HIV tests were not | (//////// | (///.//0) |
| | | finding the virus | | |
| | | No, my partner(s) was/were | XX | XX |
| | | not taking HIV medications | (XX.X%) | (XX.X%) |
| | | I do not know whether my | XX | XX |
| | | partner(s) was/were taking | (XX.X%) | (XX.X%) |
| | | HIV medications | ` ' | , |



| Question<br>Number | Question | Response | Men who have sex with men<br>(N = XX)<br>n (%) | Transgender Men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 14 | In the last 6 months, have you experienced any incidents of sexual violence, physical abuse, or any other type trauma form a partner? | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | In the last 6 | months, have you exchanged th | ings like money or drugs for sex with a | a sexual partner? |
| | | Yes, I have a sexual partner<br>things like drugs or money<br>for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave<br>me things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged<br>things like drugs or money<br>for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.101. Summary of Patient Study Participants' HIV and PrEP Knowledge (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 5 | Do you personally know of someone living with HIV? | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.102. Summary of Patient Study Participants' HIV and PrEP Knowledge (Month 6/7), N=XX, Scale Questions, Study Arms

| | | | Total | Dynamic | Routine |
|---|---|---|---|---|---|
| Question<br>Number | Question | Response | (N = XX)<br>n (%) | Implementation<br>(N = XX)<br>n (%) | Implementation<br>(N = XX)<br>n (%) |
| 6 | Please answer true or false to the following s | tatements abo | out HIV. | (/2/ | (1.5) |
| А | A person who has HIV can look healthy. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | There is a vaccine that can stop you from getting HIV. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | A person will NOT get HIV if they are taking antibiotics. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | If you only have sex once with a partner, you cannot get HIV from them. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Е | People living with HIV on HIV medications cannot spread HIV. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Everybody who has HIV knows that they have HIV. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | A natural (lamb skin) condom works better against HIV than a latex condom. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | When using condoms during sex, it is safer to use water-based lubricants than oilbased lubricants. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.103. Distributional Characteristics of Patient Study Participants' HIV and PrEP Knowledge (Month 6/7), N=XX, Scale Questions, Overall Score

| 6. Please answer true or false to the following statements about HIV. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | 0.xx |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Gender | | | | | | | | |
| Men who have<br>sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Transgender<br>Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Not Hispanic<br>or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| | | | Dyna | mic Implement | ation | | | |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Gender | | | | | | | | |
| Men who<br>have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |



| 6. Please answer true or false to the following statements about HIV. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Transgender<br>Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Black or<br>African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Not Hispanic<br>or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| | | | Rout | ine Implementa | ation | | | |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Gender | | | | | | | | |
| Men who<br>have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Transgender<br>Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Black or<br>African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Not Hispanic<br>or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |

Mean score = mean of correct responses to all of the items under 8 save for A and E; 'Don't know' responses coded as incorrect. Correct answers were 'False' for items B, C, D, F, and G and 'True' for item H



Table 6.104. Summary of Patient Study Participants' Perception of Stigma Associated with PrEP Usage (Month 6/7), N=XX, Stigma, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 7 | To what extent do you agree with eac | h of the following : | statements about | PrEP? | |
| А | My <i>friends</i> would be supportive of me taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | People experience problems when they tell their sexual partner(s) they are taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | People experience negative judgement because they take PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | My <i>family</i> would be supportive of me taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Completely<br>agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | People taking PrEP receive praise for being responsible. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | I would feel ashamed to take PrEP in front of others. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | Someone taking PrEP would be seen by others as having sex with a lot of different people. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | People on PrEP are taking care of their health. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| I | People talking PrEP experience verbal harassment. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| J | I would not want others to know if I was taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| K | Someone taking PrEP should keep their pills hidden. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| L | I would feel proud to take PrEP every day. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| M | I would have sex with someone who is taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.105. Distributional Characteristics of Patient Study Participants' Perception of Stigma Associated with PrEP Usage (Month 6/7), N=XX, Stigma, Overall Score

| 13. To what extent do | | | | | Observed | | | |
|---|---|---|---|---|---|---|---|---|
| you agree with each of<br>the following<br>statements about PrEP? | n | Mean | SD | Median<br>(Q1, Q3) | Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach'<br>s α |
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | 0.xx |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Gender | | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Not Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Dynamic Implementation | | | | | | | | |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Gender | | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |



| 13. To what extent do<br>you agree with each of<br>the following<br>statements about PrEP? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach'<br>s α |
|---|---|---|---|---|---|---|---|---|
| Transgender<br>Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Not Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Routine Implementation | | | | | | | | |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Gender | | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Transgender<br>Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Not Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |

Mean score = mean of responses to all of the items under 13 save for J with the following items are reverse scored: A, D, E, H, L,& M. Higher total score indicates higher stigma.



Table 6.106. Summary of Patient Study Participants' Choice of APRETUDE (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 16 | Do you have any concerns ab | out APRETUDE? | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 17 | What concerns do you have a | about APRETUDE? | | | |
| | | Pain or soreness from the injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other side effects from<br>APRETUDE | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Fear of needles | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Change in my insurance coverage for APRETUDE | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Possible long-term effects of the injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | How it affects other medications I take | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Scheduling or rescheduling injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Forgetting my appointment for the injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Missing an injection visit and then getting HIV | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Missing work for the injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Making time to go to the clinic/practice for the injection every 2 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Travelling to the clinic/practice for the injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Limited clinic/practice hours for injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Childcare/caregiver responsibilities during injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Lack of privacy at injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | My dignity not being respected during injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | People asking why I go to<br>the clinic/doctor every 2<br>months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | My hectic lifestyle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | My travel or holiday schedules | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Taking medication during times when I am not having sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The medication not being effective at preventing HIV | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Worrying people would think<br>I have HIV | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Worrying that people would<br>think I have a lot of sexual<br>partners because I am on<br>CAB LA for PrEP | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Worrying about my privacy because I live with someone | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Worrying about my privacy<br>because I'm on my parent's<br>health insurance | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 18 | How often are you worried th | at people may find out that you a | are taking APF | RETUDE? | |
| | | Never | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Rarely | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Sometimes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Often | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | All the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 19 | How often are you worried ab | out forgetting your APRETUDE in | | | |
| | | Never | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Rarely | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Sometimes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Often | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | All the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |


Table 6.107. Summary of Knowledge of APRETUDE and Utility of Implementation Strategies (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 73 | Overall, how much do you kno | ow about APRETUDE? | | | |
| | | A lot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Nothing | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 74 | How confident are you with yo | our current level of knowledge abo | ut APRETU[ | DE? | |
| | | Extremely confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 75 | How helpful was the information, if any, shared by the medical staff about APRETUDE? | | | | |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not receive any<br>information from medical staff | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 76 | How helpful has each of the fo | ollowing materials been in learning | about APRE | TUDE? | |
| А | Getting Started Brochure –<br>the brochure that gives you<br>an overview of how to get<br>started with APRETUDE | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Patient Brochure – this<br>brochure helps you<br>understand the process of<br>receiving APRETUDE<br>injections, including side<br>effects and insurance<br>information | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | Let's talk about HIV & PrEP<br>video – the video giving key<br>facts about HIV and PrEP<br>options (DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| D | The APRETUDE Myths and Facts video – the game show video addressing common myths about APRETUDE (DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| E | The What to Expect video which shows you what to expect during the APRETUDE process (DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| F | The ViiV Connect Video,<br>which tells you about the<br>ViiV Connect program and<br>frequently asked questions<br>(DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| G | The study website where you access APRETDUE information (RI) | Very helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| Н | The study app/website<br>where you access<br>APRETUDE information —<br>the Pillar Spot (DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| I | Important safety information – This document details important safety information relating to APRETUDE | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| J docume | Important facts – This<br>document details important<br>facts relating to APRETUDE | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| К | A flyer on PrEP options (DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |



Table 6.108. Attitude Regarding APRETUDE and Utility of Implementation Strategies (Month 6/7), N=XX

| Question | | | | | | |
|---|---|---|---|---|---|---|
| 83. Overall, ho<br>taking APRETU | ow are you feeling about<br>JDE? | Very positive | Somewhat positive | Neither<br>positive nor<br>negative | Somewhat<br>negative | Very<br>negative |
| Study Arms Total | | | | | | |
| | Total<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Routine<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynamio | : Implementation | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routine | Implementation | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | Response | | | | | |
|---|---|---|---|---|---|---|
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Dyna | mic Implementation | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Rout | ine Implementation | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Total | | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Total | ' | | | | | |
| | Men who have sex<br>with men<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Transgender men<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.109. Summary of Patient Study Participant Acquisition Process (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 77 | Have you ever heard of ViiV C | onnect? | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 78 | Where did you learn about Vii | V Connect? | | | |
| | | My healthcare provider/healthcare clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The ViiV Connect video on the study app/website (DI) | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | ViiV Connect brochure | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A friend/family member told me | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The ViiV Connect website | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.110. Summary of Patient Study Participant Acquisition Process, Insurance (Month 6/7), N=XX

| Question | | | | Response | | |
|---|---|---|---|---|---|---|
| | xtent do you agree with<br>ollowing statements? | Completely Agree | Agree | Neither<br>agree nor<br>disagree | Disagree | Completely<br>disagree |
| A. The staff | at the clinic helped me un | derstand the insurance a | pproval proces | SS | | |
| Study Arms | | | | | | |
| | Total<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Routine<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynami | c Implementation | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routine | Implementation | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | | | Response | esponse | |
|---|---|---|---|---|---|---|
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Dynar | nic Implementation | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Routir | ne Implementation | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Total | | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Total | | | | | | |
| | Men who have sex<br>with men<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Transgender men | XX | XX | XX | XX | XX |



| Question | Response | | | | | |
|---|---|---|---|---|---|---|
| | Total<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Routine<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynami | ic Implementation | | -1 | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routine | Implementation | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Total | | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | Response | | | | | |
|---|---|---|---|---|---|---|
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Dyn | amic Implementation | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Rou | tine Implementation | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Tota | al | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Total | | | | | | |
| | Men who have sex<br>with men<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Transgender men<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| C. My copa | y for APRETUDE is acceptable | | | | | |
| Study Arms | | | | | | |
| | Total<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | Response | | | | |
|---|---|---|---|---|---|---|
| | Routine<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynamic I | mplementation | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routine Ir | mplementation | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Total | | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | Response | | | | |
|---|---|---|---|---|---|---|
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Rou | tine Implementation | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Tota | al | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Total | | | | | | |
| | Men who have sex<br>with men<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Transgender men<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D. I am wor | ried about insurance coverag | e long-term | · | | | |
| Study Arms | | | | | | _ |
| | Total<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Routine<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynami | c Implementation | | 1 | | | 1 |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | | Response | | | |
|---|---|---|---|---|---|---|
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routine | Implementation | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Total | | | -1 | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Dyna | amic Implementation | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | Response | | | | | |
|---|---|---|---|---|---|---|
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Total | | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Total | | | | | | |
| | Men who have sex<br>with men<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Transgender men N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E. The insura | ance approval process was s | imple | | | | |
| Study Arms | | | | | | |
| | Total<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Routine<br>Implementation<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynamic | Implementation | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | | | Response | | |
|---|---|---|---|---|---|---|
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routine I | mplementation | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Total | | | | | | |
| | Asian<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White N = XX n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Dyna | mic Implementation | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Routi | ine Implementation | | | | | |
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Total | | | 1 | | | 1 |



| Question | | Response | | | | |
|---|---|---|---|---|---|---|
| | Hispanic or Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Total | | | | | | |
| | Men who have sex<br>with men<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Transgender men<br>N = XX<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.201. Distributional Characteristics of Acceptability of Intervention (AIM) (APRETUDE) (PSP) (Month 6/7), N=XX

| 20. AIM APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX (XX.X%) |
| Routine Implementation | XX | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX (XX.X%) |
| T-test<br>Degrees of Freedom<br>P-value | | X.XXX<br>XX<br>O.XXX | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Dynamic Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 20. AIM APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the Mean |
|---|---|---|---|---|---|---|---|
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African Americar | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African Americar | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |



| 20. AIM APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% Cl<br>for the Mean |
|---|---|---|---|---|---|---|---|
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



Table 6.202. Distributional Characteristics of Feasibility of Intervention (FIM) (APRETUDE) (PSP) (Month 6/7), N=XX

| | | | | | Observed | | 95% CI |
|---|---|---|---|---|---|---|---|
| 21. FIM APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | for the<br>Mean |
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| T-test | | | | X.XXX | | | |
| Degrees of Freedom | | | | XX | | | |
| P-value | | | | 0.XXX | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Dynamic Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 21. FIM APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Gender | | | | | | | |
| Men who have sex with<br>men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with<br>men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 21. FIM APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



Table 6.203. Distributional Characteristics of Accessibility of Intervention (AIM) (Telehealth) (PSP) (Month 6/7), N=XX

| | | | 45 | | | | |
|---|---|---|---|---|---|---|---|
| 22. AIM TELEHEALTH. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| T-test | | X.XXX | | | | | |
| Degrees of Freedom | | XX | | | | | |
| P-value | | | | 0.XXX | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Dynamic Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 22. AIM TELEHEALTH. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Gender | | | | | | | |
| Men who have sex with<br>men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with<br>men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 22. AIM TELEHEALTH. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



Table 6.204. Distributional Characteristics of Feasibility of Intervention (FIM) (Telehealth) (PSP) (Month 6/7), N=XX

| 24. FIM TELEHEALTH. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| T-test | | X.XXX | | | | | |
| Degrees of Freedom | | XX | | | | | |
| P-value | | 0.XXX | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Dynamic Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 24. FIM TELEHEALTH. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Gender | | | | | | | |
| Men who have sex with<br>men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with<br>men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 24. FIM TELEHEALTH. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



Table 6.205. Summary of Acceptability of Intervention (AIM) (APRETUDE) (PSP) (Month 6/7), N=XX

| Question | Question | Response | Total<br>(N = XX) | Dynamic<br>Implementation | Routine<br>Implementation |
|---|---|---|---|---|---|
| Number | Question | Пезропас | n (%) | (N = XX)<br>n (%) | (N = XX)<br>n (%) |
| 20 | Please indicate how much you a | gree or disagree with ( | each statemen | t based on your <b>experie</b> i | nces with APRETUDE. |
| | APRETUDE <b>meets my approval</b> for preventing HIV. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | APRETUDE for the prevention of HIV is appealing to me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I <b>like</b> APRETUDE for the prevention of HIV. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I welcome APRETUDE for the prevention of HIV | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.206. Summary of Feasibility of Intervention (FIM) (APRETUDE) (PSP) (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 21 | Please indicate how much you | u agree with each statem | nent based on y | our current expectation | ns of APRETUDE. |
| | Receiving APRETUDE injection every 2-months seems workable in my life | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Receiving APRETUDE injection every 2-months seems possible in my life | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Receiving APRETUDE injection every 2-months seems doable in my life | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Receiving APRETUDE injection every 2-months seems easy in my life | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.207. Summary of Acceptability of Intervention (AIM) (Telehealth) (PSP) (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 23 | Please indicate how much y with telehealth. | ou agree with each sta | atement based | on your current percep | tions and experience |
| | Using telehealth for APRETUDE services <b>meets my approval</b> . | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Using telehealth for APRETUDE services is appealing to me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I <b>like</b> using telehealth for APRETUDE services. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I welcome using telehealth for APRETUDE services. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.208. Summary of Feasibility of Intervention (FIM) (Telehealth) (PSP) (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 23 | Please indicate how much you | ou agree with each sta | atement based | on your current percep | tions and experience |
| | Using telehealth for APRETUDE services <b>seems</b> workable in my life. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Using telehealth for APRETUDE services <b>seems possible</b> in my life. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Using telehealth for APRETUDE services <b>seems doable</b> in my life. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Using telehealth for APRETUDE services <b>seems easy</b> in my life. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |


| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.209. Changes from Baseline to Acceptability of Intervention Measure (AIM - APRETUDE) and Feasibility of Intervention Measure (FIM - APRETUDE) (Month 6/7), N=XX

| Measure | Study Arm | n | Mean | SD | Median (Q1, Q3) | Observed Range<br>(min, max) | Missing<br>n (%) | 95% CI<br>for the Mean |
|---|---|---|---|---|---|---|---|---|
| AIM - APRETUDE Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| AIM - APRETUDE Month 6/7 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| AIM - APRETUDE Change from Baseline to<br>Month 6/7 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| FIM - APRETUDE Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| FIM - APRETUDE Month 6/7 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| FIM - APRETUDE Change from Baseline to<br>Month 6/7 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |



Table 6.210. Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – APRETUDE) (Month 6/7), N= XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 6.211. Mixed-effects Modeling of the Changes from Baseline to Month 6/7 in Acceptability of Intervention Measure (AIM – APRETUDE), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 6.212. Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – APRETUDE) (Month 6/7), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 6.213. Mixed-effects Modeling of the Changes from Baseline to Month 6/7 in Feasibility of Intervention Measure (FIM – APRETUDE), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site



Table 6.214. Changes from Baseline for Acceptability of Intervention Measure (AIM - Telehealth) and Feasibility of Intervention Measure (FIM - Telehealth) (Month 6/7), N=XX

| Measure | Study Arm | n | Mean | SD | Median (Q1, Q3) | Observed Range<br>(min, max) | Missing<br>n (%) | 95% CI<br>for the Mean |
|---|---|---|---|---|---|---|---|---|
| AIM - Telehealth Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| AIM - Telehealth Month 6/7 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| AIM - Telehealth Change from Baseline to<br>Month 6/7 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| FIM - Telehealth Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| FIM - Telehealth Month 6/7 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| FIM - Telehealth Change from Baseline to<br>Month 6/7 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |



Table 6.215. Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – Telehealth) (Month 6/7), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 6.216. Mixed-effects Modeling of the Changes from Baseline to Month 6/7 in Acceptability of Intervention Measure (AIM – Telehealth), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 6.217. Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – Telehealth) (Month 6/7), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 6.218. Mixed-effects Modeling of the Changes from Baseline to Month 6/7 in Feasibility of Intervention Measure (FIM – Telehealth), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 6.219. Summary of Pain/Activities After Injection (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 65 | Did you experience an redness, itching, swelli | y local reaction(s) following an injecti<br>ing, bruising. | on appointment | ? Examples of local r | eactions are |
| | | Yes | XX | XX | XX |
| | | 103 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX |
| | | 110 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX |
| | | T don't know | (XX.X%) | (XX.X%) | (XX.X%) |
| 66 | How acceptable was/v bruising. | vere your local reaction(s)? Examples | of local reaction | s are redness, itching | g, swelling, |
| | | Totally acceptable | XX | XX | XX |
| | | Totally acceptable | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Very acceptable | XX | XX | XX |
| | | very acceptable | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Moderately acceptable | XX | XX | XX |
| | | Moderately acceptable | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A little acceptable | XX | XX | XX |
| | | A little acceptable | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Not at all acceptable | XX | XX | XX |
| | | Not at all acceptable | (XX.X%) | (XX.X%) | (XX.X%) |
| 67 | The state of the s | e to return to your usual daily activiti<br>ck to work, social events, exercise, dr | | following an injection | appointment |
| | | Nover | XX | XX | XX |
| | | Never | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Rarely | XX | XX | XX |
| | | Nately | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Sometimes | XX | XX | XX |
| | | Joineumes | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Often | XX | XX | XX |
| | | Often | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Always | XX | XX | XX |
| | | 7 HWays | (XX.X%) | (XX.X%) | (XX.X%) |
| 68 | How bothered were yo | ou by <b>pain <u>DURING</u> the injection</b> ? | | | |
| | | Not at all | XX | XX | XX |
| | | INUL AL AII | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A little | XX | XX | XX |
| | | A IILLIC | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Moderately | XX | XX | XX |
| | | iviouerately | (XX.X%) | (XX.X%) | (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Very | XX | XX | XX |
| | | VCIY | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Extremely | XX | XX | XX |
| | | Extremely | (XX.X%) | (XX.X%) | (XX.X%) |
| 69 | Think back to your <b>first</b> injection, please rate the amount of pain/discomfort you experienced <b>AFTER</b> receiving your <b>first</b> APRETUDE injection | | | | |
| | | O (No main) | XX | XX | XX |
| | | 0 (No pain) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | _ | XX | XX | XX |
| | | 1 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | _ | XX | XX | XX |
| | | 2 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 3 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 4 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 5 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 6 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 7 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 8 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 9 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | 1 | XX | XX |
| | | 10 (Extreme pain) | XX<br>(XX.X%) | (XX.X%) | ^^<br>(XX.X%) |
| | Navateialaalaantuuruulaat/a | | | | |
| 70 | AFTER receiving your most r | nost recent injection. Please ra<br>recent APRETUDE injection | te the amount of | pain/discorniort you | experienced |
| | | 0 (No pain) | XX | XX | XX |
| | | O (NO pairi) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 1 | XX | XX | XX |
| | | 1 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 2 | XX | XX | XX |
| | | 2 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 3 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 4 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 5 | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 6 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 7 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 8 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 9 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 10 (Extreme pain) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 71 | How acceptable was your pair | n? | | | |
| | | Totally acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Moderately acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 72 | Which of the following things | have you tried to reduce the p | ain/discomfort f | ollowing your inject | ions? |
| | | Took over-the-counter pain relievers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Used a hot compress | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Used a cold compress | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Avoided sitting for long periods of time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Light stretching and exercise | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.220. Summary of Patient Study Participants' Labs and Missed Doses (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 53 | Have you missed any of your APRETUDE injection visits in the last 6 months? This means not receiving an injection within your injection window. | | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 54 | Was missing your APRETUDE in | jection visits planned or unplann | ed? | • | |
| | | All the injection visits I<br>missed were planned | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the injection visits I missed were planned and some were unplanned | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | All the injection visits I missed were unplanned | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 55 | Did you start oral PrEP after missing any of your injection visits? | | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 56 | How easy or difficult was it to s | tart oral PrEP after a missed injec | ction visit? | | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 57 | How acceptable was it to start | oral PrEP after a missed injection | visit? | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.301. Summary of Feasibility and Acceptability of Telehealth (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 22 | Have you used telehealth for any APRETUDE services in the last 6 months, such as completing forms online, video chatting with your provider, getting reminders about your injection, or scheduling injection appointments online? | | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 25 | What APRETUDE services do/o | I<br>did you receive via telehealth? | | (7.5.15.75) | (7007) |
| А | Completing relevant clinic visit forms online | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Your doctor ordering an HIV test at a lab near your home where you can go to take the test | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | A nurse coming to your<br>home to give you an HIV<br>test | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | Video chatting with your doctor | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | Receiving reminders (e.g.,<br>text, email) about your<br>scheduled injection<br>appointment | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | Scheduling your injection appointment online to go to your clinic/doctor's office for the injection | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Scheduling your injection appointment online for a nurse to come to your home and to give you the injection | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | A nurse coming to your<br>home to give you the<br>injection | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | Sending messages to your doctor online | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| I | Reviewing your health documents, such as test results, online | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 26 | How <b>comfortable</b> is/was it to | use each of the following tele | ehealth services fo | or APRETUDE? | 1 |
| А | Completing relevant clinic visit forms online | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Your doctor ordering an HIV test at a lab near your home where you can go to take the test | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | A nurse coming to your home to give you an HIV test | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | Video chatting with your doctor | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| E | Receiving reminders (e.g.,<br>text, email) about your<br>scheduled injection<br>appointment | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Scheduling your injection appointment online to go to your clinic/doctor's office for the injection | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | A nurse coming to your home to give you the injection | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | Sending messages to your doctor online | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| I | Reviewing your health documents, such as test results, online | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 27 | How <u>convenient</u> is/was it to u<br>well with your life activities ar | se each of the telehealth servior<br>and plans, with little trouble. | ces for APRETUD | E? By convenient, w | re mean fitting in |
| А | Completing relevant clinic visit forms online | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Your doctor ordering an HIV test at a lab near your home where you can go to take the test | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | A nurse coming to your home to give you a HIV test | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | Video chatting with your doctor | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | Receiving reminders (e.g.,<br>text, email) about your<br>scheduled injection<br>appointment | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Scheduling your injection appointment online to go to your clinic/doctor's office for the injection | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| G | A nurse coming to your home to give you the injection | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | Sending messages to your doctor online | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| l | Reviewing your health documents, such as test results, online | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 28 | On average, how long did you | u wait to connect to a doctor fo | or video chat? | | |
| | | Up to 5 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 6 to 10 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 11 to 15 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 16 to 30 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | More than 30 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 29 | I would recommend telehealt | h services for APRETUDE to oth | ner people. | | |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.302. Summary of Quality of Care for Patient Study Participants (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 80 | To what extent do you agree v<br>clinic/provider? | vith each of the following sta | tements regardinį | g your experience w | ith your |
| А | My provider explained<br>medical words that were<br>used so that I could<br>understand them. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | My provider encouraged me to ask questions. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | My provider really respected me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | My provider gave me<br>enough time to say what I<br>though was important. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | My provider listened carefully to what I had to say. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | - | Agree | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | Disagree | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | Completely disagree | (XX.X%) | (XX.X%) | (XX.X%) |
| F | My provider explained why tests were being done. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | My provider made me feel comfortable talking about personal things. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | My privacy was respected. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| I | My provider does not judge<br>me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| J | The provider had a respectful attitude towards my sexual orientation. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Agree | XX | XX | XX |
| | | 7.8.00 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | (\text{\text{XX}} | (\times.\times/\dots) | (XX.X/6) |
| | | Completely disagree | (XX.X%) | (XX.X%) | (XX.X%) |
| K | The staff at the clinic does not judge me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| L | The staff at this clinic is kind and respectful to me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| М | I sometimes felt insulted<br>when the clinic staff spoke<br>to me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| N | I felt judged by the clinic staff for being on PrEP. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 0 | I felt judged by my provider for being on PrEP. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.303. Summary of Quality of Care for Patient Study Participants (Month 6/7), N=XX, Non-Score Questions

| Question | | | Re | sponse | |
|---|---|---|---|---|---|
| each of the | t extent do you agree with following statements our experience with your vider? | Completely Agree | Agree | Neither agree nor<br>disagree | Disagree |
| I. My provid | der does not judge me. | | | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynar | mic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routii | ne Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | | | Response | | |
|---|---|---|---|---|---|
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, D | ynamic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, R | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | otal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | | Response | | | |
|---|---|---|---|---|---|
| n (%) | | | | | |
| Gender, Total | ' | | | | |
| Men who<br>with men | have sex | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Transgen | der men | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| J. The provider had a resp | ectful attitude to | wards my sexual or | entation. | | |
| Study Arms | | | | | |
| Total | | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Dynamic<br>Implemer | ntation | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Routine<br>Implemer | ntation | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Race, Dynamic Implemer | tation | | | | |
| Asian | | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Black or <i>A</i><br>American | | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| White | | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Other | | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Race, Routine Implement | ation | | | | |
| Asian | | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |



| Question | | | Response | | |
|---|---|---|---|---|---|
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | ı |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | utine Implementation | | | | ı |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | tal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tot | al | | | | |
| | Men who have sex<br>with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| K. The staff | at the clinic does not judge me | • | | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynar | nic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African | XX | XX | XX | XX |
| | American | | | | |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | ynamic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | 1 | 1 | I |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | . , | , | , | , , |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | | | Response | | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| Ethnicity, 7 | | | I | I | I |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, To | otal | | I | I | |
| | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | · | | | - |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| L. The staf | f at this clinic is kind and respect | ful to me. | 1 | 1 | |
| Study Arm | S | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dyna | amic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| (N = X | X) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Race, Routine Implem | entation | | | | |
| Asian | | XX | XX | XX | XX |
| (N = X | X) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Black<br>Ameri | or African<br>can | XX | XX | XX | XX |
| (N = X | X) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| White | | XX | XX | XX | XX |
| (N = X | X) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Other | | XX | XX | XX | XX |
| (N = X | X) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Race, Total | | | | | |
| Asian | | XX | XX | XX | XX |
| (N = X | X) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Black<br>Ameri | or African<br>can | XX | XX | XX | XX |
| (N = X | X) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| White | | XX | XX | XX | XX |
| (N = X | X) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Other | | XX | XX | XX | XX |
| (N = X | X) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Ethnicity, Dynamic Im | plementation | | | | |
| Hispar | nic or Latino | XX | XX | XX | XX |
| (N = X | X) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Not H | ispanic or Latino | XX | XX | XX | XX |
| (N = X | X) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Ethnicity, Routine Imp | lementation | | | | |
| Hispar | nic or Latino | XX | XX | XX | XX |
| (N = X | X) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |


| Question | | onse | | | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, 1 | Total | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, To | otal | | | | |
| | Men who have sex<br>with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| M. I somet | times felt insulted when the clini | c staff spoke to me. | | | |
| Study Arm | S | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (NI )(V) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | (N = XX) | , , | | | (////////////////////////////////////// |
| | n (%) | , | | | (///.///0) |
| Race, Dyna | | · , , | | | (777.776) |
| Race, Dyna | n (%) | XX | XX | XX | XX |
| Race, Dyna | n (%)<br>amic Implementation | | | XX<br>(XX.X%) | |
| Race, Dyna | n (%) amic Implementation Asian | XX | XX | | XX |
| Race, Dyna | n (%) amic Implementation Asian (N = XX) | XX | XX | | XX |
| Race, Dyna | n (%) amic Implementation Asian (N = XX) n (%) Black or African | XX<br>(XX.X%) | XX<br>(XX.X%) | (XX.X%) | XX<br>(XX.X%) |
| Race, Dyna | n (%) amic Implementation Asian (N = XX) n (%) Black or African American | XX<br>(XX.X%) | XX<br>(XX.X%) | (XX.X%) | XX<br>(XX.X%) |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routi | ne Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, D | ynamic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| Ethnicity, | Routine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, | Total | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, T | otal | | | | |
| | Men who have sex<br>with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| N. I felt ju | dged by the clinic staff for being | on PrEP. | | 1 | |
| Study Arn | | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | , | , , | , | , , |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dyn | amic Implementation | | 1 | 1 | I |
| . , | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | , , | , , | , , | ,, |
| | Black or African<br>American | XX | XX | XX | XX |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routin | e Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | otal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tot | al | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| O. I felt judg | ged by my provider for being or | n PrEP. | | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynar | nic Implementation | | 1 | 1 | 1 |
| | Asian | XX | XX | XX | XX |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routir | ne Implementation | | | | ı |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | ı |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | | onse | | | |
|---|---|---|---|---|---|
| Ethnicity, Dynamic Implementation | | | | | |
| Hi | spanic or Latino | XX | XX | XX | XX |
| (N | = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n ( | %) | | | | |
| No | ot Hispanic or Latino | XX | XX | XX | XX |
| (N | = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n ( | %) | | | | |
| Ethnicity, Routine | Implementation | | | | |
| His | spanic or Latino | XX | XX | XX | XX |
| (N | = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n ( | %) | | | | |
| No | ot Hispanic or Latino | XX | XX | XX | XX |
| (N | = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n ( | %) | | | | |
| Ethnicity, Total | | | | | |
| His | spanic or Latino | XX | XX | XX | XX |
| (N | = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n ( | %) | | | | |
| No | ot Hispanic or Latino | XX | XX | XX | XX |
| (N | = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n ( | %) | | | | |
| Gender, Total | · | | | | |
| | en who have sex<br>th men | XX | XX | XX | XX |
| (N | = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n ( | %) | | | | |
| Tra | ansgender men | XX | XX | XX | XX |
| (N | = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n ( | %) | | | | |



Table 6.304. Summary of Quality of Care for Patient Study Participants (Month 6/7), N=XX, Score Questions

| Question | | Re | esponse | |
|---|---|---|---|---|
| 80. To what extent do you agree with<br>each of the following statements<br>regarding your experience with your<br>clinic/provider? | n<br>Completely Agree | Agree | Neither agree nor<br>disagree | Disagree |
| A. My provider explained medical words that were used so that I could understand them. | | | | |
| Study Arms | | | | |
| Total | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Dynamic<br>Implementation | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Routine<br>Implementation | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Race, Dynamic Implementation | | | | |
| Asian | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Black or African<br>American | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| White | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Other | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Race, Routine Implementation | | | | |
| Asian | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Black or African<br>American | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | tal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | | Response | | |
|---|---|---|---|---|
| n (%) | | | | |
| Gender, Total | | ' | | |
| Men who l<br>with men | nave sex XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Transgend | er men XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| B. My provider encourage | d me to ask questions. | | | |
| Study Arms | | | | |
| Total | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Dynamic<br>Implement | tation XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Routine<br>Implement | tation | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Race, Dynamic Implement | ation | | | |
| Asian | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Black or Af<br>American | rican XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| White | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Other | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Race, Routine Implementa | ition | | | |
| Asian | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | 1 | ı |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dyn | amic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Rou | tine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Tota | al | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tot | tal | | | | |
| | Men who have sex<br>with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | <u> </u> | | | · |
| C. My provi | der really respected me. | | 1 | 1 | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynar | mic Implementation | | I | I | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | • | , | | , |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | , |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | . , | . , | | , , |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | ı |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | 1 | 1 | 1 |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| Ethnicity, T | otal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, To | tal | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| D. My prov | ider gave me enough time to sa | y what I though was | s important. | | |
| Study Arms | i | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dyna | mic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | xx |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |



| Question | | Response | | | |
|---|---|---|---|---|---|
| (N = | XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | ) | | | | |
| Race, Routine Imple | mentation | | | | |
| Asia | ı | XX | XX | XX | XX |
| (N = | XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | ) | | | | |
| | k or African<br>rican | XX | XX | XX | XX |
| (N = | XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | ) | | | | |
| Whit | e | XX | XX | XX | XX |
| (N = | XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | ) | | | | |
| Othe | er | XX | XX | XX | XX |
| (N = | XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | ) | | | | |
| Race, Total | | | | | |
| Asiaı | ı | XX | XX | XX | XX |
| (N = | XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | ) | | | | |
| | k or African<br>rican | XX | XX | XX | XX |
| (N = | XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | ) | | | | |
| Whit | e | XX | XX | XX | XX |
| (N = | XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | ) | | | | |
| Othe | er | XX | XX | XX | XX |
| (N = | XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | ) | | | | |
| Ethnicity, Dynamic I | mplementation | | | | |
| Hisp | anic or Latino | XX | XX | XX | XX |
| (N = | XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | ) | | | | |
| Not | Hispanic or Latino | XX | XX | XX | XX |
| (N = | XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (% | ) | | | | |
| Ethnicity, Routine In | plementation | | | | |
| Hisp | anic or Latino | XX | XX | XX | XX |
| (N = | XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, T | Гotal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, To | otal | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| E. My prov | ider listened carefully to what I | had to say. | | | |
| Study Arms | S | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | amic Implementation | | | | |
| Race, Dyna | anne imprementation | | | | |
| Race, Dyna | Asian | XX | XX | XX | XX |
| Race, Dyna | | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | (XX.X%) |
| Race, Dyna | Asian | | | | |
| Race, Dyna | Asian (N = XX) | | | | |
| Race, Dyna | Asian (N = XX) n (%) Black or African | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Race, Dyna | Asian (N = XX) n (%) Black or African American | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| luestion | | Response | | | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routir | ne Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | ynamic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | · | | | · |



| Question | n Response | | | | |
|---|---|---|---|---|---|
| Ethnicity, | Routine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, | Total | | | | ı |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | <u> </u> | | | |
| Gender, T | | | ı | 1 | I |
| , | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| F. My prov | vider explained why tests were b | eing done. | | I | |
| Study Arm | | - | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | - | | | · |
| Race, Dyn | amic Implementation | | 1 | 1 | I |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | . , | . , | . , | , , |
| | Black or African<br>American | XX | XX | XX | XX |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routin | e Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | otal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tot | al | | - | | |
| | Men who have sex<br>with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| G. My provi | der made me feel comfortable | talking about perso | nal things. | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynan | nic Implementation | | I | ı | I |
| · • | Asian | XX | XX | XX | XX |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Rou | tine Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Tota | al | | 1 | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | , | | | . , |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| Ethnicity, Dynamic Implementation | | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | utine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | tal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tota | al . | | | | |
| | Men who have sex<br>with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| H. My privac | y was respected. | | | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |



| Question | | | | | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynai | mic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routi | ne Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question Response | | | | | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, D | ynamic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, R | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, T | otal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, To | tal | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



Table 6.305. Summary of Utility of Proposed Implementation Strategies (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 49 | Have you used any of the follo | wing while taking APRETUC | E? | | |
| А | Brochures and other print<br>materials to educate you on<br>APRETUDE | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Videos to educate you on<br>HIV, PrEP, APRETUDE<br>materials (DI) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| С | A digital calendar specifically<br>made for APRETUDE to help<br>you plan your injections –<br>found on PillarSpot (DI) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| D | Reminders about your injections | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Е | Having video or telephone appointments with your doctor | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Sending chats or texts to<br>your doctor on the Pillar<br>Spot (DI) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| G | Having a nurse come to your<br>home to conduct your HIV<br>tests (DI) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| Н | Having a nurse come to your home to give your injection (DI) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| I | Receiving transportation to<br>the clinic/doctor's office for<br>your injection (DI) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| J | A website/app where you access APRETUDE information – the Pillar Spot (DI) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| K | The website where you access APRETUDE information (RI) | Yes | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| 50 | How useful has each of these | been in supporting you while | taking APRETUDI | Ξ? | |
| А | Brochures and other print<br>materials to educate you on<br>APRETUDE | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Videos to educate you on<br>HIV, PrEP, APRETUDE<br>materials (DI) | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| С | A digital calendar specifically<br>made for APRETUDE to help<br>you plan your injections –<br>found on PillarSpot (DI) | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| D | Reminders about your injections | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| E | Having video or telephone appointments with your doctor | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Sending chats or texts to<br>your doctor on the Pillar<br>Spot (DI) | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| G | Having a nurse come to your home to conduct your HIV test (DI) | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| Н | Having a nurse come to your home to give your injection (DI) | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| I | Receiving transportation to<br>the clinic/doctor's office for<br>your injection (DI) | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| J | A website/app where you<br>access APRETUDE<br>information – the Pillar Spot<br>(DI) | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| K | The website where you access APRETUDE information (RI) | Not at all useful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| 51 | Did your clinic or doctor offer | the following for APRETUD | E visits? | | |
| Α | Injections on specific days of the week | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| В | Ability to show up for your injection without an appointment | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | Appointments where you only get your injection and leave | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | Schedule out your injection appointments for 6 months or more | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | You and your doctor discussing the pros and cons (e.g., side effects, switching) of different PrEP options and together deciding which one is right for you. | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 52 | How useful has each of these | been in supporting you while | e taking APRETUDI | ? | |
| А | Injections on specific days of the week | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| В | Ability to show up for your injection without an appointment | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | Appointments where you only get your injection and leave | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | Schedule out your injection appointments for 6 months or more | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Е | You and your doctor discussing the pros and cons (e.g., side effects, switching) of different PrEP options and together deciding which one is right for you. | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.306. Summary of Patient Study Participants' Preferences/Acceptability of APRETUDE Information, Appointment Reminders, and Locations (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 61 | If you have questions about APRETUDE, where do you find information? | | | | |
| | | Product website | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Written materials such<br>as the study handbook<br>from my healthcare<br>provider | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Speaking to a healthcare provider | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Social Media | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Internet search | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Friends | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Family | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The study app/website | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not had any questions so far | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not find answers<br>to my questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 62 | How did you receive reminders abou | t your injection appointmer | nts? | | |
| | | Phone calls | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Texts/SMS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Existing clinic app reminder | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | E-mails | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Reminder in the postal mail | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Face-to-face reminder<br>from a healthcare<br>provider | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Written reminder/appointment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | card with date and time | | | |
| | | The study app/website | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Another type of reminder (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not received any reminders | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 63 | Which type(s) of appointment remin | ders are most helpful in kee | ping your ap | pointment? | |
| | | Phone calls | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Texts/SMS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Existing clinic app reminder | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | E-mails | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Reminder in the postal mail | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Face-to-face reminder<br>from a healthcare<br>provider | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Written<br>reminder/appointment<br>card with date and<br>time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The study app/website (DI) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Another type of reminder (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not think any of<br>the reminders are<br>helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 64 | Where else would you consider recei | ving your injections? | | | |
| | | Retail pharmacy clinic<br>(e.g., Minute Clinic,<br>CVS) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other pharmacy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Hospital outpatient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Infusion center | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Community-based organization | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | STD/STI clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Department of Health clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | PrEP clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Community health center | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Mobile van | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Nurse coming to your home | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.307. Summary of Appointment Scheduling (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 58 | How easy or difficult is it to schedule appointments at the clinic/practice for your injections? | | | | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not scheduled<br>any appointments at<br>the clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 59 | How easy or difficult is it to reschedule appointments at the clinic/practice for your injections? | | | | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not needed to reschedule any appointments | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 60 | How did you <u>reschedule</u> your app | ointment? | | | |
| | | I called the clinic/doctor's office | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I emailed the clinic/doctor's office | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I texted the clinic/doctor's office | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I scheduled the appointment online | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I sent a message on the online portal of the clinic/doctor's office | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |


| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | I went to the clinic/doctor's office | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.401. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 36 | On average, how lon when you leave? | g have you spent at the clinic/practice for \ | your injection | visit from arrival at | the clinic to |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not gotten any of my injections at a clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | How acceptable is co | oming to the clinic every 2 months for an in | jection? | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | How convenient are with little trouble. | your clinic's hours? By convenient, we mea | n fitting well | with your life activit | ies and plans, |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 39 | How easy or difficult | has it been to get to the clinic every 2 mor | | | <u>'</u> |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Very easy | XX | XX | XX |
| | | , , | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 40 | Approximately how lor | ng has it taken you to get to the clinic/pra | ctice from yo | ur home to receive | your injection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | How did you get to the | clinic/practice for your injections? | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drove a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 43 | | transportation provided by your clinic/pr<br>itting in well with your life activities and p | | | ry 2 months? <i>By</i> |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please provide your op | inion of the transportation provided by the | | (************************************** | (* * |
| | The transportation helped me keep my appointments. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The transportation service was easy to use. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Have you needed to se injection visits? | ek additional childcare/eldercare/other c | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 46 | Have you taken ar | ny time off from work to receive injections? | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How much time di | id you take off work to receive your injection | s? | | |
| | | I needed to take a whole day off work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a whole day off work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | Was your time off | work for injections generally paid or unpaid? | ) | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.402. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Race, Dynamic Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 36 | On average, how you leave? | w long have you spent at the clinic/prac | ctice for your in | jection visit fror | m arrival at th | e clinic to when |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not gotten any of my<br>injections at a clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | How acceptable | e is coming to the clinic every 2 months | for an injectior | 1? | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | How convenien with little troub | t are your clinic's hours? <i>By convenient,</i><br>le. | , we mean fittir | ng well with you | r life activities | and plans, |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 39 | How easy or dif | ficult has it been to get to the clinic eve | ry 2 months fo | r your injection | ? | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 40 | Approximately h | now long has it taken you to get to the o | clinic/practice f | rom your home | to receive y | our injection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | How did you ge | t to the clinic/practice for your injection | s? | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drove a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 43 | | t is the transportation provided by your mean fitting in well with your life activit | clinic/practice | for your injection | n visit every | |
| | , | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please provide y | our opinion of the transportation provi | ded by the clin | ic | | |
| | The<br>transportation<br>helped me<br>keep my<br>appointments. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The transportation service was easy to use. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Have you neede injection visits? | d to seek additional childcare/eldercare | e/other care to | come to the cli | nic/practice fo | or your |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 46 | Have you taken | any time off from work to receive inject | tions? | 1 | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How much time | did you take off work to receive your i | njections? | | | |
| | | I needed to take a whole day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a whole day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | Was your time o | off work for injections generally paid or | unpaid? | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.403. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Race, Routine Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 36 | On average, ho you leave? | w long have you spent at the clinic/prac | tice for your in | jection visit froi | m arrival at th | e clinic to when |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not gotten any of my injections at a clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | How acceptable | e is coming to the clinic every 2 months | for an injection | 1? | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | How convenient are your clinic's hours? By convenient, we mean fitting well with your life activities and plans, with little trouble. | | | | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 39 | How easy or di | fficult has it been to get to the clinic eve | ry 2 months fo | r your injection | ? | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 40 | Approximately l | how long has it taken you to get to the c | clinic/practice f | rom your home | to receive yo | our injection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | How did you ge | t to the clinic/practice for your injection | ıs? | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drove a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 43 | | t is the transportation provided by your<br>mean fitting in well with your life activit | clinic/practice | for your injection | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please provide y | our opinion of the transportation provi | ded by the clin | ic | | |
| | The<br>transportation<br>helped me<br>keep my<br>appointments. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The<br>transportation<br>service was<br>easy to use. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Have you neede injection visits? | d to seek additional childcare/eldercare | e/other care to | come to the cli | inic/practice f | or your |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 46 | Have you taken | any time off from work to receive inject | ions? | | 1 | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How much time | did you take off work to receive your i | njections? | | | |
| | | I needed to take a whole day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a whole day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | Was your time o | off work for injections generally paid or | unpaid? | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.404. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Race, Total

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 36 | On average, how you leave? | w long have you spent at the clinic/prac | tice for your in | jection visit fror | n arrival at th | e clinic to when |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not gotten any of my<br>injections at a clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | How acceptable | is coming to the clinic every 2 months | for an injectior | 1? | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | How convenient with little troubl | t are your clinic's hours? <i>By convenient,</i><br>le. | we mean fittir | ng well with you | r life activities | and plans, |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 39 | How easy or diff | ficult has it been to get to the clinic eve | ry 2 months fo | r your injection | ? | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 40 | Approximately how long has it taken you to get to the clinic/practice from your home to receive your injection? | | | | | |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | How did you ge | t to the clinic/practice for your injection | s? | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drove a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 43 | | t is the transportation provided by your<br>mean fitting in well with your life activiti | clinic/practice | for your injection | n visit every | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please provide y | our opinion of the transportation provi | ded by the clin | ic | | |
| | The<br>transportation<br>helped me<br>keep my<br>appointments. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The<br>transportation<br>service was<br>easy to use. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Have you neede injection visits? | d to seek additional childcare/eldercare | e/other care to | come to the cli | inic/practice f | or your |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 46 | Have you taken | any time off from work to receive inject | ions? | | 1 | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How much time | did you take off work to receive your i | njections? | | | |
| | | I needed to take a whole day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a whole day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | Was your time o | off work for injections generally paid or | unpaid? | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.405. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Ethnicity, Study Arms

| | | Response | Dynamic Implementation | | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | | Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic<br>or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| 36 | On average, ho you leave? | ow long have you spent at the clinic/prac | ctice for your i | njection visit fror | m arrival at t | he clinic to when |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not gotten any of my<br>injections at a clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | How acceptable is coming to the clinic every 2 months for an injection? | | | | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | How convenier with little troul | nt are your clinic's hours? <i>By convenient,</i><br>ble. | we mean fitt | ing well with you | r life activitie | es and plans, |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 39 | How easy or di | ifficult has it been to get to the clinic eve | ry 2 months f | or your injection | ? | |



| | | | Dynamic Implementation | | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic<br>or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic o<br>Latino<br>(N = XX)<br>n (%) |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 40 | Approximately | how long has it taken you to get to the o | clinic/practice | from your home | to receive y | our injection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | How did you ge | t to the clinic/practice for your injection | s? | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drove a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic II | mplementation | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic<br>or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please provide yo | our opinion of the transportation pro | ovided by the cl | inic | | |
| | The<br>transportation<br>helped me<br>keep my<br>appointments. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The transportation service was easy to use. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Have you needed injection visits? | d to seek additional childcare/elderca | | co come to the cli | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic II | mplementation | Routine | Implementation |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | n Response | Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic<br>or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 46 | Have you taken | any time off from work to receive injec | tions? | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How much time | e did you take off work to receive your ir | njections? | | | |
| | | I needed to take a whole day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a whole day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | Was your time | off work for injections generally paid or | unpaid? | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.406. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Ethnicity, Total

| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 36 | On average, how | w long have you spent at the clinic/pract<br>? | ice for your injection visit fi | om arrival at the clinic to |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not gotten any of my<br>injections at a clinic | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | How acceptable | is coming to the clinic every 2 months f | or an injection? | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | How convenient are your clinic's hours? By convenient, we mean fitting well with your life activities and plans, with little trouble. | | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 39 | How easy or diff | ficult has it been to get to the clinic ever | y 2 months for your injection | on? |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 40 | Approximately injection? | how long has it taken you to get to the cl | inic/practice from your ho | me to receive your |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | How did you g | et to the clinic/practice for your injections | ? | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drove a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 43 | | nt is the transportation provided by your o<br>we mean fitting in well with your life activ | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please provide y | your opinion of the transportation provid | | |
| | The<br>transportation<br>helped me<br>keep my<br>appointments. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The transportation service was easy to use. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Have you neede injection visits? | ed to seek additional childcare/eldercare | other care to come to the | clinic/practice for your |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 46 | Have you taken | any time off from work to receive inject | ions? | 1 |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 47 | How much tim | e did you take off work to receive your in | jections? | |
| | | I needed to take a whole day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a whole day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | Was your time | off work for injections generally paid or u | ınpaid? | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.407. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Gender, Total

| | | | Dynamic Im | plementation | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Men who<br>have sex<br>with men<br>(N = XX)<br>n (%) | Transgender<br>Men<br>(N = XX)<br>n (%) | Men who have sex with men (N = XX) n (%) | Transgender<br>Men<br>(N = XX)<br>n (%) |
| 36 | On average, how<br>when you leave | w long have you spent at the clinic/prac? | tice for your i | njection visit fror | m arrival at the | e clinic to |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not gotten any of my<br>injections at a clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | How acceptable | e is coming to the clinic every 2 months | for an injectio | n? | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | How convenien | t are your clinic's hours? <i>By convenient,</i><br>le. | we mean fitti | ing well with you | r life activities | and plans, |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 39 | How easy or dif | ficult has it been to get to the clinic eve | ry 2 months f | or your injection | ? | |



| | | | Dynamic Im | plementation | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Men who have sex with men (N = XX) n (%) | Transgender<br>Men<br>(N = XX)<br>n (%) | Men who have sex with men (N = XX) n (%) | Transgender<br>Men<br>(N = XX)<br>n (%) |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 40 | Approximately | how long has it taken you to get to the o | clinic/practice | from your home | to receive you | ur injection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | How did you ge | t to the clinic/practice for your injection | s? | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drove a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic In | plementation | plementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Men who have sex with men (N = XX) n (%) | Transgender<br>Men<br>(N = XX)<br>n (%) | Men who have sex with men (N = XX) n (%) | Transgender<br>Men<br>(N = XX)<br>n (%) |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please provide y | our opinion of the transportation pro | vided by the cli | nic | | |
| | The transportation helped me keep my appointments. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The transportation service was easy to use. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Have you neede injection visits? | d to seek additional childcare/elderca | are/other care t | o come to the cli | inic/practice fo | or your |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic Im | plementation | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Men who<br>have sex<br>with men<br>(N = XX)<br>n (%) | Transgender<br>Men<br>(N = XX)<br>n (%) | Men who<br>have sex<br>with men<br>(N = XX)<br>n (%) | Transgender<br>Men<br>(N = XX)<br>n (%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 46 | Have you taken | any time off from work to receive injec | tions? | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How much time did you take off work to receive your injections? | | | | | |
| | | I needed to take a whole day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a whole day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | Was your time o | off work for injections generally paid or | unpaid? | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.408. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 30 | Did you complete a Sexua | l Health Assessment from your p | orovider or cli | nic/practice in the last | 6 months? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 31 | Did your provider or anoth | ner person at the clinic/practice | discuss the re | sults of the assessmer | nt with you? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't remember | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 32 | Who discussed the results | of the assessment with you? | | | |
| | | My healthcare provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 33 | How helpful was discussin | g the results with your provider | or another pe | erson at the clinic/prac | ctice? |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 34 | Please rate your experience | ce with the Sexual Health Assess | ment | | |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | It was easy to take the<br>Sexual Health Assessment<br>on my digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor sent<br>the assessment before my<br>appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about<br>the privacy of my<br>answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor was assessing my sexual health. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not complete t | he assessment? | | | |
| | | I did not receive a Sexual<br>Health Assessment from<br>my provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made me feel uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned about the privacy of my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share<br>sexual health information<br>with my doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand why<br>my doctor or clinic was<br>asking me to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.409. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Race, Dynamic Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 30 | Did you complete a Sex | kual Health Assessment fro | om your provi | ider or clinic/praction | ce in the last 6 mo | onths? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 31 | Did your provider or ar | other person at the clinic, | practice disc | uss the results of th | ie assessment wit | th you? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't remember | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 32 | Who discussed the res | ults of the assessment wit | h you? | | | |
| | | My healthcare provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 33 | How helpful was discus | sing the results with your | provider or a | nother person at th | ne clinic/practice? | > |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 34 | Please rate your experi | ence with the Sexual Heal | th Assessmer | nt | | |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | It was easy to take<br>the Sexual Health<br>Assessment on my<br>digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor<br>sent the assessment<br>before my<br>appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor<br>was assessing my<br>sexual health. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment<br>made me feel<br>uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not comp | ete the assessment? | | | | |
| | | I did not receive a<br>Sexual Health<br>Assessment from my<br>provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX | XX | XX | XX |


| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made<br>me feel<br>uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned<br>about the privacy of<br>my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to<br>share sexual health<br>information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand<br>why my doctor or<br>clinic was asking me<br>to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.410. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Race, Routine Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 30 | Did you complete a Se | exual Health Assessment fro | om your provi | ider or clinic/praction | ce in the last 6 mo | onths? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 31 | Did your provider or a | nother person at the clinic, | /practice disc | uss the results of th | ie assessment wi | th you? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't remember | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 32 | Who discussed the res | sults of the assessment wit | h you? | | | |
| | | My healthcare provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 33 | How helpful was discu | issing the results with your | provider or a | nother person at th | ne clinic/practice? | ) |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 34 | Please rate your experience with the Sexual Health Assessment | | | | | |
| | It was easy to take<br>the Sexual Health<br>Assessment on my<br>digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor<br>sent the assessment<br>before my<br>appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned<br>about the privacy of<br>my answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor<br>was assessing my<br>sexual health. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment<br>made me feel<br>uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not comp | lete the assessment? | | | | |
| | | I did not receive a<br>Sexual Health<br>Assessment from my<br>provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | l forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made<br>me feel<br>uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned<br>about the privacy of<br>my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to<br>share sexual health<br>information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand<br>why my doctor or<br>clinic was asking me<br>to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.411. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Race, Total

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 30 | Did you complete a Sex | kual Health Assessment fro | om your provi | ider or clinic/praction | ce in the last 6 mo | onths? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 31 | Did your provider or ar | other person at the clinic, | practice disc | uss the results of th | ie assessment wit | th you? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't remember | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 32 | Who discussed the res | ults of the assessment wit | h you? | | | |
| | | My healthcare provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 33 | How helpful was discus | sing the results with your | provider or a | nother person at th | ne clinic/practice? | ) |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 34 | Please rate your experi | ence with the Sexual Heal | th Assessmer | nt | | |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | It was easy to take<br>the Sexual Health<br>Assessment on my<br>digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor<br>sent the assessment<br>before my<br>appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor<br>was assessing my<br>sexual health. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Agree | XX | XX | XX | XX |
| | | - C | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment<br>made me feel<br>uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not comp | lete the assessment? | | | | |
| | | I did not receive a<br>Sexual Health<br>Assessment from my<br>provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX | XX | XX | XX |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made<br>me feel<br>uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned<br>about the privacy of<br>my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to<br>share sexual health<br>information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand<br>why my doctor or<br>clinic was asking me<br>to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.412. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Ethnicity, Study Arms

| | | | Dynamic Imp | olementation | Routine Imp | olementation |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| 30 | Did you complete a S | Sexual Health Assessment f | rom your provic | ler or clinic/prad | ctice in the last 6 | months? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 31 | Did your provider or | another person at the clini | c/practice discu | ss the results of | the assessment | with you? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't remember | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 32 | Who discussed the r | esults of the assessment wi | ith you? | | | |
| | | My healthcare provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 33 | How helpful was disc | cussing the results with you | ır provider or an | | | |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX (XX.X%) | XX | XX | XX |



| | Question | Response | Dynamic Implementation | | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | | | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| | | | | (XX.X%) | (XX.X%) | (XX.X%) |
| 34 | Please rate your expe | rience with the Sexual He | alth Assessment | -<br>- | I | |
| | It was easy to take<br>the Sexual Health<br>Assessment on my<br>digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor | XX | XX | XX | XX |
| | | disagree | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX | XX | XX | XX |
| | | Completely agree | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | I like that my doctor<br>sent the assessment<br>before my<br>appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX | XX | XX | XX |
| | | Disagree | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned<br>about the privacy of<br>my answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor<br>was assessing my<br>sexual health. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | Response | Dynamic Implementation | | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| | | Disagrap | XX | XX | XX | XX |
| | | Disagree | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not comp | lete the assessment? | | | | |
| | | I did not receive a<br>Sexual Health<br>Assessment from my<br>provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic Implementation | | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made me feel uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned<br>about the privacy of<br>my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to<br>share sexual health<br>information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand<br>why my doctor or<br>clinic was asking me<br>to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.413. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Ethnicity, Total

| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 30 | Did you complete a Sexual He | ealth Assessment from your provide | r or clinic/practice in the | last 6 months? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 31 | Did your provider or another | person at the clinic/practice discuss | s the results of the assess | ment with you? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't remember | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 32 | Who discussed the results of | the assessment with you? | | |
| | | My healthcare provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 33 | How helpful was discussing th | ne results with your provider or ano | ther person at the clinic/p | practice? |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 34 | Please rate your experience v | vith the Sexual Health Assessment | | |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | It was easy to take the Sexual<br>Health Assessment on my<br>digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor sent the assessment before my appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor was assessing my sexual health. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX | XX |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not complete the assessment? | | | |
| | | I did not receive a Sexual<br>Health Assessment from my<br>provider or clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | l forgot | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made me feel uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | I was concerned about the privacy of my answers | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share sexual<br>health information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand why my<br>doctor or clinic was asking me<br>to complete the assessment | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.414. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Gender

| Question<br>Number | Question | Response | Men who have sex<br>with men<br>(N = XX)<br>n (%) | Transgender men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 30 | Did you complete a Sexual Hea | alth Assessment from your provide | r or clinic/practice in the | last 6 months? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 31 | Did your provider or another p | person at the clinic/practice discuss | the results of the assess | ment with you? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't remember | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 32 | Who discussed the results of t | he assessment with you? | | |
| | | My healthcare provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 33 | How helpful was discussing th | e results with your provider or ano | ther person at the clinic/ | practice? |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 34 | Please rate your experience w | ith the Sexual Health Assessment | | |



| Question<br>Number | Question | Response | Men who have sex<br>with men<br>(N = XX)<br>n (%) | Transgender men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | It was easy to take the Sexual<br>Health Assessment on my<br>digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor sent the assessment before my appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor was assessing my sexual health. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX | XX |



| Question<br>Number | Question | Response | Men who have sex<br>with men<br>(N = XX)<br>n (%) | Transgender men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not complete the assessment? | | | |
| | | I did not receive a Sexual<br>Health Assessment from my<br>provider or clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made me feel uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Men who have sex<br>with men<br>(N = XX)<br>n (%) | Transgender men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | I was concerned about the privacy of my answers | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share sexual<br>health information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand why my<br>doctor or clinic was asking me<br>to complete the assessment | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.415. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 6/7), N=XX, Site Volume

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | High Volume<br>(N = XX)<br>n (%) | Low Volume<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 30 | Did you complete a Sexual | id you complete a Sexual Health Assessment from your provider or clinic/practice in the last 6 months? | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 31 | Did your provider or anoth | er person at the clinic/practice | , , | , , | ` ' |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't remember | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 32 | Who discussed the results | of the assessment with you? | | | |
| | | My healthcare<br>provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 33 | How helpful was discussing | the results with your provider | or another pe | rson at the clinic/prac | tice? |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 34 | Please rate your experience | e with the Sexual Health Assess | ment | | |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | High Volume<br>(N = XX)<br>n (%) | Low Volume<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | It was easy to take the<br>Sexual Health Assessment<br>on my digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor sent<br>the assessment before my<br>appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor was assessing my sexual health. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | High Volume<br>(N = XX)<br>n (%) | Low Volume<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not complete the assessment? | | | | |
| | | I did not receive a Sexual<br>Health Assessment from<br>my provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | High Volume<br>(N = XX)<br>n (%) | Low Volume<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | The assessment made me feel uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned about the privacy of my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share<br>sexual health information<br>with my doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand why<br>my doctor or clinic was<br>asking me to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 6.416. Distributional Characteristics of Estimated Amount of Money Spent on Transportation for Each Injection Visit (Month 6/7), N=XX

| 42. On average, how much did transportation cost round trip for each injection visit? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex<br>with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | | Dynan | nic Impleme | ntation | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 42. On average, how much did transportation cost round trip for each injection visit? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | | Routir | ne Implemer | ntation | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



## Table Shells for Month 12/13 Analysis

| Table 7.000. | Demographic Characteristics of Patient Study Participants Completing Surveys (Month 12/13), N=XX | 424 |
|---|---|---|
| Table 7.001. | Summary of Demographic Characteristics of Patient Study Participants (Month 12/13), N=XX | 426 |
| Table 7.002. | Summary of Behaviors of Patient Study Participants (Month 12/13), N=XX | 429 |
| Table 7.003. | Summary of Patient Study Participants' Sexual History and Behaviors (Month 12/13), N=XX, Study Arms | 431 |
| Table 7.004. | Summary of Patient Study Participants' Sexual History and Behaviors (Month 12/13), N=XX, Race, Dynamic Implementation | 434 |
| Table 7.005. | Summary of Patient Study Participants' Sexual History and Behaviors (Month 12/13), N=XX, Race, Routine Implementation | 437 |
| Table 7.006. | Summary of Patient Study Participants' Sexual History and Behaviors (Month 12/13), N=XX, Race, Total | 440 |
| Table 7.007. | Summary of Patient Study Participants' Sexual History and Behaviors (Month 12/13), | 443 |
| Table 7.008. | Summary of Patient Study Participants' Sexual History and Behaviors (Month 12/13), N=XX, Ethnicity, Total | 446 |
| Table 7.009. | Summary of Patient Study Participants' Sexual History and Behaviors (Month 12/13), | 449 |
| Table 7.010. | Summary of How Patient Study Participants Learned About PILLAR (Month 12/13), N=XX. | 452 |
| Table 7.101. | Summary of Patient Study Participants' HIV and PrEP Knowledge (Month 12/13), N=XX | 453 |
| Table 7.102. | Summary of Patient Study Participants' HIV and PrEP Knowledge (Month 12/13), N=XX, Scale Questions, Study Arms | 454 |
| Table 7.103. | Distributional Characteristics of Patient Study Participants' HIV and PrEP Knowledge (Month 12/13), N=XX, Scale Questions, Overall Score | 456 |
| Table 7.104. | Summary of Patient Study Participants' Perception of Stigma Associated with PrEP Usage (Month 12/13), N=XX, Stigma, Study Arms | 459 |
| Table 7.105. | Distributional Characteristics of Patient Study Participants' Perception of Stigma Associated with PrEP Usage (Month 12/13), N=XX, Stigma, Overall Score | 463 |
| Table 7.106. | Summary of Patient Study Participants' Choice of APRETUDE (Month 12/13), N=XX | 466 |
| Table 7.107. | Summary of Knowledge of APRETUDE and Utility of Implementation Strategies (Month 12/13), N=XX | 469 |
| Table 7.108. | Attitude Regarding APRETUDE and Utility of Implementation Strategies (Month 12/13), N=XX | 474 |
| Table 7.109. | Summary of Patient Study Participant Acquisition Process (Month 12/13), N=XX | 476 |
| Table 7.110. | Summary of Patient Study Participant Acquisition Process, Insurance (Month 12/13), N=XX | 477 |
| Table 7.201. | Distributional Characteristics of Acceptability of Intervention (AIM) (APRETUDE) (PSP) | 487 |



| Table 7.202. | Distributional Characteristics of Feasibility of Intervention (FIM) (APRETUDE) (PSP) (Month 12/13), N=XX | 490 |
|---|---|---|
| Table 7.203. | Distributional Characteristics of Accessibility of Intervention (AIM) (Telehealth) (PSP) (Month 12/13), N=XX | 493 |
| Table 7.204. | Distributional Characteristics of Feasibility of Intervention (FIM) (Telehealth) (PSP) (Month 12/13), N=XX | 496 |
| Table 7.205. | Summary of Acceptability of Intervention (AIM) (APRETUDE) (PSP) (Month 6/7), N=XX | 499 |
| Table 7.206. | Summary of Feasibility of Intervention (FIM) (APRETUDE) (PSP) (Month 6/7), N=XX | 501 |
| Table 7.207. | Summary of Acceptability of Intervention (AIM) (Telehealth) (PSP) (Month 6/7), N=XX | 503 |
| Table 7.208. | Summary of Feasibility of Intervention (FIM) (Telehealth) (PSP) (Month 6/7), N=XX | 505 |
| Table 7.209. | Changes from Baseline for Acceptability of Intervention Measure (AIM - APRETUDE) and Feasibility of Intervention Measure (FIM - APRETUDE) (Month 12/13), N=XX | 507 |
| Table 7.210. | Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – APRETUDE) (Month 12/13), N=XX | 508 |
| Table 7.211. | Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Acceptability of Intervention Measure (AIM – APRETUDE), N=XX | 509 |
| Table 7.212. | Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – APRETUDE) (Month 12/13), N=XX | 510 |
| Table 7.213. | Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Feasibility of Intervention Measure (FIM – APRETUDE), N=XX | 511 |
| Table 7.214. | Changes from Baseline for Acceptability of Intervention Measure (AIM - Telehealth) and Feasibility of Intervention Measure (FIM - Telehealth) (Month 12/13), N=XX | 512 |
| Table 7.215. | Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – Telehealth) (Month 12/13), N=XX | 513 |
| Table 7.216. | Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Acceptability of Intervention Measure (AIM – Telehealth), N=XX | 514 |
| Table 7.217. | Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – Telehealth) (Month 12/13), N=XX | 515 |
| Table 7.218. | Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Feasibility of Intervention Measure (FIM – Telehealth), N=XX | 516 |
| Table 7.219. | Summary of Pain/Activities After Injection (Month 12/13), N=XX | 517 |
| Table 7.220. | Summary of Patient Study Participants' Labs and Missed Doses (Month 12/13), N=XX | 520 |
| Table 7.301. | Summary of Feasibility and Acceptability of Telehealth (Month 12/13), N=XX | 522 |
| Table 7.302. | Summary of Quality of Care for Patient Study Participants (Month 12/13), N=XX | 530 |
| Table 7.303. | Summary of Quality of Care for Patient Study Participants (Month 12/13), N=XX, Non-Score Questions | 534 |
| Table 7.304. | Summary of Quality of Care for Patient Study Participants (Month 12/13), N=XX, Score Questions | 549 |
| Table 7.305. | Distributional Characteristics of Quality of Care for Patient Study Participants (Month 12/13), N=XX, Score Questions, Overall Score | 566 |
| Table 7.306. | Summary of Utility of Proposed Implementation Strategies (Month 12/13), N=XX | 569 |



| Table 7.307. | Summary of Patient Study Participants' Preferences/Acceptability of APRETUDE Information, Appointment Reminders, and Locations (Month 12/13), N=XX | 577 |
|---|---|---|
| Table 7.308. | Summary of Appointment Scheduling (Month 12/13), N=XX | . 581 |
| Table 7.401. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 12/13), N=XX, Study Arms | 583 |
| Table 7.402. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Race, Dynamic Implementation | 587 |
| Table 7.403. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Race, Routine Implementation | 591 |
| Table 7.404. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Race, Total | 595 |
| Table 7.405. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Ethnicity, Study Arms | 599 |
| Table 7.406. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Ethnicity, Total | 603 |
| Table 7.407. | Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Gender, Total | 607 |
| Table 7.408. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Study Arms | . 611 |
| Table 7.409. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Race, Dynamic Implementation | 615 |
| Table 7.410. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Race, Routine Implementation | |
| Table 7.411. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Race, Total | |
| Table 7.412. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Ethnicity, Study Arms | |
| Table 7.413. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Ethnicity, Total | |
| Table 7.414. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Gender | |
| Table 7.415. | Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Site Volume | |
| Table 7.416. | Proportion of PSP Taking the Sexual Health Assessment through Month 13 | |
| | Distributional Characteristics of Estimated Amount of Money Spent on Transportation for Each Injection Visit (Month 12/13), N=XX | |
| Table 7.501. | Test for Differences of Implementation Arm by Site Volume on Feasibility of Intervention Measure, APRETUDE (Month 12/13), N=XX | |
| Table 7.502 | Test for Differences of Implementation Arm by Site Volume on Feasibility of | 0-10 |
| | Intervention Measure, Telehealth (Month 12/13), N=XX | . 646 |



| Table 7.503. | Test for Differences of Implementation Arm by Site Volume on Acceptability of | |
|---|---|---|
| | Intervention Measure, APRETUDE (Month 12/13), N=XX | . 646 |
| Table 7.504. | Test for Differences of Implementation Arm by Site Volume on Acceptability of | |
| | Intervention Measure, Telehealth (Month 12/13), N=XX | . 646 |



Table 7.000. Demographic Characteristics of Patient Study Participants Completing Surveys (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N=XX)<br>n (%) | Dynamic<br>Implementation<br>(N=XX)<br>n (%) | Routine<br>Implementation<br>(N=XX)<br>n (%) |
|---|---|---|---|---|---|
| DM1 | Age (years) | N | XX | XX | XX |
| | | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| DM2 | Age (years), High Volume | N | XX | XX | XX |
| | | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| DM3 | Age (years), Low Volume | N | XX | XX | XX |
| | | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| DM4 | Age | | | | |
| | | 18-25 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 26-35 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 36-49 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 50+ | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| DM5 | Study Arm | | | | |
| | | Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| DM6 | Site Volume | | | | |
| | | High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| DM7 | Gender | | | | |
| | | Men who have sex with men | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Transgender men | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| DM8 | Race | | | | |
| | | Asian | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Black or African American | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | White | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Missing/Unknown | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | | Response | Total<br>(N=XX)<br>n (%) | Dynamic<br>Implementation<br>(N=XX)<br>n (%) | Routine<br>Implementation<br>(N=XX)<br>n (%) |
|---|---|---|---|---|---|
| DM9 | Ethnicity | | | | |
| | | Hispanic or Latino | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Hispanic or Latino | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Missing/Unknown | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 7.001. Summary of Demographic Characteristics of Patient Study Participants (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 1 | Which of the following best describes | s your <u>current</u> relationship : | status? | | |
| | | Single, never married | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Single, widowed | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Single, separated or divorced | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dating, but not living with a partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dating and living with a partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Domestic<br>partnership/civil union | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Married | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 2 | How would you describe your <u>curren</u> | t living situation? | | | |
| | | I live in my own house<br>or apartment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I live in my parent's<br>house or apartment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I live in a family<br>member's house or<br>apartment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I live in a friend's house or apartment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I sleep on various<br>friends' or relatives'<br>couches | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am homeless or am living in a shelter | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I live in<br>motel(s)/hotel(s) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 3 | What <u>best</u> describes your current em | ployment status? | | | |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Employed for wages<br>full-time (1 employer) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Employed for wages<br>full-time (2 or more<br>employers) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Employed for wages part-time (1 employer) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Employed for wages<br>part-time (2 or more<br>employers) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Self-employed | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A homemaker | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Student | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Retired | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not employed | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unable to work<br>(disabled) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 4 | What type of medical insurance do y | ou currently have? | | | |
| | | My parents' insurance | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | My partner's/spouse's insurance | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Private insurance<br>provided by my<br>workplace | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Private insurance I<br>purchased through an<br>exchange (e.g.,<br>Obamacare, Affordable<br>Care Act) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Federal insurance (e.g., VA, TRICARE) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Medicare or Medicaid | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Some other health care | XX | XX | XX |
| | | plan | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't have any health | XX | XX | XX |
| | | insurance currently | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |


Table 7.002. Summary of Behaviors of Patient Study Participants (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 87 | How often do you have a drink containing alcohol? | | | | |
| | | Never | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Monthly or less | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 2 to 4 times a month | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 2 to 3 times a week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 4 or more times a week | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 88 | On days when you drink alcoho<br>bottle/ can of beer, 1 glass of v | ol, how many drinks containing a<br>vine, 1 mixed drink, or 1 shot of | | u typically have? (1 o | drink=1 standard |
| | | 1 or 2 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 3 to 4 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 5 to 6 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 7 to 9 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 10 or more | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 89 | In the last 6 months, have you provider, such as speedball, he needle, either by mainlining, sk | roin, or crack? By shooting up, i | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 90 | In the last 6 months, have you substances), <u>that</u> were not pre cocaine? | | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |



Table 7.003. Summary of Patient Study Participants' Sexual History and Behaviors (Month 12/13), N=XX, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 8 | Have you h<br>oral sex. | and sex in the last 6 months? This could be vaginal sex | κ (penis in va | gina) OR anal sex (p | enis in butt) OR |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 9 | How would | you describe your sexual behaviors in the last 6 mor | nths? | | |
| | | I have had vaginal sex (penis in vagina) with only<br>1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex (penis in vagina) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a bottom (penis in butt as a bottom) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a bottom (penis in butt as a bottom) with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top (penis in butt as a<br>top) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top (penis in butt as a<br>top) with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth, tongue, or lips on a vagina, penis, or butt) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth, tongue, or lips on a vagina, penis, or butt) with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 10 | How often | did you use a condom when you had sex in the last 6 | months? | | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 11 | In the last ( | 6 months, how would you describe the HIV status of | your sexual p | partner(s)? | |
| | | I know that none of my sexual partners from the last 6 months have HIV/AIDS | | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one sexual partner from the last 6 months is living with HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 12 | | Du know, were any of your sexual partner(s) from the<br>PrEP is a medication that prevents HIV. | | , , | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 13 | | oned that you had a least one partner in the last 6 m<br>e any of your partners taking HIV medications (antire | | | |
| | | Yes, my partner(s) was/were taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s) was/were taking HIV medications and was/were undetectable, meaning HIV tests were not finding the virus | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, my partner(s) was/were not taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether my partner(s) was/were<br>taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 14 | | 6 months, have you experienced any incidents of sex<br>m a partner? | cual violence, | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | In the last ( | 6 months, have you exchanged things like money or | drugs for sex | with a sexual partne | er? |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Yes, I have a sexual partner things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave me things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.004. Summary of Patient Study Participants' Sexual History and Behaviors (Month 12/13), N=XX, Race, Dynamic Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 8 | Have you ha | nd sex in the last 6 months? <i>Thi</i> | is could be vagin | al sex (penis in vag | nina) OR anal sex | (penis in butt) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 9 | How would | you describe your sexual beha | viors in the last 6 | 5 months? | | |
| | | I have had vaginal sex<br>(penis in vagina) with only<br>1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex<br>(penis in vagina) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a top)<br>with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a top)<br>with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips on<br>a vagina, penis, or butt)<br>with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips on<br>a vagina, penis, or butt)<br>with more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 11 | In the last 6 | months, how would you descr | ribe the HIV state | us of your sexual p | artner(s)? | |
| | | I know that none of my<br>sexual partners from the<br>last 6 months have<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one<br>sexual partner from the<br>last 6 months is living with<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual<br>partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 12 | As far as you know, were any of your sexual partner(s) from the last 6 months taking PrEP to prevent HIV infection? PrEP is a medication that prevents HIV. | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 13 | | oned that you had a least one peany of your partners taking Hi | | | | |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications and<br>was/were undetectable, | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | meaning HIV tests were not finding the virus | | | | |
| | | No, my partner(s)<br>was/were not taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether my<br>partner(s) was/were<br>taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 14 | | 5 months, have you experience form a partner? | d any incidents o | f sexual violence, | physical abuse, o | any other type |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | In the last 6 | months, have you exchanged | things like mone | y or drugs for sex | with a sexual part | ner? |
| | | Yes, I have a sexual<br>partner things like drugs<br>or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave<br>me things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged<br>things like drugs or money<br>for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.005. Summary of Patient Study Participants' Sexual History and Behaviors (Month 12/13), N=XX, Race, Routine Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 8 | Have you ha | ad sex in the last 6 months? <i>T</i> | his could be vagin | al sex (penis in vag | gina) OR anal sex | (penis in butt) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 9 | How would | you describe your sexual beh | aviors in the last 6 | 5 months? | | |
| | | I have had vaginal sex<br>(penis in vagina) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex<br>(penis in vagina) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as<br>a bottom) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as<br>a bottom) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a<br>top) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a<br>top) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips<br>on a vagina, penis, or<br>butt) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips<br>on a vagina, penis, or<br>butt) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 10 | How often | did you use a condom when y | ou had sex in the | last 6 months? | | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 11 | In the last 6 | months, how would you des | cribe the HIV stat | us of your sexual p | artner(s)? | |
| | | I know that none of my<br>sexual partners from the<br>last 6 months have<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one<br>sexual partner from the<br>last 6 months is living<br>with HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual<br>partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 12 | | u know, were any of your sex<br>PrEP is a medication that preve | | m the last 6 month | s taking PrEP to p | revent HIV |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 13 | | ned that you had a least one any of your partners taking H | | | | |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications and | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | was/were undetectable,<br>meaning HIV tests were<br>not finding the virus | | | | |
| | | No, my partner(s)<br>was/were not taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether<br>my partner(s) was/were<br>taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 14 | | 5 months, have you experience form a partner? | ed any incidents c | of sexual violence, | physical abuse, or | any other type |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | In the last 6 months, have you exchanged things like money or drugs for sex with a sexual partner? | | | | | |
| | | Yes, I have a sexual partner things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner<br>gave me things like drugs<br>or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.006. Summary of Patient Study Participants' Sexual History and Behaviors (Month 12/13), N=XX, Race, Total

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 8 | Have you ha<br>OR oral sex. | ad sex in the last 6 months? <i>Ti</i> | his could be vagin | al sex (penis in vag | gina) OR anal sex | (penis in butt) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 9 | How would | you describe your sexual beh | aviors in the last 6 | months? | | |
| | | I have had vaginal sex<br>(penis in vagina) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex<br>(penis in vagina) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as<br>a bottom) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as<br>a bottom) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a<br>top) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>top (penis in butt as a<br>top) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips<br>on a vagina, penis, or<br>butt) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex<br>(mouth, tongue, or lips<br>on a vagina, penis, or<br>butt) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | | Black or | | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
| 10 | How often | did you use a condom when y | ou had sex in the | last 6 months? | | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 11 | In the last 6 months, how would you describe the HIV status of your sexual partner(s)? | | | | | |
| | | I know that none of my<br>sexual partners from the<br>last 6 months have<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one<br>sexual partner from the<br>last 6 months is living<br>with HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual<br>partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 12 | As far as you know, were any of your sexual partner(s) from the last 6 months taking PrEP to prevent HIV infection? PrEP is a medication that prevents HIV. | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 13 | | oned that you had a least one pe<br>any of your partners taking H | | | | |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s)<br>was/were taking HIV<br>medications and | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | was/were undetectable,<br>meaning HIV tests were<br>not finding the virus | | | | |
| | | No, my partner(s)<br>was/were not taking HIV<br>medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether<br>my partner(s) was/were<br>taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 14 | | 5 months, have you experience form a partner? | ed any incidents c | of sexual violence, | physical abuse, or | any other type |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | In the last 6 months, have you exchanged things like money or drugs for sex with a sexual partner? | | | | | |
| | | Yes, I have a sexual partner things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner<br>gave me things like drugs<br>or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged things like drugs or money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.007. Summary of Patient Study Participants' Sexual History and Behaviors (Month 12/13), N=XX, Ethnicity, Study Arms

| | | | Dynamic Implementation | | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) |
| 8 | Have you had sex in the last 6 months? This could be vaginal sex (penis in vagina) OR anal sex (penis in butt) OR oral sex. | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 9 | How would | you describe your sexual behavio | ors in the last 6 m | onths? | | |
| | | I have had vaginal sex (penis<br>in vagina) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex (penis<br>in vagina) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic Implementation | | Routine Imp | lementation |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanio<br>or Latino<br>(N = XX)<br>n (%) |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Most of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | None of the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 11 | In the last 6 | months, how would you describ | e the HIV status o | of your sexual partr | ner(s)? | |
| | | I know that none of my<br>sexual partners from the last<br>6 months have HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I know that at least one<br>sexual partner from the last<br>6 months is living with<br>HIV/AIDS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know my sexual<br>partners' HIV status | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 12 | As far as you know, were any of your sexual partner(s) from the last 6 months taking PrEP to prevent HIV infection? PrEP is a medication that prevents HIV. | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 13 | | oned that you had a least one part<br>e any of your partners taking HIV I | | | | |
| | | Yes, my partner(s) was/were taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, my partner(s) was/were taking HIV medications and was/were undetectable, meaning HIV tests were not finding the virus | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic Imp | Dynamic Implementation | | Routine Implementation |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) |
| | | No, my partner(s) was/were not taking HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not know whether my<br>partner(s) was/were taking<br>HIV medications | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 14 | In the last 6 months, have you experienced any incidents of sexual violence, physical abuse, or any other type trauma form a partner? | | | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | In the last 6 months, have you exchanged things like money or drugs for sex with a sexual partner? | | | | | |
| | | Yes, I have a sexual partner<br>things like drugs or money<br>for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave<br>me things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged<br>things like drugs or money<br>for sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.008. Summary of Patient Study Participants' Sexual History and Behaviors (Month 12/13), N=XX, Ethnicity, Total

| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 8 | Have you h | ad sex in the last 6 months? <i>This co</i> | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 9 | How would you describe your sexual behaviors in the last 6 months? | | | |
| | | I have had vaginal sex (penis<br>in vagina) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex (penis<br>in vagina) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 10 | How often | did you use a condom when you ha | d sex in the last 6 months? | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) |



| 11 | In the last 6 | Most of the time Some of the time A little of the time None of the time I prefer not to answer months, how would you describe to the time of my sexual partners from the last 6 months have HIV/AIDS | XX | n (%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) |
|---|---|---|---|---|
| 11 | In the last 6 | Some of the time A little of the time None of the time I prefer not to answer months, how would you describe to the time the second | (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) AXX (XX.X%) he HIV status of your sexual par | (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) |
| 11 | In the last 6 | A little of the time None of the time I prefer not to answer months, how would you describe to the last of the time. | XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) AX (XX.X%) AX (XX.X%) AX XX XX XX XX XX XX | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%) |
| 11 | In the last 6 | A little of the time None of the time I prefer not to answer months, how would you describe to the last of the time. | XX (XX.X%) XX (XX.X%) XX (XX.X%) he HIV status of your sexual par | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>XX<br>(XX.X%) |
| 11 | In the last 6 | None of the time I prefer not to answer months, how would you describe t I know that none of my sexual partners from the last | (XX.X%) XX (XX.X%) XX (XX.X%) he HIV status of your sexual par | (XX.X%) XX (XX.X%) XX (XX.X%) tner(s)? |
| 11 | In the last 6 | None of the time I prefer not to answer months, how would you describe t I know that none of my sexual partners from the last | XX<br>(XX.X%)<br>XX<br>(XX.X%)<br>he HIV status of your sexual par | XX<br>(XX.X%)<br>XX<br>(XX.X%) |
| 11 | In the last 6 | I prefer not to answer months, how would you describe t I know that none of my sexual partners from the last | (XX.X%) XX (XX.X%) he HIV status of your sexual par XX | (XX.X%) XX (XX.X%) ther(s)? |
| 11 | In the last 6 | months, how would you describe t I know that none of my sexual partners from the last | XX<br>(XX.X%)<br>he HIV status of your sexual par<br>XX | XX<br>(XX.X%)<br>tner(s)? |
| 11 | In the last 6 | months, how would you describe t I know that none of my sexual partners from the last | (XX.X%)<br>he HIV status of your sexual par<br>XX | (XX.X%) |
| 11 | In the last 6 | I know that none of my<br>sexual partners from the last | he HIV status of your sexual par | tner(s)? |
| | | I know that none of my<br>sexual partners from the last | XX | |
| | | sexual partners from the last | | XX |
| | | 6 months have HIV/AIDS | /VV V0/\ | /VV V0/\ |
| | | | (XX.X%) | (XX.X%) |
| | | I know that at least one | | |
| | | sexual partner from the last | XX | XX |
| | | 6 months is living with<br>HIV/AIDS | (XX.X%) | (XX.X%) |
| | | I do not know my sexual | XX | XX |
| | | partners' HIV status | (XX.X%) | (XX.X%) |
| | | I profer not to answer | XX | XX |
| | | I prefer not to answer | (XX.X%) | (XX.X%) |
| | | u know, were any of your sexual pa<br>rEP is a medication that prevents H | | taking PrEP to prevent HIV |
| | | No | XX | XX |
| | | INO | (XX.X%) | (XX.X%) |
| | | Yes | XX | XX |
| | | | (XX.X%) | (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | · · · · · · | · · · |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 1 4 | You mentioned that you had a least one partner in the last 6 months who is living with HIV/AIDS. As far as you know, were any of your partners taking HIV medications (antiretrovirals) to treat their HIV infection? | | | |
| | | Yes, my partner(s) was/were | XX | XX |
| | | taking HIV medications | (XX.X%) | (XX.X%) |
| | | Yes, my partner(s) was/were | | |
| | | taking HIV medications and | XX | XX |
| | | was/were undetectable,<br>meaning HIV tests were not | (XX.X%) | (XX.X%) |
| | | finding the virus | | |
| | | No, my partner(s) was/were | XX | XX |
| | | not taking HIV medications | (XX.X%) | (XX.X%) |
| | | I do not know whether my | XX | XX |
| | | partner(s) was/were taking<br>HIV medications | (XX.X%) | (XX.X%) |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 14 | In the last 6 months, have you experienced any incidents of sexual violence, physical abuse, or any other type of trauma form a partner? | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | In the last 6 | months, have you exchanged thing | gs like money or drugs for sex wi | th a sexual partner? |
| | | Yes, I have a sexual partner<br>things like drugs or money<br>for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave<br>me things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged<br>things like drugs or money<br>for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.009. Summary of Patient Study Participants' Sexual History and Behaviors (Month 12/13), N=XX, Gender, Total

| Question<br>Number | Question | Response | Men who have sex with men<br>(N = XX)<br>n (%) | Transgender Men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 8 | Have you h | ad sex in the last 6 months? <i>This</i> | could be vaginal sex (penis in vagina) ( | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 9 | How would you describe your sexual behaviors in the last 6 months? | | | |
| | | I have had vaginal sex (penis<br>in vagina) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had vaginal sex (penis<br>in vagina) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a<br>bottom (penis in butt as a<br>bottom) with more than 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>only 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had anal sex as a top<br>(penis in butt as a top) with<br>more than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with only 1<br>partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have had oral sex (mouth,<br>tongue, or lips on a vagina,<br>penis, or butt) with more<br>than 1 partner | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 10 | How often | did you use a condom when you l | had sex in the last 6 months? | |
| | | All of the time | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Men who have sex with men (N = XX) | Transgender Men<br>(N = XX) |
|---|---|---|---|---|
| Number | | | n (%) | n (%) |
| | | | XX | XX |
| | | Most of the time | (XX.X%) | (XX.X%) |
| | | - 6.1 | XX | XX |
| | | Some of the time | (XX.X%) | (XX.X%) |
| | | | XX | XX |
| | | A little of the time | (XX.X%) | (XX.X%) |
| | | | XX | XX |
| | | None of the time | (XX.X%) | (XX.X%) |
| | | | XX | XX |
| | | I prefer not to answer | (XX.X%) | (XX.X%) |
| 11 | In the last 6 | months how would you describe | e the HIV status of your sexual partne | r(s)? |
| .1 | III the last c | | the fire status of your sexual partite | 1(5). |
| | | I know that none of my sexual partners from the last | XX | XX |
| | | 6 months have HIV/AIDS | (XX.X%) | (XX.X%) |
| | | I know that at least one | | |
| | | sexual partner from the last | XX | XX |
| | | 6 months is living with | (XX.X%) | (XX.X%) |
| | | HIV/AIDS | (************************************** | ( ) |
| | | I do not know my sexual | XX | XX |
| | | partners' HIV status | (XX.X%) | (XX.X%) |
| | | | XX | XX |
| | | I prefer not to answer | (XX.X%) | (XX.X%) |
| 12 | | u know, were any of your sexual per<br>PrEP is a medication that prevents | partner(s) from the last 6 months taki | ng PrEP to prevent HIV |
| | comer. | | XX | XX |
| | | No | (XX.X%) | (XX.X%) |
| | | | XX | XX |
| | | Yes | (XX.X%) | (XX.X%) |
| | | | | · |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX X8/) | XX<br>(VV V0/) |
| | | | (XX.X%) | (XX.X%) |
| 13 | You mentioned that you had a least one partner in the last 6 months who is living with HIV/AIDS. As far as yo know, were any of your partners taking HIV medications (antiretrovirals) to treat their HIV infection? | | | |
| | | Yes, my partner(s) was/were | XX | XX |
| | | taking HIV medications | (XX.X%) | (XX.X%) |
| | | Yes, my partner(s) was/were | | |
| | | taking HIV medications and | XX | XX |
| | | was/were undetectable, | (XX.X%) | (XX.X%) |
| | | meaning HIV tests were not finding the virus | | , , |
| | | | \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | 107 |
| | | No, my partner(s) was/were | XX<br>(VV V0/) | XX<br>(VX V0/) |
| | | not taking HIV medications | (XX.X%) | (XX.X%) |
| | | I do not know whather my | | |
| | | I do not know whether my partner(s) was/were taking | XX | XX |



| Question<br>Number | Question | Response | Men who have sex with men<br>(N = XX)<br>n (%) | Transgender Men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 14 | In the last 6 months, have you experienced any incidents of sexual violence, physical abuse, or any other type o trauma form a partner? | | | |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 15 | In the last 6 | months, have you exchanged th | ings like money or drugs for sex with a | a sexual partner? |
| | | Yes, I have a sexual partner<br>things like drugs or money<br>for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Yes, a sexual partner gave<br>me things like drugs or<br>money for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No, I have not exchanged<br>things like drugs or money<br>for sex | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.010. Summary of How Patient Study Participants Learned About PILLAR (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 91 | How did you learn about the PILL | .AR study? | | | |
| | | A discussion with my healthcare provider | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A flyer or poster in my clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A friend/family told<br>me | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Social media | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | An event in my community | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.101. Summary of Patient Study Participants' HIV and PrEP Knowledge (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 5 | Do you personally know of | someone living with HIV? | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.102. Summary of Patient Study Participants' HIV and PrEP Knowledge (Month 12/13), N=XX, Scale Questions, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 6 | Please answer true or false to the following st | tatements abo | out HIV. | | |
| А | A person who has HIV can look healthy. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | There is a vaccine that can stop you from getting HIV. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | A person will NOT get HIV if they are taking antibiotics. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | If you only have sex once with a partner, you cannot get HIV from them. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | People living with HIV on HIV medications cannot spread HIV. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Everybody who has HIV knows that they have HIV. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | A natural (lamb skin) condom works better against HIV than a latex condom. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | When using condoms during sex, it is safer to use water-based lubricants than oil-based lubricants. | True | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | False | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't<br>know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.103. Distributional Characteristics of Patient Study Participants' HIV and PrEP Knowledge (Month 12/13), N=XX, Scale Questions, Overall Score

| | • | | | | • | | | |
|---|---|---|---|---|---|---|---|---|
| 6. Please answer true or false to the following statements about HIV. | n | Mean | SD | Median<br>(Q1, Q3) | Observe<br>d Range<br>(Minimu<br>m,<br>Maximu<br>m) | Missing<br>n (%) | 95% Cl<br>for the<br>Mean | Cronbach's<br>α |
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | 0.xx |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Gender | | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Ethnicity | | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Not Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| | | | Dynamic Ir | nplementation | | | | |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Gender | | | | | | | | |



| 6. Please answer true or false to the following statements about HIV. | n | Mean | SD | Median<br>(Q1, Q3) | Observe<br>d Range<br>(Minimu<br>m,<br>Maximu<br>m) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Ethnicity | | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Not Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| | | | Routine In | nplementation | | | | |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Gender | | | | | | | | |
| Men who have<br>sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |



| 6. Please answer true or false to the following statements about HIV. | n | Mean | SD | Median<br>(Q1, Q3) | Observe<br>d Range<br>(Minimu<br>m,<br>Maximu<br>m) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Not Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X (X.X,<br>X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |

Mean score = mean of correct responses to all of the items under 8 save for A and E; 'Don't know' responses coded as incorrect. Correct answers were 'False' for items B, C, D, F, and G and 'True' for item H.



Table 7.104. Summary of Patient Study Participants' Perception of Stigma Associated with PrEP Usage (Month 12/13), N=XX, Stigma, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 7 | To what extent do you agree with eac | h of the following s | statements about | PrEP? | |
| А | My <i>friends</i> would be supportive of me taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | People experience problems when they tell their sexual partner(s) they are taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | People experience negative judgement because they take PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | My <i>family</i> would be supportive of me taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Completely<br>agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | People taking PrEP receive praise for being responsible. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | I would feel ashamed to take PrEP in front of others. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | Someone taking PrEP would be seen by others as having sex with a lot of different people. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | People on PrEP are taking care of their health. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| I | People talking PrEP experience verbal harassment. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| J | I would not want others to know if I was taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| K | Someone taking PrEP should keep their pills hidden. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| L | I would feel proud to take PrEP every day. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| M | I would have sex with someone who is taking PrEP. | Completely<br>Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.105. Distributional Characteristics of Patient Study Participants' Perception of Stigma Associated with PrEP Usage (Month 12/13), N=XX, Stigma, Overall Score

| Mean Score XX | | | | <u> </u> | ' '' | , 0 | , | | |
|---|---|---|---|---|---|---|---|---|---|
| Study Arm | you agree with each of the following statements about | n | Mean | SD | | Range<br>(Minimum, | | for the | Cronbach's<br>α |
| Dynamic Implementation | Mean Score | XX | X.XX | X.XXX | | | | | 0.xx |
| Manufaction | Study Arm | | | | | | | | |
| Implementation | • | XX | X.XX | X.XXX | | | | | - |
| High | | XX | X.XX | X.XXX | | | | , | - |
| High | Site Volume | | | | | | | | |
| Company | High | XX | X.XX | X.XXX | | | | , , | _ |
| Men who have sex with men XX X.XX X.XXX X.XX X.XX X.XX XX X.XXX X.XXX X.XXX X.XXX X.XXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX X.XXXX <td>Low</td> <td>XX</td> <td>X.XX</td> <td>X.XXX</td> <td></td> <td></td> <td></td> <td>,</td> <td>_</td> | Low | XX | X.XX | X.XXX | | | | , | _ |
| sex with men XX XXXX XXXXX (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Gender | | | | | | | | |
| Men XX X.XX X.XXX (X.X, X.XX) (X.X, X.X) (XX, X.XX) X.XXXX Race XX X.XX X.XXX X.XX X.XX XX XX X.XXXX X.XXXXX X.XXXXXX X.XXXXX X.XXXXX X.XXXXX X.XXXXX X.XXXXXXXX X.XXXXXX X.XXXXX X.XXXXX X.XXXXX X.XXXXXX X.XXXXX X.XXXXXX X.XXXXX X.XXXXX X.XXXXX X.XXXXXXX X.XXXXXXX X.XXXXXX X.XXXXXX | | XX | X.XX | X.XXX | | | | | _ |
| Asian XX XXXX XXXXX XXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | · · | XX | X.XX | X.XXX | | | | , , | _ |
| Asian | Race | | | | | | | | |
| American XX X.XXX X.XXX (X.XX, X.XX) (X.X, X.X) (X.XXX) X.XXXX White XX X.XX X.XXX X.XX X.XX X.XX (X.XXX, X.XX) (X.XXX, X.XX) (X.XXX, X.XX) X.XXX X.XXXX X.XXX X.XXXX (X.XXX, X.XX) (X.XXX, X.XX) X.XXXX (X.XXX, X.XX) X.XXXX (X.XXX, X.XX) (X.XXX, X.XXX) (X.XXX, X | Asian | XX | X.XX | X.XXX | | | | | _ |
| White XX X.XXX X.XXX (X.X, X.XX) (X.X, X.X) (X.X, X.X) X.XXXX Other XX X.XX X.XXX X.XX X.X X.X (X.XXX, X.XX) X.X XX X.XXXX X.XXXX X.XXX X.XXXX X.XXXXX X.XXXXXXX X.XXXXXX X.XXXXX X.XXXXX X.XXXXX X.XXXXXXXX X.XXXXXXXX X.XXXXXXXXXX X.XXXXXXXXXXX X.XXXXXXXXXXX X.XXXXXXXXXX X.XXXXXXXXXXXXXXXXX X.XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | XX | X.XX | X.XXX | | | | | _ |
| Other XX X.XX X.XXX (X.XX, X.XX) (X.X, X.X) (XX.XX) X.XXXX Hispanic or Latino XX X.XX X.XXX X.XXX X.XX X.XXX (X.XXX, X.XX) (X.XXX, X.XX) (X.XXX, X.XX) (X.XXX, X.XXX) (X.XXX, X.XXXX) (X.XXX, X.XXX) (X.XXX, X.XXXX) (X.XXX, X.XXXX) (X.XXX, X.XXXX) (X.XXX, X.XXXXX) (X.XXX, X.XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | White | XX | X.XX | X.XXX | | | | , , | _ |
| Hispanic or | Other | XX | X.XX | X.XXX | | | | , , | _ |
| Latino XX X.XX X.XXX (X.XX, X.XX) (X.X, X.X) (XX.XX) X.XXXX Not Hispanic or Latino XX X.XX X.XXX X.XX X.XX XX (X.XXX, X.XX) (X.XXX, X.XX) (XX.XXX) X.XXXX X.XXXX (X.XXX, X.XX) (X.XXX, X.XX) XXXXX (X.XXX, X.XX) XXXXX (X.XXX, X.XX) (X.XXX, X.XX) (X.XXX, X.XX) (X.XXX, X.XX) (X.XXX, X.XX) (X.XXX, X.XXX) (X.XXX, X.XXXX) (X.XXX, X.XXXX) (X.XXX, X.XXXX) (X.XXX, X.XXXX) (X.XXX, X.XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Ethnicity | | | | | | | | |
| Or Latino XX X.XXX X.XXX (X.XX, X.XX) (X.X, X.X) (XX.XX) X.XXXX Dynamic Implementation Site Volume XX X.XXX X.XXX X.XX X.XX XXX XXXX XXXXX XXXXX XXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | • | XX | X.XX | X.XXX | | | | | - |
| Site Volume XX X.XXX X.XXXX X.XXXX X.XXXX X.XXXXX X.XXXXX X.XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | XX | X.XX | X.XXX | | | | , , | - |
| High XX X.XX X.XXX X.XX X.XX X.XX X.XX X.XXX X.XXX X.XXXX X.XXXX X.XXXX X.XXXXX X.XXXXX X.XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | Dyna | mic Implement | ation | | | |
| High XX X.XX X.XXX (X.XX, X.XX) (X.X, X.X) (XX.XX) X.XXXX Low XX X.XX X.XXX X.XX XX XX (X.XXX, XXX) | Site Volume | | | | | | | | |
| Low XX X.XX X.XXX (X.XX, X.XX) (X.X, X.X) (XX.XX) X.XXX) | High | XX | X.XX | X.XXX | | | | | _ |
| Gender | Low | XX | X.XX | X.XXX | | | | | _ |
| | Gender | | | | | | | | |



| 7. To what extent do you agree with each of the following statements about PrEP? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Men who<br>have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Transgender<br>Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Black or<br>African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Not Hispanic<br>or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| | | | Rout | tine Implementa | ation | | | |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Gender | | | | | | | | |
| Men who<br>have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Transgender<br>Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Black or<br>African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |


| 7. To what extent do you agree with each of the following statements about PrEP? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Not Hispanic<br>or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |

Mean score = mean of responses to all of the items under 13 save for J with the following items are reverse scored: A, D, E, H, L,& M. Higher total score indicates higher stigma.



Table 7.106. Summary of Patient Study Participants' Choice of APRETUDE (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 16 | Do you have any concer | ns about APRETUDE? | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 17 | What concerns do you h | ave about APRETUDE? | | | |
| | | Pain or soreness from the injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other side effects from APRETUDE | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Fear of needles | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Change in my insurance coverage for APRETUDE | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Possible long-term effects of the injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | How it affects other medications I take | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Scheduling or rescheduling injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Forgetting my appointment for the injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Missing an injection visit and then getting HIV | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Missing work for the injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Making time to go to the clinic/practice for the injection every 2 months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Travelling to the clinic/practice for the injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Limited clinic/practice hours for injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Childcare/caregiver responsibilities during injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Lack of privacy at injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | My dignity not being respected during injection visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | People asking why I go to<br>the clinic/doctor every 2<br>months | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | My hectic lifestyle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | My travel or holiday schedules | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Taking medication during times when I am not having sex | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The medication not being effective at preventing HIV | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Worrying people would think<br>I have HIV | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Worrying that people would<br>think I have a lot of sexual<br>partners because I am on<br>CAB LA for PrEP | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Worrying about my privacy because I live with someone | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Worrying about my privacy<br>because I'm on my parent's<br>health insurance | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 18 | How often are you worried that people may find out that you are taking APRETUDE? | | | | |
| | | Never | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Rarely | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Sometimes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Often | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | All the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 19 | How often are you worried ak | out forgetting your APRETUDE in | jection visits | ) | |
| | | Never | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Rarely | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Sometimes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Often | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | All the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.107. Summary of Knowledge of APRETUDE and Utility of Implementation Strategies (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 75 | Overall, how much do you kno | ow about APRETUDE? | | | |
| | | A lot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Nothing | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 76 | How confident are you with yo | our current level of knowledge a | bout APRETU[ | DE? | |
| | | Extremely confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all confident | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 77 | How helpful is the information | n, if any, shared by the medical s | taff about APF | RETUDE? | |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not receive any<br>information from medical<br>staff | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 78 | How helpful has each of the fo | bllowing materials been in learni | ng about APRI | TUDE? | |
| А | Getting Started Brochure –<br>the brochure that gives you<br>an overview of how to get<br>started with APRETUDE | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Did not receive/Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Patient Brochure – this brochure helps you understand the process of receiving APRETUDE injections, including side effects and insurance information | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Did not receive/Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | Let's talk about HIV & PrEP<br>video – the video giving key<br>facts about HIV and PrEP<br>options (DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not receive/Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| D | The APRETUDE Myths and Facts video – the game | Very helpful | XX | XX | N/A |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | show video addressing<br>common myths about<br>APRETUDE (DI) | | (XX.X%) | (XX.X%) | |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not receive/Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| E | The What to Expect video which shows you what to expect during the APRETUDE process (DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not receive/Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| F | The ViiV Connect Video,<br>which tells you about the<br>ViiV Connect program and<br>frequently asked questions<br>(DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not receive/Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| G | The study website where you access APRETDUE information (RI) | Very helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Did not receive/Did not use it | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| Н | The study app/website<br>where you access<br>APRETUDE information —<br>the Pillar Spot (DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not receive/Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| I | Important safety<br>information – This<br>document details important<br>safety information<br>relating to APRETUDE | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Did not receive/Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| J | Important facts — This<br>document details important<br>facts relating to APRETUDE | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Did not receive/Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| K | A flyer on PrEP options (DI) | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Did not receive/Did not use it | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |



Table 7.108. Attitude Regarding APRETUDE and Utility of Implementation Strategies (Month 12/13), N=XX

| Question | | | | | | |
|---|---|---|---|---|---|---|
| 86. Overall, ho<br>taking APRETI | ow are you feeling about<br>JDE? | Very positive | Somewhat positive | Neither<br>positive nor<br>negative | Somewhat<br>negative | Very<br>negative |
| Study Arms | | | | | | |
| | Total<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Routine<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynami | c Implementation | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routine | Implementation | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | | Response | | |
|---|---|---|---|---|---|
| Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Dynamic Implementation | | | | | |
| Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Routine Implementation | | | | | |
| Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Total | ' | | | | |
| Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Total | ' | | | | |
| Men who have sex<br>with men<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Transgender men<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.109. Summary of Patient Study Participant Acquisition Process (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 79 | Have you ever heard of ViiV C | onnect? | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 80 | Where did you learn about Vii | V Connect? | | | |
| | | My healthcare provider/healthcare clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The ViiV Connect video on the study app/website (DI) | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | ViiV Connect brochure | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A friend/family member told me | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The ViiV Connect website | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.110. Summary of Patient Study Participant Acquisition Process, Insurance (Month 12/13), N=XX

| Question | | | | Response | | |
|---|---|---|---|---|---|---|
| | extent do you agree with ollowing statements? | Completely Agree | Agree | Neither<br>agree nor<br>disagree | Disagree | Completely disagree |
| A. The staf | f at the clinic helped me und | derstand the insurance a | pproval proces | S | | |
| Study Arms | | | | | | |
| | Total<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Routine<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynam | ic Implementation | | | | | _ |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routine | e Implementation | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | Response | | | | |
|---|---|---|---|---|---|---|
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Dynam | ic Implementation | | | | | |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Routine | Implementation | | | | | |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Total | | | | | | |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Total | | | | | | |
| | Men who have sex<br>with men<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Transgender men<br>(N = XX) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | | | Response | | |
|---|---|---|---|---|---|---|
| | Total<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Routine<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynami | ic Implementation | | -1 | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routine | e Implementation | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Total | | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | Response | | | | |
|---|---|---|---|---|---|---|
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Dyna | amic Implementation | | | | | |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Rout | tine Implementation | | | | | |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Tota | ıl | | | | | |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Total | | | | | | |
| | Men who have sex<br>with men<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Transgender men<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| C. My copay | for APRETUDE is acceptable | | | | | |
| Study Arms | | | | | | |
| | Total<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | Response | | | | |
|---|---|---|---|---|---|---|
| | Routine<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynamic | Implementation | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routine I | mplementation | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Total | | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | Response | | | | | |
|---|---|---|---|---|---|---|
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Rou | tine Implementation | | • | | | • |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Tota | al | | | | | |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Total | | | | | | |
| | Men who have sex<br>with men<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Transgender men<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D. I am wor | ried about insurance coverag | e long-term | | | | |
| Study Arms | | | | | | _ |
| | Total<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Routine<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynami | c Implementation | | | | | 1 |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | | | Response | | |
|---|---|---|---|---|---|---|
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routine | e Implementation | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Total | | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Dyr | namic Implementation | | | | | |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | Response | | | | | |
|---|---|---|---|---|---|---|
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Total | | | | | | |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Total | | | | | | |
| | Men who have sex<br>with men<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Transgender men<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E. The insura | ance approval process was s | mple | | | | |
| Study Arms | | | | | | |
| | Total<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Routine<br>Implementation<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Dynamic | Implementation | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | Response | | | | |
|---|---|---|---|---|---|---|
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Routine | Implementation | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Race, Total | | | | | | |
| | Asian<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Black or African<br>American<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | White<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Other<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Dyn | amic Implementation | | | | | |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Ethnicity, Rou | tine Implementation | | ı | 1 | | |
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question | | | | Response | | |
|---|---|---|---|---|---|---|
| | Hispanic or Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Gender, Total | | | | | | |
| | Men who have sex<br>with men<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Transgender men<br>(N = XX)<br>n (%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.201. Distributional Characteristics of Acceptability of Intervention (AIM) (APRETUDE) (PSP) (Month 12/13), N=XX

| 20. AIM APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| T-test | X.XXX | | | | | | |
| Degrees of Freedom | | XX | | | | | |
| P-value | | 0.XXX | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Dynamic Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 20. All | M APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|---|
| Gende | er | | | | | Waximami | | |
| men | Men who have sex with | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | | |
| | Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnic | ity | | | | | | | |
| | Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routir | ne Implementation | | | | | | | |
| Site V | olume | | | | | | | |
| | High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gende | er | | | | | | | |
| men | Men who have sex with | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | | |
| | Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnic | ity | | | | | | | |
| | Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 20. AIM APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



Table 7.202. Distributional Characteristics of Feasibility of Intervention (FIM) (APRETUDE) (PSP) (Month 12/13), N=XX

| 21. FIM APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| T-test | | | | X.XXX | | | |
| Degrees of Freedom | | | | XX | | | |
| P-value | | | | 0.XXX | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Dynamic Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 21. FIN | M APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|---|
| Gende | er | | | | | | | |
| men | Men who have sex with | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | | |
| | Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnic | ity | | | | | | | |
| | Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routin | ne Implementation | | | | | | | |
| Site Vo | olume | | | | | | | |
| | High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gende | er | | | | | | | |
| men | Men who have sex with | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | | |
| | Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnic | ity | | | | | | | |
| | Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 21. FIM APRETUDE. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



Table 7.203. Distributional Characteristics of Accessibility of Intervention (AIM) (Telehealth) (PSP) (Month 12/13), N=XX

| (1 51 ) (141611611 12) | ** | | | | | | |
|---|---|---|---|---|---|---|---|
| 23. AIM TELEHEALTH. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| T-test | | | | X.XXX | | | |
| Degrees of Freedom | | | | XX | | | |
| P-value | | | | 0.XXX | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Dynamic Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 23. AIM | TELEHEALTH. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|---|
| Gender | | | | | | | | |
| Men N | Men who have sex with | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| T | ransgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | | |
| F | Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| E | Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| ١ | White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| ( | Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | / | | | | | | | |
| ŀ | Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| ١ | Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine | Implementation | | | | | | | |
| Site Volu | ıme | | | | | | | |
| ŀ | High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| L | ow | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | | |
| Men | Men who have sex with | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Т | ransgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | | |
| A | Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| E | Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| ١ | White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| ( | Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | , | | | | | | | |
| | Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 23. AIM TELEHEALTH. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



Table 7.204. Distributional Characteristics of Feasibility of Intervention (FIM) (Telehealth) (PSP) (Month 12/13), N=XX

| (141011111 12/ 13/), 14 | | | | | | | |
|---|---|---|---|---|---|---|---|
| 24. FIM TELEHEALTH. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| T-test | | | | X.XXX | | | |
| Degrees of Freedom | | | | XX | | | |
| P-value | | | | 0.XXX | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Dynamic Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 24. FIN | VI TELEHEALTH. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|---|
| Gende | er | | | | | | | |
| men | Men who have sex with | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | | |
| | Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnic | ity | | | | | | | |
| | Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routir | ne Implementation | | | | | | | |
| Site Vo | olume | | | | | | | |
| | High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gende | er | | | | | | | |
| men | Men who have sex with | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Transgender Men | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | | |
| | Asian | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Black or African American | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | White | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| | Other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnic | ity | | | | | | | |
| | Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



| 24. FIM TELEHEALTH. | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



Table 7.205. Summary of Acceptability of Intervention (AIM) (APRETUDE) (PSP) (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 20 | Please indicate how much you | ı agree with each st | atement based | on your current expecta | ations of APRETUDE. |
| | APRETUDE <b>meets my approval</b> for preventing HIV. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | APRETUDE for the prevention of HIV is appealing to me. | Completely<br>agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I <b>like</b> APRETUDE for the prevention of HIV. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I welcome APRETUDE for the prevention of HIV | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree<br>nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |


Table 7.206. Summary of Feasibility of Intervention (FIM) (APRETUDE) (PSP) (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 21 | Please indicate how much y | ou agree with each sta | atement based | on your experiences wi | th APRETUDE. |
| | Receiving APRETUDE injection every 2-months seems workable in my life | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Receiving APRETUDE injection every 2-months seems possible in my life | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Receiving APRETUDE injection every 2-months seems doable in my life | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Receiving APRETUDE injection every 2-months seems easy in my life | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.207. Summary of Acceptability of Intervention (AIM) (Telehealth) (PSP) (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 23 | Please indicate how much y with telehealth. | ou agree with each sta | u agree with each statement based on your current perceptions and experi | | |
| | Using telehealth for APRETUDE services <b>meets my approval</b> . | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Using telehealth for APRETUDE services <b>is</b> appealing to me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I <b>like</b> using telehealth for APRETUDE services. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I welcome using telehealth for APRETUDE services. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.208. Summary of Feasibility of Intervention (FIM) (Telehealth) (PSP) (Month 6/7), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 24 | Please indicate how much you with telehealth. | ou agree with each sta | itement based | on your current percep | tions and experience |
| | Using telehealth for APRETUDE services <b>seems</b> workable in my life. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Using telehealth for APRETUDE services <b>see possible</b> in my life. | APRETUDE services seems | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Using telehealth for APRETUDE services <b>seems doable</b> in my life. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | Using telehealth for APRETUDE services <b>seems easy</b> in my life. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely<br>disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.209. Changes from Baseline for Acceptability of Intervention Measure (AIM - APRETUDE) and Feasibility of Intervention Measure (FIM - APRETUDE) (Month 12/13), N=XX

| Measure | Study Arm | n | Mean | SD | Median (Q1, Q3) | Observed Range<br>(min, max) | Missing<br>n (%) | 95% CI<br>for the Mean |
|---|---|---|---|---|---|---|---|---|
| AIM - APRETUDE Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| AIM - APRETUDE Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| AIM - APRETUDE Change from Baseline to<br>Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| FIM - APRETUDE Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| FIM - APRETUDE Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| FIM - APRETUDE Change from Baseline to<br>Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |



Table 7.210. Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – APRETUDE) (Month 12/13), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 7.211. Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Acceptability of Intervention Measure (AIM – APRETUDE), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 7.212. Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – APRETUDE) (Month 12/13), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 7.213. Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Feasibility of Intervention Measure (FIM – APRETUDE), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 7.214. Changes from Baseline for Acceptability of Intervention Measure (AIM - Telehealth) and Feasibility of Intervention Measure (FIM - Telehealth) (Month 12/13), N=XX

| Measure | Study Arm | n | Mean | SD | Median (Q1, Q3) | Observed Range<br>(min, max) | Missing<br>n (%) | 95% CI<br>for the Mean |
|---|---|---|---|---|---|---|---|---|
| AIM - Telehealth Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| AIM - Telehealth Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| AIM - Telehealth Change from Baseline to<br>Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| FIM - Telehealth Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| FIM - Telehealth Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| FIM - Telehealth Change from Baseline to<br>Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |



Table 7.215. Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – Telehealth) (Month 12/13), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 7.216. Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Acceptability of Intervention Measure (AIM – Telehealth), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 7.217. Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – Telehealth) (Month 12/13), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 7.218. Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Feasibility of Intervention Measure (FIM – Telehealth), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 7.219. Summary of Pain/Activities After Injection (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 67 | Did you experience any redness, itching, swellin | local reaction(s) following an injecting, bruising. | on appointment | ? Examples of local r | eactions are |
| | | Yes | XX | XX | XX |
| | | Tes | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX |
| | | IVO | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX |
| | | 1 don't know | (XX.X%) | (XX.X%) | (XX.X%) |
| 68 | How acceptable was/wabruising. | ere your local reaction(s)? Examples | of local reaction | s are redness, itching | g, swelling, |
| | | Tatally, a constabile | XX | XX | XX |
| | | Totally acceptable | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Varyaccantable | XX | XX | XX |
| | | Very acceptable | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Madarataly assentable | XX | XX | XX |
| | | Moderately acceptable | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A little acceptable | XX | XX | XX |
| | | A little acceptable | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Not at all acceptable | XX | XX | XX |
| | | Not at all acceptable | (XX.X%) | (XX.X%) | (XX.X%) |
| 69 | How often are you able to return to your usual daily activities immediately following an injection appointment (for example, going back to work, social events, exercise, driving)? | | | | |
| | | Never | XX | XX | XX |
| | | Nevel | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Rarely | XX | XX | XX |
| | | Nately | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Sometimes | XX | XX | XX |
| | | סטוויכנווווביז | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Often | XX | XX | XX |
| | | Oiteii | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Always | XX | XX | XX |
| | | Aiways | (XX.X%) | (XX.X%) | (XX.X%) |
| 70 | How bothered were yo | u by pain <u>DURING</u> the injection? | | | |
| | | Not at all | XX | XX | XX |
| | | Not at all | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Λ ;++ - | XX | XX | XX |
| | | A little | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Moderately | XX | XX | XX |
| | | Moderately | (XX.X%) | (XX.X%) | (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Von | XX | XX | XX |
| | | Very | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Extremely | XX | XX | XX |
| | | Extremely | (XX.X%) | (XX.X%) | (XX.X%) |
| 71 | Think back to your <b>first</b> inje<br>your <b>first</b> APRETUDE injecti | ection, please rate the amount<br>ion | of pain/discomfort | you experienced <u>AF</u> | TER receiving |
| | | O (No noin) | XX | XX | XX |
| | | 0 (No pain) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 1 | XX | XX | XX |
| | | 1 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 2 | XX | XX | XX |
| | | 2 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 3 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 4 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 5 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 6 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 7 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 8 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 9 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 10 (Extreme pain) | (XX.X%) | (XX.X%) | (XX.X%) |
| 72 | | most recent injection. Please r<br>recent APRETUDE injection | | | |
| | | - 4 | XX | XX | XX |
| | | 0 (No pain) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 1 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 2 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 3 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | 4 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 5 | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 6 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 7 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 8 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 9 | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 10 (Extreme pain) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 73 | How acceptable was your pair | i? | | | |
| | | Totally acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Moderately acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 74 | Which of the following things | have you tried to reduce the p | , , | i i | |
| | | Took over-the-counter pain relievers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Used a hot compress | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Used a cold compress | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Avoided sitting for long periods of time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Light stretching and exercise | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.220. Summary of Patient Study Participants' Labs and Missed Doses (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 53 | Have you missed any of your APRETUDE injection visits in the last 6 months? This means not receiving an injection within your injection window. | | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 54 | Was missing your APRETUDE in | njection visits planned or unplan | ned? | | |
| | | All the injection visits I<br>missed were planned | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Some of the injection visits I missed were planned and some were unplanned | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | All the injection visits I missed were unplanned | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I prefer not to answer | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 55 | Did you start oral PrEP after m | issing any of your injection visits | ? | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 56 | How easy or difficult was it to start oral PrEP after a missed injection visit? | | | | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 57 | How acceptable was it to start | oral PrEP after a missed injectio | n visit? | 1 | 1 |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.301. Summary of Feasibility and Acceptability of Telehealth (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 22 | Have you used telehealth for any APRETUDE services in the last 6 months, such as completing forms online, video chatting with your provider, getting reminders about your injection, or scheduling injection appointments online? | | | | |
| | | Yes | XX | XX | XX |
| | | 163 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | XX | XX | XX |
| | | I don't know | (XX.X%) | (XX.X%) | (XX.X%) |
| 25 | What APRETUDE services do/ | did you receive via telehealth? | | | |
| ^ | Completing relevant clinic | Yes | XX | XX | XX |
| А | visit forms online | res | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| В | Your doctor ordering an HIV test at a lab near your home where you can go to take the test | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX | XX | XX |
| | | INO | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX |
| | | 1 2 2 1 2 1 1 1 2 1 | (XX.X%) | (XX.X%) | (XX.X%) |
| С | A nurse coming to your home to give you an HIV test | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | (\(\lambda.\(\lambda\)\) | (\lambda.\lambda/\delta) XX | (\lambda \tau \tau \tau \tau \tau \tau \tau \ta |
| | | I don't know | (XX.X%) | (XX.X%) | (XX.X%) |
| D | Video chatting with your doctor | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | Receiving reminders (e.g., text, email) about your scheduled injection appointment | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | I don't know | (XX.X%) | (XX.X%) | (XX.X%) |
| F | Scheduling your injection appointment online to go to your clinic/doctor's office for the injection | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | A nurse coming to your home to give you the injection | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | Sending messages to your doctor online | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| I | Reviewing your health documents, such as test results, online | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| J | A nurse coming to your home to conduct your labs (e.g., STI tests) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 26 | How <u>comfortable</u> is/was it to | use each of the following teleh | ealth services fo | r APRETUDE? | |
| А | Completing relevant clinic visit forms online | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Neither comfortable nor | XX | XX | XX |
| | | uncomfortable | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Your doctor ordering an HIV test at a lab near your home where you can go to take the test | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | A nurse coming to your home to give you an HIV test | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | Video chatting with your doctor | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | Receiving reminders (e.g., text, email) about your | Very comfortable | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | scheduled injection<br>appointment | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Scheduling your injection appointment online to go to your clinic/doctor's office for the injection | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | A nurse coming to your home to give you the injection | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | Sending messages to your doctor online | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| I | Reviewing your health<br>documents, such as test<br>results, online | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| J | A nurse coming to your home to conduct your labs (e.g., STI tests) | Very comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat comfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither comfortable nor uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not comfortable at all | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 27 | How <u>convenient</u> is/was it to u<br>well with your life activities an | se each of the telehealth servior<br>and plans, with little trouble. | ces for APRETUD | E? By convenient, w | e mean fitting in |
| А | Completing relevant clinic visit forms online | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Your doctor ordering an HIV test at a lab near your home where you can go to take the test | Very convenient | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat convenient | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | A nurse coming to your<br>home to give you an HIV<br>test | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | Video chatting with your doctor | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | Receiving reminders (e.g.,<br>text, email) about your<br>scheduled injection<br>appointment | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Scheduling your injection appointment online to go to your clinic/doctor's office for the injection | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Neither convenient nor | XX | XX | XX |
| | | inconvenient | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat inconvenient | XX | XX | XX |
| | | Joinewhat inconvenient | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | A nurse coming to your home to give you the injection | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | (XX.X%)<br>XX<br>(XX.X%) | XX<br>(XX.X%) | (XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | Sending messages to your doctor online | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 1 | Reviewing your health documents, such as test results, online | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| J | A nurse coming to your home to conduct your labs (e.g., STI tests) | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither convenient nor inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very inconvenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 28 | On average, how long did you | wait to connect to a doctor fo | r video chat? | | |
| | | Up to 5 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 6 to 10 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 11 to 15 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 16 to 30 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 30 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 29 | I would recommend telehealt | h services for APRETUDE to oth | ner people. | | |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.302. Summary of Quality of Care for Patient Study Participants (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 82 | To what extent do you agree v<br>clinic/provider? | vith each of the following sta | tements regarding | g your experience w | ith your |
| А | My provider explained<br>medical words that were<br>used so that I could<br>understand them. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | My provider encouraged me to ask questions. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | My provider really respected me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | My provider gave me<br>enough time to say what I<br>though was important. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | My provider listened carefully to what I had to say. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | Disagree | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | XX | XX | XX |
| | | Completely disagree | (XX.X%) | (XX.X%) | (XX.X%) |
| F | My provider explained why tests were being done. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| G | My provider made me feel comfortable talking about personal things. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Н | My privacy was respected. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| I | My provider does not judge me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| J | The provider had a respectful attitude towards my sexual orientation. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Agree | XX | XX | XX |
| | | 7.8.00 | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | (\text{\text{XX}} | (\times.\times/\dots) | (XX.X/6) |
| | | Completely disagree | (XX.X%) | (XX.X%) | (XX.X%) |
| K | The staff at the clinic does not judge me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| L | The staff at this clinic is kind and respectful to me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| М | I sometimes felt insulted<br>when the clinic staff spoke<br>to me. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| N | I felt judged by the clinic staff for being on PrEP. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 0 | I felt judged by my provider for being on PrEP. | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.303. Summary of Quality of Care for Patient Study Participants (Month 12/13), N=XX, Non-Score Questions

| Question | | Response | | |
|---|---|---|---|---|
| 82. To what extent do you agree wit each of the following statements regarding your experience with you clinical/provider? | Completely Agree | Agree | Neither agree nor<br>disagree | Disagree |
| I. My provider does not judge me. | | | | |
| Study Arms | | | | |
| Total | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Dynamic<br>Implementation | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Routine<br>Implementation | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Race, Dynamic Implementation | | | | |
| Asian | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Black or African<br>American | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| White | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Other | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Race, Routine Implementation | | | | |
| Asian | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Black or African<br>American | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |



| Question | | | Resp | Response | |
|---|---|---|---|---|---|
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | utine Implementation | | I | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | - | | | · |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | · · · · · · | | | . , |
| Ethnicity, To | 1 1 | | I. | <u>I</u> | |
| • | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | . , | , | . , | , , |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| Gender, Tot | al | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| J. The provi | der had a respectful attitude | towards my sexual or | ientation. | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynar | nic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routir | ne Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |


| Question | | Response | | | |
|---|---|---|---|---|---|
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | I | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dyna | mic Implementation | | | | ı |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Routi | ne Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Total | | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tot | tal | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| K. The staff | at the clinic does not judge me | | | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynar | mic Implementation | | | 1 | ı |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | <u> </u> | | | · |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | <u> </u> | | | · |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | . , | , | , | ` ' |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | ı |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | 1 | 1 | 1 |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| Ethnicity, T | Total | | | 1 | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, To | otal | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| L. The staff | f at this clinic is kind and respect | ful to me. | | | |
| Study Arms | S | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dyna | amic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routine I | mplementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dyna | mic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Rout | ine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, 1 | Total | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, To | otal | | | | |
| | Men who have sex<br>with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| M. I somet | times felt insulted when the clini | c staff spoke to me. | | | |
| Study Arm | S | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (NI )(V) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | (N = XX) | , , | | | (////////////////////////////////////// |
| | n (%) | , | | | (///.///0) |
| Race, Dyna | | · , , | | | (777.776) |
| Race, Dyna | n (%) | XX | XX | XX | XX |
| Race, Dyna | n (%)<br>amic Implementation | | | XX<br>(XX.X%) | |
| Race, Dyna | n (%) amic Implementation Asian | XX | XX | | XX |
| Race, Dyna | n (%) amic Implementation Asian (N = XX) | XX | XX | | XX |
| Race, Dyna | n (%) amic Implementation Asian (N = XX) n (%) Black or African | XX<br>(XX.X%) | XX<br>(XX.X%) | (XX.X%) | XX<br>(XX.X%) |
| Race, Dyna | n (%) amic Implementation Asian (N = XX) n (%) Black or African American | XX<br>(XX.X%) | XX<br>(XX.X%) | (XX.X%) | XX<br>(XX.X%) |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routi | ne Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, D | ynamic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| Ethnicity, Routine Implementation | | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, | Total | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, T | otal | | | | |
| | Men who have sex<br>with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| N. I felt ju | idged by the clinic staff for being | on PrEP. | | | |
| Study Arn | ns | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | <u> </u> | - | - | · |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | <u> </u> | | | , |
| Race, Dyn | namic Implementation | | 1 | 1 | I |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | . , | . , | . , | , |
| | Black or African<br>American | XX | XX | XX | XX |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routin | e Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | otal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tot | al | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| O. I felt judg | ged by my provider for being or | n PrEP. | | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynar | nic Implementation | | 1 | 1 | 1 |
| | Asian | XX | XX | XX | XX |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routi | ine Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| Ethnicity, Dynami | c Implementation | | | | |
| Hi | spanic or Latino | XX | XX | XX | XX |
| (N | I = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| N | ot Hispanic or Latino | XX | XX | XX | XX |
| (1) | I = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| Ethnicity, Routine | Implementation | | | | |
| Hi | spanic or Latino | XX | XX | XX | XX |
| (1) | I = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| N | ot Hispanic or Latino | XX | XX | XX | XX |
| (1) | I = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| Ethnicity, Total | | | | | |
| Hi | spanic or Latino | XX | XX | XX | XX |
| (1) | I = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| N | ot Hispanic or Latino | XX | XX | XX | XX |
| (1) | I = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| Gender, Total | | | | | |
| | len who have sex<br>ith men | XX | XX | XX | XX |
| 7) | I = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| Tr | ansgender men | XX | XX | XX | XX |
| (1) | I = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |



Table 7.304. Summary of Quality of Care for Patient Study Participants (Month 12/13), N=XX, Score Questions

| Question | | Response | | |
|---|---|---|---|---|
| 82. To what extent do you agree wit each of the following statements regarding your experience with your clinic/provider? | Completely Agree | Agree | Disagree | Completely<br>Disagree |
| A. My provider explained medical wo | ords that were used so that I | could understand | them. | |
| Study Arms | | | | |
| Total | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Dynamic<br>Implementation | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Routine<br>Implementation | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Race, Dynamic Implementation | | | | |
| Asian | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Black or African<br>American | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| White | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Other | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Race, Routine Implementation | | | | |
| Asian | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |
| Black or African<br>American | XX | XX | XX | XX |
| (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | utine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | tal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| Gender, Tot | al | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| B. My provi | der encouraged me to ask qu | estions. | | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynar | nic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routin | ne Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | | | Resp | Response | |
|---|---|---|---|---|---|
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | 1 | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | 1 | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | utine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | | | 1 | 1 | 1 |
| | Hispanic or Latino | XX | XX | XX | XX |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tot | al | | | | |
| | Men who have sex<br>with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| C. My provid | der really respected me. | | | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynar | nic Implementation | | | 1 | I |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | <u> </u> | | | · |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | · |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | . , | . , | , | , , |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | ı |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | 1 | 1 | 1 |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | Response | | | | |
|---|---|---|---|---|---|
| n (%) | | | | | |
| Ethnicity, Total | <u>'</u> | | | | ı |
| Hispanio | or Latino | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Not Hisp | anic or Latino | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Gender, Total | ' | | | | |
| Men wh<br>with me | o have sex<br>n | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Transge | nder men | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| D. My provider gave me | enough time to sa | y what I though was | important. | | |
| Study Arms | | | | | |
| Total | | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Dynamio<br>Implemo | | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Routine<br>Impleme | entation | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Race, Dynamic Impleme | entation | | | | |
| Asian | | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Black or<br>America | | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| White | | XX | XX | XX | XX |
| (N = XX) | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n (%) | | | | | |
| Other | | XX | XX | XX | XX |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| 1) | N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| Race, Routine Im | plementation | | | | |
| А | sian | XX | XX | XX | XX |
| 1) | N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| | lack or African<br>merican | XX | XX | XX | XX |
| 1) | N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| V | Vhite | XX | XX | XX | XX |
| 1) | N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| С | ther | XX | XX | XX | XX |
| 1) | N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| Race, Total | | | | | |
| А | sian | XX | XX | XX | XX |
| 1) | N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| | lack or African<br>merican | XX | XX | XX | XX |
| 1) | V = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| V | Vhite | XX | XX | XX | XX |
| 1) | V = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| C | ther | XX | XX | XX | XX |
| 1) | N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| Ethnicity, Dynam | ic Implementation | | | | |
| Н | lispanic or Latino | XX | XX | XX | XX |
| 1) | N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| Ν | lot Hispanic or Latino | XX | XX | XX | XX |
| 1) | N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| n | (%) | | | | |
| Ethnicity, Routin | e Implementation | | | | |
| Н | lispanic or Latino | XX | XX | XX | XX |
| 1) | V = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, T | Гotal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, To | otal | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| E. My prov | ider listened carefully to what I | had to say. | | | |
| Study Arms | S | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | amic Implementation | | | | |
| Race, Dyna | anne imprementation | | | | |
| Race, Dyna | Asian | XX | XX | XX | XX |
| Race, Dyna | | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | (XX.X%) |
| Race, Dyna | Asian | | | | |
| Race, Dyna | Asian (N = XX) | | | | |
| Race, Dyna | Asian (N = XX) n (%) Black or African | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Race, Dyna | Asian (N = XX) n (%) Black or African American | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routi | ne Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | ı |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, D | ynamic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | Response | | | | |
|---|---|---|---|---|---|
| Ethnicity, | Routine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, | Total | | | | ı |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | <u> </u> | | | |
| Gender, T | | | ı | 1 | I |
| , | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| F. My prov | vider explained why tests were b | eing done. | | I | |
| Study Arm | | - | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | - | | | · |
| Race, Dyn | amic Implementation | | 1 | 1 | I |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | . , | . , | . , | , , |
| | Black or African<br>American | XX | XX | XX | XX |



| Question | | | Resp | onse | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routin | e Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Dy | namic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | otal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tot | al | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| G. My provi | der made me feel comfortable | talking about perso | nal things. | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynar | nic Implementation | | 1 | 1 | 1 |
| <u> </u> | Asian | XX | XX | XX | XX |



| Question | Response | | | | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routir | ne Implementation | • | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | ı |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



| Question | | Resp | Response | | |
|---|---|---|---|---|---|
| Ethnicity, Dynamic Implementation | | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, Ro | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, To | otal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, Tot | al | | | | |
| | Men who have sex<br>with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| H. My privad | cy was respected. | | | | |
| Study Arms | | | | | |
| | Total | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Dynamic<br>Implementation | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Routine<br>Implementation | XX | XX | XX | XX |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Dynai | mic Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Routi | ne Implementation | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Race, Total | | | | | |
| | Asian | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Black or African<br>American | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | White | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| Question | | Response | | | |
|---|---|---|---|---|---|
| | n (%) | | | | |
| | Other | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, D | ynamic Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, R | outine Implementation | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Ethnicity, T | otal | | | | |
| | Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Not Hispanic or Latino | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| Gender, To | tal | | | | |
| | Men who have sex with men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |
| | Transgender men | XX | XX | XX | XX |
| | (N = XX) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | n (%) | | | | |



Table 7.305. Distributional Characteristics of Quality of Care for Patient Study Participants (Month 12/13), N=XX, Score Questions, Overall Score

| 82. To what extent do you agree with each of the following statements regarding your experience with your clinic/provider? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | 0.xx |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Gender | | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Transgender<br>Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Black or African<br>American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Not Hispanic<br>or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| | | | Dyna | mic Implementa | ation | | | |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |



| 82. To what extent<br>do you agree with<br>each of the<br>following<br>statements<br>regarding your<br>experience with<br>your clinic/provider? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Gender | | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Black or<br>African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Not Hispanic<br>or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| | | | Rout | ine Implementa | tion | | | |
| Site Volume | | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Gender | | | | | | | | |
| Men who<br>have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Transgender<br>Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Race | | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Black or<br>African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | - |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |



| 82. To what extent do you agree with each of the following statements regarding your experience with your clinic/provider? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean | Cronbach's<br>α |
|---|---|---|---|---|---|---|---|---|
| Ethnicity | | | | | | | | |
| Hispanic or<br>Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |
| Not Hispanic<br>or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) | _ |

Mean score = mean of responses of items A-H. Responses were scored on a scale of 1-4 with higher scores indicating higher quality of care.



Table 7.306. Summary of Utility of Proposed Implementation Strategies (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 49 | Have you used any of the follo | wing while taking APRETUD | E? | | |
| А | Brochures and other print<br>materials to educate you on<br>APRETUDE | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Videos to educate you on<br>HIV, PrEP, APRETUDE<br>materials (DI) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| С | A digital calendar specifically<br>made for APRETUDE to help<br>you plan your injections –<br>found on PillarSpot (DI) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| D | Reminders about your injections | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | Having video or telephone appointments with your doctor | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Sending chats or texts to<br>your doctor on the Pillar<br>Spot (DI) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| G | Having a nurse come to your<br>home to conduct your HIV<br>tests (DI) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| Н | Having a nurse come to your home to give your injection (DI) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| I | Receiving transportation to I the clinic/doctor's office for your injection (DI) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| J | A website/app where you access APRETUDE information – the Pillar Spot (DI) | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| K | The website where you access APRETUDE information (RI) | Yes | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| 50 | How useful has each of these | been in supporting you while | taking APRETUDI | E? | |
| А | Brochures and other print<br>materials to educate you on<br>APRETUDE | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| В | Videos to educate you on<br>HIV, PrEP, APRETUDE (DI) | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| С | A digital calendar specifically<br>made for APRETUDE to help<br>you plan your injections –<br>found on PillarSpot (DI) | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| D | Reminders about your injections | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| E | Having video or telephone appointments with your doctor | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| F | Sending chats or texts to<br>your doctor on the Pillar<br>Spot (DI) | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| G | Having a nurse come to your home to conduct your HIV tests (DI) | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| Н | Having a nurse come to your home to give your injection (DI) | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |


| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| 1 | Receiving transportation to<br>the clinic/doctor's office for<br>your injection (DI) | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| J | A website/app where you access APRETUDE information – the Pillar Spot (DI) | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | N/A |
| К | The website where you access APRETUDE information (RI) | Not at all useful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | N/A | XX<br>(XX.X%) |
| 51 | Did your clinic or doctor offer | the following for APRETUDE | visits? | | |
| А | Injections on specific days of the week | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| В | Ability to show up for your injection without an appointment | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | Appointments where you only get your injection and leave | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | Schedule out your injection appointments for 6 months or more | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | You and your doctor discussing the pros and cons (e.g., side effects, switching) of different PrEP options and together deciding which one is right for you | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 52 | How useful has each of these | been in supporting you whi | le taking APRETUDE | ? | |
| А | Injections on specific days of the week | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| В | Ability to show up for your injection without an appointment | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| С | Appointments where you only get your injection and leave | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D | Schedule out your injection appointments for 6 months or more | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E | You and your doctor discussing the pros and cons (e.g., side effects, switching) of different PrEP options and together deciding which one is right for you | Not at all useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not very useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Extremely useful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 85 | I am happy I switched from or | ral PrEP to APRETUDE. | | | |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not use oral PrEP<br>before receiving<br>APRETUDE | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 84 | I would recommend APRETU | DE to other people who could b | enefit from it. | | |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.307. Summary of Patient Study Participants' Preferences/Acceptability of APRETUDE Information, Appointment Reminders, and Locations (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 61 | If you have questions about AF | PRETUDE, where do you fin | d information? | | |
| | | I did not find answers<br>to my questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Product website | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Written materials such as the study handbook | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Speaking to a healthcare provider | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Social Media | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Internet search | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Friends | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Family | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The study app/website | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not had any questions so far | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 62 | How did you receive reminder | s about your injection appo | intments? | | |
| | | Phone calls | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Texts/SMS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Existing clinic app reminder | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | E-mails | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Reminder in the postal mail | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Face-to-face reminder<br>from a healthcare<br>provider | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Written<br>reminder/appointment | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | card with date and time | (XX.X%) | (XX.X%) | (XX.X%) |
| | | The study app/website | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Another type of reminder (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not received any reminders | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 63 | Which type(s) of appointment | t reminders are most helpfu | ll in keeping your ap | ppointment? | |
| | | Phone calls | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Texts/SMS | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Existing clinic app reminder | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | E-mails | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Reminder in the postal mail | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Face-to-face reminder<br>from a healthcare<br>provider | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Written<br>reminder/appointment<br>card with date and<br>time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The study app/website | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Another type of reminder (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I do not think any of<br>the reminders are<br>helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 64 | Have you received APRETUDE | injections at any locations of | other than your clin | ic in the past 12 mo | nths? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 65 | Which of the following location | ons have you received APRE | TUDE injections in t | he past 12 months? | |
| | | Nurse coming to your home | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | In face in a contract | XX | XX | XX |
| | | Infusion center | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Retail pharmacy clinic (e.g., Minute Clinic, | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | CVS) | | | |
| | | Other pharmacy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Hospital outpatient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Community-based | XX | XX | XX |
| | | organization | (XX.X%) | (XX.X%) | (XX.X%) |
| | | STD/STI clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Department of Health | XX | XX | XX |
| | | clinic | (XX.X%) | (XX.X%) | (XX.X%) |
| | | PrEP clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Community health | XX | XX | XX |
| | | center | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Mobile van | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 66 | Where else would you consid- | er receiving your injections? | ( / | (* ) | (* 1, 2) |
| | | Retail pharmacy clinic | | | |
| | | (e.g., Minute Clinic, | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other pharmacy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Hospital outpatient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Infusion center | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Community-based organization | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | STD/STI clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Department of Health clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | PrEP clinic | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Community health center | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Mobile van | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Nurse coming to your home | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.308. Summary of Appointment Scheduling (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX) | Routine<br>Implementation<br>(N = XX) |
|---|---|---|---|---|---|
| 58 | How easy or difficult is it to schedule appointments at the clinic/practice for your injections? | | | | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not scheduled any appointments at the clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 59 | How easy or difficult is it to reschedule appointments at the clinic/practice for your | | | | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not needed to<br>reschedule any<br>appointments | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 60 | How did you <u>reschedule</u> your app | pointment? | | | |
| | | I called the clinic/doctor's office | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I emailed the clinic/doctor's office | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I texted the clinic/doctor's office | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I scheduled the appointment online | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I sent a message on the online portal of the clinic/doctor's office | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX) | Routine<br>Implementation<br>(N = XX) |
|---|---|---|---|---|---|
| | | I went to the clinic/doctor's office | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.401. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 12/13), N=XX, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 36 | On average, how long h<br>when you leave? | nave you spent at the clinic/practice for y | our injection | visit from arrival at | the clinic to |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not gotten any of my injections at a clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | How acceptable is coming to the clinic every 2 months for an injection? | | | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | How convenient are yo with little trouble. | ur clinic's hours? By convenient, we mea | n fitting well | with your life activit | ies and plans, |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 39 | How easy or difficult ha | as it been to get to the clinic every 2 mor | | | <u> </u> |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Very easy | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 40 | Approximately how lo | ng has it taken you to get to the clinic/pra | ctice from yo | ur home to receive | your injection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | How did you get to th | e clinic/practice for your injections? | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drove a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 43 | | e transportation provided by your clinic/pr<br>fitting in well with your life activities and p | | | ry 2 months? <i>By</i> |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Convenient | XX<br>(VV V0/) | XX<br>(VV V9/) | XX<br>(VX V9/) |
| | | | (XX.X%)<br>XX | (XX.X%)<br>XX | (XX.X%)<br>XX |
| | | Somewhat convenient | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please provide your op | inion of the transportation provided by t | he clinic | | |
| | The transportation helped me keep my appointments. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The transportation service was easy to use. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Have you needed to se injection visits? | ek additional childcare/eldercare/other c | are to come | to the clinic/practice | e for your |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 46 | Have you taken any tim | ne off from work to receive injections? | | | |
| | | Yes | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How much time did yo | ou take off work to receive your injections | s? | | |
| | | I needed to take a whole day off work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a whole day off work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | Was your time off wor | rk for injections generally paid or unpaid? | ) | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.402. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Race, Dynamic Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 36 | On average, how long have you spent at the clinic/practice for your injection visit from arrival at the clinic to when you leave? | | | | | |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not gotten any of my injections at a clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | How acceptable is coming to the clinic every 2 months for an injection? | | | | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | How convenient are your clinic's hours? By convenient, we mean fitting well with your life activities and plans, with little trouble. | | | | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 39 | How easy or di | fficult has it been to get to the clinic eve | ry 2 months fo | r your injection | ? | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 40 | Approximately l | how long has it taken you to get to the c | clinic/practice f | rom your home | to receive yo | our injection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | How did you ge | t to the clinic/practice for your injection | ıs? | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drove a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 43 | | t is the transportation provided by your<br>mean fitting in well with your life activit | clinic/practice | for your injection | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please provide your opinion of the transportation provided by the clinic | | | | | |
| | The<br>transportation<br>helped me<br>keep my<br>appointments. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The transportation service was easy to use. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Have you neede injection visits? | d to seek additional childcare/eldercare | e/other care to | come to the cli | nic/practice fo | or your |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 46 | Have you taken | any time off from work to receive inject | tions? | 1 | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How much time | did you take off work to receive your i | njections? | | | |
| | | I needed to take a whole day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a whole day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | Was your time off work for injections generally paid or unpaid? | | | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.403. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Race, Routine Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 36 | On average, how long have you spent at the clinic/practice for your injection visit from arrival at the clinic to when you leave? | | | | | |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not gotten any of my<br>injections at a clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | How acceptable is coming to the clinic every 2 months for an injection? | | | | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | How convenient are your clinic's hours? By convenient, we mean fitting well with your life activities and plans, with little trouble. | | | | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 39 | How easy or dif | ficult has it been to get to the clinic eve | ry 2 months fo | r your injection | ? | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 40 | Approximately l | how long has it taken you to get to the c | linic/practice f | rom your home | to receive yo | our injection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | How did you get to the clinic/practice for your injections? | | | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drove a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 43 | | t is the transportation provided by your<br>mean fitting in well with your life activiti | clinic/practice | for your injection | n visit every | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please provide y | our opinion of the transportation provi | ded by the clin | ic | | |
| | The<br>transportation<br>helped me<br>keep my<br>appointments. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The<br>transportation<br>service was<br>easy to use. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Have you neede injection visits? | d to seek additional childcare/eldercare | e/other care to | come to the cli | inic/practice f | or your |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 46 | Have you taken | any time off from work to receive inject | ions? | | 1 | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How much time | did you take off work to receive your i | njections? | | | |
| | | I needed to take a whole day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a whole day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | Was your time off work for injections generally paid or unpaid? | | | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.404. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Race, Total

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 36 | On average, how you leave? | w long have you spent at the clinic/prac | tice for your in | jection visit fror | n arrival at th | e clinic to when |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not gotten any of my<br>injections at a clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | How acceptable is coming to the clinic every 2 months for an injection? | | | | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | How convenient are your clinic's hours? By convenient, we mean fitting well with your life activities and plans, with little trouble. | | | | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 39 | How easy or diff | ficult has it been to get to the clinic eve | ry 2 months fo | r your injection | ? | |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 40 | Approximately l | how long has it taken you to get to the c | linic/practice f | rom your home | to receive yo | our injection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | How did you get to the clinic/practice for your injections? | | | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drove a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 43 | | t is the transportation provided by your<br>mean fitting in well with your life activiti | clinic/practice | for your injection | n visit every | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please provide your opinion of the transportation provided by the clinic | | | | | |
| | The<br>transportation<br>helped me<br>keep my<br>appointments. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The transportation service was easy to use. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Have you neede injection visits? | d to seek additional childcare/eldercare | e/other care to | come to the cli | nic/practice f | or your |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 46 | Have you taken | any time off from work to receive injec | tions? | <u> </u> | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How much time | did you take off work to receive your i | njections? | | | |
| | | I needed to take a whole day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a whole day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | Was your time o | off work for injections generally paid or | unpaid? | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.405. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Ethnicity, Study Arms

| | | | Dynamic Implementation | | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic<br>or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| 36 | On average, how long have you spent at the clinic/practice for your injection visit from arrival at the clinic to when you leave? | | | | | |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not gotten any of my<br>injections at a clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | How acceptabl | le is coming to the clinic every 2 months | for an injection | on? | • | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | How convenier | nt are your clinic's hours? <i>By convenient,</i><br>ble. | we mean fitt | ing well with you | r life activitie | es and plans, |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 39 | How easy or di | ifficult has it been to get to the clinic eve | ry 2 months f | or your injection | ? | |



| | | | Dynamic Implementation | | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic<br>or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic o<br>Latino<br>(N = XX)<br>n (%) |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 40 | Approximately | how long has it taken you to get to the o | clinic/practice | from your home | to receive y | our injection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | How did you ge | t to the clinic/practice for your injection | s? | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drove a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic Ir | mplementation | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic<br>or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please provide y | our opinion of the transportation pro | vided by the cl | inic | | |
| | The transportation helped me keep my appointments. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The transportation service was easy to use. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Have you needed injection visits? | d to seek additional childcare/elderca | are/other care t | co come to the cli | nic/practice | for your |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic II | mplementation | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Not Hispanic<br>or Latino<br>(N = XX)<br>n (%) | Hispanic<br>or<br>Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 46 | Have you taken | any time off from work to receive injec | tions? | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How much time | e did you take off work to receive your ir | njections? | | | |
| | | I needed to take a whole day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a whole day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | Was your time | off work for injections generally paid or | unpaid? | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.406. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Ethnicity, Total

| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 36 | On average, h<br>when you leav | ow long have you spent at the clinic/pract<br>/e? | ice for your injection visit f | |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not gotten any of my<br>injections at a clinic | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | How acceptab | ole is coming to the clinic every 2 months f | or an injection? | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | How convenient are your clinic's hours? By convenient, we mean fitting well with your life activities and plans, with little trouble. | | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 39 | How easy or d | lifficult has it been to get to the clinic ever | y 2 months for your injecti | on? |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 40 | Approximately injection? | how long has it taken you to get to the cl | inic/practice from your hor | me to receive your |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | How did you get to the clinic/practice for your injections? | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drove a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 43 | | It is the transportation provided by your of<br>we mean fitting in well with your life activ | | |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please provide y | our opinion of the transportation provic | led by the clinic | |
| | The<br>transportation<br>helped me<br>keep my<br>appointments. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The transportation service was easy to use. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Have you neede injection visits? | d to seek additional childcare/eldercare, | other care to come to the | e clinic/practice for your |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 46 | Have you taken | any time off from work to receive injecti | ons? | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 47 | How much tim | e did you take off work to receive your in | jections? | |
| | | I needed to take a whole day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a whole day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | Was your time | off work for injections generally paid or u | unpaid? | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.407. Summary of Acceptability and Feasibility of APRETUDE Injection Visits (Month 6/7), N=XX, Gender, Total

| | | | Dynamic Im | plementation | Routine Im | plementation |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Men who<br>have sex<br>with men<br>(N = XX)<br>n (%) | Transgender<br>Men<br>(N = XX)<br>n (%) | Men who have sex with men (N = XX) n (%) | Transgender<br>Men<br>(N = XX)<br>n (%) |
| 36 | On average, how<br>when you leave | w long have you spent at the clinic/prac? | ctice for your i | njection visit fror | m arrival at the | e clinic to |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I have not gotten any of my<br>injections at a clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 37 | How acceptable | e is coming to the clinic every 2 months | for an injectio | n? | | |
| | | Very acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all acceptable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 38 | How convenien | t are your clinic's hours? <i>By convenient,</i><br>le. | we mean fitti | ing well with you | r life activities | and plans, |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 39 | How easy or dif | ficult has it been to get to the clinic eve | ry 2 months f | or your injection | ? | • |



| | | | Dynamic Implementation | | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Men who have sex with men (N = XX) n (%) | Transgender<br>Men<br>(N = XX)<br>n (%) | Men who have sex with men (N = XX) n (%) | Transgende<br>Men<br>(N = XX)<br>n (%) |
| | | Very easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Easy | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither easy nor difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Very difficult | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 40 | Approximately | how long has it taken you to get to the o | clinic/practice | from your home | to receive you | ur injection? |
| | | Up to 20 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 21-40 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 41-60 minutes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | 61-90 minutes (1hr-1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | More than 90 minutes (more than 1.5hrs) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 41 | How did you ge | et to the clinic/practice for your injection | ıs? | | | |
| | | Taxi/transportation service | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Ride-share service (e.g., Uber, Lyft) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Dropped off by someone else | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Drove a private vehicle | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Public transportation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Bicycle/scooter/skateboard/walking | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Transportation provided by clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |


| | | | Dynamic Im | nplementation | Routine Im | plementation |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Men who<br>have sex<br>with men<br>(N = XX)<br>n (%) | Transgender<br>Men<br>(N = XX)<br>n (%) | Men who<br>have sex<br>with men<br>(N = XX)<br>n (%) | Transgende<br>Men<br>(N = XX)<br>n (%) |
| | | Very convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all convenient | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 44 | Please provide y | our opinion of the transportation pro | ovided by the cli | nic | | 1 |
| | The<br>transportation<br>helped me<br>keep my<br>appointments. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The transportation service was easy to use. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 45 | Have you needed injection visits? | d to seek additional childcare/elderca | are/other care t | o come to the cli | nic/practice fo | or your |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic Im | plementation | Routine Im | olementation |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Men who have sex with men (N = XX) n (%) | Transgender<br>Men<br>(N = XX)<br>n (%) | Men who<br>have sex<br>with men<br>(N = XX)<br>n (%) | Transgender<br>Men<br>(N = XX)<br>n (%) |
| | | I am not caring for others right now (N/A) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 46 | Have you taker | any time off from work to receive injec | tions? | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I am not working right now | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 47 | How much time | e did you take off work to receive your ir | njections? | | | |
| | | I needed to take a whole day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a whole day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for each injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I needed to take a partial day off<br>work for some injections | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 48 | Was your time | off work for injections generally paid or | unpaid? | | | |
| | | Paid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Unpaid | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.408. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Study Arms

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 30 | Did you complete a Sexual Health Assessment from your provider or clinic/practice in the last 6 months? | | | | |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 31 | Did your provider or anot | her person at the clinic/practice | discuss the re | sults of the assessmer | nt with you? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't remember | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 32 | Who discussed the result | s of the assessment with you? | | | |
| | | My healthcare provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 33 | How helpful was discussir | ng the results with your provider | or another pe | erson at the clinic/prac | ctice? |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 34 | Please rate your experien | ce with the Sexual Health Assess | ment | | 1 |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | It was easy to take the<br>Sexual Health Assessment<br>on my digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor sent<br>the assessment before my<br>appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about<br>the privacy of my<br>answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor was<br>assessing my sexual<br>health | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not complete t | he assessment? | | | |
| | | I did not receive a Sexual<br>Health Assessment from<br>my provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made me feel uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned about the privacy of my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share<br>sexual health information<br>with my doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand why<br>my doctor or clinic was<br>asking me to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.409. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Race, Dynamic Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 30 | Did you complet | e a Sexual Health Assessmen | t from your provi | der or clinic/pract | ice in the last 6 m | onths? |
| | | V. | XX | XX | XX | XX |
| | | Yes | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX | XX |
| | | NO | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX | XX |
| | | TUOITERIOW | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 31 | Did your provide | er or another person at the cl | inic/practice discu | uss the results of t | he assessment wi | th you? |
| | | Vos | XX | XX | XX | XX |
| | | Yes | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX | XX |
| | | No | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't remember | XX | XX | XX | XX |
| | | r don t remember | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 32 | Who discussed t | he results of the assessment | with you? | | | |
| | | My healthcare | XX | XX | XX | XX |
| | | provider/doctor | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Apurco | XX | XX | XX | XX |
| | | A nurse | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A social worker | XX | XX | XX | XX |
| | | A Social Worker | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A peer educator | XX | XX | XX | XX |
| | | A peer educator | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Other (please | XX | XX | XX | XX |
| | | specify) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 33 | How helpful was | discussing the results with y | our provider or ar | nother person at t | he clinic/practice? | ? |
| | | Very helpful | XX | XX | XX | XX |
| | | very neipiui | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat helpful | XX | XX | XX | XX |
| | | Somewhat helpful | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A little helpful | XX | XX | XX | XX |
| | | , these fierprof | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Not at all helpful | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 34 | Please rate your | experience with the Sexual F | Health Assessmen | t | | |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | It was easy to take<br>the Sexual Health<br>Assessment on my<br>digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my<br>doctor sent the<br>assessment before<br>my appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my<br>doctor was<br>assessing my sexual<br>health | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not com | plete the assessment? | | | | |
| | | I did not receive a<br>Sexual Health<br>Assessment from<br>my provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment<br>made me feel<br>uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned<br>about the privacy of<br>my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to<br>share sexual health<br>information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand<br>why my doctor or<br>clinic was asking me<br>to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.410. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Race, Routine Implementation

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 30 | Did you complete | e a Sexual Health Assessmen | t from your provid | der or clinic/practi | ce in the last 6 m | onths? |
| | | Yes | XX | XX | XX | XX |
| | | 165 | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX | XX |
| | | 110 | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 31 | Did your provide | r or another person at the cl | inic/practice discu | iss the results of t | he assessment wi | th you? |
| | | Yes | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't remember | XX | XX | XX | XX |
| | | li Cil | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 32 | Who discussed th | ne results of the assessment | | | | |
| | | My healthcare provider/doctor | XX<br>(xx, x0/) | XX (222 222) | XX<br>()()() ()() | XX<br>(xx, x0/) |
| | | provider/doctor | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | | (XX.X70)<br>XX | (XX.X70)<br>XX | (XX.X70)<br>XX | (XX.X/0)<br>XX |
| | | A social worker | ^^<br>(XX.X%) | ^^<br>(XX.X%) | ^^<br>(XX.X%) | ^^<br>(XX.X%) |
| | | | XX | XX | XX | XX |
| | | A peer educator | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Other (please | XX | XX | XX | XX |
| | | specify) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | 1.1/4.1. | XX | XX | XX | XX |
| | | I don't know | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 33 | How helpful was | discussing the results with y | | nother person at t | he clinic/practice? | ? |
| | | Von boleful | XX | XX | XX | XX |
| | | Very helpful | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat helpful | XX | XX | XX | XX |
| | | Somewhat Helpful | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A little helpful | XX | XX | XX | XX |
| | | / thede helpful | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Not at all helpful | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 34 | Please rate your | experience with the Sexual F | lealth Assessment | t | | |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | It was easy to take<br>the Sexual Health<br>Assessment on my<br>digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my<br>doctor sent the<br>assessment before<br>my appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my<br>doctor was<br>assessing my sexual<br>health | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Neither agree nor disagree | XX | XX | XX | XX |
| | | Agree | (XX.X%)<br>XX<br>(XX.X%) | (XX.X%)<br>XX<br>(XX.X%) | (XX.X%)<br>XX<br>(XX.X%) | (XX.X%)<br>XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment<br>made me feel<br>uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not com | plete the assessment? | | | | |
| | | I did not receive a<br>Sexual Health<br>Assessment from<br>my provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | l forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment<br>made me feel<br>uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned<br>about the privacy of<br>my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to<br>share sexual health<br>information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand why my doctor or clinic was asking me to complete the assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.411. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Race, Total

| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| 30 | Did you complet | e a Sexual Health Assessmen | t from your provid | der or clinic/practi | ice in the last 6 m | onths? |
| | | Vas | XX | XX | XX | XX |
| | | Yes | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX | XX |
| | | NO | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX | XX |
| | | T GOTT E KNOW | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 31 | Did your provide | er or another person at the cl | inic/practice discu | iss the results of t | he assessment wi | th you? |
| | | Yes | XX | XX | XX | XX |
| | | Tes | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX | XX |
| | | 140 | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't remember | XX | XX | XX | XX |
| | | r don t remember | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 32 | Who discussed t | he results of the assessment | with you? | | | |
| | | My healthcare | XX | XX | XX | XX |
| | | provider/doctor | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A nurse | XX | XX | XX | XX |
| | | Atturse | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A social worker | XX | XX | XX | XX |
| | | 7.000.a. Werker | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A peer educator | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Other (please | XX | XX | XX | XX |
| | | specify) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 33 | How helpful was | discussing the results with y | | | | |
| | | Very helpful | XX | XX | XX | XX |
| | | , , | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Somewhat helpful | XX | XX | XX | XX |
| | | · | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A little helpful | XX | XX | XX | XX |
| | | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Not at all helpful | XX (V/ V0/) | XX (V/V V0/) | XX (V/V V0/) | XX (V// V0/) |
| 0. | 51 | | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| 34 | Please rate your | experience with the Sexual F | Health Assessment | t | | |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | It was easy to take<br>the Sexual Health<br>Assessment on my<br>digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my<br>doctor sent the<br>assessment before<br>my appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my<br>doctor was<br>assessing my sexual<br>health | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | Neither agree nor | XX | XX | XX | XX |
| | | disagree | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment<br>made me feel<br>uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not com | plete the assessment? | | | | |
| | | I did not receive a<br>Sexual Health<br>Assessment from<br>my provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I forgot | l forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Asian<br>(N = XX)<br>n (%) | Black or<br>African<br>American<br>(N = XX)<br>n (%) | White<br>(N = XX)<br>n (%) | Other<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|---|
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment<br>made me feel<br>uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned<br>about the privacy of<br>my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to<br>share sexual health<br>information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand<br>why my doctor or<br>clinic was asking me<br>to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.412. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Ethnicity, Study Arms

| | | | Dynamic Imp | olementation | Routine Imp | lementation |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| 30 | Did you complete a S | exual Health Assessment f | rom your provic | ler or clinic/prac | ctice in the last 6 | months? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 31 | Did your provider or | another person at the clini | c/practice discu | ss the results of | the assessment | with you? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't remember | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 32 | Who discussed the re | esults of the assessment wi | ith you? | | | |
| | | My healthcare provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 33 | How helpful was disc | ussing the results with you | ır provider or an | other person at | the clinic/practi | ce? |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX (XX.X%) | XX | XX | XX |



| | | | Dynamic Imp | olementation | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| | | | | (XX.X%) | (XX.X%) | (XX.X%) |
| 34 | Please rate your expe | rience with the Sexual He | alth Assessment | -<br>- | I | |
| | It was easy to take<br>the Sexual Health<br>Assessment on my<br>digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor | XX | XX | XX | XX |
| | | disagree | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX | XX | XX | XX |
| | | Completely agree | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | I like that my doctor<br>sent the assessment<br>before my<br>appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX | XX | XX | XX |
| | | Disagree | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned<br>about the privacy of<br>my answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor<br>was assessing my<br>sexual health. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic Im | olementation | Routine Implementation | |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| | | Disagrap | XX | XX | XX | XX |
| | | Disagree | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not comp | lete the assessment? | | | | |
| | | I did not receive a<br>Sexual Health<br>Assessment from my<br>provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| | | | Dynamic Im | plementation | Routine Imp | olementation |
|---|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Hispanic or<br>Latino<br>(N = XX)<br>n (%) | Not<br>Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment<br>made me feel<br>uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned<br>about the privacy of<br>my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to<br>share sexual health<br>information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand<br>why my doctor or<br>clinic was asking me<br>to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.413. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Ethnicity, Total

| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 30 | Did you complete a Sexual He | alth Assessment from your provide | r or clinic/practice in the | last 6 months? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 31 | Did your provider or another | person at the clinic/practice discuss | s the results of the assess | ment with you? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't remember | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 32 | Who discussed the results of | the assessment with you? | | |
| | | My healthcare provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 33 | How helpful was discussing th | ne results with your provider or ano | ther person at the clinic/ | oractice? |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 34 | Please rate your experience w | vith the Sexual Health Assessment | | |



| Question<br>Number | Question | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | It was easy to take the Sexual<br>Health Assessment on my<br>digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor sent the assessment before my appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor was assessing my sexual health. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX | XX |



| Question<br>Question<br>Number | | Response | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not complete the assessment? | | | |
| | | I did not receive a Sexual<br>Health Assessment from my<br>provider or clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | l forgot | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made me feel uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question Response | | Hispanic or Latino<br>(N = XX)<br>n (%) | Not Hispanic or<br>Latino<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | I was concerned about the privacy of my answers | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share sexual<br>health information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand why my<br>doctor or clinic was asking me<br>to complete the assessment | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.414. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Gender

| Question<br>Number | Question | Response | Men who have sex<br>with men<br>(N = XX)<br>n (%) | Transgender men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| 30 | Did you complete a Sexua | l Health Assessment from your provid | er or clinic/practice in the | last 6 months? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 31 | Did your provider or anot | her person at the clinic/practice discus | ss the results of the assess | ment with you? |
| | | Yes | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | No | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't remember | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 32 | Who discussed the results | s of the assessment with you? | | |
| | | My healthcare provider/doctor | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A nurse | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A social worker | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A peer educator | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 33 | How helpful was discussir | ng the results with your provider or an | other person at the clinic/ | practice? |
| | | Very helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Not at all helpful | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 34 | Please rate your experien | ce with the Sexual Health Assessment | • | |



| Question<br>Number | Question | Response | Men who have sex<br>with men<br>(N = XX)<br>n (%) | Transgender men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | It was easy to take the Sexual<br>Health Assessment on my<br>digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | a.g.rai aerreer | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor sent the assessment before my appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor was assessing my sexual health. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX | XX |



| Question<br>Number | Question | Response | Men who have sex<br>with men<br>(N = XX)<br>n (%) | Transgender men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not complete th | <u> </u> | | |
| | | I did not receive a Sexual<br>Health Assessment from my<br>provider or clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment made me feel uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Men who have sex<br>with men<br>(N = XX)<br>n (%) | Transgender men<br>(N = XX)<br>n (%) |
|---|---|---|---|---|
| | | I was concerned about the privacy of my answers | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share sexual<br>health information with my<br>doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand why my<br>doctor or clinic was asking me<br>to complete the assessment | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.415. Summary of Reach and Perceptions of Sexual Health Assessment Tool (Month 12/13), N=XX, Site Volume

| Question<br>Number | Question | Response | Total<br>(N = XX) | High Volume<br>(N = XX) | Low Volume<br>(N = XX) |
|---|---|---|---|---|---|
| Number | | | n (%) | n (%) | n (%) |
| 30 | Did you complete a Sexual Health Assessment from your provider or clinic/practice in the last 6 months? | | | | |
| | | V | XX | XX | XX |
| | | Yes | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX |
| | | No | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX |
| | | T don't know | (XX.X%) | (XX.X%) | (XX.X%) |
| 31 | Did your provider or a | nother person at the clinic/practice | discuss the res | ults of the assessmer | nt with you? |
| | | Vec | XX | XX | XX |
| | | Yes | (XX.X%) | (XX.X%) | (XX.X%) |
| | | No | XX | XX | XX |
| | | INO | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't remember | XX | XX | XX |
| | | r don't remember | (XX.X%) | (XX.X%) | (XX.X%) |
| 32 | Who discussed the results of the assessment with you? | | | | |
| | | My healthcare | XX | XX | XX |
| | | provider/doctor | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Apura | XX | XX | XX |
| | | A nurse | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A social worker | XX | XX | XX |
| | | A Social Worker | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A poor adjuster | XX | XX | XX |
| | | A peer educator | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Other (please specify) | XX | XX | XX |
| | | Other (please specify) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | I don't know | XX | XX | XX |
| | | T don't know | (XX.X%) | (XX.X%) | (XX.X%) |
| 33 | How helpful was discu | ussing the results with your provider | or another per | rson at the clinic/prac | ctice? |
| | | Very helpful | XX | XX | XX |
| | | very neipiul | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Samowhat halaful | XX | XX | XX |
| | | Somewhat helpful | (XX.X%) | (XX.X%) | (XX.X%) |
| | | A little helpful | XX | XX | XX |
| | | A little helpful | (XX.X%) | (XX.X%) | (XX.X%) |
| | | Not at all leaderful | XX | XX | XX |
| | | Not at all helpful | (XX.X%) | (XX.X%) | (XX.X%) |
| 34 | Please rate vour expe | rience with the Sexual Health Assess | ment | | |



| Question<br>Number | Question Response | | Total<br>(N = XX)<br>n (%) | High Volume<br>(N = XX)<br>n (%) | Low Volume<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | It was easy to take the<br>Sexual Health Assessment<br>on my digital device. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor sent<br>the assessment before my<br>appointment. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I was concerned about the privacy of my answers. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I like that my doctor was assessing my sexual health. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | High Volume<br>(N = XX)<br>n (%) | Low Volume<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | | (XX.X%) | (XX.X%) | (XX.X%) |
| | The assessment asked the right questions to help my doctor and me determine whether PrEP was right for me. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | The assessment made me feel uncomfortable. | Completely disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| 35 | Why did you not complete the assessment? | | | | |
| | | I did not receive a Sexual<br>Health Assessment from<br>my provider or<br>clinic/practice | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I forgot | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not know how to complete it | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The link my doctor sent did not work | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | I didn't have the time | I didn't have the time | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment took too long to complete | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | The assessment included too many personal questions | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | High Volume<br>(N = XX)<br>n (%) | Low Volume<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | The assessment made me feel uncomfortable | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I was concerned about the privacy of my answers | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not want to share<br>sexual health information<br>with my doctor or clinic | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I did not understand why<br>my doctor or clinic was<br>asking me to complete the<br>assessment | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | Other (please specify) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 7.416. Proportion of PSP Taking the Sexual Health Assessment through Month 13

| Proportion Taking the Sexual Health Assessment through Month 13 | N=XX<br>n | % |
|---|---|---|
| Study Arm | | |
| Dynamic Implementation | XX | X.XX% |
| Routine Implementation | XX | X.XX% |
| Site Volume | | |
| High | XX | X.XX% |
| Low | XX | X.XX% |
| Gender | | |
| Men who have sex with men | XX | X.XX |
| Transgender Men | XX | X.XX% |
| Race | | |
| Asian | XX | X.XX% |
| Black or African American | XX | X.XX% |
| White | XX | X.XX% |
| Other | XX | X.XX% |
| Ethnicity | | |
| Hispanic or Latino | XX | X.XX% |
| Not Hispanic or Latino | XX | X.XX% |
| Setting of administration | | |
| Face-to-face | XX | X.XX% |
| Telehealth | XX | X.XX% |
| Dynamic Implementation | | |
| Race | | |
| Asian | XX | X.XX% |
| Black or African American | XX | X.XX% |
| White | XX | X.XX% |
| Other | XX | X.XX% |
| Ethnicity | | |
| Hispanic or Latino | XX | X.XX% |
| Not Hispanic or Latino | XX | X.XX% |
| Routine Implementation | | |
| Race | | |
| Asian | XX | X.XX% |
| Black or African American | XX | X.XX% |
| White | XX | X.XX% |
| Other | XX | X.XX% |
| Ethnicity | | |
| Hispanic or Latino | XX | X.XX% |
| Not Hispanic or Latino | XX | X.XX% |



Table 7.417. Distributional Characteristics of Estimated Amount of Money Spent on Transportation for Each Injection Visit (Month 12/13), N=XX

| 42. On average, how much did transportation cost round trip for each injection visit? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Dynamic Implementation | | | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |


| 42. On average, how much did transportation cost round trip for each injection visit? | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Routine Implementation | | 1 | | 1 | | ı | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Gender | | | | | | | |
| Men who have sex with men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Transgender Men | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Race | | | | | | | |
| Asian | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Black or African American | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| White | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Other | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Ethnicity | | | | | | | |
| Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |
| Not Hispanic or Latino | XX | X.XX | X.XXX | X.XX<br>(X.XX, X.XX) | X.X<br>(X.X, X.X) | XX<br>(XX.X%) | (X.XXX,<br>X.XXX) |



Table 7.501. Test for Differences of Implementation Arm by Site Volume on Feasibility of Intervention Measure, APRETUDE (Month 12/13), N=XX

| Source | DF | MS | F | р |
|----------------------------|------|-------|----|--------|
| Study Arm (DI vs. RI) | X.XX | X.XXX | XX | 0.XXXX |
| Volume (High vs. Low) | X.XX | X.XXX | XX | 0.XXXX |
| Interaction, Arm by Volume | X.XX | X.XXX | XX | 0.XXXX |
| Error | X.XX | X.XXX | - | - |

Table 7.502. Test for Differences of Implementation Arm by Site Volume on Feasibility of Intervention Measure, Telehealth (Month 12/13), N=XX

| Source | DF | MS | F | p |
|----------------------------|------|-------|----|--------|
| Study Arm (DI vs. RI) | X.XX | X.XXX | XX | 0.XXXX |
| Volume (High vs. Low) | X.XX | X.XXX | XX | 0.XXXX |
| Interaction, Arm by Volume | X.XX | X.XXX | XX | 0.XXXX |
| Error | X.XX | X.XXX | - | - |

Table 7.503. Test for Differences of Implementation Arm by Site Volume on Acceptability of Intervention Measure, APRETUDE (Month 12/13), N=XX

| Source | DF | MS | F | p |
|----------------------------|------|-------|----|--------|
| Study Arm (DI vs. RI) | X.XX | X.XXX | XX | 0.XXXX |
| Volume (High vs. Low) | X.XX | X.XXX | XX | 0.XXXX |
| Interaction, Arm by Volume | X.XX | X.XXX | XX | 0.XXXX |
| Error | X.XX | X.XXX | - | - |

Table 7.504. Test for Differences of Implementation Arm by Site Volume on Acceptability of Intervention Measure, Telehealth (Month 12/13), N=XX

| Source | DF | MS | F | р |
|----------------------------|------|-------|----|--------|
| Study Arm (DI vs. RI) | X.XX | X.XXX | XX | 0.XXXX |
| Volume (High vs. Low) | X.XX | X.XXX | XX | 0.XXXX |
| Interaction, Arm by Volume | X.XX | X.XXX | XX | 0.XXXX |
| Error | X.XX | X.XXX | - | - |

A Phase 4, Randomized, Open-label, Two-arm Study Evaluating Implementation Strategies for the Delivery of Cabotegravir in Low- and High-volume Pre-exposure Prophylaxis (PrEP) Sites in the US for HIV Uninfected MSM and Transgender Men ≥18: 217710 PILLAR

Statistical Analysis Plan: Staff Study Participants Questionnaire

### EVA-32399 | October 4, 2024 | Version 2.0

#### Prepared For:



#### Prepared By:

PPD , MA | Senior Research Scientist, Patient Centered Research | PPD , MPH | Research Scientist, Patient Centered Research | PPD , MSc | Lead Data Analyst, Patient Centered Research | PPD , MPH | Research Associate III, Patient Centered Research Associate III, Patient Centered

#### Project Contact:

PPD , MS, PMP | Tel: PPD







### **Table of Contents**

| 1 | INTRODUCTION | 1 |
|---|---|---|
| 2 | PILLAR STUDY DESIGN | 1 |
| | 2.1 Feasibility of Intervention Measure | 3 |
| | 2.2 Acceptability of Intervention Measure | 4 |
| | 2.3 SSP Additional Questionnaire Items | 4 |
| | 2.4 Summary of Feasibility | 4 |
| | 2.5 Analysis Population | 5 |
| | 2.6 Missing Data Handling Scheme | 5 |
| | 2.7 Significance Levels and Multiplicity | 5 |
| 3 | STATISTICAL METHODS | 5 |
| | 3.1 Cross-sectional Distributional Characteristics of Study Variables and Features of Score Distributions | 6 |
| | 3.2 Feasibility and Acceptability of APRETUDE, Implementation Support, and Telehealth | |
| | 3.2.1 Cross-sectional Descriptive Statistics by Visits | 6 |
| | 3.2.2 Assessment of Variability Within vs. Between ClustersError! Bookmark not | defined. |
| | 3.2.3 Mixed-effects Models at M4/5 and M12/13 | 6 |
| | 3.2.4 Change from Baseline Mixed Models | 7 |
| | 3.3 SSP Perception of Facilitators and Barriers to Feasibility and Acceptability of APRETUDE | 7 |
| | 3.4 Acceptability and Utility of DI Compared with RI for APRETUDE Administration | 8 |
| | 3.5 Fidelity and Reach of Client Sexual Health Assessment | |
| | 3.5.1 SSP Perceptions of Sexual Health Assessment | 8 |
| | 3.5.2 Fidelity and Reach of Client Sexual Health Assessment | |
| | 3.6 Feasibility of Implementation of APRETUDE | 8 |
| | 3.7 Summaries of Site-level Characteristics | |
| | 3.8 Differences by Implementation Arm and Site Volume, FIM APRETUDE, FIM Implementati Support, and FIM Telehealth | |
| 4 | REFERENCES | 10 |
| 5 | TABLE SHELLS FOR BASELINE ANALYSIS | 11 |
| 6 | TABLES FOR MONTH 4/5 ANALYSIS | 104 |
| 7 | TABLES FOR MONTH 12/13 ANALYSIS | 262 |
| 8 | MULTIPLE TIMEPOINT TABLES | 439 |



### **List of Abbreviations**

| Abbreviation | Definition |
|--------------|--------------------------------------------------------|
| AIM | Acceptability of Intervention Measure |
| САВ | Cabotegravir |
| FIM | Feasibility of Intervention Measure |
| DTI | Direct to injection |
| LA | Long-acting |
| ISQ | Implementation science questionnaire |
| MSM | Men who have sex with men |
| PrEP | Pre-exposure prophylaxis |
| PSP | Patient Study Participant |
| RE-AIM | Reach, Efficacy, Adoption, Implementation, Maintenance |
| OLI | Oral lead-in |
| REML | Residual maximum likelihood |
| SAP | Statistical analysis plan |
| RI | Routine implementation |
| SD | Standard deviation |
| SSP | Staff Study Participant |
| SSI | Semi-structured interviews |
| TGM | Transgender Men |



### 1 Introduction

The study is conducted following the FDA approval and commercial availability of cabotegravir long-acting for pre-exposure prophylaxis (CAB LA for PrEP) in the U.S. This is an open-label, phase 4, two-arm (dynamic implementation and routine implementation) study of the delivery of CAB LA for PrEP in low and high-volume sites in the U.S. for men who have sex with men (MSM) and transgender (TGM) men greater than or equal to 18 years of age. About eighteen clinics (~9 high and ~9 low volume) have been randomized 2:1 to either dynamic implementation (DI) or routine implementation (RI) (protocol # 217710/ Amendment 1.0).

This statistical analysis plan (SAP) describes the analysis of the Staff Study Participant (SSP) questionnaire, which includes the analyses assessing the study personnel's responses to questions regarding acceptability and feasibility of implementing cabotegravir (CAB, GKS1265744) long-acting (CAB LA, APRETUDE), as well as their assessments of the process of delivering APRETUDE to Patient Study Participants (PSPs).

### 2 Pillar Study Design

The phase 4 study is designed to evaluate dynamic implementation (DI) versus routine implementation (RI) strategies on the feasibility of delivering APRETUDE within a variety of study sites—e.g., high versus low volume PrEP centers—over 12 months. The patient population includes MSM and TGM, but the focus of the current SAP is on the study staff at the PrEP sites. Approximately 18 sites were randomized 2:1 in the DI or RI implementation arms with approximately five staff members designated at each of these sites as SSPs. The key comparison of interest is the DI vs RI comparison, and since the randomization is at the site level, SSPs are nested within the randomization, i.e., the study is cluster-randomized. This may affect the interpretation of certain outcomes as the independence of responses may not hold. The implementation outcomes for this phase of data analysis will be assessed from the perspective of the SSPs.<sup>1</sup>

Objectives/endpoints relevant to the current SAP are listed in Table A.



### Table A. Study objectives for SSP data

| Objective Type | Objectives | Endpoints |
|---|---|---|
| Primary | To evaluate feasibility of dynamic implementation (DI) compared to routine implementation (RI) for APRETUDE administration. | Staff study participants' (SSPs) mean Feasibility of<br>Intervention Measure (FIM) score at M13. <sup>1</sup> |
| | To evaluate change in feasibility of RI and DI for APRETUDE administration | Change from baseline in SSPs' FIM score at M5 and M13. |
| | To evaluate change in feasibility of RI and DI for APRETUDE administration | SSPs perceptions of facilitators and barriers to RI and DI and overall implementation of PrEP into routine care assessed through M13. |
| | To evaluate feasibility and acceptability of telehealth delivery for APRETUDE administration by clinical staff. | SSPs' mean FIM and AIM scores as well as ISQ responses for telehealth delivery at BL, M5 and M13. |
| | To evaluate feasibility and acceptability of telehealth delivery for APRETUDE administration by clinical staff. | Change from baseline in SSPs' FIM and AIM score as well as ISQ responses for telehealth delivery at M5 and M13. |
| | To evaluate feasibility and acceptability of telehealth delivery for APRETUDE administration by clinical staff. | SSPs perception of facilitators and barriers to feasibility and acceptability of telehealth use through M13. |
| | To evaluate acceptability and utility of DI compared to RI for APRETUDE administration | SSPs' mean AIM score and ISQ responses at BL, M5 and M13. |
| | To evaluate acceptability and utility of DI compared to RI for APRETUDE administration | Change from baseline in SSPs' AIM score and ISQ responses at M5 and M13. |
| Secondary | To evaluate acceptability and utility of DI compared to RI for APRETUDE administration | Proportion of SSPs that respond in agreement on relevant items on the ISQ that each implementation strategy is fit for use through M13. |
| | To evaluate acceptability and utility of DI compared to RI for APRETUDE administration | SSPs perceptions of utility of implementation strategies and facilitators and barriers to acceptability of RI and DI through M13. |
| | To evaluate fidelity to injection and dosing window | SSPs perception of barriers and facilitators to fidelity to injections through M13. |
| | To evaluate fidelity and reach of client Sexual<br>Health Assessment | Proportion of site staff who administer Sexual Health<br>Assessment through M13. |
| | To evaluate fidelity and reach of client Sexual<br>Health Assessment | SSPs perceptions of Sexual Health Assessment through M13. |
| | To evaluate adaptations to any implementation strategies used in clinics to include but not limited to modifications to toolkits, RI and DI to support APRETUDE implementation | SSPs perceptions of adaptations to implementation strategies through M13. |
| | To evaluate perceptions, barriers and facilitators with SSPs | SSPs perception of barriers and facilitators through M13. |
| Tertiary | CCI | |





<sup>1</sup>If the site has only DTI patients, endpoints will be a month prior for SSPs

### 2.1 Feasibility of Intervention Measure

The Feasibility of Intervention Measure (FIM) is employed to evaluate the extent to which an intervention can be carried out. This four-item measure assesses perceived intervention feasibility by employing a standard item stem to various aspects of feasibility. The items are measured on a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The FIM has been validated with other implementation outcome measures.<sup>2</sup> Higher scores for FIM indicate greater feasibility. There are no reverse-scored items on the FIM and the mean score for feasibility of the intervention is calculated by averaging the responses from four items. The FIM has been adapted to measure SSPs' assessments of implementation of APRETUDE, implementation support, and telehealth. Mean scores for the FIM are derived by averaging the four items at each administration where at least two of four item responses are available. This mechanism for handling scoring in the presence of missing item-level responses has been used widely in patient- and clinician-reported outcomes.<sup>3</sup>



### 2.2 Acceptability of Intervention Measure

The Acceptability of Intervention Measure (AIM) is employed to evaluate the perception that a given intervention or treatment is satisfactory. It is similar to the FIM as it is a four-item measure, but it assesses perceived intervention acceptability instead of feasibility. The items are measured on a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The AIM was validated with a suite of implementation outcome measures. Higher scores for AIM indicate greater acceptability. As with the FIM, there are no reverse-scored items on the AIM, and the mean score for acceptability of the intervention is calculated by averaging the responses from four items, provided at least two of the four items have viable responses. The AIM has been adapted to measure SSPs' assessments of the implementation of: APRETUDE, implementation support, and telehealth.

### 2.3 SSP Additional Questionnaire Items

The tailored SSP questionnaire was developed specifically for this study and contains items regarding the SSP's role at the study site, as well as their attitudes, concerns, and anticipated/implemented procedures regarding the use of APRETUDE. The baseline SSP questionnaire has 78 items plus subitems including the FIM and AIM. The Month 4/5 and Month 12/13 questionnaires have 98 and 103 items including the FIM and AIM, respectively, plus subitems that employ several different response options.

### 2.4 Summary of Feasibility

Feasibility will be systematically evaluated and summarized using the RE-AIM Framework (Reach, Efficacy, Adoption, Implementation, Maintenance). This is adapted from Brant (2020).<sup>4</sup> Feasibility will be summarized across different data streams. Assessment will entail summarizing the following:

- Reach: 1) number of PrEP seeking individuals taken from the Clinic Demographic Questionnaires administered quarterly; 2) number of SSP administered sexual health assessments; 3) number of PSPs who receive sexual health assessments
- Effectiveness: 1) percent of initiated oral PrEP vs. APRETUDE taken from Clinic Demographic Questionnaires administered quarterly; 2) percent of individuals on APRETUDE taken from the Clinic Demographic Questionnaires administered quarterly; 3) SSP skill level with PrEP
- Adoption: Data from the implementation science questionnaire on perceptions of barriers and facilitators
- Implementation: Summary for FRAME-IS results and pre-screening or screening records.
- Maintenance: SSP satisfaction and assessment of APRETUDE implementation from implementation science question

SSP-supplied data to support the RE-AIM Framework include data listed above that come from the quarterly Clinic Demographic Questionnaire and the SSP-administered implementation science questionnaire.



### 2.5 Analysis Population

The study population in this analysis will be all the respondents who complete any item on the SSP questionnaire at any time point.

### 2.6 Missing Data Handling Scheme

Missing data at the item level are anticipated to be rare. However, in some cases, the SSP may terminate before completing the survey in its entirety. The scoring algorithm and handling the missing values for FIM and AIM are described in Sections 2.1, 2.2, and 3.2.1. If a participant decides to withdraw from the study, the data will be handled according to the protocol: "If the SSP is changing roles, the individual assuming the role will be enrolled in the study. An SSP will be considered lost to follow-up only if that SSP role in the clinic is eliminated. Otherwise, an SSP who leaves their role will be replaced with the SSP who assumes the role to complete subsequent assessments." SSPs will be analyzed according to the data given, no data imputation will be implemented. Replacement SSPs will be included in any cross-sectional analyses. Although it is not anticipated that any replacement SSPs will have baseline data and thus will not be included in change from baseline analyses, should a replacement SSP have baseline data, those individuals would be included in change from baseline analyses.

### 2.7 Significance Levels and Multiplicity

Any statistical significance tests will be two-tailed and will be conducted with Type I error probability fixed at 0.05. Statistical significance, then, will be determined if the p-value is less than 0.05. No multiplicity adjustment will be performed. The general null and alternative hypotheses for statistical tests will be for a given parameter  $(\theta)$ —e.g., mean:

 $H_0: \theta = 0$ 

Versus

 $H_A: \theta \neq 0$ 

### 3 Statistical Methods

Continuous and interval-like variables will be summarized using descriptive statistics (e.g., n, mean, standard deviation [SD], minimum, first quartile, median, third quartile, and maximum). Means and quartiles will be summarized to one decimal place beyond the data values, SD will be reported to two decimal places more than the source data, and minima and maxima will be reported to the same precision level as the source data. Categorical variables will be reported as frequency counts as whole numbers and percentages with one decimal (e.g., 10.1%), the percentage of SSPs in corresponding categories. Continuous outcomes will be evaluated depending on the number of group comparisons being made. Grouping variables with two levels will be compared with t-tests. Grouping variables with three or more categories will be evaluated with F-tests and pairwise comparisons will be calculated to aid in interpretation of main effects. Categorical variables will be analyzed with Cochran-Mantel-Haenszel tests or Fisher's Exact Test depending on data availability per category, i.e., if any cell of a given contingency table has a cell with incidence of five or less. Summaries by clinic/practice type will be stratified by the following groupings based on Question 1 from the Site Questionnaire:



University/Academia/Research; Federally Qualified Health Center / Department of Health; Nonprofit; Private.

# 3.1 Cross-sectional Distributional Characteristics of Study Variables and Features of Score Distributions

For questions with ordinal responses, a univariate distribution of every item will be tabulated. Standard distributional statistics will be tabulated for interval-like (ordinal) variables, including mean, SD, median, percentage missing, minimum, and maximum of responses, percentage of the sample at the ceiling and floor, first and third quartiles, and 95% confidence intervals. For questions with categorical responses, a frequency distribution of all responses will be presented with the number and percentage of a given response.

# 3.2 Feasibility and Acceptability of APRETUDE, Implementation Support, and Telehealth

### 3.2.1 Cross-sectional Descriptive Statistics by Visits

SSPs' mean FIM and AIM scores focusing on APRETUDE, Implementation Support, and telehealth at baseline, M4/M5, and M12/M13 will be evaluated by the study arms by both descriptive statistics and using the mixed-effects modeling approaches described below. Descriptive statistics of scores and coded item response will include those listed in Section 3.1 for continuous variables. Additionally, item response frequencies and percentages will be produced for individual items to further assess the distribution of responses.

### 3.2.2 Mixed-effects Models at M4/5 and M12/13

Cross-sectional mixed-effects models will be fit to the FIM and AIM mean scores at M4/5 and M12/13. These mixed-effects models will be fit using residual maximum likelihood (REML) and will assume data are missing at random. All data will be included regardless of early cessation from the implementation arm. The dependent variables will be the FIM and AIM mean scores, respectively. In the model, implementation arm (DI versus RI), site volume (high versus low) and the implementation arm by site volume interaction will be fitted as fixed terms, with separate random intercepts fitted to allow for clustering within sites, and for variability within the sites. Site volume was categorized as high versus low according to the reported estimate of PrEP patient seen monthly. These data were split at the median of 50; values above 50 were considered high and those below 50 were considered low. The baseline scores centered around their site mean will be fitted as both fixed and random covariates. An unstructured covariance structure will be fitted to account for the dependence of the residuals within the provider. Should the unstructured covariance structure cause model fitting problems (e.g., nonconvergence), heterogenous compound symmetry will be considered followed by homogenous compound symmetry. Should model fitting problems persist, the random effect on centered mean baseline score will be removed and models will be fit according to the same order of covariance structures (unstructured, then heterogenous compound symmetry, then homogenous compound symmetry).



The corresponding multilevel model for the FIM and AIM scores,  $Y_{ij}$ , for the  $i^{th}$  individual at the  $j^{th}$  site is expressed as:

$$\begin{split} Y_{ij} &= \beta_{00} + \beta_{01}I_j + \beta_{02}V_j + \beta_{03}I_jV_j + \beta_{10}\big(B_{ij} - \bar{B}_j\big) + u_{0j} + u_{1j}\big(B_{ij} - \bar{B}_j\big) + e_{ij} \\ & e_{ij} \sim N(0, \sigma^2) \\ \begin{pmatrix} u_{0j} \\ u_{1j} \end{pmatrix} \sim N\begin{bmatrix} \begin{pmatrix} 0 \\ 0 \end{pmatrix}, \begin{pmatrix} \tau_{00} & \tau_{01} \\ \tau_{10} & \tau_{11} \end{pmatrix} \end{bmatrix} \end{split}$$

With fixed effects for baseline score  $(B_{ij} - \bar{B}_j)$ , implementation arm  $(I_j)$ , site volume  $(V_j)$ , and the arm by volume interaction. The parameter  $\beta_{00}$  is the fixed mean for the RI arm with low volume. The parameters  $\beta_{01}$ ,  $\beta_{02}$ ,  $\beta_{03}$ , and  $\beta_{10}$  are regression weights for the fixed effects of DI arm, high volume, arm by volume, and baseline score, respectively. Random effects for sites  $(u_{0j})$ , baseline scores across sites  $(u_{1j})$ , and the residual error  $(e_{ij})$  are also included. All random effects and the error term are assumed to be independent. Coding of the mixed-effects models will be done as suggested by Singer (1998). It is worth noting that there is likely a range restriction on both FIM and AIM endpoints given that the measures are fairly discrete (i.e., on a 1-5 scale with 0.25 increments) and so adjustment of the mixed-effects models may be necessary if the model fits are determined to be affected by this range restriction. The study implementation arms and specific timepoint contrasts will be calculated within the mixed-effects modeling framework.

### 3.2.3 Change from Baseline Mixed Models

Change from baseline in SSPs' AIM and FIM scores at M4/5, and M12/M13 will be modeled similarly to those described in Section 3.2.2. The dependent variables in this case, however, will be the change from baseline in FIM and AIM mean scores, respectively.

The corresponding multilevel model for the changes from baseline in FIM and AIM scores,  $(Y_{ij} - B_{ij})$ , for the  $i^{th}$  individual at the  $j^{th}$  site is expressed as:

$$\begin{split} \left(Y_{ij} - B_{ij}\right) &= \beta_{00} + \beta_{01}I_j + \beta_{02}V_j + \beta_{03}I_jV_j + \beta_{10}\left(B_{ij} - \bar{B}_j\right) + u_{0j} + u_{1j}\left(B_{ij} - \bar{B}_j\right) + e_{ij} \\ &\qquad \qquad e_{ij} \sim N\left(0, \sigma^2\right) \\ \left(\begin{matrix} u_{0j} \\ u_{1j} \end{matrix}\right) \sim N\left[\begin{pmatrix} 0 \\ 0 \end{matrix}\right], \begin{pmatrix} \tau_{00} & \tau_{01} \\ \tau_{10} & \tau_{11} \end{pmatrix}\right] \end{split}$$

Similar to the model in Section 3.2.2, we include the same fixed and random effects. All random effects and the error term are assumed to be independent and random effects will be fit with an unstructured covariance matrix at the outset. Model fitting will be attempted until an adequately fitting model is found according to the hierarchy of covariance structures and model specifications described in section 3.2.2. REML will be used to estimate the model's parameters.

# 3.3 SSP Perception of Facilitators and Barriers to Feasibility and Acceptability of APRETUDE

The SSP perception of facilitators and barriers to feasibility and acceptability of APRETUDE will be tabulated by implementation arm and site volume. Descriptive analyses of the facilitators and barriers will



be conducted at all time points. Additionally, post-baseline—i.e., at M4/5 and M12/M13—Cochran—Mantel—Haenszel tests of these categorical outcomes by arm and subgroup will be completed with a p-value less than 0.05 considered to be statistically significant. Also, Fisher's Exact test may be used if any cell in the cross-tabulation of categorical variables is five or less.

## 3.4 Acceptability and Utility of DI Compared with RI for APRETUDE Administration

Proportion of SSPs responded in agreement on relevant items that each implementation strategy is fit for use, e.g., if a strategy is used and whether that strategy was found to be useful, at M12/M13 will be estimated. It will be compared between the two study arms, site volume, and SSP type as a stratification factor using a Cochran–Mantel–Haenszel test. Baseline responses will be summarized descriptively.

### 3.5 Fidelity and Reach of Client Sexual Health Assessment

### 3.5.1 SSP Perceptions of Sexual Health Assessment

SSP perceptions of Sexual Health Assessment through M4/5 and M12/M13 will be tabulated by implementation arm and site volume. Cochran–Mantel–Haenszel tests will be computed comparing implementation arms at M12/13. A p-value of less than 0.05 will be considered statistically significant.

#### 3.5.2 Fidelity and Reach of Client Sexual Health Assessment

Proportions of the site staff who administer the Sexual Health Assessment through M12/M13 and by clinic characteristics and their 95% confidence interval will be estimated. The difference between the proportions by clinic characteristics will be assessed using a two-sided 95% confidence intervals, and a Cochran–Mantel–Haenszel statistic will be provided.

### 3.6 Feasibility of Implementation of APRETUDE

SSP evaluations of feasibility measured as reach, effectiveness, adoption, implementation, and maintenance through M13 will be tabulated by study arm and clinic characteristics, and a Cochran—Mantel—Haenszel test of these categorical outcomes of the subgroups will be completed. A p-value less than 0.05 will be considered statistically significant. The subgroups will include study arm and clinic characteristics. The analysis will be completed at M4/5 and M12/M13.

### 3.7 Summaries of Site-level Characteristics

Responses by the site designee for the 17-item overall site-level questionnaire will be summarized at baseline.



# 3.8 Differences by Implementation Arm and Site Volume, AIM/FIM APRETUDE, AIM/FIM Implementation Support, and AIM/FIM Telehealth

Difference for AIM/FIM means scores in SSP by implementation arm (RI, DI), site volume (high, low), and the interaction of these variables will be tested using a 2 x 2 between-subjects analysis of variance. The AIM/FIM for APRETUDE, implementation support and telehealth will be tested, separately, in all analyses all factors will be fixed. Significant interactions will be followed up with appropriate simple effects.



### 4 References

- 1. A Phase 4, randomized, open-label, two-arm study evaluating implementation strategies for the delivery of Cabotegravir in low and high-volume pre-exposure prophylaxis (PrEP) sites in the U.S. for HIV uninfected MSM and transgender men ≥18. Study protocol 217710/Amendment 1.0. ViiV Healthcare Company, Research Triangle Park, NC.
- 2. Weiner BJ, Lewis CC, Stanick C, et al. Psychometric assessment of three newly developed implementation outcome measures. *Implement Sci.* 2017;12(1):108.
- 3. Cella D. Manual of the Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System—Version 4. Evanston, IL: Center on Outcomes, Research & Education (CORE), Evanston Northwestern Healthcare and Northwestern University; 1997.
- 4. Brant AR, Dhillon P, Hull S, et al. Integrating HIV Pre-Exposure Prophylaxis into Family Planning Care: A RE-AIM Framework Evaluation. *AIDS Patient Care STDS*. 2020;34(6):259-266.
- 5. Singer JD. Using SAS PROC MIXED to fit multilevel models, hierarchical models, and individual growth models. *J Educational Behavioral Stat.* 1998;24(4):323-355.



### **5** Table shells for Baseline Analysis

| Table 1.001 | Demographic Characteristics of Staff Study Participants (Month 1), N=XX | . 13 |
|---|---|---|
| Table 1.002 | Characteristics of Staff Study Participants (Month 1), N=XX | . 15 |
| Table 1.003 | Summary of Confidence with Skills (Month 1), N=XX | . 17 |
| Table 1.004 | Summary of Staff Study Participants' Perceptions Regarding APRETUDE (Month 1), N=XX | . 19 |
| Table 1.005 | Summary of Experiences with the Acquisition Process (Month 1), N=XX | . 23 |
| Table 1.101 | Summary of Acceptability of Intervention Measure (AIM - APRETUDE) and Feasibility of Intervention Measure (FIM - APRETUDE) Items (Month 1), N=XX | . 30 |
| Table 1.102 | Distributional Characteristics of the Acceptability of Intervention Measure (AIM – APRETUDE) (Month 1), N=XX | . 31 |
| Table 1.103 | Distributional Characteristics of the Feasibility of Intervention Measure (FIM - APRETUDE) (Month 1), N=XX | . 33 |
| Table 1.201 | Summary of Acceptability of Intervention Measure (AIM - IMPLEMENTATION SUPPORT) and Feasibility of Intervention Measure (FIM - IMPLEMENTATION SUPPORT) Items (Month 1), N=XX | . 35 |
| Table 1.202 | Distributional Characteristics of the Acceptability of Intervention Measure (AIM – IMPLEMENTATION SUPPORT) (Month 1), N=XX | . 36 |
| Table 1.203 | Distributional Characteristics of the Feasibility of Intervention Measure (FIM - IMPLEMENTATION SUPPORT) (Month 1), N=XX | . 38 |
| Table 1.301 | Summary of Acceptability of Intervention Measure (AIM - TELEHEALTH) and Feasibility of Intervention Measure (FIM - TELEHEALTH) Items (Month 1), N=XX | . 40 |
| Table 1.302 | Distributional Characteristics of the Acceptability of Intervention Measure (AIM – TELEHEALTH) (Month 1), N=XX | . 41 |
| Table 1.303 | Distributional Characteristics of the Feasibility of Intervention Measure (FIM - TELEHEALTH) (Month 1), N=XX | . 43 |
| Table 1.304 | Summary of Feasibility and Acceptability of Telehealth (Month 1), N=XX | |
| Table 1.401 | Summary of Utility of Proposed Implementation Strategies (Month 1), N=XX | .50 |
| Table 1.501 | Summary of Perceived Barriers to Delivering APRETUDE to Patients (Month 1), N=XX | .54 |
| Table 1.502 | Summary of Perceptions of Administering APRETUDE (Month 1), N=XX | . 57 |
| Table 1.503 | Summary of Perceived Barriers to Managing Delivery of APRETUDE (Month 1), N=XX | . 59 |
| Table 1.504 | Summary of Perceived Resourcing Barriers to Support Delivery of APRETUDE (Month 1), N=XX | . 62 |
| Table 1.505 | Summary of Perceptions of Clinic/Practice Culture and Environment | . 65 |
| Table 1.506 | Summary of Barriers to PrEP Provisioning (Month 1), N=XX | . 67 |
| Table 1.601 | Summary of the Sexual Health Assessment Tool (Month 1), N=XX | . 69 |
| Table 1.602 | Summary of the PrEP Communication Tool (Month 1), N=XX | .72 |
| Table 1.701 | Summary of the Optional Oral Lead-in Phase of APRETUDE (Month 1), N=XX | . 74 |
| Table 1.702 | Summary of Study Staff Participants' Injectable Cabotegrevir Experience (Month 1), N=XX | . 76 |



| Table 1.801 | Summary of Perceived Number of APRETUDE Patients Clinic/Practice Can Manage Per Week on an Ongoing Basis (Month 1), N=XX | . 80 |
|---|---|---|
| Table 1.802 | Distributional Characteristics of Reported Number of People in Clinic Trained and Prepared to Give APRETUDE Injections (Month 1), N=XX | .81 |
| Table 1.803 | Distributional Characteristics of Estimated Number of Staff Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25 People (Month 1), N=XX | .82 |
| Table 1.804 | Summary of Estimated Percentage of Staff Time/Full-Time Equivalent Hours Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25 People (Month 1), N=XX | .83 |
| Table 1.805 | Summary of Plans to Create New Roles/Positions in Clinic to Coordinate the APRETUDE Program (Month 1), N=XX | . 84 |
| Table 1.806 | Summary of Number of New Roles/Positions in Clinic to Coordinate the APRETUDE Program (Month 1), N=XX | . 85 |
| Table 1.807 | Summary of How Clinic/Practice Plans to Track Patients on APRETUDE (Month 1), N=XX | .86 |
| Table 1.808 | Summary of How Clinic/Practice Responds to Patients who Do Not Show for a Regularly Scheduled Appointment (Month 1), N=XX | . 87 |
| Table 1.809 | Summary Characteristics of Whether Clinic/Practice has Specific Person in Charge of Following Up on No-Shows (Month 1), N=XX | . 88 |
| Table 1.810 | Summary of Type of Systems Clinic has in Place to Remind Patients of Upcoming Appointments (Month 1), N=XX | . 89 |
| Table 1.811 | Summary of Type of Systems Clinic has in Place to Offer Upcoming Appointments (Month 1), N=XXT | . 90 |
| Table 1.812 | Summary of Implementing APRETUDE in Practice (Month 1), N=XX | .91 |
| Table 1.901 | Distributional Characteristics of Select Study Site Characteristics (Month 1), N=XX | .93 |
| Table 1.902 | Summary of Selected Study Site Characteristics (Month 1), N=XX | 102 |



Table 1.001 Demographic Characteristics of Staff Study Participants (Month 1), N=XX

| | | | Study | / Arm |
|---|---|---|---|---|
| Question<br>Number | | Total<br>(N=XX) | Dynamic<br>Implementation<br>(N=XX) | Routine<br>Implementation<br>(N=XX) |
| | | n (%) | n (%) | n (%) |
| 69 | Gender | | | |
| | Cisgender Male | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Cisgender Female | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Transgender Man | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Transgender Woman | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Nonbinary | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Gender Queer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other Gender | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I prefer not to answer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 70 | Age (years) | | | |
| | N | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 70 | Age (years), High Volume | | | |
| | N | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 70 | Age (years), Low Volume | | | |
| | N | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 70 | Age | | | |
| | 18-25 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 26-35 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 66-49 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| | | | Study Arm | |
|---|---|---|---|---|
| Question<br>Number | | Total<br>(N=XX) | Dynamic<br>Implementation<br>(N=XX) | Routine<br>Implementation<br>(N=XX) |
| | | n (%) | n (%) | n (%) |
| | 50+ | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 71 | Race | | | |
| | White/Caucasian | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Black | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Asian | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Native American | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Pacific Islander | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Mixed Race | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other Race | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | l Prefer not to Answer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 72 | Ethnicity | | | |
| | Hispanic/Latinx | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Non-Hispanic/Latinx | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Prefer not to answer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.002 Characteristics of Staff Study Participants (Month 1), N=XX

| Question<br>Number | Characteristic | | Stud | Study Arm |
|---|---|---|---|---|
| | | Total<br>(N=XX) | | Routine<br>Implementation<br>(N=XX) |
| | | n (%) | n (%) | n (%) |
| 1 | Provider Type | | | |
| | Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Nurse Practitioner | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Physician Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Social worker/case manager | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Office administrator/clinic administrator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Laboratory staff/technician/phlebotomist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Front desk staff/ Scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 2 | Personally Administer Injections | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 3 | Prescribe Medications as part of role | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 4 | Currently Prescribing Oral PrEP[2] | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 5 | Currently Provide PrEP Counseling | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 73 | Specialty[2][3] | | | |
| | Infectious disease specialist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Internal medicine/ primary care/general doctor/<br>family practitioner | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | HIC Specialist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Immunologist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Women's health/obstetricians and gynecologists | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Endocrinologist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other[4] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Characteristic | Study Arm | | y Arm |
|---|---|---|---|---|
| 74 | Length of Time practicing Medicine | | | |
| | <1 year | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 1–5 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 6–10 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 11-15 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 16-20 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | >21 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

- [1] Other responses include: xxx
- [2] Only SSPs who responded 'Yes' to 'Do you prescribe medications as part of your role?'
- [3] Not mutually exclusive
- [4] Other responses include: xxx



Table 1.003 Summary of Confidence with Skills (Month 1), N=XX

| | | | | Study Arm | |
|---|---|---|---|---|---|
| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>( N = XX)<br>n (%) |
| 6 | Please rate your level of confiden | ce for each skill listed: | | | |
| | Talking to Patient About Sexual<br>History | Somewhat Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Extremely Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My Role | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Screening Patient to Determine CAND PrEP | Not At All Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Extremely Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My Role | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Answering Patient's Questions<br>About PrEP | A Little Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Extremely Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My Role | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Suggesting PrEP to a Patient | Not At All Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Extremely Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| | Question | Response | | Study Arm | |
|---|---|---|---|---|---|
| Question<br>Number | | | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>( N = XX)<br>n (%) |
| | | Not Applicable To My Role | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Monitoring a Patient on PrEP | Not At All Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Extremely Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My Role | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.004 Summary of Staff Study Participants' Perceptions Regarding APRETUDE (Month 1), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 7 | In your opinion, APRETUD | E is appropriate for which individuals? | | | |
| | | Are Sexually Active | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have Been Sexually Active With 1<br>Or More Partners In The Last 6<br>Months | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Are Currently Adherent On Daily<br>Oral Prep | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Are Non-Adherent On Daily Oral<br>Prep | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Use Prep On Demand (I.E., Event-<br>Based Prep, Prep 2-1-1) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Could Benefit From Prep But Do<br>Not Want To Use Daily Prep | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have Previously Used And<br>Discontinued Daily Prep | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Feel Stigmatized About Taking Oral<br>Prep | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Request APRETUDE Spontaneously | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have Sex Without A Condom | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Engage In Anal Sex | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have A Sexual Partner Living With<br>HIV | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Live In Areas With High HIV<br>Prevalence | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Currently Have Or Recently<br>(Within The Past 6 Months) Have<br>Had An Sti Other Than HIV | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Are In Monogamous Relationships | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Inject Drugs | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have Sex With A Person/People<br>Who Inject Drugs | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Experience Stigma Around Using HIV Prevention | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Are Concerned About Taking Pills<br>Every Day | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Experience Stress Or Anxiety Over<br>Adherence Of A Daily Pill Regimen | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have More Chaotic Lifestyles (E.G.,<br>Variable Work Schedules,<br>Frequent Travel, Balancing Work<br>And School) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have More Structured Lifestyles<br>(E.G., Regular Work Hours, Little<br>To No Unplanned Travels) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have Difficulty Planning Or<br>Organizing | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have Stable Income And Stable<br>Housing | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Experience Homelessness Or Are<br>Unstably Housed | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have Psychiatric Comorbidities | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have Sex With Someone Who Has<br>Recently Been In Jail/Prison | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Are Incarcerated, Temporarily<br>Incarcerated, Or Recently Released<br>From Incarcerated | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 8 | Are individuals with specific demographics more appropriate for APRETUDE? | | | | |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 9 | In your opinion, what are | the demographics of the individuals w | ho are appro | priate for APRETUD | E? |
| | | Patients <35 Years Old | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Patients 35-50 Years Old | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Patients >50 Years Old | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Black Transgender Men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Black Transgender Women | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Black Cisgender Women | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Black Cisgender Men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Black Non-Binary Individuals | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Black Men Who Have Sex With<br>Men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | White Transgender Men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | White Transgender Women | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | White Cisgender Women | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | White Cisgender Men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | White Non-Binary Individuals | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | White Men Who Have Sex With Men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Latinx Transgender Men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Latinx Transgender Women | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Latinx Cisgender Women | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Latinx Cisgender Men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Latinx Non-Binary Individuals | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Latinx Men Who Have Sex With Men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other Transgender Men Of Color | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other Transgender Women Of<br>Color | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other Cisgender Women Of Color | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other Cisgender Men Of Color | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other Non-Binary Individuals Of<br>Color | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other Men Who Have Sex With Men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 10 | Has any of the patient | s at this clinic/practice asked for (or about | | ? | I |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 11 | Are you or this clinic/pr | ractice proactively informing patients abo | ut APRETUD | Ε? | |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 12 | How are you or this clir | nic/practice informing patients about APR | ETUDE? | | |
| | | Provision Of Educational Materials | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | During Consultation With Patient | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Through Peer Educators | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Referring Patients To Prep<br>Providers | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Posters In The Clinic/Practice | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Flyers In The Clinic/Practice | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Mentions On The Clinic/Practice's<br>Website | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Mentions On Social Media | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.005 Summary of Experiences with the Acquisition Process (Month 1), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 34 | | rolved in any part of acquisition process to<br>n, claims, sending documents to insurance | | | |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 35 | How will your providers o | or clinic/practice acquire APRETUDE? | | | |
| | | Buy-And-Bill - Purchases<br>Apretude From A Wholesaler<br>Or Specialty Distributor And<br>Bills The Primary Third-Party<br>Payer | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | White Bagging - Submits Prescription To A Specialty Pharmacy Within Viiv's Specialty Pharmacy Network | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | |
| | | Clear Bagging - Internal Pharmacy Maintains Inventory Of The Medication, Processes The Claim, And Delivers The Medication | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 36 | Who in your clinic/practice is responsible for completing the insurance benefits verification process for specialty medications for patients? | | | | |
| | | Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse Practitioner/Physician<br>Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Specialty Pharmacy | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Social Worker/Case Manager | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Front Desk Staff/Scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Dedicated Administrator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Apretude Coordinator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 37 | Have you or your clinic/praction | ce used ViiV Connect previously? | | | |
| | | Yes, I Have Personally Used It | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Yes, The Clinic/Practice Has<br>Used It But I Have Not<br>Personally Used It | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 38 | For each item, please indicate how concerned you would be about each of the following based on your current expectations, understanding and knowledge of ViiV Connect. | | | | |
| | Authorization Wait Times | Extremely Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Understanding Status of<br>Authorization | Extremely Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Not At All Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Extremely Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Amount of paperwork | Extremely Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Clarity on Coverage Approval | Extremely Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Ensuring Medication Comes to Right Place | Extremely Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Potential Loss of Enthusiasm of APRETUDE | Extremely Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Moderately Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Patient Dissatisfy With Clinic<br>Staff | Extremely Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Staff Dissatisfy With<br>Acquisition Proc | Extremely Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Potential Disruption of Clinic<br>Flow | Extremely Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Time-consuming Process | Extremely Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | on Response | | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Inequitable Access for Eligible<br>Patients | Extremely Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Concerned | (XX.X%) | | XX (XX.X%) |
| 39 | "I would recommend ViiV Conne<br>medications." | ect to other providers and clinics/ | practices to | aid in the acquisitic | on of ViiV |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Agree Or Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely Disagree | YY | | XX (XX.X%) |
| | | Completely Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 40 | How helpful or unhelpful do you think each type of support would be to your clinic/practice in using ViiV Connect? | | | | |
| | ViiV Connect Services and<br>Support Info | Not At All Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Acquisition Guides | Not At All Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question Response | | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Billing, Coding and<br>Reimbursement Info | Not At All Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Benefits Verification | Not At All Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Live Support | Not At All Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Video for Patients on What<br>ViiV Connect | Not At All Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | Video for Provider Describe<br>ViiV Connect | Not At All Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Payer/Insurer List Cover Med<br>& Coverage | Not At All Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Patient Info Abt ViiV Connect<br>& Acq Proc | Not At All Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | ViiV Connect Tracker | Not At All Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.101 Summary of Acceptability of Intervention Measure (AIM - APRETUDE) and Feasibility of Intervention Measure (FIM - APRETUDE ) Items (Month 1), N=XX

| Measure | ltem | Total<br>Sample | 1<br>Completely<br>Disagree | 2<br>Disagree | 3 Neither<br>Agree<br>nor<br>Disagree | 4 Agree | 5<br>Completely<br>Agree |
|---|---|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| AIM | 1. The idea of APRETUDE in our clinic/practice meets my approval. | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 2. The idea of APRETUDE in our clinic/practice is appealing to me. | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 3. I like the idea of APRETUDE in our clinic/practice. | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 4. I welcome APRETUDE in our clinic/practice. | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| FIM | APRETUDE seems implementable in our clinic/practice | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 2. APRETUDE seems possible in our clinic/practice | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 3. APRETUDE seems doable in our clinic/practice | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | 4. APRETUDE seems easy to use in our clinic/practice | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |



Table 1.102 Distributional Characteristics of the Acceptability of Intervention Measure (AIM – APRETUDE) (Month 1), N=XX

| AIM – APRETUDE | n | Mean | SD | Median (Q1,<br>Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |


| AIM – APRETUDE | n | Mean | SD | Median (Q1,<br>Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Items | | | | | | | |
| 1. The idea of APRETUDE in our clinic/practice meets my approval. | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 2. The idea of APRETUDE in our clinic/practice is appealing to me. | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 3. I like the idea of APRETUDE in our clinic/practice. | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 4. I welcome APRETUDE in our clinic/practice. | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |

<sup>[1]</sup> Mid-level providers include nurse practitioners and physician assistants.



Table 1.103 Distributional Characteristics of the Feasibility of Intervention Measure (FIM - APRETUDE) (Month 1), N=XX

| FIM - APRETUDE | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Office administrator /clinic administrator/front desk staff/scheduler | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |



| FIM - APRETUDE | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Items | | | | | | | |
| APRETUDE seems implementable in our clinic/practice | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |
| 2. APRETUDE seems possible in our clinic/practice | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |
| 3. APRETUDE seems doable in our clinic/practice | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |
| 4. APRETUDE seems easy to use in our clinic/practice | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |

<sup>[1]</sup> Mid-level providers include nurse practitioners and physician assistants.



Table 1.201 Summary of Acceptability of Intervention Measure (AIM - IMPLEMENTATION SUPPORT) and Feasibility of Intervention Measure (FIM - IMPLEMENTATION SUPPORT) Items (Month 1), N=XX

| | 1001110 (111011011 2)) 11 701 | | | | | | |
|---|---|---|---|---|---|---|---|
| Measure | ltem | Total<br>Sample | 1<br>Completely<br>Disagree | 2<br>Disagree | 3<br>Neither<br>Agree<br>nor<br>Disagree | 4 Agree | 5<br>Completely<br>Agree |
| | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| AIM | 1. The implementation support has met my approval. | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 2. The implementation support was appealing to me. | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. I like the implementation support I have received. | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. I welcome the implementation support I have received. | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| FIM | 1. The implementation support seems implementable in our clinic/practice | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | The implementation support seems possible in our clinic/practice | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. The implementation support seems doable in our clinic/practice | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. The implementation support seems easy to use in our clinic/practice | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |



Table 1.202 Distributional Characteristics of the Acceptability of Intervention Measure (AIM – IMPLEMENTATION SUPPORT) (Month 1), N=XX

| AIM – IMPLEMENTATION SUPPORT | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP<br>educator/PrEP navigator | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Office administrator /clinic<br>administrator/front desk staff/scheduler | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X,<br>X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |



| AIM – IMPLEMENTATION SUPPORT | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Items | | | | | | | |
| 1. The implementation support has met my approval. | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |
| 2. The implementation support was appealing to me. | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |
| 3. I like the implementation support I have received | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |
| 4. I welcome the implementation support I have received. | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |

<sup>[1]</sup> Mid-level providers include nurse practitioners and physician assistants.



Table 1.203 Distributional Characteristics of the Feasibility of Intervention Measure (FIM - IMPLEMENTATION SUPPORT) (Month 1), N=XX

| FIM - IMPLEMENTATION SUPPORT | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |



| FIM - IMPLEMENTATION SUPPORT | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Items | | | | | | | |
| The implementation support seems implementable in our clinic/practice | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |
| 2. The implementation support seems possible in our clinic/practice | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |
| 3. The implementation support seems doable in our clinic/practice | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |
| 4. The implementation support seems easy to use in our clinic/practice | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |

<sup>[1]</sup> Mid-level providers include nurse practitioners and physician assistants.



Table 1.301 Summary of Acceptability of Intervention Measure (AIM - TELEHEALTH) and Feasibility of Intervention Measure (FIM - TELEHEALTH) Items (Month 1), N=XX

| Measure | ltem | Total<br>Sample | 1<br>Completely<br>Disagree | 2<br>Disagree | 3<br>Neither<br>Agree<br>nor<br>Disagree | 4<br>Agree | 5<br>Completely<br>Agree |
|---|---|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| AIM | 1. The idea of telehealth for APRETUDE in our clinic/practice meets my approval. | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 2. The idea of telehealth for APRETUDE in our clinic/practice is appealing to me. | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. I like the idea of telehealth for APRETUDE in our clinic/practice. | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. I welcome telehealth for APRETUDE in our clinic/practice. | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| FIM | 1. Telehealth for APRETUDE seems implementable in our clinic/practice | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 2. Telehealth for APRETUDE seems possible in our clinic/practice | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. Telehealth for APRETUDE seems doable in our clinic/practice | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. Telehealth for APRETUDE seems easy to use in our clinic/practice | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |



Table 1.302 Distributional Characteristics of the Acceptability of Intervention Measure (AIM – TELEHEALTH) (Month 1), N=XX

| AIM – TELEHEALTH | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/oth<br>er | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |



| AIM – TELEHEALTH | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Items | | | | | | | |
| 1. The idea of telehealth for APRETUDE in our clinic/practice meets my approval. | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |
| 2. The idea of telehealth for APRETUDE in our clinic/practice is appealing to me. | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |
| 3. I like the idea of telehealth for APRETUDE in our clinic/practice. | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |
| 4. I welcome telehealth for APRETUDE in our clinic/practice. | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |

<sup>[1]</sup> Mid-level providers include nurse practitioners and physician assistants.



Table 1.303 Distributional Characteristics of the Feasibility of Intervention Measure (FIM - TELEHEALTH) (Month 1), N=XX

| FIM - TELEHEALTH | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case<br>manager/PrEP educator/PrEP<br>navigator | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/o<br>ther | XX | X.XX | X.XXX | X.XX<br>(X.XX,X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |



| FIM - TELEHEALTH | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Items | | | | | | | |
| Telehealth for APRETUDE seems implementable in our clinic/practice | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |
| 2. Telehealth for APRETUDE seems possible in our clinic/practice | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |
| 3. Telehealth for APRETUDE seems doable in our clinic/practice | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |
| 4. Telehealth for APRETUDE seems easy to use in our clinic/practice | XX | X.X | X.XX | X.XX<br>(X.XX,X.XX) | X.X (X, X) | XX (XX.X) | (X.XX,<br>X.XX) |

<sup>[1]</sup> Mid-level providers include nurse practitioners and physician assistants.



Table 1.304 Summary of Feasibility and Acceptability of Telehealth (Month 1), N=XX

| Question | Out the | | Total<br>(N = XX) | Dynamic<br>Implementation<br>(N = XX) | Routine<br>Implementation<br>(N = XX) |
|---|---|---|---|---|---|
| Number<br>19 | Question Does your clinic/practice use any form | Response n of telehealth (i.e., use of electronic information and telecommunication | n (%) | n (%) | n (%) |
| 13 | Does your clinic/practice use any form | Yes | | XX (XX.X%) | VV (VV V0/) |
| | | No No | XX (XX.X%) | | XX (XX.X%) |
| | | 112 123 124 125 125 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 20 | What are the current telehealth service | ces and capabilities of your clinic/practice? | I | | I |
| | | Video Consultation: Using Videoconferencing Technology To Facilitate A Patient Visit With Both Physician And Patient Present At The Same Time. | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Telephone Consultation And Visits | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Remote Monitoring Of Patient Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Online Appointment Scheduling: Ability For Patients To Make<br>Appointments Without Interacting With Staff | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Patient Portal Conversations: Ability For Patients To Send<br>Messages In An Online Portal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | At-Home Testing Services: Providers Order Tests And Send To<br>Patient's Home To Complete | | | |
| | | Sending And Receiving Patient Reported Outcomes Questionnaires (E.G., Quality Of Life, Health Behaviors), Via An Online System | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Online Prescription Refill Requests | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Online Portal For Patients To Access Medical Documents, Such As<br>Visit Summaries And Test Results | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Text Messaging With Patients About Care | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Email Reminders To Patients About Upcoming Visits | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Text Reminders | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Automated Phone Call Reminder | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Staff Phone Call Reminder | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question | | | Total<br>(N = XX) | Dynamic<br>Implementation<br>(N = XX) | Routine<br>Implementation<br>(N = XX) |
|---|---|---|---|---|---|
| Number | Question | Response | n (%) | n (%) | n (%) |
| | | Sending Motivational Reminders To Adhere To Care | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 21 | Overall, how comfortable are you using | g telehealth systems to care for patients? | | | |
| | | Very Comfortable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Comfortable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Comfortable Nor Uncomfortable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Uncomfortable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Uncomfortable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Using The Telehealth Systems Is Not Part Of My Role | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 22 | Why is telehealth not used by your clin | ic/practice? | | | |
| | | Do Not Know How To Use Telehealth | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Telehealth Is Too Expensive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Telehealth Is Too Impersonal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Telehealth Does Not Allow Staff To Do The Necessary Physical Exams | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Concerns About Telehealth Privacy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Lack Of Patient Access To Computers And/Or The Internet | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 23 | How easy or difficult do you think it wo | ould be for your clinic/practice to implement the following modules via | telehealth to pro | vide APRETUDE serv | vices? |
| | Digital Assmt to Patients Before Appt | Very Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Easy Nor Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Online Schedule/Reschedule Cons/Inj<br>Appt | Very Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question | | | Total<br>(N = XX) | Dynamic<br>Implementation<br>(N = XX) | Routine<br>Implementation<br>(N = XX) |
|---|---|---|---|---|---|
| Number | Question | Response | n (%) | n (%) | n (%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Easy Nor Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | HIV Test Service: At Home Testing Kit | Very Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Easy Nor Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | HIV Test Service: Lab Testing | Very Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Easy Nor Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | HIV Test Service: Clinic Appt for Test | Very Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Easy Nor Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Video/VR Consult. for Initial/FU Visits | Very Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Easy Nor Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Insurance/Benefits Verifications | Very Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question | | | Total<br>(N = XX) | Dynamic<br>Implementation<br>(N = XX) | Routine<br>Implementation<br>(N = XX) |
|---|---|---|---|---|---|
| Number | Question | Response | n (%) | | n (%) |
| | | Neither Easy Nor Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Send Oral Lead-in to Patient's Home | Very Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Easy Nor Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Home Health Nurse to Administer Inj | Very Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Easy Nor Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Clinic Appt to Receive Only Injection | Very Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Easy Nor Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Alt Inj Site for Inj Administration | Very Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Easy Nor Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Inj Appt Reminders: Text, Digital,<br>Email | Very Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Neither Easy Nor Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Motiv Rem to Patient Persist on<br>APRETUDE | Very Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Easy Nor Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.401 Summary of Utility of Proposed Implementation Strategies (Month 1), N=XX

| Table 1.401 Summary 0 | | торозов ии | promontano | ii oti ategies ( | | |
|---|---|---|---|---|---|---|
| 24. How useful will the following be in the implementation of APRETUDE into your practice/clinic? | Total<br>Sample<br>n (%) | Not at all<br>useful<br>n (%) | A little useful<br>n (%) | Somewhat<br>useful<br>n (%) | Useful<br>n (%) | Very useful<br>n (%) |
| A. Sexual Health Assessment<br>tool: short assessment sent<br>digitally to patients before their<br>appointment <sup>1</sup> | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| B. Frequently Asked Questions<br>Brochure – designed to answer<br>questions providers may have<br>when implementing APRETUDE<br>in their practice | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| C. Readiness Consideration –<br>checklist that helps providers<br>assess readiness to prescribe<br>APRETUDE in the practice | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| D. Getting Started Overview - guide that provides initiation and administration guidance for the APRETUDE injections, along with some additional helpful resources, including information on the acquisition process | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| 24. How useful will the following be in the implementation of APRETUDE into your practice/clinic? | Total<br>Sample<br>n (%) | Not at all<br>useful<br>n (%) | A little useful<br>n (%) | Somewhat<br>useful<br>n (%) | Useful<br>n (%) | Very useful<br>n (%) |
|---|---|---|---|---|---|---|
| E. Injection Education Video –<br>walks through the process of<br>administering APRETUDE<br>injection | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. Provider Website – location where all materials and videos on APRETUDE for the study are located <sup>2</sup> | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| G. Patient materials (e.g., welcome brochure) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| H. Implementation Guidance<br>Video – guidance on how to<br>implement APRETUDE into the<br>clinic/practice | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| I. Appointment scheduler –<br>planner to help schedule<br>patient's appointment<br>accounting for target injection<br>date | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 24. How useful will the following be in the implementation of APRETUDE into your practice/clinic? | Total<br>Sample<br>n (%) | Not at all<br>useful<br>n (%) | A little useful<br>n (%) | Somewhat<br>useful<br>n (%) | Useful<br>n (%) | Very useful<br>n (%) |
|---|---|---|---|---|---|---|
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| J. Pre-scheduled appointment<br>Guidance – document on how<br>to preschedule appointments <sup>1</sup> | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| K. Designated injection days Guidance – document on how to use designated injections day(s)/specific days for patients to receive injections <sup>1</sup> | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| L. Drop-in Injection Visits<br>Guidance – document on how<br>to provide injection only/drop-in<br>visits <sup>1</sup> | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| M. Providing transportation support to patients to appointments <sup>1</sup> | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| N. One-on-one monthly implementation facilitation calls to help problem solve issues during implementation <sup>1</sup> | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| O. Group implementation facilitation calls to help problem | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 24. How useful will the following be in the implementation of APRETUDE into your practice/clinic? | Total<br>Sample<br>n (%) | Not at all<br>useful<br>n (%) | A little useful<br>n (%) | Somewhat<br>useful<br>n (%) | Useful<br>n (%) | Very useful<br>n (%) |
|---|---|---|---|---|---|---|
| solve issues during<br>implementation with other<br>clinics/practices | | | | | | |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| P. Document on how to discuss sexual health¹ | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Q. PrEP Options Communication tool – infographic to help discuss the pros and cons of PrEP options with patients to help patients decide on a PrEP option <sup>1</sup> | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| R. Information on transgender-<br>friendly care [1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

<sup>[1]</sup> Only SSPs in the Dynamic Implementation were asked this question



Table 1.501 Summary of Perceived Barriers to Delivering APRETUDE to Patients (Month 1), N=XX

| 41. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| A. Patients' ability to keep appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| B. Patients' injection-<br>related pain/soreness | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. Risk of drug resistance for patients not adherent to injections | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D. Cost of APRETUDE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 41. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| E. Keeping a patient engaged and motivated to continue APRETUDE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. Identifying eligible individuals for APRETUDE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| G. Worried that a patient will feel stigmatized if offered APRETUDE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| H. Patients' willingness to<br>travel every 2 months for<br>an injection appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| I. Patient lack of belief in the efficacy of APRETUDE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 41. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.502 Summary of Perceptions of Administering APRETUDE (Month 1), N=XX

| | | | | • | ** | |
|---|---|---|---|---|---|---|
| 42. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
| A. Difficulty of giving the gluteal medial injection | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| B. Understanding how to manage patients who miss an injection dose | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. How to transition patients off of APRETUDE who want to stop taking it (e.g., should other PrEP be offered) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D. Understanding how to use oral PrEP medication for a <u>planned</u> missed injection visit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 42. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| E. Understanding how to restart APRETUDE after a missed injection | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. Managing the oral lead-in<br>phase of APRETUDE before<br>starting injections if needed | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| G. Ability to provide adherence counseling and support, when injection dosing visits are missed | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.503 Summary of Perceived Barriers to Managing Delivery of APRETUDE (Month 1), N=XX

| 43. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| A. Management of scheduling injection appointments every 2 months during correct injection (I.e., dosing) windows | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| B. Management of rescheduling appointments during correct injection (I.e., dosing) windows | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. Ability to schedule/reschedule patients who missed APRETUDE visits within correct injection (I.e., dosing) windows | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D. Ability to identify and flag missed injection visits to providers (in a timely manner) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 43. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | , | , , | , | , , | , | , , |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| E. Ability to manage patients presenting to APRETUDE injection appointments with other care needs that need to be addressed | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. Persistence to follow up with patient on missed appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| G. Provider time to discuss<br>HIV prevention with all<br>eligible patients | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| H. Ability to provide HIV screening as indicated at each injection visit and | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 43. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| provide rapid<br>intervention/follow-up<br>based on results status | | | | | | |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| I. HIV monitoring requirements associated with APRETUDE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.504 Summary of Perceived Resourcing Barriers to Support Delivery of APRETUDE (Month 1), N=XX

| 44. Please indicate how concerned you would be about each of the following potentially being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| A. Staff resourcing to ensure appropriate clinic flow | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| B. Number of exam rooms for injections | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. Clinic staff to administer injections | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 44. Please indicate how concerned you would be about each of the following potentially being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| D. Staff preparation (i.e., education, training, inservices) to implement APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| E. Staff time to provide counseling and support to patients, such as answering questing between visit, keeping patients motivated | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. Staff belief in the efficacy of APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 44. Please indicate how concerned you would be about each of the following potentially being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total | Extremely | Moderately | Somewhat | Slightly | Not at all |
|---|---|---|---|---|---|---|
| | Sample | concerned | concerned | concerned | concerned | concerned |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



 Table 1.505
 Summary of Perceptions of Clinic/Practice Culture and Environment

| 45. How much do you agree or disagree with the following statements about your clinic/practice? | Total<br>Sample<br>n (%) | Completely<br>Disagree<br>n (%) | Disagree<br>n (%) | Neither<br>agree nor<br>disagree<br>n (%) | Agree<br>n (%) | Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|
| A. People at all levels openly talk about what is and isn't working | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| B. Most people in this clinic<br>are willing to change how<br>they do things in response to<br>feedback from others | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. It is hard to get things to change in our clinic | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D. People in this clinic operate as a real team | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | | | | | | |
| Site Volume | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | | | | | | |
| E. Staff members often show signs of stress and strain | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |



| 45. How much do you agree or disagree with the following statements about your clinic/practice? | Total<br>Sample<br>n (%) | Completely<br>Disagree<br>n (%) | Disagree<br>n (%) | Neither<br>agree nor<br>disagree<br>n (%) | Agree<br>n (%) | Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. We regularly take time to<br>consider ways to improve<br>how we do things | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| G. Leadership strongly supports clinic change efforts | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.506 Summary of Barriers to PrEP Provisioning (Month 1), N=XX

| 68. Indicate your level of agreement with the following statements: | Total<br>Sample<br>n (%) | Completely<br>Disagree<br>n (%) | Disagree<br>n (%) | Neither<br>agree nor<br>disagree<br>n (%) | Agree<br>n (%) | Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|
| A. The use of PrEP will cause patients to engage in riskier behaviors | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| B. Providing PrEP endorses the risk behaviors of users | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. Only people who engage in risky behavior need PrEP | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D. Only people with many sexual partners need PrEP | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | | | | | | |
| Site Volume | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | | | | | | |
| E. All sexually active people can benefit from PrEP | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |


| 68. Indicate your level of agreement with the following statements: | Total<br>Sample<br>n (%) | Completely<br>Disagree<br>n (%) | Disagree<br>n (%) | Neither<br>agree nor<br>disagree<br>n (%) | Agree<br>n (%) | Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. Providing PrEP will result<br>in an increase in sexually<br>transmitted diseases among<br>patients | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| G. People do not need PrEP if they act responsibly | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.601 Summary of the Sexual Health Assessment Tool (Month 1), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 25 | Has your clinic/practice started to use the Sexual Health Assessment Tool? | | | | |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 26 | Who in your clinic/prac | tice is or will be responsible for distributing | g the Sexual | Health Assessmen | t tool to patients? |
| | | Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse Practitioner/Physician<br>Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Social Worker/Case Manager | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Front Desk Staff/Scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Peer Educator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 27 | Who in your clinic/practice is or will be responsible for reviewing and discussing the results of the Sexual Health Assessment tool with patients? | | | | |
| | | Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse Practitioner/Physician<br>Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Social Worker/Case Manager | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Front Desk Staff/Scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Peer Educator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The Results Are Or Will Not Be<br>Discussed With Patients | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 28 | How often is your clinic/practice | planning to use the Sexual Health | Assessmer | nt tool with each pa | itient? |
| | | Annually With Each Patient | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | As Needed Based On Patient<br>Behaviors | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | As Needed Based On Patient<br>Demographics | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Before Every Visit With Each<br>Patient | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29 | "Please indicate your level of agreement with the following statements about the Sexual Health Tool." | | | | |
| | The Sexual Health Assessment<br>Tool is/will be easy to<br>implement in my<br>clinic/practice | Completely Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Agree Nor Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | The Sexual Health Assessment<br>Tool is/will be an easy way to<br>identify individuals interested<br>in PrEP | Completely Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Agree Nor Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | The Sexual Health Assessment<br>Tool helps/will help to<br>facilitate conversations about<br>PrEP with patients | Completely Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Agree Nor Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.602 Summary of the PrEP Communication Tool (Month 1), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 30 | Has your clinic/practice sta | arted to use PrEP Options Communicat | ion Tool? | | |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 31 | Who in your clinic/practice | e is or will be responsible for using the | PrEP Option: | s Communication To | ool with patients? |
| | | Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse<br>Practitioner/Physician<br>Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Social Worker/Case<br>Manager | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Front Desk Staff/Scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Peer Educator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 32 | How often is your clinic/practice planning to use PrEP Options Communication Tool with each patient? | | | | |
| | | Annually With Each Patient | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Before Every Visit With<br>Each Patient | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | As Needed Based On<br>Patient Demographics | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | As Needed Based On<br>Patient Behaviors | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 33 | "Please indicate your level of agre<br>Tool" | ement with the following state | ements about | t the PrEP Options ( | Communication |
| | The PrEP Options Communication Tool will be easy to implement in my clinic/practice | Completely Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Agree Nor<br>Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | The PrEP Options Communication Tool will help to facilitate conversations about PrEP with patients | Completely Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Agree Nor<br>Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.701 Summary of the Optional Oral Lead-in Phase of APRETUDE (Month 1), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 62 | What sources of informatio | What sources of information will you draw upon in assessing whether an oral lead-in is needed or not? | | | |
| | | Scientific Literature | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Independent Medical<br>Education | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Data From Viiv/Gsk | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Scientific Conferences | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Clinic Rounds | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Cdc Guidelines | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other Medical Colleagues | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 63 | What are the main factors that will drive your decision to use oral lead-in? | | | | |
| | | The Ability To Assess The<br>Safety/Tolerability Of<br>Apretude In All Patients | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The Ability To Assess The Safety/Tolerability Of Apretude In Patients With A History Of Allergy/Drug Intolerance | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The Availability Of More Data<br>From Clinical Trials Using An<br>Oral Lead-In Phase | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The Ability To Increase Drug<br>Concentration Before Starting<br>The Injections | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Being Cautious With A New<br>Medication | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Providing Patient With<br>Protection Against HIV Until<br>The Injection Arrives | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Patient Request | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 64 | How influential would you sa<br>lead-in phase? | ay the patient's preferences will be | e in the decisio | n of whether or not | to use an oral |
| | | Very Influential | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Influential | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Influential | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Very Influential | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Influential | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 65 | Are you prescribing or plann | ing to prescribe optional oral lead- | in for APRETU | DE prior to the first | injection? |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Yes, For All Patients | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Yes, For Some Patients | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Sure | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 66 | For patients who plan to miss an injection, what protection do you offer or plan on offering them until they receive their next injection? | | | | |
| | | Cabotegravir Oral Tablets | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Tdf/Ftc | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Taf/Ftc | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Provision Of Condoms | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Risk Reduction Education | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | None | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.702 Summary of Study Staff Participants' Injectable Cabotegrevir Experience (Month 1), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 60 | Does your clinic/practice currently administer CABENUVA, the long acting injectable treatment for people with HIV? | | | | |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 61 | How easy or difficult has it be | een to implement CABENUVA in you | ır clinic/pract | tice? | |
| | | Very Easy | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Easy Nor Difficult | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | l Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 67 | "Please rate how appropriate | you believe each setting would be | for administ | ering the APRETUDI | E." |
| | HIV-Specialty Clinic | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Primary Care Clinic/Private<br>Practice | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | • | • | • | • | |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Not At All Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Women's Health<br>Practice/Center | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Community Health Center | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Hospital Outpatient | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Retail Pharmacy | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other Pharmacy | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | At Home/Home-based Bare | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Community Based<br>Organization | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Infusion Center | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | STD/STI Clinic | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | PrEP Clinic | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Department of Health Clinic | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other(s), please specify | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.801 Summary of Perceived Number of APRETUDE Patients Clinic/Practice Can Manage Per Week on an Ongoing Basis (Month 1), N=XX

| 46. How many APRETUDE patients do you think your clinic/practice can manage per week on an ongoing basis? | Total | 0-10 | 11-25 | 26-50 | 51-100 | 101-200 | >200 | I don't |
|---|---|---|---|---|---|---|---|---|
| | Sample | Patients | Patients | Patients | Patients | Patients | Patients | know |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n=xx (%) |
| Total Sample | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



Table 1.802 Distributional Characteristics of Reported Number of People in Clinic Trained and Prepared to Give APRETUDE Injections (Month 1), N=XX

| • | | | | | ** | | | |
|---|---|---|---|---|---|---|---|---|
| 47. Approximately how many people in your clinic are trained and prepared to give APRETUDE injections? | Total<br>Sample<br>n (%) | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum<br>and<br>Maximum) | Missing<br>n (%) | 95% CI for the<br>Mean | l don't<br>know<br>n (%) |
| Total Sample | XX<br>(XX.X) | X.X | X.XX | X.X (X.X,X.X) | XX<br>(XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX<br>(XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX<br>(XX.X) | X.X | X.XX | X.X (X.X,X.X) | XX<br>(XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX<br>(XX.X%) |
| Routine<br>Implementation | XX<br>(XX.X) | X.X | X.XX | X.X (X.X,X.X) | XX<br>(XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX<br>(XX.X%) |
| Site Volume | | | | | | | | |
| High | XX<br>(XX.X) | X.X | X.XX | X.X (X.X,X.X) | XX<br>(XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X) | X.X | X.XX | X.X (X.X,X.X) | XX<br>(XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX<br>(XX.X%) |



Table 1.803 Distributional Characteristics of Estimated Number of Staff Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25 People (Month 1), N=XX

| 48. How much staff in total do you estimate will be needed per week to incorporate APRETUDE into your clinic/practice for approximately 25 people? | Total<br>Sample<br>n (%) | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum<br>and<br>Maximum) | Percent<br>Missing | 95% CI for<br>the Mean | I don't<br>know<br>n (%) |
|---|---|---|---|---|---|---|---|---|---|
| Total Sample | XX<br>(XX.X) | XX<br>(XX.X) | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | XX.X<br>(XX.X,<br>XX.X) | XX (XX.X%) | (X.XXX,<br>X.XXX) | XX<br>(XX.X%) |
| Study Arm | | | | | | | | | |
| Dynamic<br>Implementation | XX<br>(XX.X) | XX<br>(XX.X) | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | XX.X<br>(XX.X,<br>XX.X) | XX (XX.X%) | (X.XXX,<br>X.XXX) | XX<br>(XX.X%) |
| Routine<br>Implementation | XX<br>(XX.X) | XX<br>(XX.X) | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | XX.X<br>(XX.X,<br>XX.X) | XX (XX.X%) | (X.XXX,<br>X.XXX) | XX<br>(XX.X%) |
| Site Volume | | | | | | | | | |
| High | XX<br>(XX.X) | XX<br>(XX.X) | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | XX.X<br>(XX.X,<br>XX.X) | XX (XX.X%) | (X.XXX,<br>X.XXX) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X) | XX<br>(XX.X) | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | XX.X<br>(XX.X,<br>XX.X) | XX (XX.X%) | (X.XXX,<br>X.XXX) | XX<br>(XX.X%) |



Table 1.804 Summary of Estimated Percentage of Staff Time/Full-Time Equivalent Hours

Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25

People (Month 1), N=XX

| 49. How much staff time/full-time equivalent hours (FTE) do you estimate will be needed per week to incorporate APRETUDE into your clinic/practice for approximately 25 people? | Total<br>Sample<br>n (%) | 1-20% FTE<br>or 0.4 -<br>8hrs of<br>staff time<br>n (%) | 21-40% FTE<br>or 8.4 - 16hrs<br>of staff time<br>n (%) | 41-60% FTE<br>or 16.4 - 24<br>hrs of staff<br>time<br>n (%) | 61-80% FTE<br>or 24.4 –<br>32hrs of<br>staff time<br>n (%) | 81-100%<br>FTE or<br>32.4 -<br>40hrs of<br>staff<br>time<br>n (%) | l don't<br>know<br>n (%) |
|---|---|---|---|---|---|---|---|
| Total Sample | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic<br>Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Routine<br>Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 1.805 Summary of Plans to Create New Roles/Positions in Clinic to Coordinate the APRETUDE Program (Month 1), N=XX

| 50. Do you plan to create new role(s)/new position(s) in your clinic to coordinate the APRETUDE program? | Total Sample<br>n (%) | Yes<br>n (%) | No<br>n (%) | Maybe<br>n (%) | I don't<br>know<br>n (%) |
|---|---|---|---|---|---|
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.806 Summary of Number of New Roles/Positions in Clinic to Coordinate the APRETUDE Program (Month 1), N=XX

| 51. How many new role(s)/new position(s) are you planning to create in your clinic to coordinate the APRETUDE program? [1] | Total<br>Sample<br>n (%) | 1<br>n (%) | 2<br>n (%) | 3<br>n (%) | 4<br>n (%) | 5<br>n (%) | More<br>than 5<br>n (%) | I don't<br>know<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| Total Sample | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Routine<br>Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |

<sup>[1]</sup> Only includes SSPs who responded 'yes' or 'maybe' to 'Do you plan to create new role(s)/new position(s) in your clinic to coordinate the APRETUDE program?'



Table 1.807 Summary of How Clinic/Practice Plans to Track Patients on APRETUDE (Month 1), N=XX

| 52. How does your clinic/practice plan to track patients on APRETUDE? | Total<br>Sample<br>n (%) | Use a<br>spreadsheet<br>such as MS<br>Excel<br>n (%) | Assign<br>specific<br>staff to<br>track<br>patients<br>n (%) | Have providers track their own patients n (%) | Create<br>alerts in<br>electronic<br>medical<br>records<br>(EMRs)<br>n (%) | Other<br>[1]<br>n (%) | l don't<br>know<br>n (%) |
|---|---|---|---|---|---|---|---|
| Total Sample | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |

<sup>[1]</sup> Other responses include: xxxxx



Table 1.808 Summary of How Clinic/Practice Responds to Patients who Do Not Show for a Regularly Scheduled Appointment (Month 1), N=XX

| 53. What does your clinic/practice do if a patient does not show for a regularly scheduled appointment? | Total<br>Sample<br>n (%) | Phone the<br>patient to<br>reschedule<br>n (%) | Text the patient to reschedule n (%) | Email the<br>patient to<br>reschedule<br>n (%) | Send the<br>patient a<br>postal<br>letter to<br>reschedule<br>n (%) | Wait until the<br>patient<br>contacts the<br>clinic/practice<br>to reschedule<br>n (%) | Charge<br>the<br>patient<br>a fee<br>for not<br>showing<br>up n (%) | I don't<br>know/not<br>applicable<br>to role<br>n (%) | Other<br>[1]<br>n (%) |
|---|---|---|---|---|---|---|---|---|---|
| Total Sample | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | | | |
| Dynamic | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |

<sup>[1]</sup> Other responses include: xxxxx



Table 1.809 Summary Characteristics of Whether Clinic/Practice has Specific Person in Charge of Following Up on No-Shows (Month 1), N=XX

| 54. Is there a specific person in charge of following up on noshows? | Total Sample<br>n (%) | Yes<br>n (%) | No<br>n (%) | l don't know<br>n (%) |
|---|---|---|---|---|
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.810 Summary of Type of Systems Clinic has in Place to Remind Patients of Upcoming Appointments (Month 1), N=XX

| 55. What type of systems does your clinic have in place to remind patients of an upcoming appointment?[1] | Total<br>Sample<br>n (%) | Phone<br>Call from<br>Staff n<br>(%) | Automated<br>Phone call<br>n (%) | Text<br>Message<br>n (%) | Email<br>n (%) | Postal<br>Mail n<br>(%) | Phone App<br>Notification<br>n (%) | Other<br>[2]<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| Total Sample | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |

<sup>[1]</sup> Responses are not mutually exclusive; participants can select all that apply

<sup>[2]</sup> Other responses included: xxxxx



Table 1.811 Summary of Type of Systems Clinic has in Place to Offer Upcoming Appointments (Month 1), N=XX

| | Total Sample | Study | / Arm | Site Vol | ume |
|---|---|---|---|---|---|
| 56. How do you plan to offer appointments for APRETUDE injections? [1] | | Dynamic<br>Implementatio<br>n | Routine<br>Implementatio<br>n | High | Low |
| | n (%) | n (%) | n (%) | n (%) | n (%) |
| Appointments each day of the week | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Appointments only on certain days of the week | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Appointments spread out over the month | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Injection only appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Allow patients to drop-in for injections on any day without an appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Allow patients to drop-in with little advanced notice (e.g., 24 hour notice) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Allow patients to drop-in on<br>a specific injection day<br>without an appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| After hours appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Appointments each day of the week | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Before hours appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Weekend appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Home nursing appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mobile clinic option | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Alternate site appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Depends on the schedule of the injection nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Depends on the schedule of the APRETUDE provider | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| I don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



Table 1.812 Summary of Implementing APRETUDE in Practice (Month 1), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 57 | Does your clinic/practice currently offer the | ne following types of ap | pointments | to patients for any | of your services? |
| | After Hours | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Before Hours | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Weekend Hours | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Home Nursing | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Mobile Clinic | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Drop-in visits without prior appointment | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Drop-in visits with little advance scheduling | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 58 | How do you feel about implementing APRETUDE at your clinic/practice? | Extremely Positive | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Positive | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Positive | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Positive | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not At All Positive | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 59 | How easy or difficult will it be to implement APRETUDE into your current workflow? | Very Easy | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat Easy | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither Easy Nor<br>Difficult | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 1.901 Distributional Characteristics of Select Study Site Characteristics (Month 1), N=XX

| Question<br>Number | Question | Response | Statistics | Total<br>(N = XX) | Dynamic<br>Implementation<br>(N = XX) | Routine Implementation<br>(N = XX) |
|---|---|---|---|---|---|---|
| 2 | Please estimate | the percentage of your patients with the followi | ng types of insurand | ce/health coverage. | | |
| | % | of Medicare | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| | % | of Medicaid | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| | % | of Federal (VA, TRICARE, IHS) | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| | % | of Private/Commercial Insurance | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X |



| Question<br>Number | Question | Response | Statistics | Total<br>(N = XX) | Dynamic<br>Implementation<br>(N = XX) | Routine Implementation<br>(N = XX) |
|---|---|---|---|---|---|---|
| | | | Q3<br>Maximum | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X |
| | | % of Self-pay | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| | | % of Uninsured | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| | | % of Other | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| 4 | How many l | health care providers (e.g., MD/DO, NP, PA) does the | clinic/practice have | (including both full | -time and part-time)? | |
| | | Insert number | n<br>Mean<br>SD<br>Minimum<br>Q1 | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X |



| Question<br>Number | Question | Response | Statistics | Total<br>(N = XX) | Dynamic<br>Implementation<br>(N = XX) | Routine Implementation<br>(N = XX) |
|---|---|---|---|---|---|---|
| | | | Median | XX.X | XX.X | XX.X |
| | | | Q3 | XX.X | XX.X | XX.X |
| | | | Maximum | | | |
| 6 | Please estimate the total patient population at this clinic/practice | | | | | |
| | | | n | XX | XX | XX |
| | | | Mean | XX.X | XX.X | XX.X |
| | | | SD | XX.XX | XX.XX | XX.XX |
| | | | Minimum | XX.X | XX.X | XX.XX |
| | | Total Pt Population at Clinic/Practice | Q1 | XX.X | XX.X | XX.X |
| | | | Median | XX.X | XX.X | XX.X |
| | | | Q3 | XX.X | XX.X | XX.X |
| | | | Maximum | XX.X | XX.X | XX.X |
| | DI | Please estimate the percentage of the clinic/practice's patient population who are: | | | | |
| 7 | | | | | | |
| | | | n | XX | XX | XX |
| | | | Mean | XX.X | XX.X | XX.X |
| | | 0/ fp ii - 25 y - 011 | SD | XX.XX | XX.XX | XX.XX |
| | | | Minimum | XX.X | XX.X | XX.X |
| | | % of Patients <35 Years Old | Q1 | XX.X | XX.X | XX.X |
| | | | Median | XX.X | XX.X | XX.X |
| | | | Q3 | XX.X | XX.X | XX.X |
| | | | Maximum | XX.X | XX.X | XX.X |
| | | | n | XX | XX | XX |
| | | | Mean | XX<br>XX.X | XX<br>XX.X | XX<br>XX.X |
| | | | SD | XX.XX | XX.XX | XX.XX |
| | | | Minimum | XX.XX | XX.X | XX.X |
| | | % of Patients 35-50 Years Old | Q1 | XX.X | XX.X | XX.X |
| | | | Median | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X |
| | | | Q3 | XX.X | XX.X | XX.X |
| | | | Q3<br>Maximum | XX.X | XX.X | XX.X |
| | | | IVIdXIIIIUIII | | | |
| | | Was f Dation to a FO Verma Old | n | XX | XX | XX |
| | | % of Patients >50 Years Old | Mean | XX.X | XX.X | XX.X |
| | | | | XX.XX | XX.XX | XX.XX |



| Question<br>Number | Question | Response | Statistics | Total<br>(N = XX) | Dynamic<br>Implementation<br>(N = XX) | Routine Implementation<br>(N = XX) |
|---|---|---|---|---|---|---|
| | | | SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| 8 | Please estin | nate the percentage of the clinic/practice's patient po | pulation who are: | | | |
| | | % of Transgender Women | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| | | % of Transgender Men | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3 Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| | | % of Cisgender Heterosexual Men | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| | | % of Cisgender Heterosexual Women | n<br>Mean | XX<br>XX.X | XX<br>XX.X | XX<br>XX.X |



| Question<br>Number | Question | Response | Statistics | Total<br>(N = XX) | Dynamic<br>Implementation<br>(N = XX) | Routine Implementatior<br>(N = XX) |
|---|---|---|---|---|---|---|
| | | | SD<br>Minimum<br>Q1 | XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.XX<br>XX.X<br>XX.X<br>XX.X |
| | | | Median<br>Q3<br>Maximum | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X |
| | | % of Cisgender Men Who Have Sex With Men | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3 | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| | | | Maximum | XX.X | XX.X<br>XX.X | XX.X |
| | | % of Non-binary | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| 9 | Among pati | ients who are transgender men, please estimate the | percentage who are | : | | |
| | | % of Black/African American,Non-Hispanic | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3 | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X |
| | | | Maximum | XX.X | XX.X | XX.X |



| Question<br>Number | Question | Response | Statistics | Total<br>(N = XX) | Dynamic<br>Implementation<br>(N = XX) | Routine Implementation<br>(N = XX) |
|---|---|---|---|---|---|---|
| | | % of White, Non-Hispanic | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| | | % of Latinx/Latino | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| | | % of Other Race/Ethnicity, Non-Hispanic | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| 10 | Among pati | ients who are men who have sex with men, please | estimate the percenta | ge who are: | | |
| | | % of Black/African American,Non-Hispanic | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3 | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.XX<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X |



| Question<br>Number | Question | Response | Statistics | Total<br>(N = XX) | Dynamic<br>Implementation<br>(N = XX) | Routine Implementation<br>(N = XX) |
|---|---|---|---|---|---|---|
| | | | Maximum | | | |
| | | % of White, Non-Hispanic | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| | | % of Latinx/Latino | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| | | % of Other Race/Ethnicity, Non-Hispanic | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| 11 | In the last y | rear, what was the estimated number of HIV-negative | patients seen at yo | ur clinic/practice? | • | |
| | | Estimated HIV-negative Pt seen at Clinic | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X |



| Question<br>Number | Question | Response | Statistics | Total<br>(N = XX) | Dynamic<br>Implementation<br>(N = XX) | Routine Implementation (N = XX) |
|---|---|---|---|---|---|---|
| | | | Q3 | XX.X | XX.X | XX.X |
| | | | Maximum | XX.X | XX.X | XX.X |
| 12 | How many patients would you estimate received oral PrEP at the clinic/practice in the last year? Please provide for entire clinic/practice | | | | | |
| | | | n | XX | XX | XX |
| | | | Mean | XX.X | XX.X | XX.X |
| | | | SD | XX.XX | XX.XX | XX.XX |
| | | | Minimum | XX.X | XX.XX<br>XX.X | XX.X |
| | | HIV PrEP Seeking Persons Clinic See | Q1 | XX.X | XX.X | XX.X |
| | | | Median | XX.X | XX.X | XX.X |
| | | | Q3 | XX.X | XX.X | XX.X |
| | | | | XX.X<br>XX.X | XX.X | XX.X |
| | | | Maximum | 707.77 | 701.71 | 701.71 |
| | | | n<br>Mean | XX | XX | XX |
| | | Estimate Pt Initiated Any PrEP Oral/Inj | SD<br>Minimum<br>Q1 | XX.X<br>XX.XX<br>XX.X | XX.X<br>XX.XX<br>XX.X | XX.X<br>XX.XX<br>XX.X |
| | | Estimate Pt Initiated Any PrEP Oral/Inj | SD<br>Minimum<br>Q1 | XX.XX<br>XX.X<br>XX.X | XX.XX<br>XX.X<br>XX.X | XX.XX<br>XX.X<br>XX.X |
| | | Estimate Pt Initiated Any PrEP Oral/Inj | SD<br>Minimum<br>Q1<br>Median | XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.XX<br>XX.X<br>XX.X<br>XX.X |
| | | Estimate Pt Initiated Any PrEP Oral/Inj | SD<br>Minimum<br>Q1<br>Median<br>Q3 | XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| | | Estimate Pt Initiated Any PrEP Oral/Inj | SD<br>Minimum<br>Q1<br>Median | XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.XX<br>XX.X<br>XX.X<br>XX.X | XX.XX<br>XX.X<br>XX.X<br>XX.X |
| 14 | How many I | Estimate Pt Initiated Any PrEP Oral/Inj<br>HIV PrEP seeking persons did the clinic/practice s | SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| 14 | How many l | | SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |



| Question<br>Number | Question | Response | Statistics | Total<br>(N = XX) | Dynamic<br>Implementation<br>(N = XX) | Routine Implementation<br>(N = XX) |
|---|---|---|---|---|---|---|
| | | Estimate Pt Initiated Any PrEP Oral/Inj | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| 16 | How many patients would you estimate initiated APRETUDE in the last 3 months at the clinic/practice? Please provide for the entire clinic/practice | | | | | |
| | | Estimate Pt Initiated APRETUDE at Clinic | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X |
| 17 | | nts who have been prescribed PrEP at your clinic/prace<br>entire clinic/practice | tice, how many wo | uld you estimate hav | e completed the Sexu | al Health Assessment? Pleaso |
| | | Est. Pt prescribe PrEP/Complete Sex Asmt | n<br>Mean<br>SD<br>Minimum<br>Q1<br>Median<br>Q3<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.X<br>XX.XX<br>XX.X<br>XX.X<br>XX.X<br>XX.X<br>XX.X |



Table 1.902 Summary of Selected Study Site Characteristics (Month 1), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 1 | Which of the following best describes the | e practice setting or affiliation? | | | |
| | | AIDS HEALTHCARE FOUNDATION (AHF) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | COMMUNITY BASED-ORGANIZATION/PROVIDER | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | FEDERALLY QUALIFIED HEALTH CENTER (FQHC) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HOSPITAL - GENERAL, COMMUNITY, DISTRICT<br>GENERAL | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | NON-PROFIT/NOT-FOR-PROFIT ORGANIZATION | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | PRIVATE PRACTICE - HIV SPECIALIST (SUCH AS INFECTIOUS DISEASE OR PRIMARY CARE PHYSICIAN W/ SUB-SPECIALTY IN HIV) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | PRIVATE PRACTICE INTERNAL MEDICINE AND HIV SPECIALIST | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | RESEARCH INSTITUTION - NOT UNIVERSITY-<br>BASED | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | UNIVERSITY OR MEDICAL SCHOOL BASED HOSPITAL/ UNIVERSITY ACADEMIC SETTING | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 3 | Is the practice/clinic located in an Ending | n Ending the Epidemic (ETE) County? | | | |
| | | NO | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | YES | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 5 | What types of clinical staff are at the clin | ic/practice? | | | |
| | | CRC, PATIENT CARE COORDINATOR | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | FRONT DESK STAFF/ SCHEDULER | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | LABORATORY<br>STAFF/TECHNICIAN/PHLEBOTOMIST | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | MEDICAL ASSISTANT | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | MENTAL HEALTH THERAPIST | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | MOBILE TESTING/WELLNESS CLINIC/MOBILE CLINIC | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | NURSE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | NURSE PRACTITIONER/ PHYSICIAN ASSISTANT | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | OFFICE ADMINISTRATOR /CLINIC ADMINISTRATOR | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | PHARMACIST | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | PHYSICIAN | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | PREP EDUCATOR/PREP NAVIGATOR | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | SOCIAL WORKER/CASE MANAGER | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |


## 6 Tables for Month 4/5 Analysis

| Table 2.001 | Demographic Characteristics of New Staff Study Participants (Month 4/5), N=XX | . 107 |
|---|---|---|
| Table 2.002 | Demographic Characteristics of Longitudinal* Staff Study Participants (Month 4/5),<br>N=XX | . 109 |
| Table 2.003 | Characteristics of New Staff Study Participants (Month 4/5), N=XX | . 111 |
| Table 2.004 | Characteristics of Longitudinal* Staff Study Participants (Month 4/5), N=XX | . 113 |
| Table 2.005 | Summary of Confidence with Skills (Month 4/5), N=XX | . 115 |
| Table 2.006 | Summary of Staff Study Participants' Perceptions Regarding APRETUDE (Month 4/5), N=XX | . 117 |
| Table 2.007 | Summary of Experiences with the Acquisition Process (Month 4/5), N=XX | . 119 |
| Table 2.101 | Summary of Acceptability of Intervention Measure (AIM - APRETUDE) and Feasibility of Intervention Measure (FIM - APRETUDE ) Items (Month 4/5), N=XX | . 128 |
| Table 2.102 | Distributional Characteristics of the Acceptability of Intervention Measure (AIM – APRETUDE) (Month 4/5), N=XX | . 130 |
| Table 2.103 | Distributional Characteristics of the Feasibility of Intervention Measure (FIM - APRETUDE) (Month 4/5), N=XX | . 132 |
| Table 2.104 | Changes from Baseline to Acceptability of Intervention Measure (AIM - APRETUDE) and Feasibility of Intervention Measure (FIM - APRETUDE) (Month 4/5), N=XX Error! Bookr not defined. | mark |
| Table 2.105 | Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – APRETUDE) (Month 4/5), N=XX | . 135 |
| Table 2.106 | Mixed-effects Modeling of the Changes from Baseline to Month 4/5 in Acceptability of Intervention Measure (AIM – APRETUDE), N=XX | . 136 |
| Table 2.107 | Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – APRETUDE) (Month 4/5), N=XX | . 137 |
| Table 2.108 | Mixed-effects Modeling of the Changes from Baseline to Month 4/5 in Feasibility of Intervention Measure (FIM – APRETUDE), N=XX | . 138 |
| Table 2.201 | Summary of Acceptability of Intervention Measure (AIM - Implementation Support) and Feasibility of Intervention Measure (FIM - Implementation Support) Items (Month 4/5), N=XX. | . 139 |
| Table 2.202 | Distributional Characteristics of the Acceptability of Intervention Measure (AIM – Implementation Support) (Month 4/5), N=XX | |
| Table 2.203 | Distributional Characteristics of the Feasibility of Intervention Measure (FIM - Implementation Support) (Month 4/5), N=XX | . 143 |
| Table 2.204 | Changes from Baseline for Acceptability of Intervention Measure (AIM - Implementation Support) and Feasibility of Intervention Measure (FIM - Implementation Support) (Month 4/E) Nevy | 145 |
| Table 2.205 | Implementation Support) (Month 4/5), N=XX | . 145<br>146 |



| Table 2.206 | Mixed-effects Modeling of the Changes from Baseline to Month 4/5 in Acceptability of Intervention Measure (AIM – Implementation Support), N=XX | 147 |
|---|---|---|
| Table 2.207 | Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – Implementation Support) (Month 4/5), N=XX | 148 |
| Table 2.208 | Mixed-effects Modeling of the Changes from Baseline to Month 4/5 in Feasibility of Intervention Measure (FIM – Implementation Support), N=XX | 149 |
| Table 2.301 | Summary of Acceptability of Intervention Measure (AIM - Telehealth) and Feasibility of Intervention Measure (FIM - Telehealth ) Items (Month 4/5), N=XX | 150 |
| Table 2.302 | Distributional Characteristics of the Acceptability of Intervention Measure (AIM – Telehealth) (Month 4/5), N=XX | 152 |
| Table 2.303 | Distributional Characteristics of the Feasibility of Intervention Measure (FIM - Telehealth) (Month 4/5), N=XX | 154 |
| Table 2.304 | Changes from Baseline for Acceptability of Intervention Measure (AIM - Telehealth) and Feasibility of Intervention Measure (FIM - Telehealth ) (Month 4/5), N=XX | 156 |
| Table 2.305 | Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – Telehealth) (Month 4/5), N=XX | 157 |
| Table 2.306 | Mixed-effects Modeling of the Changes from Baseline to Month 4/5 in Acceptability of Intervention Measure (AIM – Telehealth), N=XX | 158 |
| Table 2.307 | Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – Telehealth) (Month 4/5), N=XX | 159 |
| Table 2.308 | Mixed-effects Modeling of the Changes from Baseline to Month 4/5 in Feasibility of Intervention Measure (FIM – Telehealth), N=XX | 160 |
| Table 2.309 | Summary of Feasibility and Acceptability of Telehealth (Month 4/5), N=XX | 161 |
| Table 2.310 | Summary of Telehealth Services/Systems Used (Month 4/5), N=XX | 167 |
| Table 2.311 | Summary of Ease of Use of Telehealth Services/Systems Used (Month 4/5), N=XX | 171 |
| Table 2.312 | Summary of Helpfulness of Services/Systems Used (Month 4/5), N=XX | 176 |
| Table 2.313 | Summary of Satisfaction of Services/Systems Used (Month 4/5), N=XX | 181 |
| Table 2.401 | Summary of Utility of Proposed Implementation Strategies (Month 4/5), N=XX | 186 |
| Table 2.501 | Summary of Perceived Barriers to Delivering APRETUDE to Patients (Month 4/5), N=XX | 193 |
| Table 2.502 | Summary of Perceptions of Administering APRETUDE (Month 4/5), N=XX | 202 |
| Table 2.503 | Summary of Perceived Barriers to Managing Delivery of APRETUDE (Month 4/5), N=XX | 209 |
| Table 2.504 | Summary of Perceived Resourcing Barriers to Support Delivery of APRETUDE (Month 4/5), N=XX | 218 |
| Table 2.505 | Summary of Perceptions of Clinic/Practice Culture and Environment (Month 4/5), N=XX | |
| | Summary of Barriers to PrEP Provisioning (Month 4/5), N=XX | |
| | Distributional Characteristics of Barriers to PrEP Provisioning (Month 4/5), N=XX | |
| | Shift from Baseline to Month 4/5 in Summary of Perceived Barriers to Delivering APRETUDE to Patients (Month 4/5), N=XX | |
| Table 2.509 | Shift from Baseline to Month 4/5 in Summary of Perceptions of Administering | |
| | APRETUDE (Month 4/5), N=XX | 231 |



| Table 2.510 | Shift from Baseline to Month 4/5 in Summary of Perceived Barriers to Managing Delivery of APRETUDE (Month 4/5), N=XX | 232 |
|---|---|---|
| Table 2.511 | Shift from Baseline to Month 4/5 in Summary of Perceived Resourcing Barriers to Support Delivery of APRETUDE (Month 4/5), N=XX | 232 |
| Table 2.512 | Shift from Baseline to Month 4/5 in Summary of Perceptions of Clinic/Practice Culture and Environment (Month 4/5), N=XX | 232 |
| Table 2.513 | Shift from Baseline to Month 4/5 in Summary of Barriers to PrEP Provisioning (Month 4/5), N=XX | 233 |
| Table 2.601 | Summary of the Sexual Health Assessment Tool (Month 4/5), N=XX | 234 |
| Table 2.602 | Summary of the PrEP Communication Tool (Month 4/5), N=XX | 237 |
| Table 2.701 | Summary of the Optional Oral Lead-in Phase of APRETUDE (Month 4/5), N=XX | 240 |
| Table 2.801 | Summary of Perceived Number of APRETUDE Patients Clinic/Practice Can Manage Per Week on an Ongoing Basis (Month 4/5), N=XX | 246 |
| Table 2.802 | Distributional Characteristics of People in Clinic Trained and Prepared to Give APRETUDE Injections (Month 4/5), N=XX | 247 |
| Table 2.803 | Distributional Characteristics of Estimated Number of Staff Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25 People (Month 4/5), N=XX | 248 |
| Table 2.804 | Summary of Estimated Percentage of Staff Time/Full-Time Equivalent Hours Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25 People (Month 4/5), N=XX | 249 |
| Table 2.805 | Summary of Plans to Create New Roles/Positions in Clinic to Coordinate the APRETUDE Program (Month 4/5), N=XX | 250 |
| Table 2.806 | Summary of Number of New Roles/Positions in Clinic to Coordinate the APRETUDE Program (Month 4/5), N=XX | 251 |
| Table 2.807 | Summary of How Clinic/Practice Plans to Track Patients on APRETUDE (Month 4/5), N=XX | 252 |
| Table 2.808 | Summary of How Clinic/Practice Responds to Patients who Do Not Show for a Regularly Scheduled Appointment (Month 4/5), N=XX | 253 |
| Table 2.809 | Summary of Whether Clinic/Practice has Specific Person in Charge of Following Up on No-Shows (Month 4/5), N=XX | 254 |
| Table 2.810 | Summary of Type of Systems Clinic has in Place to Remind Patients of Upcoming Appointments (Month 4/5), N=XX | 255 |
| Table 2.811 | Summary of Type of Systems Clinic has in Place to Offer Upcoming Appointments (Month 4/5), N=XX | 256 |
| Table 2.812 | Summary of Implementing APRETUDE in Practice (Month 4/5), N=XX | 258 |
| Table 2.901 | Quarterly Site Reporting. | 260 |



Table 2.001 Demographic Characteristics of New Staff Study Participants (Month 4/5), N=XX

| Question<br>Number | Characteristic | | Study | / Arm |
|---|---|---|---|---|
| | | Total<br>(N=XX) | Dynamic<br>Implementation<br>(N=XX) | Routine<br>Implementation<br>(N=XX) |
| | | n (%) | n (%) | n (%) |
| 88 | Gender | | | |
| | Cisgender Male | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Cisgender Female | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Transgender Man | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Transgender Woman | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Nonbinary | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Gender Queer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other Gender | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I prefer not to answer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 89 | Age (years) | | | |
| | N | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 89 | Age (years), High Volume | | | |
| | N | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 89 | Age (years), Low Volume | | | |
| | N | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 89 | Age | | | |
| | 18-25 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 26-35 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 66-49 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Characteristic | Characteristic | | / Arm |
|---|---|---|---|---|
| | | Total<br>(N=XX) | Dynamic<br>Implementation<br>(N=XX) | Routine<br>Implementation<br>(N=XX) |
| | | n (%) | n (%) | n (%) |
| | 50+ | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 90 | Race | | | |
| | White/Caucasian | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Black | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Asian | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Native American | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Pacific Islander | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Mixed Race | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other Race | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I Prefer not to Answer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 91 | Ethnicity | | | |
| | Hispanic/Latinx | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Non-Hispanic/Latinx | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Prefer not to answer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.002 Demographic Characteristics of Longitudinal\* Staff Study Participants (Month 4/5), N=XX

| 88 Gender XX (XX.X%) XX (XX.XX%) XX (XX.XX%) | Routine plementation (N=XX) n (%) XX (XX.X%) |
|---|---|
| 88 Gender Cisgender Male XX (XX.X%) XX (XX.X%) Cisgender Female XX (XX.X%) XX (XX.X%) Transgender Man XX (XX.X%) XX (XX.X%) Transgender Woman XX (XX.X%) XX (XX.X%) | XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) |
| Cisgender Male XX (XX.X%) XX (XX.X%) Cisgender Female XX (XX.X%) XX (XX.X%) Transgender Man XX (XX.X%) XX (XX.X%) Transgender Woman XX (XX.X%) XX (XX.X%) | XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) |
| Cisgender Female XX (XX.X%) XX (XX.X%) Transgender Man XX (XX.X%) XX (XX.X%) Transgender Woman XX (XX.X%) XX (XX.X%) | XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) |
| Transgender Man XX (XX.X%) XX (XX.X%) Transgender Woman XX (XX.X%) XX (XX.X%) | XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) |
| Transgender Woman XX (XX.X%) XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| | XX (XX.X%)<br>XX (XX.X%) |
| Nonbinary XX (XX.X%) XX (XX.X%) | XX (XX.X%) |
| , | |
| Gender Queer XX (XX.X%) XX (XX.X%) | XX (XX.X%) |
| Other Gender XX (XX.X%) XX (XX.X%) | |
| I prefer not to answer XX (XX.X%) XX (XX.X%) | XX (XX.X%) |
| 89 Age (years) | |
| N XX XX | XX |
| Mean (SD) XX.X (XX.XX) XX.X (XX.XX) X | XX.X (XX.XX) |
| Median XX.X XX.X | XX.X |
| Q1, Q3 XX, XX XX, XX | XX, XX |
| Min-Max XX.X, XX.X XX.X, XX.X | XX.X, XX.X |
| Missing XX (XX.X%) XX (XX.X%) | XX (XX.X%) |
| 89 Age (years), High Volume | |
| N XX XX | XX |
| Mean (SD) XX.X (XX.XX) XX.X (XX.XX) X | XX.X (XX.XX) |
| Median XX.X XX.X | XX.X |
| Q1, Q3 XX, XX XX, XX | XX, XX |
| Min-Max XX.X, XX.X XX.X, XX.X | XX.X, XX.X |
| Missing XX (XX.X%) XX (XX.X%) | XX (XX.X%) |
| 89 Age (years), Low Volume | |
| N XX XX | XX |
| Mean (SD) XX.X (XX.XX) XX.X (XX.XX) X | XX.X (XX.XX) |
| Median XX.X XX.X | XX.X |
| Q1, Q3 XX, XX XX, XX | XX, XX |
| Min-Max XX.X, XX.X XX.X, XX.X | XX.X, XX.X |
| Missing XX (XX.X%) XX (XX.X%) | XX (XX.X%) |
| 89 Age | |
| 18-25 | XX (XX.X%) |
| 26-35 | XX (XX.X%) |



| Question<br>Number | Characteristic | | Study Arm | |
|---|---|---|---|---|
| | | Total<br>(N=XX) | Dynamic<br>Implementation<br>(N=XX) | Routine<br>Implementation<br>(N=XX) |
| | | n (%) | n (%) | n (%) |
| | 66-49 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 50+ | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 90 | Race | | | |
| | White/Caucasian | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Black | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Asian | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Native American | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Pacific Islander | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Mixed Race | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other Race | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | l Prefer not to Answer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 91 | Ethnicity | | | |
| | Hispanic/Latinx | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Non-Hispanic/Latinx | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Prefer not to answer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

<sup>\*</sup> Longitudinal = SSPs who completed any portion of any questionnaire at Baseline and at Month 4/5



Table 2.003 Characteristics of New Staff Study Participants (Month 4/5), N=XX

| Question<br>Number | Characteristic | | Study | / Arm |
|---|---|---|---|---|
| | | Total<br>(N=XX) | Dynamic<br>Implementation<br>(N=XX) | Routine<br>Implementation<br>(N=XX) |
| | | n (%) | n (%) | n (%) |
| 1 | Provider Type | | | |
| | Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Nurse Practitioner | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Physician Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Social worker/case manager | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Office administrator/clinic administrator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Laboratory staff/technician/phlebotomist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Front desk staff/ Scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 2 | Personally Administer Injections | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 3 | Prescribe Medications as part of role | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 4 | Currently Provide PrEP Counseling | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 92 | Specialty | | | |
| | Infectious disease specialist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Internal medicine/ primary care/general doctor/<br>family practitioner | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | HIC Specialist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Immunologist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Women's health/obstetricians and gynecologists | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Endocrinologist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other[2] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 93 | Length of Time practicing Medicine | | | |
| | <1 year | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 1–5 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Characteristic | Characteristic | | |
|---|---|---|---|---|
| | 6–10 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 11-15 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 16-20 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | >21 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

 $\label{eq:constraint} \mbox{[1] Other responses include: } \mbox{xxx}$ 

[2] Other responses include: xxx



Table 2.004 Characteristics of Longitudinal\* Staff Study Participants (Month 4/5), N=XX

| Question<br>Number | Characteristic | | Stud | y Arm |
|---|---|---|---|---|
| | | Total<br>(N=XX) | Dynamic<br>Implementation<br>(N=XX) | Routine<br>Implementation<br>(N=XX) |
| | | n (%) | n (%) | n (%) |
| 1 | Provider Type | | | |
| | Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Nurse Practitioner | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Physician Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Social worker/case manager | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Office administrator/clinic administrator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Laboratory staff/technician/phlebotomist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Front desk staff/ Scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 2 | Personally Administer Injections | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 3 | Prescribe Medications as part of role | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 4 | Currently Provide PrEP Counseling | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 92 | Specialty | | | |
| | Infectious disease specialist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Internal medicine/ primary care/general doctor/<br>family practitioner | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | HIC Specialist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Immunologist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Women's health/obstetricians and gynecologists | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Endocrinologist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other[2] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 93 | Length of Time practicing Medicine | | | |
| | <1 year | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 1–5 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Characteristic | | Stud | y Arm |
|--------------------|----------------|------------|------------|------------|
| | 6–10 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 11-15 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 16-20 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | >21 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

<sup>\*</sup> Longitudinal = SSPs who completed any portion of any questionnaire at Baseline and at Month 4/5

<sup>[1]</sup> Other responses include: xxx

<sup>[2]</sup> Other responses include: xxx



Table 2.005 Summary of Confidence with Skills (Month 4/5), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 5 | "Please rate your level of confidence for each skill listed." | | | | |
| | Talking to Patient About Sexual<br>History | Not At All Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Bit Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My<br>Role | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Screening a patient to determine whether they are an appropriate candidate for PrEP | Not At All Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Bit Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My<br>Role | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Answering Patient's Questions<br>About PrEP | Not At All Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Bit Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My<br>Role | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Suggesting PrEP to a Patient | Not At All Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Bit Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My<br>Role | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | Counseling a patient about using other methods of protection (e.g., condoms) while on PrEP | Not At All Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Bit Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My<br>Role | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Monitoring a Patient on PrEP | Not At All Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Bit Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Confident | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My<br>Role | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.006 Summary of Staff Study Participants' Perceptions Regarding APRETUDE (Month 4/5), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 6 | In your opinion, APRETU | DE is appropriate for which individuals? | | | |
| | | are sexually active | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have been sexually active with 1 or more partners in the last 6 months | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | are currently adherent on daily oral PrEP | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | are non-adherent on daily oral<br>PrEP | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | use PrEP on demand (i.e., event-<br>based PrEP, PrEP 2-1-1) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | could benefit from PrEP but do<br>not want to use daily PrEP | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have previously used and discontinued daily PrEP | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | feel stigmatized about taking oral<br>PrEP | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | request APRETUDE spontaneously | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have sex without a condom | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | engage in anal sex | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have a sexual partner living with HIV | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | live in areas with high HIV prevalence | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | currently have or recently (within<br>the past 6 months) have had an<br>STI other than HIV | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | are in monogamous relationships | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | inject drugs | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have sex with a person/people who inject drugs | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | experience stigma around using HIV prevention | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | are concerned about taking pills every day | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | experience stress or anxiety over adherence of a daily pill regimen | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have more chaotic lifestyles (e.g.,<br>variable work schedules,<br>frequent travel, balancing work<br>and school) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | have more structured lifestyles<br>(e.g., regular work hours, little to<br>no unplanned travels) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have difficulty planning or organizing | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have stable income and stable housing | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | experience homelessness or are unstably housed | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have psychiatric comorbidities | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have sex with someone who has recently been in jail/prison | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | are incarcerated, temporarily incarcerated, or recently released from incarcerated | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 7 | Has any of the patients at | this clinic/practice asked for (or about) | APRETUDE? | ) | |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 8 | Are you or this clinic/prac | tice proactively informing patients abo | ut APRETUDI | E? | |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 9 | How are you or this clinic, | /practice informing patients about APR | ETUDE? | | |
| | | Provision of educational materials | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | During consultation with patient | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Through peer educators | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Referring patients to PrEP providers | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Posters in the clinic/practice | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Flyers in the clinic/practice | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Mentions on the clinic/practice's website | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Mentions on social media | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.007 Summary of Experiences with the Acquisition Process (Month 4/5), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 39 | Are you involved in any of part of the benefits verification and acquisition process for APRETUDE, such as completing enrollment forms, sending documents to insurance companies, purchasing APRETUDE? | | | | |
| | | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 40 | Is your clinic/practice | using ViiV Connect to acquire APRETUDE? | | | |
| | | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 41 | Do You Personally Use | ViiV Connect? | 1 | | |
| | | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 42 | How are your provide | rs or clinic/practice acquiring APRETUDE? | | | |
| | | Buy-and-Bill - purchases<br>APRETUDE from a wholesaler<br>or specialty distributor and<br>bills the primary third-party<br>payer. | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | White Bagging - submits prescription to a specialty pharmacy within ViiV's specialty pharmacy network and the specialty pharmacy processes the claim and ships APRETUDE for administration. | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Clear Bagging - internal pharmacy maintains inventory of the medication, processes the claim, and delivers the medication. | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 43 | Who in your clinic/pra<br>APRETUDE? | ctice is primarily responsible for completir | ng the insuranc | e benefits verificati | on process for |
| | | Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse practitioner/physician assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Speciality pharmacy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Medical assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Social worker/case manager | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Front desk staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Dedicated administrator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | APRETUDE coordinator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 44 | On average, how long d | oes it take to complete the APRETUDE e | nrollment form | 1? | |
| | | 1-5 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 6-10 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 11-15 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 16-20 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 21-25 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 26-30 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 31+ minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I have not completed this form | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 45 | On average, how long has it taken to receive confirmation of benefits verification for APRETUDE? | | | | |
| | | 1-2 days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 3-4 days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 5-6 days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 7-8 days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 9-10 days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 11-15 days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 16-20 days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 20+ days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 46 | On average, how long h | as it taken for patients to receive APRET | UDE from the p | oint of benefits ver | ification? |
| | | 1-2 days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 3-4 days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 5-6 days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 7-8 days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 9-10 days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 11-15 days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 16-20 days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 20+ days | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 47 | "For each item, please indicate how concerned you are about each of the following based on your current expectations, understanding and knowledge of ViiV Connect." | | | | |
| | Authorization wait times | Extremely concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Understanding status of authorization | Extremely concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Understanding how to seek assistance | Extremely concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Amount of paperwork | Extremely concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Clarity on coverage approval | Extremely concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Ensuring medication comes to the right place (e.g., clinic/practice, pharmacy) | Extremely concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Potential loss of enthusiasm for APRETUDE by patients | Extremely concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Potential patient<br>dissatisfaction with clinic staff | Extremely concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Staff dissatisfaction with the acquisition process | Extremely concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Potential disruption of clinic flow | Extremely concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Time-consuming process | Extremely concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Inequitable access for eligible patients | Extremely concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 48 | "Please indicate how much | you agree or disagree with eac | h of the follo | wing statements. | " |
| | I understand how to use ViiV<br>Connect (skip applicable if<br>Q41=yes) | Completely disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Completely agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I understand how to<br>complete the APRETUDE<br>forms in ViiV Connect (skip<br>applicable if Q41=yes) | Completely disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Completing the benefits enrollment forms is easy | Completely disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | The live support for ViiV<br>Connect is helpful | Completely disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I am knowledgeable about<br>the patient savings card for<br>APRETUDE for patients | Completely disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | The benefits verification process of ViiV Connect is time consuming (RC) (skip applicable if Q41=yes) | Completely disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I am satisfied with the benefits verification process | Completely disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | It has been easy to acquire<br>APRETUDE for patients | Completely disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I know what to do if I am<br>having trouble acquiring<br>APRETUDE for patients | Completely disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I am knowledgeable about<br>the patient assistance<br>program for APRETUDE | Completely disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 49 | How helpful or unhelpful has each type of support been to your clinic/practice in using ViiV Connect?" | | | | |
| | ViiV Connect Services and<br>Support information (e.g.,<br>ViiV Connect Brochure,<br>Provider Portal Brochure) | Not at all helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | ViiV Connect Enrollment information (annotated enrollment forms, enrollment form) | Not at all helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Did not use it | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Acquisition Guides (e.g., ordering guide, buy and bill checklist, specialty pharmacy checklist) | Not at all helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Billing, Coding and reimbursement information (e.g., prior authorization checklist, reimbursement guide) | Not at all helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Benefits Verification –<br>understanding summary of<br>benefits (illustrated form<br>highlights patient benefit<br>summary and how to read it) | Not at all helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Live support (e.g., access coordinators) | Not at all helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Video for patients on what is<br>ViiV Connect (DI) | Not at all helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | A video for providers<br>describing what is ViiV<br>Connect (DI) | Not at all helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Patient informational material about ViiV Connect and the acquisition process | Not at all helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Medication Acquisition Tracker – web-based tool to track patients' benefits acquisition journey from enrollment to medication receipt at the clinic/practice (DI) | Not at all helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | APRETUDE Payer Information found on the PILLAR Spot: spreadsheet updated on a weekly basis and gives providers information on which payers are covering APRETUDE and under what type of benefit | Not at all helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Very helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 50 | How helpful or unhelpful has re<br>began has been to your clinic/p | ceiving the list of payers/insurers ractice? | who cover the | e medication and w | hen coverage |
| | | Not at all helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 51 | I would recommend ViiV Conne<br>medications. | ect to other providers and clinics/p | oractices to aid | in the acquisition o | of ViiV |
| | | Completely agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely Disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.101 Summary of Acceptability of Intervention Measure (AIM - APRETUDE) and Feasibility of Intervention Measure (FIM - APRETUDE ) Items (Month 4/5), N=XX

| Measure | ltem | Study Arm | Total<br>Sample | 1<br>Completely<br>Disagree | 2<br>Disagree | 3<br>Neither<br>Agree<br>nor<br>Disagree | 4<br>Agree | 5<br>Completel<br>y Agree |
|---|---|---|---|---|---|---|---|---|
| | 4 4 9 9 5 7 4 9 5 1 | l | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| AIM | <ol> <li>APRETUDE in our clinic/practice meets my approval.</li> </ol> | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 2. APRETUDE in our clinic/practice is appealing to me. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. I like APRETUDE in our clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. I welcome<br>APRETUDE in our<br>clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| FIM | 1. APRETUDE seems implementable in our clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 2.APRETUDE seems<br>possible in our<br>clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |



| Measure | ltem | Study Arm | Total<br>Sample | 1<br>Completely<br>Disagree | 2<br>Disagree | 3<br>Neither<br>Agree<br>nor<br>Disagree | 4<br>Agree | 5<br>Completel<br>y Agree |
|---|---|---|---|---|---|---|---|---|
| | | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | | Implementation | | | | | | |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. APRETUDE seems<br>doable in our<br>clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. APRETUDE seems<br>easy to use in our<br>clinic/practice | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |



Table 2.102 Distributional Characteristics of the Acceptability of Intervention Measure (AIM – APRETUDE) (Month 4/5), N=XX

| AIM – APRETUDE | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXX | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXX | | | | | |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |



| AIM – APRETUDE | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% Cl<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Items | | | | | | | |
| 1. APRETUDE in our clinic/practice meets my approval. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 2. APRETUDE in our clinic/practice is appealing to me. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 3. I like APRETUDE in our clinic/practice. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 4. I welcome APRETUDE in our clinic/practice. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |

<sup>[1]</sup> Mid-level providers include nurse practitioners and physician assistants.



Table 2.103 Distributional Characteristics of the Feasibility of Intervention Measure (FIM - APRETUDE) (Month 4/5), N=XX

| FIM - APRETUDE | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXX | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXX | | | | | |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |



| FIM - APRETUDE | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% Cl<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Items | | | | | | | |
| 1. APRETUDE seems implementable in our clinic/practice. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 2.APRETUDE seems possible in our clinic/practice. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 3. APRETUDE seems doable in our clinic/practice. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 4. APRETUDE seems easy to use in our clinic/practice | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |

<sup>[1]</sup> Mid-level providers include nurse practitioners and physician assistants.



Table 2.104 Changes from Baseline to Acceptability of Intervention Measure (AIM - APRETUDE) and Feasibility of Intervention Measure (FIM - APRETUDE) (Month 4/5), N=XX

| Measure | Study Arm | n | Mean | SD | Median (Q1, Q3) | Observed Range<br>(min, max) | Missing<br>n (%) | 95% CI<br>for the Mean |
|---|---|---|---|---|---|---|---|---|
| AIM - APRETUDE Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| AIM - APRETUDE Month 4/5 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| AIM - APRETUDE Change from Baseline to<br>Month 4/5 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| FIM - APRETUDE Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| FIM - APRETUDE Month 4/5 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| FIM - APRETUDE Change from Baseline to<br>Month 4/5 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |



Table 2.105 Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – APRETUDE) (Month 4/5), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 2.106 Mixed-effects Modeling of the Changes from Baseline to Month 4/5 in Acceptability of Intervention Measure (AIM – APRETUDE), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 2.107 Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – APRETUDE) (Month 4/5), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 2.108 Mixed-effects Modeling of the Changes from Baseline to Month 4/5 in Feasibility of Intervention Measure (FIM – APRETUDE), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 2.201 Summary of Acceptability of Intervention Measure (AIM - Implementation Support) and Feasibility of Intervention Measure (FIM - Implementation Support) Items (Month 4/5), N=XX

| Measure | ltem | Study Arm | Total<br>Sample<br>n (%) | 1<br>Completely<br>Disagree<br>n (%) | 2<br>Disagree<br>n (%) | 3<br>Neither<br>Agree<br>nor<br>Disagree<br>n (%) | 4<br>Agree<br>n (%) | 5<br>Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| | 1. The implementation | | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) |
| AIM | support has met my approval. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 2. The implementation support was appealing to me. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. I like the implementation support I have received. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. I welcome the implementation support I have received. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| FIM | The implementation support seems implementable in our clinic/practice | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |


| Measure | ltem | Study Arm | Total<br>Sample<br>n (%) | 1<br>Completely<br>Disagree<br>n (%) | 2<br>Disagree<br>n (%) | 3<br>Neither<br>Agree<br>nor<br>Disagree<br>n (%) | 4<br>Agree<br>n (%) | 5<br>Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| | 2. The implementation support seems possible in our clinic/practice | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. The implementation support seems doable in our clinic/practice | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. The implementation support seems easy to use in our clinic/practice | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |



Table 2.202 Distributional Characteristics of the Acceptability of Intervention Measure (AIM – Implementation Support) (Month 4/5), N=XX

| | 7. | | | Median | Observed<br>Range | Missing | 95% CI |
|---|---|---|---|---|---|---|---|
| AIM – Implementation Support | n | Mean | SD | (Q1, Q3) | (Minimum,<br>Maximum) | n (%) | for the<br>Mean |
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test | | XX.XX | | | | | |
| Degrees of Freedom<br>P-Value | | 0.XXXX | | | | | |
| Site Volume | | 0.7777 | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test | | XX.XX | | | | | |
| Degrees of Freedom | | XX | | | | | |
| P-Value | | 0.XXXX | | | | | |
| Clinic Type | | | | X.XX (X.XX, | | XX | (X.XXX, |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | (XX.X) | X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |



| AIM – Implementation Support | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Items | | | | | | | |
| The implementation support has met my approval. | XX | X.X | X.XX | X.X (X.X,<br>X.X) | X (X, X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |
| 2. The implementation support was appealing to me. | XX | X.X | X.XX | X.X (X.X,<br>X.X) | X (X, X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |
| 3. I like the implementation support I have received. | XX | X.X | X.XX | X.X (X.X,<br>X.X) | X (X, X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |
| 4. I welcome the implementation support I have received. | XX | X.X | X.XX | X.X (X.X,<br>X.X) | X (X, X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |

<sup>[1]</sup> Mid-level providers include nurse practitioners and physician assistants.



Table 2.203 Distributional Characteristics of the Feasibility of Intervention Measure (FIM - Implementation Support) (Month 4/5), N=XX

| | 1.1 | | | | | | |
|---|---|---|---|---|---|---|---|
| FIM - Implementation Support | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | XX.XX<br>XX<br>0.XXXX | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | XX.XX<br>XX<br>0.XXXX | | | | | |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |



| FIM - Implementation Support | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Items | | | | | | | |
| The implementation support seems implementable in our clinic/practice | XX | X.X | X.XX | X.X (X.X, X.X) | X (X.X, X.X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 2. The implementation support seems possible in our clinic/practice | XX | X.X | X.XX | X.X (X.X, X.X) | X (X.X, X.X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 3. The implementation support seems doable in our clinic/practice | XX | X.X | X.XX | X.X (X.X, X.X) | X (X.X, X.X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 4. The implementation support seems easy to use in our clinic/practice | XX | X.X | X.XX | X.X (X.X, X.X) | X (X.X, X.X) | XX<br>(XX.X) | (X.XX, X.XX) |



Table 2.204 Changes from Baseline for Acceptability of Intervention Measure (AIM - Implementation Support) and Feasibility of Intervention Measure (FIM - Implementation Support) (Month 4/5), N=XX

| Measure | Study Arm | n | Mean | SD | Median (Q1, Q3) | Observed Range<br>(min, max) | Missing<br>n (%) | 95% CI<br>for the Mean |
|---|---|---|---|---|---|---|---|---|
| AIM - Implementation Support Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| AIM – Implementation Support Month 4/5 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| AIM - Implementation Support Change from Baseline to Month 4/5 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| FIM - Implementation Support Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| FIM - Implementation Support Month 4/5 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| FIM - Implementation Support Change from Baseline to Month 4/5 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |



Table 2.205 Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – Implementation Support) (Month 4/5), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 2.206 Mixed-effects Modeling of the Changes from Baseline to Month 4/5 in Acceptability of Intervention Measure (AIM – Implementation Support), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 2.207 Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – Implementation Support) (Month 4/5), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 2.208 Mixed-effects Modeling of the Changes from Baseline to Month 4/5 in Feasibility of Intervention Measure (FIM – Implementation Support), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 2.301 Summary of Acceptability of Intervention Measure (AIM - Telehealth) and Feasibility of Intervention Measure (FIM - Telehealth) Items (Month 4/5), N=XX

| | | i intervention measa | ( | referredit | | | | |
|---|---|---|---|---|---|---|---|---|
| Measure | ltem | Study Arm | Total<br>Sample | 1<br>Completely<br>Disagree | 2<br>Disagree | 3<br>Neither<br>Agree<br>nor<br>Disagree | 4<br>Agree | 5<br>Completely<br>Agree |
| | | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| AIM | 1. Telehealth for APRETUDE delivery in our clinic/practice meets my approval. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 2. Telehealth for APRETUDE delivery in our clinic/practice is appealing to me. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. I like using<br>telehealth for<br>APRETUDE<br>delivery in our<br>clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. I welcome<br>telehealth for<br>APRETUDE<br>delivery in our<br>clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| FIM | 1. Telehealth<br>for APRETUDE<br>delivery seems<br>implementable | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |



| Measure | ltem | Study Arm | Total<br>Sample | 1<br>Completely<br>Disagree | 2<br>Disagree | 3<br>Neither<br>Agree<br>nor<br>Disagree | 4<br>Agree | 5<br>Completely<br>Agree |
|---|---|---|---|---|---|---|---|---|
| | | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | in our<br>clinic/practice. | | | | | | | |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 2. Telehealth<br>for APRETUDE<br>delivery seems<br>possible in our<br>clinic/practice | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. Telehealth<br>for APRETUDE<br>delivery seems<br>doable in our<br>clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. Telehealth for APRETUDE delivery seems easy to use in our clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |



Table 2.302 Distributional Characteristics of the Acceptability of Intervention Measure (AIM – Telehealth) (Month 4/5), N=XX

| AIM – TELEHEALTH | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXX | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXX | | | | | |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |



| AIM – TELEHEALTH | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% Cl<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Items | | | | | | | |
| 1. Telehealth for APRETUDE in our clinic/practice meets my approval. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 2. Telehealth for APRETUDE in our clinic/practice is appealing to me. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 3. I like using telehealth for APRETUDE in our clinic/practice. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 4. I welcome telehealth for APRETUDE in our clinic/practice. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |

<sup>[1]</sup> Mid-level providers include nurse practitioners and physician assistants.



Table 2.303 Distributional Characteristics of the Feasibility of Intervention Measure (FIM - Telehealth) (Month 4/5), N=XX

| | | | | | Observed | d 05% SI | |
|---|---|---|---|---|---|---|---|
| FIM - TELEHEALTH | n | Mean | SD | Median<br>(Q1, Q3) | Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXX | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXX | | | | | |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |



| FIM - TELEHEALTH | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Items | | | | | | | |
| 1. Telehealth for APRETUDE seems implementable in our clinic/practice | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 2. Telehealth for APRETUDE seems possible in our clinic/practice | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 3. Telehealth for APRETUDE seems doable in our clinic/practice | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 4. Telehealth for APRETUDE seems easy to use in our clinic/practice | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |



Table 2.304 Changes from Baseline for Acceptability of Intervention Measure (AIM - Telehealth) and Feasibility of Intervention Measure (FIM - Telehealth ) (Month 4/5), N=XX

| Measure | Study Arm | n | Mean | SD | Median (Q1, Q3) | Observed Range<br>(min, max) | Missing<br>n (%) | 95% CI<br>for the Mean |
|---|---|---|---|---|---|---|---|---|
| AIM - Telehealth Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| AIM - Telehealth Month 4/5 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| AIM - Telehealth Change from Baseline to<br>Month 4/5 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| FIM - Telehealth Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| FIM - Telehealth Month 4/5 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| FIM - Telehealth Change from Baseline to<br>Month 4/5 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | X (X.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |



Table 2.305 Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – Telehealth) (Month 4/5), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 2.306 Mixed-effects Modeling of the Changes from Baseline to Month 4/5 in Acceptability of Intervention Measure (AIM – Telehealth), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 2.307 Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – Telehealth) (Month 4/5), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | τ | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 2.308 Mixed-effects Modeling of the Changes from Baseline to Month 4/5 in Feasibility of Intervention Measure (FIM – Telehealth), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | τ | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ²) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 2.309 Summary of Feasibility and Acceptability of Telehealth (Month 4/5), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 14 | Does your clinic/practice use | any form of telehealth for APRE | TUDE delivery? | | |
| | | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 17 | What telehealth services does your clinic/practice provide for APRETUDE? | | | | |
| | | Video consultation: using videoconferencing technology to facilitate a patient visit with both physician and patient present at the same time. | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Telephone consultation and visits | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Remote monitoring of patient health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Online appointment scheduling: ability for patients to make appointments without interacting with staff | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Patient portal conversations: ability for patients to send messages in an online portal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | At-home testing services: providers order tests and send to patient's home to complete | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sending and receiving patient reported outcomes questionnaires (e.g., quality of life, health behaviors), via an online system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Online prescription refill requests | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Online portal for patients<br>to access medical<br>documents, such as visit<br>summaries and test results | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Text messaging with patients about care | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Email reminders to patients about upcoming visits | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Text reminders | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Automated phone call reminder | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Staff phone call reminder | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sending motivational reminders to help patients persist on APRETUDE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sending cabotegravir oral lead in to patient's home | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Insurance/benefits verification | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 18 | "How easy or difficult is it to<br>patients?" | o use the following telehealth syst | ems to provide | APRETUDE services | to your |
| | Video consultation | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Telephone consultation | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Remote monitoring of patients | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Online appointment scheduling | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Patient portal conversations:<br>ability for patients to send<br>messages to providers | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | At-home testing services | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Send and receiving patient reported outcomes questionnaires (e.g., quality of life, health behaviors), via an online system | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Online prescription refills | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Online portal for patients to access medical documents, such as visit summaries and test results | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Text messaging with patients about care | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Email reminders to patient about upcoming visits | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Text reminders | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Automated phone call reminders | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Staff phone call reminder | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Sending motivational reminders to help patients persist on APRETUDE | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Sending cabotegravir oral lead in to patient's home | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Insurance/benefits verification | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 19 | In the last 6 months, what pr consults, video)? | oportion of your APRETUDE visit | s would you est | imate were via tele | health (e.g., tele- |
| | | None (0%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Few (1-30%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Some (31-65%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Most (66%-99%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All (100%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 20 | Why is telehealth not used b | y your clinic/practice? | | | |
| | | Do not know how to use telehealth | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Telehealth is too expensive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Telehealth is too impersonal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Telehealth does not allow<br>staff to do the necessary<br>physical exams | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Concerns about telehealth privacy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Lack of patient access to computers and/or the internet | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.310 Summary of Telehealth Services/Systems Used (Month 4/5), N=XX

| | | <u>*</u> | | | |
|---|---|---|---|---|---|
| 21. Which of the following telehealth services/systems is your clinic/practice using to deliver APRETUDE during the PILLAR study? A. Online system for | Total<br>Sample<br>n (%) | Yes, my clinic's<br>service/system<br>n (%) | Yes,<br>services/systems<br>offered through<br>PILLAR study<br>n (%) | No<br>n (%) | l don't<br>know<br>n (%) |
| scheduling/rescheduling consultations and injection appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Study Arm | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | |
| University/Academia/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Social worker/case manager/PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Laboratory<br>staff/technician/phlebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| B. Video/virtual consultations for initial and follow-up visits | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Study Arm | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | |
| University/Academia/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| 21. Which of the following telehealth services/systems is your clinic/practice using to deliver APRETUDE during the PILLAR study? | Total<br>Sample<br>n (%) | Yes, my clinic's<br>service/system<br>n (%) | Yes,<br>services/systems<br>offered through<br>PILLAR study<br>n (%) | No<br>n (%) | l don't<br>know<br>n (%) |
|---|---|---|---|---|---|
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. Injection Administration: home health nurse to administer injection | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | |
| University/Academia/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 21. Which of the following telehealth services/systems is your clinic/practice using to deliver APRETUDE during the PILLAR study? | Total<br>Sample<br>n (%) | Yes, my clinic's<br>service/system<br>n (%) | Yes,<br>services/systems<br>offered through<br>PILLAR study<br>n (%) | No<br>n (%) | l don't<br>know<br>n (%) |
|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D. Injection appointment reminders: text, digital, email | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | |
| University/Academia/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| E. HIV testing services: at home nurse testing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 21. Which of the following telehealth services/systems is your clinic/practice using to deliver APRETUDE during the PILLAR study? | Total<br>Sample<br>n (%) | Yes, my clinic's<br>service/system<br>n (%) | Yes,<br>services/systems<br>offered through<br>PILLAR study<br>n (%) | No<br>n (%) | l don't<br>know<br>n (%) |
|---|---|---|---|---|---|
| Clinic Type | | | | | |
| University/Academia/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.311 Summary of Ease of Use of Telehealth Services/Systems Used (Month 4/5), N=XX

| 22. How easy or difficult has each of the telehealth services/systems been for your clinic/practice to implement for the delivery of APRETUDE? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| A. Online system for scheduling/rescheduling consultations and injection appointments | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



| 22. How easy or difficult has each of the telehealth services/systems been for your clinic/practice to implement for the delivery of APRETUDE? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| B. Video/virtual consultations for initial and follow-up visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| C. Injection Administration: home health nurse to administer injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |



| 22. How easy or difficult has each of<br>the telehealth services/systems been<br>for your clinic/practice to implement<br>for the delivery of APRETUDE? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| D. Injection appointment reminders: text, digital, email | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



| 22. How easy or difficult has each of the telehealth services/systems been for your clinic/practice to implement for the delivery of APRETUDE? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | , | , | | , | | | , , |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| E. HIV testing services: at home nurse testing | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |



| 22. How easy or difficult has each of<br>the telehealth services/systems been<br>for your clinic/practice to implement<br>for the delivery of APRETUDE? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |


Table 2.312 Summary of Helpfulness of Services/Systems Used (Month 4/5), N=XX

| 23. How helpful or unhelpful has each of the telehealth services/systems been to the delivery of APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| A. Online system for scheduling/rescheduling consultations and injection appointments | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



| 23. How helpful or unhelpful has each of the telehealth services/systems been to the delivery of APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| B. Video/virtual consultations for initial and follow-up visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| C. Injection Administration: home health nurse to administer injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |



| 23. How helpful or unhelpful has each of the telehealth services/systems been to the delivery of APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| D. Injection appointment reminders: text, digital, email | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



| 23. How helpful or unhelpful has each of the telehealth services/systems been to the delivery of APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| E. HIV testing services: at home nurse testing | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |



| 23. How helpful or unhelpful has each of the telehealth services/systems been to the delivery of APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



Table 2.313 Summary of Satisfaction of Services/Systems Used (Month 4/5), N=XX

| 24. How satisfied or dissatisfied have you been with each of the telehealth services/systems for delivering APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>satisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Neither<br>satisfied<br>nor<br>dissatisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Very<br>satisfied<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| A. Online system for scheduling/rescheduling consultations and injection appointments | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |



| 24. How satisfied or dissatisfied have you been with each of the telehealth services/systems for delivering APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>satisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Neither<br>satisfied<br>nor<br>dissatisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Very<br>satisfied<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| B. Video/virtual consultations for initial and follow-up visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| C. Injection Administration: home health nurse to administer injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |



| 24. How satisfied or dissatisfied have you been with each of the telehealth services/systems for delivering APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>satisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Neither<br>satisfied<br>nor<br>dissatisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Very<br>satisfied<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| D. Injection appointment reminders: text, digital, email | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |



| 24. How satisfied or dissatisfied have you been with each of the telehealth services/systems for delivering APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>satisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Neither<br>satisfied<br>nor<br>dissatisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Very<br>satisfied<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| E. HIV testing services: at home nurse testing | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |



| 24. How satisfied or dissatisfied have you been with each of the telehealth services/systems for delivering APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>satisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Neither<br>satisfied<br>nor<br>dissatisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Very<br>satisfied<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |



Table 2.401 Summary of Utility of Proposed Implementation Strategies (Month 4/5), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 25 | Have you used the following in the imple | ementation of AF | PRETUDE into your p | oractice/clinic? | |
| 25A | Frequently Asked Questions Brochure | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 25B | Readiness Consideration | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 25C | Get Started Overview-Init/Adm Guide | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 25D | Injection Education Video | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 25E | Provider Website – location where all<br>materials and videos on APRETUDE for<br>the study is located | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 25F | Patient Materials | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 25G | Implementation Guidance Video | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 25H | Appointment Scheduler | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 251 | Pre-scheduled Appointment Guidance | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 25J | Designated Injection Days Guidance | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 25K | Drop-in Injection Visits Guidance | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 25L | Transport Support to Patient Appt | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 25M | Monthly Implement Facilitation Call | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 25N | Group Implement Facilitation Calls | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 250 | Document on How Discuss Sex Health | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 25P | PILLAR Spot | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 26 | How often have you used the following | in the implement | tation of APRETUDE | into your practice/o | clinic? |
| 26A | Frequent Ask Question Brochure | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 26B | Readiness Consideration | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 26C | Getting Started Overview | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 26D | Injection Education Video | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 26F | Patient Materials | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 26G | Implementation Guidance Video | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 26H | Appointment Scheduler | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 261 | Pre-scheduled Appt Guidance | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 26J | Designated Inj Days Guidance | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 26K | Drop-in Inj Visits Guidance | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 26L | Transport Support to Pt Appt | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 26M | Monthly Implement Facilit Call | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 26N | Group Implement Facilit Calls | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 260 | Doc on How Discuss Sex Health | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 26P | PILLAR Spot | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 27 | How useful are the following in the impl | ementation of Al | PRETUDE into your | practice/clinic? | |
| 27A | Frequently Asked Questions Brochure | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 27B | Readiness Consideration | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 27C | Getting Started Overview-Init/Adm<br>Guide | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 27D | Injection Education Video | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 27E | Provider Website | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 27F | Patient Materials | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 27G | 27G Implementation Guidance Video | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 27H | 27H Appointment Scheduler | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 271 | Pre-scheduled Appointment Guidance | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 27J | Designated Injection Days Guidance | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 27K | Drop-in Injection Visits Guidance | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 27L | Provide Transport Support to Patient Appt | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 27M | Monthly Implementation Facilitation<br>Call | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 27N | Group Implementation Facilitation Calls | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 270 | Document on How to Discuss Sexual<br>Health | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 27P | PILLAR Spot | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.501 Summary of Perceived Barriers to Delivering APRETUDE to Patients (Month 4/5), N=XX

| 52. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| A. Patients' ability to keep appointments | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic administrator/front desk staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 52. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| B. Patients' injection-related pain/soreness | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. Risk of drug resistance for patients not adherent to injections | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 52. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D. Cost of APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |



| 52. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| E. Keeping a patient engaged and motivated to continue APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 52. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. Identifying eligible individuals for<br>APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 52. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic administrator/front desk staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| G. Worried that a patient will feel stigmatized if offered APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |



| 52. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| H. Patients' willingness to travel every<br>2 months for an injection<br>appointment | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 52. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| I. Patient lack of belief in the efficacy of APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 52. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.502 Summary of Perceptions of Administering APRETUDE (Month 4/5), N=XX

| 53. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| your current expectations and knowledge. | | | | | | |
| A. Difficulty of giving the gluteal medial injection | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 53. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| B. Understanding how to manage patients who miss an injection dose | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. How to transition patients off of APRETUDE who want to stop taking it (e.g., should other PrEP be offered) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 53. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D. Understanding how to use oral<br>PrEP medication for a <u>planned</u> missed<br>injection visit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |



| 53. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| E. Understanding how to restart<br>APRETUDE after a missed injection | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 53. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. Managing the oral lead-in phase of<br>APRETUDE before starting injections if<br>needed | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 53. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| G. Ability to provide adherence counseling and support when injection dosing visits are missed | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |



| 53. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.503 Summary of Perceived Barriers to Managing Delivery of APRETUDE (Month 4/5), N=XX

| 54. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| A. Management of scheduling injection appointments every 2 months during correct injection (I.e., dosing) windows | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 54. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| B. Management of rescheduling appointments during correct injection (I.e., dosing) windows | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 54. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| C. Ability to schedule/reschedule patients who missed APRETUDE visits within correct injection (I.e., dosing) windows | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |


| 54. Please indicate how concerned you would be about each of the | Total<br>Sample | Extremely concerned | Moderately concerned | Somewhat concerned | Slightly concerned | Not at all concerned |
|---|---|---|---|---|---|---|
| following being a barrier or challenge<br>to APRETUDE delivery based on your<br>current expectations and knowledge. | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| D. Ability to identify and flag missed injection visits to providers (in a timely manner) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| E. Ability to manage patients presenting to APRETUDE injection | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 54. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| appointments with other care needs that need to be addressed | | | | | | |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. Persistence to follow up with patient on missed appointments | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |



| 54. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| G. Provider time to discuss HIV prevention with all eligible patients | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 54. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| H. Ability to provide HIV screening as indicated at each injection visit and provide rapid intervention/follow-up based on results status | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 54. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| I. HIV monitoring requirements associated with APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 54. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.504 Summary of Perceived Resourcing Barriers to Support Delivery of APRETUDE (Month 4/5), N=XX

| (101011611 1/3), 14 700 | | | | | | |
|---|---|---|---|---|---|---|
| 55. Please indicate how concerned you would be about each of the following potentially being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
| A. Staff resourcing to ensure appropriate clinic flow | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| you would be about each of the following potentially being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| B. Number of exam rooms for injections | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| C. Clinic staff to administer injections | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| you would be about each of the following potentially being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| D. Staff preparation (i.e., education,<br>training, in-services) to implement<br>APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| 55. Please indicate how concerned you would be about each of the following potentially being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| E. Staff time to provide counseling and support to patients, such as answering questing between visit, keeping patients motivated | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |



| 55. Please indicate how concerned you would be about each of the following potentially being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| F. Staff belief in the efficacy of<br>APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| 55. Please indicate how concerned you would be about each of the following potentially being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.505 Summary of Perceptions of Clinic/Practice Culture and Environment (Month 4/5), N=XX

| 56. How much do you agree or disagree with the following statements about your clinic/practice? | Total<br>Sample<br>n (%) | Completely<br>Disagree<br>n (%) | Disagree<br>n (%) | Neither<br>agree nor<br>disagree<br>n (%) | Agree<br>n (%) | Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|
| A. People at all levels openly talk about what is and isn't working | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| B. Most people in this clinic<br>are willing to change how<br>they do things in response to<br>feedback from others | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. It is hard to get things to change in our clinic | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D. People in this clinic operate as a real team | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | | | | | | |
| Site Volume | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | | | | | | |
| E. Staff members often show signs of stress and strain | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 56. How much do you agree or disagree with the following statements about your clinic/practice? | Total<br>Sample<br>n (%) | Completely<br>Disagree<br>n (%) | Disagree<br>n (%) | Neither<br>agree nor<br>disagree<br>n (%) | Agree<br>n (%) | Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. We regularly take time to consider ways to improve how we do things | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| G. Leadership strongly supports clinic change efforts | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.506 Summary of Barriers to PrEP Provisioning (Month 4/5), N=XX

| 87. Indicate your level of agreement with the following statements: | Total<br>Sample<br>n (%) | Completely<br>Disagree<br>n (%) | Disagree<br>n (%) | Neither<br>agree nor<br>disagree<br>n (%) | Agree<br>n (%) | Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|
| A. The use of PrEP will cause patients to engage in riskier behaviors | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| B. Providing PrEP endorses the risk behaviors of users | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. Only people who engage in risky behavior need PrEP | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D. Only people with many sexual partners need PrEP | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | | | | | | |
| Site Volume | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | | | | | | |
| E. All sexually active people can benefit from PrEP | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 87. Indicate your level of agreement with the following statements: | Total<br>Sample<br>n (%) | Completely<br>Disagree<br>n (%) | Disagree<br>n (%) | Neither<br>agree nor<br>disagree<br>n (%) | Agree<br>n (%) | Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. Providing PrEP will result<br>in an increase in sexually<br>transmitted diseases among<br>patients | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| G. People do not need PrEP if they act responsibly | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.507 Distributional Characteristics of Barriers to PrEP Provisioning (Month 4/5), N=XX

| 87. Indicate your level of agreement with the following statements: | Study Arm | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|---|
| | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| A. The use of PrEP<br>will cause patients<br>to engage in | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| riskier behaviors | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| B. Providing PrEP<br>endorses the risk<br>behaviors of users | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| C. Only people<br>who engage in<br>risky behavior | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| need PrEP | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| D. Only people<br>with many sexual<br>partners need | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| PrEP | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| E. All sexually<br>active people can<br>benefit from PrEP | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |



| 87. Indicate your level of agreement with the following statements: | Study Arm | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|---|
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| F. Providing PrEP | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| will result in an<br>increase in<br>sexually<br>transmitted | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| diseases among | T-test | | X.XXX | | | | | |
| patients | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| G. People do not<br>need PrEP if they<br>act responsibly | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| acticsponsibly | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Total Score | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX<br>(X.XX,<br>X.XX) | X.X (X.X, X.X) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |



Table 2.508 Shift from Baseline to Month 4/5 in Summary of Perceived Barriers to Delivering APRETUDE to Patients (Month 4/5), N=XX

52. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge.

#### A. Patients' ability to keep appointments

| | | | | | | M4/5 | | | |
|---|---|---|---|---|---|---|---|---|---|
| Study Arm | y Arm N Baseline | Extremely<br>Concerned | Moderately<br>Concerned | Somewhat<br>Concerned | Slightly<br>Concerned | Not at all<br>Concerned | Missing | Total | |
| | | Extremely<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| | | Moderately<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| | | Somewhat<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| DI | XX | Slightly Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| | | Not at all<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| | | Missing | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| | | Total | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| RI | XX | Extremely<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |



| Moderately<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
|---|---|---|---|---|---|---|---|
| Somewhat<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| Slightly Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| Not at all<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| Missing | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| Total | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |

Note 1: Shift tables will be created as above for items 52b through 52i.

Missing: BL = missing item at BL. M 4/5 = missing item at M 4/5.

Percentage calculations:

Column total %: numerator= number selecting respective response at M 4/5, denominator = number responding at M 4/5

Row total %: numerator= number selecting respective response at BL, denominator = number responding at BL

Cell %: numerator = number selecting respective combination of BL and M 4/5 responses, denominator=number of participants responding at BL.

Total: N = number of participants that completed the question at either BL or M 4/5

### Table 2.509 Shift from Baseline to Month 4/5 in Summary of Perceptions of Administering APRETUDE (Month 4/5), N=XX

Note 1: Shift tables will be created as shown for Table 2.508 for items 53a through 53g.

Missing: BL = missing item at BL. M 4/5 = missing item at M 4/5.

Percentage calculations:

Column total %: numerator= number selecting respective response at M 4/5, denominator = number responding at M 4/5

Row total %: numerator= number selecting respective response at BL, denominator = number responding at BL

Cell %: numerator = number selecting respective combination of BL and M 4/5 responses, denominator=number of participants responding at BL.

Total: N = number of participants that completed the question at either BL or M 4/5



## Table 2.510 Shift from Baseline to Month 4/5 in Summary of Perceived Barriers to Managing Delivery of APRETUDE (Month 4/5), N=XX

Note 1: Shift tables will be created as shown for Table 2.508 for items 54a through 54i.

Missing: BL = missing item at BL. M 4/5 = missing item at M 4/5.

Percentage calculations:

Column total %: numerator= number selecting respective response at M 4/5, denominator = number responding at M 4/5

Row total %: numerator= number selecting respective response at BL, denominator = number responding at BL

Cell %: numerator = number selecting respective combination of BL and M 4/5 responses, denominator=number of participants responding at BL.

Total: N = number of participants that completed the question at either BL or M 4/5

# Table 2.511 Shift from Baseline to Month 4/5 in Summary of Perceived Resourcing Barriers to Support Delivery of APRETUDE (Month 4/5), N=XX

Note 1: Shift tables will be created as shown for Table 2.508 for items 55a through 55f.

Missing: BL = missing item at BL. M 4/5 = missing item at M 4/5.

Percentage calculations:

Column total %: numerator= number selecting respective response at M 4/5, denominator = number responding at M 4/5

Row total %: numerator= number selecting respective response at BL, denominator = number responding at BL

Cell %: numerator = number selecting respective combination of BL and M 4/5 responses, denominator=number of participants responding at BL.

Total: N = number of participants that completed the question at either BL or M 4/5

## Table 2.512 Shift from Baseline to Month 4/5 in Summary of Perceptions of Clinic/Practice Culture and Environment (Month 4/5), N=XX

Note 1: Shift tables will be created as shown for Table 2.508 for items 56a through 56g.

.

Missing: BL = missing item at BL. M 4/5 = missing item at M 4/5.

Percentage calculations:

Column total %: numerator= number selecting respective response at M 4/5, denominator = number responding at M 4/5

Row total %: numerator= number selecting respective response at BL, denominator = number responding at BL

Cell %: numerator = number selecting respective combination of BL and M 4/5 responses, denominator=number of participants responding at BL.

Total: N = number of participants that completed the question at either BL or M 4/5



### Table 2.513 Shift from Baseline to Month 4/5 in Summary of Barriers to PrEP Provisioning (Month 4/5), N=XX

Note 1: Shift tables will be created as shown for Table 2.508 for items 87a through 87g.

Missing: BL = missing item at BL. M 4/5 = missing item at M 4/5.

Percentage calculations:

Column total %: numerator= number selecting respective response at M 4/5, denominator = number responding at M 4/5

Row total %: numerator= number selecting respective response at BL, denominator = number responding at BL

Cell %: numerator = number selecting respective combination of BL and M 4/5 responses, denominator=number of participants responding at BL.

Total: N = number of participants that completed the question at either BL or M 4/5



Table 2.601 Summary of the Sexual Health Assessment Tool (Month 4/5), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 28 | Has your clinic/practice started | to use the Sexual Health Assessm | nent? | | |
| | | No And Not Planning To Use<br>The Sexual Health Assessment | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No But Planning To Use The<br>Sexual Health Assessment | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29 | Who in your clinic/practice is c | Who in your clinic/practice is or will be responsible for distributing the Sexual Health Assessment to patients? | | | |
| | | Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse practitioner/physician assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Medical assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Social worker/case manager | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Front desk staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Peer educator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 30 | Who in your clinic/practice is c<br>Assessment with patients? | or will be responsible for reviewing | and discussi | ng the results of th | e Sexual Health |
| | | Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse practitioner/physician assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Medical assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Social worker/case manager | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Front desk staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Peer educator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The results are or will not be discussed with patients | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 31 | How often have you used the S | Sexual Health Assessment in your | clinic/practic | e? | |
| | | Rarely | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 32 | "Please indicate your level of agreement with the following statements about the Sexual Health Assessment." | | | | |
| | The Sexual Health Assessment is/will be easy to implement in my clinic/practice | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | The Sexual Health<br>Assessment is/will be an easy<br>way to identify individuals<br>interested in PrEP | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | The Sexual Health Assessment helps/will help to facilitate conversations about PrEP with patients | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 33 | Why is the Sexual Health<br>Assessment not used by your<br>clinic/practice? | Already have a similar assessment | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Does not integrate with the EMR | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The assessment is difficult to administer | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Concerns about patient privacy | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The assessment does not ask the right questions | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The assessment takes too much time | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The assessment is not needed | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.602 Summary of the PrEP Communication Tool (Month 4/5), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 34 | Has your clinic, | /practice started to use PrEP Options Communi | cation Tool? | | |
| | | No and not planning to use the PrEP Options Communication Tool | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No but planning to use the PrEP Options<br>Communication Tool | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 35 | Who in your cl<br>patients? | Who in your clinic/practice is or will be responsible for using the PrEP Options Communication Tool with patients? | | | |
| | | Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse practitioner/physician assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Medical assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Social worker/case manager | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Front desk staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Peer educator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 36 | How often hav | How often have you used the PrEP Options Communication Tool in your clinic/practice? | | | |
| | | Rarely | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 37 | Please indicate<br>Tool | your level of agreement with the following sta | tements abo | ut the PrEP Options | Communication |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | The PrEP Options Communication Tool is/will be easy to implement in my clinic/practice | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | The PrEP Options Communication Tool helps/will help to facilitate conversations about PrEP with patients | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 38 | Why is the PrEP<br>Options<br>Communication<br>Tool not used by<br>your<br>clinic/practice? | Already have a similar tool | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Do not have time in a clinical visit to use the tool | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Do not understand the information in the tool | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Tool does not provide the right information | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Tool is not needed | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.701 Summary of the Optional Oral Lead-in Phase of APRETUDE (Month 4/5), N=XX

| Question<br>Number | Question | uestion Response | | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N= XX)<br>n (%) |
|---|---|---|---|---|---|
| 73 | How do you start your patients with APRETUDE? | | | | |
| | | Directly with injection | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | With optional oral lead-in using oral cabotegravir | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | With oral PrEP (TDF/FTC or TAF/FTC) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 74 | "Of all your patients who ha | "Of all your patients who have been prescribed APRETUDE, please estimate the percentage that started:" | | | |
| | Directly with injection<br>who switched from oral<br>PrEP | N | XX | XX | XX |
| | | Mean (SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | X.X, X.X | X.X, X.X | X.X, X.X |
| | | Range (Min, Max) | XX (XX, XX) | XX (XX, XX) | XX (XX, XX) |
| | Directly with injection who are new to PrEP | N | XX | XX | XX |
| | | Mean (SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | X.X, X.X | X.X, X.X | X.X, X.X |
| | | Range (Min, Max) | XX (XX, XX) | XX (XX, XX) | XX (XX, XX) |
| | With optional oral lead-in (oral Cabotegravir) | N | XX | XX | XX |
| | | Mean (SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | X.X, X.X | X.X, X.X | X.X, X.X |
| | | Range (Min, Max) | XX (XX, XX) | XX (XX, XX) | XX (XX, XX) |
| | With oral PrEP (TDF/FTC or TAF/FTC) | N | XX | XX | XX |
| | | Mean (SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | X.X, X.X | X.X, X.X | X.X, X.X |
| | | Range (Min, Max) | XX (XX, XX) | XX (XX, XX) | XX (XX, XX) |
| | Other | N | XX | XX | XX |



| Question<br>Number | Ouestion Response | | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N= XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Mean (SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | X.X, X.X | X.X, X.X | X.X, X.X |
| | | Range (Min, Max) | XX (XX, XX) | XX (XX, XX) | XX (XX, XX) |
| 75 | What sources of info | ormation have you drawn upon in assessing | whether oral | lead-in is needed o | r not? |
| | | Scientific literature | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Independent Medical Education | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Data from ViiV/GSK | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Scientific conferences | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Clinic rounds | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | CDC guidelines | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other medical colleagues | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other sources | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 76 | What are the main f | actors that drive your decision to use oral l | ead-in or not? | | |
| | | The ability to assess the safety/tolerability of APRETUDE in all patients | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The ability to assess the safety/tolerability of APRETUDE in patients with a history of allergy/drug intolerance | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The availability of more data from clinical trials using an oral lead-in phase | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The ability to increase drug concentration before starting the injections | | XX (XX.X%) | XX (XX.X%) |
| | | Being cautious with a new medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Providing patient with protection against HIV until the injection arrives | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Patient request | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Enough data exists from clinical trials to start patients with injection without oral lead in | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Provide patients with immediate protection with a long acting method by not using oral lead in | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N= XX)<br>n (%) |
|---|---|---|---|---|---|
| 77 | How influential are patient preferences in the decision of whether or not to use an oral lead-in phase? | | | | |
| | | Very influential | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Influential | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat influential | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not very influential | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all influential | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 78 | Have any of your pa | tients missed injection visit(s)? | | | |
| | | No, none of my patients have missed their injection visits | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Yes, some of my patients have had planned missed visits | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Yes, some of my patients have had unplanned missed visits | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 79 | For patients who have missed an injection visit, what protection were they given/offered until they received their next injection? | | | | |
| | | Cabotegravir oral tablets | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | TDF/FTC | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | TAF/FTC | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Provision of condoms | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Risk reduction education | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | None | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Do not know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 80 | For patients who planext injection? | an to miss an injection, what protection do Cabotegravir oral tablets | you plan on of | fering them until th | xx (xx.x%) |
| | | TDF/FTC | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | TAF/FTC | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Provision of condoms | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Risk reduction education | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| | | None | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Do not know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 81 | How easy or difficult | t was it to start patients on oral PrEP for a | , , | ` ′ | // (///.//0) |
| 01 | 110W Casy of difficult | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | very easy | // (///.//o) | /// (///.//o) | /// (///.//u) |
| | | Somewhat easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N= XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Somewhat difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 82 | Ho | w acceptable was it to start patients on oral | PrEP after a m | nissed injection visit | :? |
| | | Very acceptable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Acceptable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Acceptable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Acceptable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Acceptable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 83 | Before initiating a p | patient on PrEP, what type of HIV test do you | ı primarily use | ? | |
| | Oral PrEP | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4 <sup>th</sup> gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/ antibody test<br>(rapid test) 4 <sup>th</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test) 3 <sup>rd</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | APRETUDE | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4 <sup>th</sup> gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/ antibody test<br>(rapid test) 4 <sup>th</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test) 3 <sup>rd</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 84 | Before initiating a patient on PrEP, what type of HIV test have you ever used? | | | | |
| | Oral PrEP | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4 <sup>th</sup> gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/ antibody test<br>(rapid test) 4 <sup>th</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test) 3 <sup>rd</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | APRETUDE | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question Response | | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N= XX)<br>n (%) |
|---|---|---|---|---|---|
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4 <sup>th</sup> gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/ antibody test<br>(rapid test) 4 <sup>th</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test) 3 <sup>rd</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 85 | For follow-up visits for p | patients who are on PrEP, what type of I | HIV test do you | u primarily use? | |
| | Oral PrEP | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4 <sup>th</sup> gen lab | HIV antigen/antibody test | | XX (XX.X%) |
| | | HIV antigen/ antibody test<br>(rapid test) 4 <sup>th</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test) 3 <sup>rd</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | APRETUDE | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4 <sup>th</sup> gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/ antibody test<br>(rapid test) 4 <sup>th</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test) 3 <sup>rd</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 86 | For follow-up visits for p | patients who are on PrEP, what type of I | HIV test have y | ou ever used? | |
| | Oral PrEP | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4 <sup>th</sup> gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/ antibody test<br>(rapid test) 4 <sup>th</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test) 3 <sup>rd</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | APRETUDE | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N= XX)<br>n (%) |
|---|---|---|---|---|---|
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4 <sup>th</sup> gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/ antibody test<br>(rapid test) 4 <sup>th</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test) 3 <sup>rd</sup> gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.801 Summary of Perceived Number of APRETUDE Patients Clinic/Practice Can Manage Per Week on an Ongoing Basis (Month 4/5), N=XX

| 57. How many APRETUDE patients do you think your clinic/practice can manage per week on an ongoing basis? | Total | 0-10 | 11-25 | 26-50 | 51-100 | 101-200 | >200 | I don't |
|---|---|---|---|---|---|---|---|---|
| | Sample | Patients | Patients | Patients | Patients | Patients | Patients | know |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n=xx (%) |
| Total Sample | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



Table 2.802 Distributional Characteristics of People in Clinic Trained and Prepared to Give APRETUDE Injections (Month 4/5), N=XX

| | | | <u> </u> | | | | | |
|---|---|---|---|---|---|---|---|---|
| 58. Approximately how many people in your clinic are trained and prepared to give APRETUDE injections? | Total<br>Sample<br>n (%) | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum<br>and<br>Maximum) | Percent<br>Missing | 95%<br>Confidence<br>Interval | l don't know<br>n (%) |
| Total Sample | XX<br>(XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX<br>(XX, XX) | XX.X% | X.XX (X.XX,<br>X.XX) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX<br>(XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX<br>(XX, XX) | XX.X% | X.XX (X.XX,<br>X.XX) | XX (XX.X%) |
| Routine<br>Implementation | XX<br>(XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX<br>(XX, XX) | XX.X% | X.XX (X.XX,<br>X.XX) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX<br>(XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX<br>(XX, XX) | XX.X% | X.XX (X.XX,<br>X.XX) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX<br>(XX, XX) | XX.X% | X.XX (X.XX,<br>X.XX) | XX (XX.X%) |


Table 2.803 Distributional Characteristics of Estimated Number of Staff Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25 People (Month 4/5), N=XX

| 48. How much staff in total do you estimate is/will be needed per week to incorporate APRETUDE into your clinic/practice for approximately 25 people? | Total<br>Sample<br>n (%) | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum<br>and<br>Maximum) | Percent<br>Missing | 95%<br>Confidence<br>Interval | l don't know<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| Total Sample | XX<br>(XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX<br>(XX, XX) | XX.X% | X.XX (X.XX,<br>X.XX) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX<br>(XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX<br>(XX, XX) | XX.X% | X.XX (X.XX,<br>X.XX) | XX (XX.X%) |
| Routine<br>Implementation | XX<br>(XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX<br>(XX, XX) | XX.X% | X.XX (X.XX,<br>X.XX) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX<br>(XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX<br>(XX, XX) | XX.X% | X.XX (X.XX,<br>X.XX) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX<br>(XX, XX) | XX.X% | X.XX (X.XX,<br>X.XX) | XX (XX.X%) |



Table 2.804 Summary of Estimated Percentage of Staff Time/Full-Time Equivalent Hours

Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25

People (Month 4/5), N=XX

| 60. How much staff time/full-time equivalent hours (FTE) do you estimate is/will be needed per week to incorporate APRETUDE into your clinic/practice for approximately 25 people? | Total<br>Sample<br>n (%) | 1-20% FTE<br>or 0.4 –<br>8hrs of<br>staff time<br>n (%) | 21-40% FTE<br>or 8.4 –<br>16hrs of staff<br>time<br>n (%) | 41-60% FTE<br>or 16.4 – 24<br>hrs of staff<br>time<br>n (%) | 61-80% FTE<br>or 24.4 –<br>32hrs of<br>staff time<br>n (%) | 81-100%<br>FTE or<br>32.4 –<br>40hrs of<br>staff<br>time<br>n (%) | l don't<br>know<br>n (%) |
|---|---|---|---|---|---|---|---|
| Total Sample | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic<br>Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Routine<br>Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 2.805 Summary of Plans to Create New Roles/Positions in Clinic to Coordinate the APRETUDE Program (Month 4/5), N=XX

| 61. Have you created or do you plan to create new role(s)/new position(s) in your clinic to coordinate the APRETUDE program? | Total Sample<br>n (%) | Yes<br>n (%) | No<br>n (%) | Maybe<br>n (%) | l don't know<br>n (%) |
|---|---|---|---|---|---|
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | |
| Dynamic<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.806 Summary of Number of New Roles/Positions in Clinic to Coordinate the APRETUDE Program (Month 4/5), N=XX

| 62. How many new role(s)/new position(s) have been created or will be created in your clinic to coordinate the APRETUDE program? [1] | Total<br>Sample<br>n (%) | 1<br>n (%) | 2<br>n (%) | 3<br>n (%) | 4<br>n (%) | 5<br>n (%) | More<br>than 5 n<br>(%) | l don't<br>know<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| Total Sample | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Routine<br>Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |

<sup>[1]</sup> Only includes SSPs who responded 'yes' or 'maybe' to 'Do you plan to create new role(s)/new position(s) in your clinic to coordinate the APRETUDE program?'



Table 2.807 Summary of How Clinic/Practice Plans to Track Patients on APRETUDE (Month 4/5), N=XX

| 63. How is the clinic/practice tracking patients on APRETUDE? | Total<br>Sample<br>n (%) | Use a<br>spreadsheet<br>such as MS<br>Excel<br>n (%) | Assign<br>specific<br>staff to<br>track<br>patients<br>n (%) | Have providers track their own patients n (%) | Create<br>alerts in<br>electronic<br>medical<br>records<br>(EMRs)<br>n (%) | Other<br>[1]<br>n (%) | l don't<br>know<br>n (%) |
|---|---|---|---|---|---|---|---|
| Total Sample | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |

<sup>[1]</sup> Other responses include: xxxxx



Table 2.808 Summary of How Clinic/Practice Responds to Patients who Do Not Show for a Regularly Scheduled Appointment (Month 4/5), N=XX

| 64. What does your clinic/practice do if a patient does not show for a APRETUDE visit? | Total<br>Sample<br>n (%) | Phone the<br>patient to<br>reschedule<br>n (%) | Text the patient to reschedule n (%) | Email the<br>patient to<br>reschedule<br>n (%) | Send the<br>patient a<br>postal<br>letter to<br>reschedule<br>n (%) | Wait until the patient contacts the clinic/practice to reschedule n (%) | Charge<br>the<br>patient<br>a fee<br>for not<br>showing<br>up n (%) | I don't<br>know/not<br>applicable<br>to role<br>n (%) | Other<br>[1]<br>n (%) |
|---|---|---|---|---|---|---|---|---|---|
| Total Sample | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Total Sample | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | | | |
| Dynamic | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | | | |
| ∐iah | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| High | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| LOW | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |

<sup>[1]</sup> Other responses include: xxxxx



Table 2.809 Summary of Whether Clinic/Practice has Specific Person in Charge of Following Up on No-Shows (Month 4/5), N=XX

| 65. Is there a specific person in charge of following up on no-shows for APRETUDE appointments? | Total Sample<br>n (%) | Yes<br>n (%) | No<br>n (%) | l don't know<br>n (%) |
|---|---|---|---|---|
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.810 Summary of Type of Systems Clinic has in Place to Remind Patients of Upcoming Appointments (Month 4/5), N=XX

| 69. How do you remind patients of an upcoming APRETUDE appointment?[1] | Total<br>Sample<br>n (%) | Phone<br>Call from<br>Staff n<br>(%) | Automated<br>Phone call<br>n (%) | Text<br>Message<br>n (%) | Email<br>n (%) | Postal<br>Mail n<br>(%) | Phone App<br>Notification<br>n (%) | Other<br>[2]<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| Total Sample | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |

<sup>[1]</sup> Responses are not mutually exclusive; participants can select all that apply

<sup>[2]</sup> Other responses included: xxxxx



Table 2.811 Summary of Type of Systems Clinic has in Place to Offer Upcoming Appointments (Month 4/5), N=XX

| | Total Sample | Stud | y Arm | Site V | olume |
|---|---|---|---|---|---|
| 70. How do you plan to offer appointments for APRETUDE injections? | | Dynamic | Routine | High Volume | Low Volume |
| ioi /ii Nerobe injections. | n (%) | n (%) | n (%) | n (%) | n (%) |
| Appointments each day of the week | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Appointments only on certain days of the week | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Appointments spread out over the month | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Injection only appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Allow patients to drop-in for injections on any day without an appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Allow patients to drop-in with little advanced notice (e.g., 24 hour notice) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Allow patients to drop-in on a specific injection day without an appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| After hours appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Appointments each day of the week | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Before hours appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Weekend appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Home nursing appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mobile clinic option | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Alternate site appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Depends on the schedule of the injection nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Depends on the schedule of the APRETUDE provider | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| I don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



- [1] Responses are not mutually exclusive; participants can select all that apply
- [2] Other responses include: xxxxx



Table 2.812 Summary of Implementing APRETUDE in Practice (Month 4/5), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 67 | APRETUDE must be administe | red within a two-week injectior | n window every | two months after th | ne loading doses. |
| | | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have not rescheduled any injections thus far | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 68 | How easy or difficult has it be | en to reschedule appointments | for APRETUDE i | njections? | |
| | | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have not rescheduled any injections thus far | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 69 | How do you remind patients o | of an upcoming APRETUDE appo | ointment? | | |
| | | Phone call from Staff | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Automated phone call | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Text message | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Email | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Postal Mail | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Phone app notification | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 70 | How does your practice/clinic | currently offer appointments for | or APRETUDE inj | ections? | |
| | | Appointments each day of the week | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appointments only on certain days of the week | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appointments spread out over the month | XX (XX.X%) | XX XX.X%) | XX (XX.X%) |
| | | Injection-only appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Allow patients to drop-in for injections on any day without an appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Allow patients to drop-in with little advance notice (e.g., 24 hr notice) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Allow patients to drop-in on a specific injection day without an appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | After hours appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Before hours appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Weekend appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Home nursing appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Mobile clinic option | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Alternate site appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Depends on the schedule of the injection nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Depends on the schedule of the APRETUDE provider | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Unsure | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 71 | How easy or difficult has it be | en to implement APRETUDE int | o your current w | vorkflow? | |
| | | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have not rescheduled any injections thus far | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 72 | How do you feel about impler | nenting APRETUDE at your clini | c/practice? | | |
| | | Extremely positive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Positive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat positive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little positive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all positive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 2.901 Quarterly Site Reporting

| Question | | Total | Dynamic<br>Implementation | Routine<br>Implementation |
|---|---|---|---|---|
| 14. How many HIV PrEP seeking persons did the clinic/practice see in the last 3 months? | | | | |
| Baseline | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |
| Quarter X* | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |
| 15. How many patients would you estimate initiated any type of PrEP – oral or injectable – at the clinic/practice in the last 3 months? | | | | |
| Baseline | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |
| Quarter X* | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |
| 16. How many patients would you estimate initiated APRETUDE in the last 3 months at the clinic/practice? | | | | |
| Baseline | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |



| Question | | Total | Dynamic<br>Implementation | Routine<br>Implementation |
|---|---|---|---|---|
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |
| Quarter X* | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |
| 17. Of all patients who have been prescribed PrEP at your clinic/practice, how many would you estimate have completed the Sexual Health Assessment provided by the PILLAR study? | | | | |
| Baseline | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |
| Quarter X* | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |

NOTE: reporting is not compiled on schedule with Month 4/5 or Month 12/13 collections, but is instead collected quarterly \*To be populated for each quarter separately depending on available of quarterly data.



## 7 Tables for Month 12/13 Analysis

| Table 3.001 | Demographic Characteristics of New Staff Study Participants (Month 12/13), N=XX | . 266 |
|---|---|---|
| Table 3.002 | Demographic Characteristics of Longitudinal* Study Participants (Month 12/13), N=XX | . 268 |
| Table 3.003 | Characteristics of New Staff Study Participants (Month 12/13), N=XX | . 269 |
| Table 3.004 | Characteristics of Longitudinal* Staff Study Participants (Month 12/13), N=XX | . 271 |
| Table 3.005 | Summary of Confidence with Skills (Month 12/13), N=XX | . 273 |
| Table 3.006 | Staff Study Participants' Perceptions Regarding APRETUDE (Month 12/13), N=XX | . 275 |
| Table 3.007 | Summary of Experiences with the Acquisition Process (Month 12/13), N=XX | . 279 |
| Table 3.101 | Summary of Acceptability of Intervention Measure (AIM – APRETUDE) and Feasibility of Intervention Measure (FIM – APRETUDE) Items (Month 12/13), N=XX | . 293 |
| Table 3.102 | Distributional Characteristics of the Acceptability of Intervention Measure (AIM – APRETUDE) (Month 12/13), N=XX | . 295 |
| Table 3.103 | Distributional Characteristics of the Feasibility of Intervention Measure (FIM – APRETUDE) (Month 12/13), N=XX | . 297 |
| Table 3.104 | Changes from Baseline for Acceptability of Intervention Measure (AIM – APRETUDE) and Feasibility of Intervention Measure (FIM – APRETUDE) (Month 12/13), N=XX | . 299 |
| Table 3.105 | Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – APRETUDE) (Month 12/13), N=XX | . 300 |
| Table 3.106 | Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Acceptability of Intervention Measure (AIM – APRETUDE), N=XX | . 301 |
| Table 3.107 | Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – APRETUDE) (Month 12/13), N=XX | . 302 |
| Table 3.108 | Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Feasibility of Intervention Measure (FIM – APRETUDE), N=XX | . 303 |
| Table 3.201 | Summary of Acceptability of Intervention Measure (AIM – Implementation Support) and Feasibility of Intervention Measure (FIM – Implementation Support) Items (Month 12/13), N=XX | . 304 |
| Table 3.202 | Distributional Characteristics of the Acceptability of Intervention Measure (AIM – Implementation Support) (Month 12/13), N=XX | . 306 |
| Table 3.203 | Distributional Characteristics of the Feasibility of Intervention Measure (FIM – Implementation Support) (Month 12/13), N=XX | . 308 |
| Table 3.204 | Changes from Baseline to Acceptability of Intervention Measure (AIM – Implementation Support) and Feasibility of Intervention Measure (FIM – Implementation Support ) (Month 12/13), N=XX | . 310 |
| Table 3.205 | Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – Implementation Support) (Month 12/13), N=XX | . 311 |
| Table 3.206 | Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Acceptability of Intervention Measure (AIM – Implementation Support), N=XX | . 312 |
| Table 3.207 | Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – Implementation Support) (Month 12/13), N=XX | 313 |



| Table 3.208 | Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Feasibility of Intervention Measure (FIM – Implementation Support), N=XX | 314 |
|---|---|---|
| Table 3.301 | Summary of Acceptability of Intervention Measure (AIM – Telehealth) and Feasibility of Intervention Measure (FIM – Telehealth) Items (Month 12/13), N=XX | 315 |
| Table 3.302 | Distributional Characteristics of the Acceptability of Intervention Measure (AIM – Telehealth) (Month 12/13), N=XX | 317 |
| Table 3.303 | Distributional Characteristics of the Feasibility of Intervention Measure (FIM – Telehealth) (Month 12/13), N=XX | 319 |
| Table 3.304 | Changes from Baseline for Acceptability of Intervention Measure (AIM – Telehealth) and Feasibility of Intervention Measure (FIM – Telehealth) (Month 12/13), N=XX | 321 |
| Table 3.305 | Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – Telehealth) (Month 12/13), N=XX | 322 |
| Table 3.306 | Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Acceptability of Intervention Measure (AIM – Telehealth), N=XX | 323 |
| Table 3.307 | Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – Telehealth) (Month 12/13), N=XX | 324 |
| Table 3.308 | Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Feasibility of Intervention Measure (FIM – Telehealth), N=XX | 325 |
| Table 3.309 | Summary of Feasibility and Acceptability of Telehealth (Month 12/13), N=XX | 326 |
| Table 3.310 | Summary of Telehealth Services/Systems Used (Month 12/13), N=XX | 332 |
| Table 3.311 | Summary of Ease of Use of Telehealth Services/Systems Used (Month 12/13), N=XX | 336 |
| Table 3.312 | Summary of Helpfulness of Services/Systems Used (Month 12/13), N=XX | 342 |
| Table 3.313 | Summary of Satisfaction of Services/Systems Used (Month 12/13), N=XX | 348 |
| Table 3.401 | Summary of Utility of Proposed Implementation Strategies (Month 12/13), N=XX | 353 |
| Table 3.501 | Summary of Perceived Barriers to Delivering APRETUDE to Patients (Month 12/13), N=XX | 359 |
| Table 3.502 | Summary of Perceptions of Administering APRETUDE (Month 12/13), N=XX | 368 |
| Table 3.503 | Summary of Perceived Barriers to Managing Delivery of APRETUDE (Month 12/13), N=XX | 376 |
| Table 3.504 | Summary of Perceived Resourcing Barriers to Support Delivery of APRETUDE (Month 12/13), N=XX | 387 |
| Table 3.505 | Summary of Perceptions of Clinic/Practice Culture and Environment (Month 12/13), N=XX | 394 |
| Table 3.506 | Summary of Barriers to PrEP Provisioning (Month 12/13), N=XX | 396 |
| Table 3.507 | Distributional Characteristics of Barriers to PrEP Provisioning (Month 12/13), N=XX | 398 |
| Table 3.508 | Shift from Month 4/5 to Month 12/13 in Summary of Perceived Barriers to Delivering APRETUDE to Patients (Month 12/13), N=XX | 400 |
| Table 3.509 | Shift from Month 4/5 to Month 12/13 in Summary of Perceptions of Administering APRETUDE (Month 12/13), N=XX | |
| Table 3.510 | Shift from Month 4/5 to Month 12/13 in Summary of Perceived Barriers to Managing | 402 |



| Table 3.511 | Shift from Month 4/5 to Month 12/13 in Summary of Perceived Resourcing Barriers to Support Delivery of APRETUDE (Month 12/13), N=XX | 402 |
|---|---|---|
| Table 3.512 | Shift from Month 4/5 to Month 12/13 in Summary of Perceptions of Clinic/Practice Culture and Environment (Month 12/13), N=XX | 402 |
| Table 3.513 | Shift from Month 4/5 to Month 12/13 in Summary of Barriers to PrEP Provisioning (Month 12/13), N=XX | 403 |
| Table 3.601 | Summary of the Sexual Health Assessment Tool (Month 12/13), N=XX | 404 |
| Table 3.602 | Summary of the PrEP Communication Tool (Month 12/13), N=XX | 407 |
| Table 3.701 | Summaries of the Optional Oral Lead-in Phase of APRETUDE (Month 12/13), N=XX | 409 |
| Table 3.702 | Assessment of Alternate Sites of Administration of APRETUDE (Month 12/13), N=XX | 415 |
| Table 3.801 | Summary of Perceived Number of APRETUDE Patients Clinic/Practice Can Manage Per Week on an Ongoing Basis (Month 12/13), N=XX | 421 |
| Table 3.802 | Distributional Characteristics of Reported Number of People in Clinic Trained and Prepared to Give APRETUDE Injections (Month 12/13), N=XX | 422 |
| Table 3.803 | Distributional Characteristics of Estimated Number of Staff Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25 People (Month 12/13), N=XX | 423 |
| Table 3.804 | Summary of Estimated Percentage of Staff Time/Full-Time Equivalent Hours Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25 People (Month 12/13), N=XX | 424 |
| Table 3.805 | Summary of Plans to Create New Roles/Positions in Clinic to Coordinate the APRETUDE Program (Month 12/13), N=XX | 425 |
| Table 3.806 | Summary of Number of New Roles/Positions in Clinic to Coordinate the APRETUDE Program (Month 12/13), N=XX | 426 |
| Table 3.807 | Summary of How Clinic/Practice Plans to Track Patients on APRETUDE (Month 12/13), N=XX | 427 |
| Table 3.808 | Summary of How Clinic/Practice Responds to Patients who Do Not Show for a Regularly Scheduled Appointment (Month 12/13), N=XX | 428 |
| Table 3.809 | Summary of Whether Clinic/Practice has Specific Person in Charge of Following Up on No-Shows (Month 12/13), N=XX | 429 |
| Table 3.810 | Summary of Type of Systems Clinic has in Place to Remind Patients of Upcoming Appointments (Month 12/13), N=XX | 430 |
| Table 3.811 | Summary of Type of Systems Clinic has in Place to Offer Upcoming Appointments (Month 12/13), N=XX | 431 |
| Table 3.812 | Summary of Implementing APRETUDE in Practice (Month 12/13), N=XX | 432 |
| Table 3.813. | Test for Differences of Implementation Arm by Site Volume on Feasibility of Intervention Measure, APRETUDE (Month 12/13), N=XX | 435 |
| Table 3.814. | Test for Differences of Implementation Arm by Site Volume on Feasibility of Intervention Measure, Implementation Support (Month 12/13), N=XX | 435 |
| Table 3.815. | Test for Differences of Implementation Arm by Site Volume on Feasibility of Intervention Measure, Telehealth (Month 12/13), N=XX | 435 |



| Table 3.816. | Test for Differences of Implementation Arm by Site Volume on Acceptability of | |
|---|---|---|
| | Intervention Measure, APRETUDE (Month 12/13), N=XX | 435 |
| Table 3.817. | Test for Differences of Implementation Arm by Site Volume on Acceptability of | |
| | Intervention Measure, Implementation Support (Month 12/13), N=XX | 435 |
| Table 3.818. | Test for Differences of Implementation Arm by Site Volume on Acceptability of | |
| | Intervention Measure, Telehealth (Month 12/13), N=XX | 436 |



Table 3.001 Demographic Characteristics of New Staff Study Participants (Month 12/13), N=XX

| Question<br>Number | Characteristic | | Stud | / Arm |
|---|---|---|---|---|
| | | Total<br>(N=XX) | Dynamic<br>Implementation<br>(N=XX) | Routine<br>Implementation<br>(N=XX) |
| | | n (%) | n (%) | n (%) |
| 99 | Gender | | | |
| | Cisgender Male | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Cisgender Female | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Transgender Man | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Transgender Woman | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Nonbinary | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Gender Queer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other Gender | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I prefer not to answer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 100 | Age (years) | | | |
| | N | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 100 | Age (years), High Volume | | | |
| | N | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 100 | Age (years), Low Volume | | | |
| | N | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 100 | Age | , , | , | , , |
| | 18-25 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 26-35 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | . (, 3) | ( / | \ |



| Question<br>Number | Characteristic | | / Arm | |
|---|---|---|---|---|
| | | Total<br>(N=XX) | Dynamic<br>Implementation<br>(N=XX) | Routine<br>Implementation<br>(N=XX) |
| | | n (%) | n (%) | n (%) |
| | 66-49 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 50+ | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 101 | Race | | | |
| | White/Caucasian | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Black | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Asian | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Native American | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Pacific Islander | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Mixed Race | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other Race | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | l Prefer not to Answer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 102 | Ethnicity | | | |
| | Hispanic/Latinx | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Non-Hispanic/Latinx | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Prefer not to answer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.002 Demographic Characteristics of Longitudinal\* Study Participants (Month 12/13), N=XX

| Question<br>Number | Characteristic | | Study | / Arm |
|---|---|---|---|---|
| Number | | Total<br>(N=XX) | Dynamic<br>Implementation<br>(N=XX) | Routine<br>Implementation<br>(N=XX) |
| | | n (%) | n (%) | n (%) |
| 99 | Gender | | | |
| | Cisgender Male | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Cisgender Female | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Transgender Man | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Transgender Woman | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Nonbinary | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Gender Queer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other Gender | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I prefer not to answer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 100 | Age (years) | | | |
| | N | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 100 | Age (years), High Volume | | | |
| | N | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 100 | Age (years), Low Volume | | | |
| | N | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX, XX | XX, XX | XX, XX |
| | Min-Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 100 | Age | | | |
| | 18-25 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 1 | I to the second | |



| Question<br>Number | Characteristic | | Study Arm | |
|---|---|---|---|---|
| Number | | Total<br>(N=XX) | Dynamic<br>Implementation<br>(N=XX) | Routine<br>Implementation<br>(N=XX) |
| | | n (%) | n (%) | n (%) |
| | 66-49 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 50+ | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 101 | Race | | | |
| | White/Caucasian | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Black | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Asian | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Native American | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Pacific Islander | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Mixed Race | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other Race | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I Prefer not to Answer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 102 | Ethnicity | | | |
| | Hispanic/Latinx | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Non-Hispanic/Latinx | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Prefer not to answer | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

<sup>\*</sup> Longitudinal = SSPs who completed any portion of any questionnaire at Baseline, Month 4/5 and Month 12/13

Table 3.003 Characteristics of New Staff Study Participants (Month 12/13), N=XX

| Question<br>Number | Characteristic | | Study Arm | |
|---|---|---|---|---|
| | Total<br>(N=XX) | | Dynamic<br>Implementation<br>(N=XX) | Routine<br>Implementation<br>(N=XX)<br>n (%) |
| | | n (%) | n (%) | |
| 1 | Provider Type | | | |
| | Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Nurse Practitioner | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Physician Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Social worker/case manager | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Office administrator/clinic administrator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Laboratory staff/technician/phlebotomist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | | | Study Arm | |
|---|---|---|---|---|
| | Front desk staff/ Scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 2 | Personally Administer Injections | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 3 | Prescribe Medications as part of role | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 4 | Currently Provide PrEP Counseling | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 103 | Specialty | | | |
| | Infectious disease specialist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Internal medicine/ primary care/general doctor/<br>family practitioner | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | HIC Specialist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Immunologist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Women's health/obstetricians and gynecologists | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Endocrinologist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other[2] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 104 | Length of Time practicing Medicine | | | |
| | <1 year | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 1–5 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 6–10 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 11-15 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 16-20 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | >21 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

<sup>[1]</sup> Other responses include: xxx

<sup>[2]</sup> Other responses include: xxx



Table 3.004 Characteristics of Longitudinal\* Staff Study Participants (Month 12/13), N=XX

| Question<br>Number | Characteristic | | Stud | y Arm |
|---|---|---|---|---|
| | | Total<br>(N=XX) | Dynamic<br>Implementation<br>(N=XX) | Routine<br>Implementation<br>(N=XX) |
| | | n (%) | n (%) | n (%) |
| 1 | Provider Type | | | |
| | Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Nurse Practitioner | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Physician Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Social worker/case manager | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Office administrator/clinic administrator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Laboratory staff/technician/phlebotomist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Front desk staff/ Scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 2 | Personally Administer Injections | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 3 | Prescribe Medications as part of role | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 4 | Currently Provide PrEP Counseling | | | |
| | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 103 | Specialty | | | |
| | Infectious disease specialist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Internal medicine/ primary care/general doctor/<br>family practitioner | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | HIC Specialist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Immunologist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Women's health/obstetricians and gynecologists | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Endocrinologist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other[2] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 104 | Length of Time practicing Medicine | | | |
| | <1 year | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 1–5 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | * | • | • |



| Question<br>Number | Characteristic | | Study Arm | |
|--------------------|----------------|------------|------------|------------|
| | 6–10 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 11-15 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | 16-20 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | >21 years | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

<sup>\*</sup> Longitudinal = SSPs who completed any portion of any questionnaire at Baseline, Month 4/5 and Month 12/13

<sup>[1]</sup> Other responses include: xxx

<sup>[2]</sup> Other responses include: xxx



Table 3.005 Summary of Confidence with Skills (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 5 | "Please rate your level of confidence for each skill listed." | | | | |
| | Talking to Patient About Sexual<br>History | Not At All Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Bit Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My<br>Role | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Screening a patient to determine whether they are an appropriate candidate for PrEP | Not At All Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Bit Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My<br>Role | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Answering Patient's Questions<br>About PrEP | Not At All Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Bit Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My<br>Role | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Suggesting PrEP to a Patient | Not At All Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Bit Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My<br>Role | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Counseling Pt Other Method of protection | Not At All Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Bit Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Very Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My<br>Role | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Monitoring a Patient on PrEP | Not At All Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A Little Bit Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Confident | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not Applicable To My<br>Role | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.006 Staff Study Participants' Perceptions Regarding APRETUDE (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 6 | In your opinion, APRETU[ | DE is appropriate for which individuals? | | | |
| | | Are sexually active | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have been sexually active with 1 or more partners in the last 6 months | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | are currently adherent on daily oral PrEP | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | are non-adherent on daily oral<br>PrEP | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | use PrEP on demand (i.e., event-<br>based PrEP, PrEP 2-1-1) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | could benefit from PrEP but do<br>not want to use daily PrEP | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have previously used and discontinued daily PrEP | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | feel stigmatized about taking oral<br>PrEP | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | request APRETUDE spontaneously | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have sex without a condom | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | engage in anal sex | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have a sexual partner living with HIV | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | live in areas with high HIV prevalence | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | currently have or recently (within<br>the past 6 months) have had an<br>STI other than HIV | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | are in monogamous relationships | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | inject drugs | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have sex with a person/people who inject drugs | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | experience stigma around using HIV prevention | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | are concerned about taking pills every day | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | experience stress or anxiety over adherence of a daily pill regimen | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have more chaotic lifestyles (e.g., variable work schedules, frequent travel, balancing work and school) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have more structured lifestyles<br>(e.g., regular work hours, little to<br>no unplanned travels) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have difficulty planning or organizing | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have stable income and stable housing | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | experience homelessness or are unstably housed | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have psychiatric comorbidities | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | have sex with someone who has recently been in jail/prison | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | are incarcerated, temporarily incarcerated, or recently released from incarcerated | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 7 | Are Individuals with specif | ic demographics more appropriate for | APRETUDE | ? | |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 8 | In your opinion, what are t | he demographics of the individuals w | ho are appro | ppriate for APRETU | DE? |
| | | Patients <35 years old | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Patients 35-50 years old | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Patients >50 years old | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Black transgender men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Black transgender women | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Black cisgender women | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|
| Black cisgender men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Black non-binary individuals | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Black men who have sex with men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| White transgender men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| White transgender women | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| White cisgender women | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| White cisgender men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| White non-binary individuals | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| White men who have sex with men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Latinx transgender men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Latinx transgender women | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Latinx cisgender women | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Latinx cisgender men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Latinx non-binary individuals | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Latinx men who have sex with men | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other transgender men of color | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other transgender women of color | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other cisgender women of color | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other cisgender men of color | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other non-binary individuals of color | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other men who have sex with men of color | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| tier | color Other men who have sex with men of color | color (XX.X%) Other men who have sex with XX (XX.X%) | color (XX.X%) XX (XX.X%) Other men who have sex with XX YY (XY.Y%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 10 | Are you or this clinic/pract | ice proactively informing patients abo | ut APRETUD | E? | |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 11 | How are you or this clinic/ | practice informing patients about APR | ETUDE? | | |
| | | Provision of educational materials | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | During consultation with patient | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Through peer educators | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Referring patients to PrEP providers | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Posters in the clinic/practice | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Flyers in the clinic/practice | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Mentions on the clinic/practice's website | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Mentions on social media | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.007 Summary of Experiences with the Acquisition Process (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 42 | | y of part of the benefits verification and<br>t forms, sending documents to insuranc | | | |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 43 | Is your clinic/practice ι | using ViiV Connect to acquire APRETUDE | Ξ? | | |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 44 | Do You Personally Use | ViiV Connect? | | | |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 45 | How are your provider | s or clinic/practice acquiring APRETUDE | ? | | |
| | | Buy-and-Bill — purchases<br>APRETUDE from a<br>wholesaler or specialty<br>distributor and bills the<br>primary third-party payer. | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | White Bagging — submits prescription to a specialty pharmacy within ViiV's specialty pharmacy network and the specialty pharmacy processes the claim and ships APRETUDE for administration. | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Clear Bagging – internal pharmacy maintains inventory of the medication, processes the claim, and delivers the medication. | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 46 | Who in your clinic/pra<br>APRETUDE? | Who in your clinic/practice is primarily responsible for completing the insurance benefits verification process for APRETUDE? | | | |
| | | Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse practitioner/physician assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Speciality pharmacy | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Medical assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Social worker/case manager | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Front desk staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Dedicated administrator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | APRETUDE coordinator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 47 | On average, how long | does it take to complete the APRETUDE | enrollment fo | orm? | |
| | | 1-5 minutes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 6-10 minutes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 11-15 minutes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 16-20 minutes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 21-25 minutes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 26-30 minutes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 31+ minutes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | I have not completed this form | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 48 | On average, how long has it t | aken to receive confirmation of b | enefits verific | cation for APRETUD | E? |
| | | 1-2 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 3-4 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 5-6 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 7-8 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 9-10 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 11-15 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 16-20 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 20-30 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 31-40 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 41-60 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 61+ days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 49 | On average, how long has it t | aken for patients to receive APRE | TUDE from th | ne point of benefits | verification? |
| | | 1-2 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 3-4 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 5-6 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 7-8 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 9-10 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 11-15 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 16-20 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | 21-30 days | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 50 | | e how concerned you are about<br>and knowledge of ViiV Connect." | each of the fo | ollowing based on yo | our current |
| | Authorization wait times | Extremely concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Understanding status of authorization | Extremely concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Understanding how to seek assistance | Extremely concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Amount of paperwork | Extremely concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Slightly concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Clarity on coverage approval | Extremely concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Ensuring medication comes to the right place (e.g., clinic/practice, pharmacy) | Extremely concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Potential loss of enthusiasm for APRETUDE by patients | Extremely concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Potential patient<br>dissatisfaction with clinic<br>staff | Extremely concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |


| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Slightly concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Staff dissatisfaction with the acquisition process | Extremely concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Potential disruption of clinic flow | Extremely concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Time-consuming process | Extremely concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Inequitable access for eligible patients | Extremely concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Moderately concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Slightly concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Not at all concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 51 | "Please indicate how much yo | u agree or disagree with each of the following statements." | | | |
| | I understand how to use ViiV<br>Connect (skip applicable if<br>Q44=yes) | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I understand how to<br>complete the APRETUDE<br>forms in ViiV Connect (skip<br>applicable if Q44=yes) | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Completing the benefits enrollment forms is easy (skip applicable if Q42=yes) | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Connec | The live support for ViiV<br>Connect is helpful (skip<br>applicable if Q43=yes) | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I am knowledgeable about<br>the patient savings card for<br>APRETUDE for patients (skip<br>applicable if Q42=yes) | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | The benefits verification process of ViiV Connect is time consuming (RC) (skip applicable if Q43=yes) | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I am satisfied with the<br>benefits verification process<br>(skip applicable if Q42=yes) | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | It has been easy to acquire<br>APRETUDE for patients (skip<br>applicable if Q42=yes) | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I know what to do if I am<br>having trouble acquiring<br>APRETUDE for patients (skip<br>applicable if Q42=yes) | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | I am knowledgeable about<br>the patient assistance<br>program for APRETUDE (skip<br>applicable if Q42=yes) | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 52 | How helpful or unhelpful has e | each type of support been to yo | ur clinic/pract | ice in using ViiV Cor | inect?" |
| | ViiV Connect Services and<br>Support information (e.g.,<br>ViiV Connect Brochure,<br>Provider Portal Brochure) | Not at all helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Did not use it | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | ViiV Connect Enrollment information (annotated enrollment forms, enrollment form) | Not at all helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Acquisition Guides (e.g.,<br>ordering guide, buy and bill<br>checklist, specialty<br>pharmacy checklist) | Not at all helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Billing, Coding and reimbursement information (e.g., prior authorization checklist, reimbursement guide) | Not at all helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Did not use it | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Benefits Verification —<br>understanding summary of<br>benefits (illustrated form<br>highlights patient benefit<br>summary and how to read<br>it) | Not at all helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Live support (e.g., access coordinators) | Not at all helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Video for patients on what is<br>ViiV Connect (DI) | Not at all helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | A video for providers<br>describing what is ViiV<br>Connect (DI) | Not at all helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Patient informational<br>material about ViiV Connect<br>and the acquisition process | Not at all helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Medication Acquisition Tracker – web-based tool to track patients' benefits acquisition journey from enrollment to medication receipt at the clinic/practice (DI) | Not at all helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | APRETUDE Payer Information found on the PILLAR Spot: spreadsheet updated on a weekly basis and gives providers information on which payers are covering APRETUDE and under what type of benefit | Not at all helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 53 | How helpful or unhelpful has r<br>began has been to your clinic/ | eceiving the list of payers/insur-<br>practice? | ers who cover | the medication and | d when coverage |
| | | Not at all helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very helpful | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Did not use it | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 54 | I would recommend ViiV Conn<br>medications. | ect to other providers and clinic | s/practices to | aid in the acquisition | on of ViiV |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |





Table 3.101 Summary of Acceptability of Intervention Measure (AIM – APRETUDE) and Feasibility of Intervention Measure (FIM – APRETUDE ) Items (Month 12/13), N=XX

| Measure | ltem | Study Arm | Total<br>Sample | 1<br>Completely<br>Disagree | 2<br>Disagree | 3<br>Neither<br>Agree<br>nor<br>Disagree | 4<br>Agree | 5<br>Completely<br>Agree |
|---|---|---|---|---|---|---|---|---|
| | | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| AIM | APRETUDE in our clinic/practice meets my approval. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 2. APRETUDE in our clinic/practice is appealing to me. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. I like APRETUDE in our clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. I welcome<br>APRETUDE in our<br>clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| FIM | APRETUDE seems implementable in our clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 2.APRETUDE seems possible in our clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |



| Measure | ltem | Study Arm | Total<br>Sample | 1<br>Completely<br>Disagree | 2<br>Disagree | 3<br>Neither<br>Agree<br>nor<br>Disagree | 4<br>Agree | 5<br>Completely<br>Agree |
|---|---|---|---|---|---|---|---|---|
| | | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. APRETUDE seems<br>doable in our<br>clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. APRETUDE seems easy to use in our clinic/practice | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |



Table 3.102 Distributional Characteristics of the Acceptability of Intervention Measure (AIM – APRETUDE) (Month 12/13), N=XX

| AIM – APRETUDE | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Intervention | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Routine Intervention | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test Degrees of Freedom P-Value | | X.XXX<br>XX<br>0.XXXX | | | | | |
| Site Volume<br>High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXXX | | | | | |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |



| AIM – APRETUDE | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | xx | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Items | | | | | | | |
| 1. APRETUDE in our clinic/practice meets my approval. | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |
| 2. APRETUDE in our clinic/practice is appealing to me. | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |
| 3. I like APRETUDE in our clinic/practice. | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |
| 4. I welcome APRETUDE in our clinic/practice. | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |

<sup>[1]</sup> Mid-level providers include nurse practitioners and physician assistants.



Table 3.103 Distributional Characteristics of the Feasibility of Intervention Measure (FIM – APRETUDE) (Month 12/13), N=XX

| FIM – APRETUDE | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Intervention | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Routine Intervention | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXXX | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Low | xx | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXXX | | | | | |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | xx | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |



| FIM – APRETUDE | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | xx | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Items | | | | | | | |
| 1. APRETUDE seems implementable in our clinic/practice. | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |
| 2.APRETUDE seems possible in our clinic/practice. | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |
| 3. APRETUDE seems doable in our clinic/practice. | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |
| 4. APRETUDE seems easy to use in our clinic/practice | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XX,<br>X.XX) |

<sup>[1]</sup> Mid-level providers include nurse practitioners and physician assistants.



Table 3.104 Changes from Baseline for Acceptability of Intervention Measure (AIM – APRETUDE) and Feasibility of Intervention Measure (FIM – APRETUDE) (Month 12/13), N=XX

| Measure | Study Arm | n | Mean | SD | Median (Q1, Q3) | Observed Range<br>(Minimum, Maximum) | Missing<br>n (%) | 95% CI<br>for the Mean |
|---|---|---|---|---|---|---|---|---|
| AIM - APRETUDE Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| AIM - APRETUDE Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| AIM - APRETUDE Change from Baseline to<br>Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| FIM - APRETUDE Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| FIM - APRETUDE Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| FIM - APRETUDE Change from Baseline to<br>Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |



Table 3.105 Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – APRETUDE) (Month 12/13), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 3.106 Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Acceptability of Intervention Measure (AIM – APRETUDE), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 3.107 Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – APRETUDE) (Month 12/13), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 3.108 Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Feasibility of Intervention Measure (FIM – APRETUDE), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 3.201 Summary of Acceptability of Intervention Measure (AIM – Implementation Support) and Feasibility of Intervention Measure (FIM – Implementation Support) Items (Month 12/13), N=XX

| Measure | ltem | Study Arm | Total<br>Sample<br>n (%) | 1<br>Completely<br>Disagree<br>n (%) | 2<br>Disagree<br>n (%) | 3<br>Neither<br>Agree<br>nor<br>Disagree<br>n (%) | 4<br>Agree<br>n (%) | 5<br>Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| | 1. The impulsor embedies | | 11 (70) | 11 (70) | 11 (70) | 11 (76) | 11 (70) | 11 (70) |
| AIM | The implementation support has met my approval. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 2. The implementation support was appealing to me. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. I like the implementation support I have received. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. I welcome the implementation support I have received. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| FIM | The implementation support seems implementable in our clinic/practice | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |



| Measure | ltem | Study Arm | Total<br>Sample<br>n (%) | 1<br>Completely<br>Disagree<br>n (%) | 2<br>Disagree<br>n (%) | 3<br>Neither<br>Agree<br>nor<br>Disagree<br>n (%) | 4<br>Agree<br>n (%) | 5<br>Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| | 2. The implementation support seems possible in our clinic/practice | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. The implementation support seems doable in our clinic/practice | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. The implementation support seems easy to use in our clinic/practice | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |



Table 3.202 Distributional Characteristics of the Acceptability of Intervention Measure (AIM – Implementation Support) (Month 12/13), N=XX

| AIM – Implementation Support | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXX | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXX | | | | | |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |



| AIM – Implementation Support | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Items | | | | | | | |
| 1. The implementation support has met my approval. | XX | X.X | X.XX | X.X (X.X, X.X) | X.X (X, X.) | XX<br>(XX.X) | (X.XX, X.XX) |
| 2. The implementation support was appealing to me. | XX | X.X | X.XX | X.X (X.X, X.X) | X.X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 3. I like the implementation support I have received. | XX | X.X | X.XX | X.X (X.X, X.X) | X.X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 4. I welcome the implementation support I have received. | XX | X.X | X.XX | X.X (X.X, X.X) | X.X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |

<sup>[1]</sup> Mid-level providers include nurse practitioners and physician assistants.



Table 3.203 Distributional Characteristics of the Feasibility of Intervention Measure (FIM – Implementation Support) (Month 12/13), N=XX

| FIM — Implementation Support | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXX | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXX | | | | | |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |



| FIM – Implementation Support | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% Cl<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Items | | | | | | | |
| The implementation support seems implementable in our clinic/practice | XX | X.X | X.XX | X.X (X.X, X.X) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XX, X.XX) |
| 2. The implementation support seems possible in our clinic/practice | XX | X.X | X.XX | X.X (X.X, X.X) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XX, X.XX) |
| 3. The implementation support seems doable in our clinic/practice | XX | X.X | X.XX | X.X (X.X, X.X) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XX, X.XX) |
| 4. The implementation support seems easy to use in our clinic/practice | XX | X.X | X.XX | X.X (X.X, X.X) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XX, X.XX) |



Table 3.204 Changes from Baseline to Acceptability of Intervention Measure (AIM – Implementation Support) and Feasibility of Intervention Measure (FIM – Implementation Support ) (Month 12/13), N=XX

| Measure | Study Arm | n | Mean | SD | Median (Q1, Q3) | Observed Range<br>(Minimum, Maximum) | Missing<br>n (%) | 95% Cl<br>for the Mean |
|---|---|---|---|---|---|---|---|---|
| AIM – Implementation Support Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| AIM - Implementation Support Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| AIM - Implementation Support Change from<br>Baseline to Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| FIM - Implementation Support Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| FIM - Implementation Support Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| FIM - Implementation Support Change from Baseline to Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |



Table 3.205 Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – Implementation Support) (Month 12/13), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 3.206 Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Acceptability of Intervention Measure (AIM – Implementation Support), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 3.207 Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – Implementation Support) (Month 12/13), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 3.208 Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Feasibility of Intervention Measure (FIM – Implementation Support), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 3.301 Summary of Acceptability of Intervention Measure (AIM – Telehealth) and Feasibility of Intervention Measure (FIM – Telehealth) Items (Month 12/13), N=XX

| Measure | ltem | Study Arm | Total<br>Sample | 1 2<br>Completely<br>Disagree Disagree | | 3<br>Neither<br>Agree<br>nor<br>Disagree | 4<br>Agree | 5<br>Completely<br>Agree |
|---|---|---|---|---|---|---|---|---|
| | | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| AIM | 1. Telehealth for<br>APRETUDE delivery in<br>our clinic/practice<br>meets my approval. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 2. Telehealth for APRETUDE delivery in our clinic/practice is appealing to me. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. I like using telehealth<br>for APRETUDE delivery<br>in our clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. I welcome telehealth<br>for APRETUDE delivery<br>in our clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| FIM | 1. Telehealth for<br>APRETUDE delivery<br>seems implementable<br>in our clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 2. Telehealth for<br>APRETUDE delivery | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |



| Measure | ltem | Study Arm | Total<br>Sample | 1<br>Completely<br>Disagree | 2<br>Disagree | 3<br>Neither<br>Agree<br>nor<br>Disagree | 4<br>Agree | 5<br>Completely<br>Agree |
|---|---|---|---|---|---|---|---|---|
| | | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | seems possible in our clinic/practice | | | | | | | |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 3. Telehealth for<br>APRETUDE delivery<br>seems doable in our<br>clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | 4. Telehealth for<br>APRETUDE delivery<br>seems easy to use in<br>our clinic/practice. | Overall | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Dynamic<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |
| | | Routine<br>Implementation | XX<br>(XX.X) | XX (XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX<br>(XX.X) | XX (XX.X) |



Table 3.302 Distributional Characteristics of the Acceptability of Intervention Measure (AIM – Telehealth) (Month 12/13), N=XX

| AIM – TELEHEALTH | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXX | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXX | | | | | |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |



| AIM – TELEHEALTH | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.X, X.X) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Items | | | | | | | |
| 1. Telehealth for APRETUDE in our clinic/practice meets my approval. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 2. Telehealth for APRETUDE in our clinic/practice is appealing to me. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 3. I like using telehealth for APRETUDE in our clinic/practice. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 4. I welcome telehealth for APRETUDE in our clinic/practice. | XX | X.X | X.XX | X.X (X.X, X.X) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |

<sup>[1]</sup> Mid-level providers include nurse practitioners and physician assistants.



Table 3.303 Distributional Characteristics of the Feasibility of Intervention Measure (FIM – Telehealth) (Month 12/13), N=XX

| FIM — TELEHEALTH | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Mean Score | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Routine Implementation | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXXX | | | | | |
| Site Volume | | | | | | | |
| High | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Low | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| T-test<br>Degrees of Freedom<br>P-Value | | X.XXX<br>XX<br>0.XXXX | | | | | |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| FQHC/Department of Health | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nonprofit | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Private | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Provider Type | | | | | | | |
| Physician | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Mid-level providers[1] | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Nurse | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Medical Assistant | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Pharmacist | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Social worker/case manager/PrEP<br>educator/PrEP navigator | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |


| FIM – TELEHEALTH | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Laboratory<br>staff/technician/phlebotomist/other | XX | X.XX | X.XXX | X.XX (X.XX,<br>X.XX) | X.X (X.XX, X.XX) | XX<br>(XX.X) | (X.XXX,<br>X.XXX) |
| Items | | | | | | | |
| 1. Telehealth for APRETUDE seems implementable in our clinic/practice | XX | X.X | X.XX | X.X (X.XX, X.XX) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 2. Telehealth for APRETUDE seems possible in our clinic/practice | XX | X.X | X.XX | X.X (X.XX, X.XX) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 3. Telehealth for APRETUDE seems doable in our clinic/practice | XX | X.X | X.XX | X.X (X.XX, X.XX) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |
| 4. Telehealth for APRETUDE seems easy to use in our clinic/practice | XX | X.X | X.XX | X.X (X.XX, X.XX) | X (X, X) | XX<br>(XX.X) | (X.XX, X.XX) |



Table 3.304 Changes from Baseline for Acceptability of Intervention Measure (AIM – Telehealth) and Feasibility of Intervention Measure (FIM – Telehealth) (Month 12/13), N=XX

| Measure | Study Arm | n | Mean | SD | Median (Q1, Q3) | Observed Range<br>(Minimum, Maximum) | Missing<br>n (%) | 95% CI<br>for the Mean |
|---|---|---|---|---|---|---|---|---|
| AIM – Telehealth Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| AIM - Telehealth Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| AIM - Telehealth Change from Baseline to<br>Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |
| FIM - Telehealth Baseline | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| FIM - Telehealth Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| FIM - Telehealth Change from Baseline to<br>Month 12/13 | Dynamic<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | Routine<br>Implementation | XX | X.XX | X.XXX | X.XX (X.XX, X.XX) | X.X (X.X, X.X) | XX (XX.X%) | (X.XXX, X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | 0.XXX | | | | | |



Table 3.305 Mixed-effects Modeling of the Acceptability of Intervention Measure (AIM – Telehealth) (Month 12/13), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 3.306 Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Acceptability of Intervention Measure (AIM – Telehealth), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | Т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 3.307 Mixed-effects Modeling of the Feasibility of Intervention Measure (FIM – Telehealth) (Month 12/13), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 3.308 Mixed-effects Modeling of the Changes from Baseline to Month 12/13 in Feasibility of Intervention Measure (FIM – Telehealth), N=XX

| Fixed effects | | | | | |
|---|---|---|---|---|---|
| Parameter | Estimate | Standard Error | Denominator<br>Degrees of<br>Freedom | т | p-Value |
| Intercept (RI, Low) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm (DI) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Volume (High) | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Study Arm by Volume | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Baseline Mean Score[1] | X.XX | X.XXX | XX | X.XX | 0.XXXX |
| Random Effects | | | | | |
| Covariance Parameter | Estimate | Standard Error | | Z | p-Value |
| Site Variance (τ(0,0)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Covariance (τ(0,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Baseline Variance (τ(1,1)) | X.XX | X.XXX | - | X.XX | 0.XXXX |
| Residual Variance (σ2) | X.XX | X.XXX | - | X.XX | 0.XXXX |

<sup>[1]</sup> Baseline mean score centered by site.



Table 3.309 Summary of Feasibility and Acceptability of Telehealth (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 16 | Does your clinic/prac | tice use any form of telehealth for APRE | TUDE delivery? | | |
| | | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 19 | What telehealth serv | ices does your clinic/practice provide fo | r APRETUDE? | _ | |
| | | Video consultation: using videoconferencing technology to facilitate a patient visit with both physician and patient present at the same time. | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Telephone consultation and visits | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Remote monitoring of patient health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Online appointment scheduling: ability for patients to make appointments without interacting with staff | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Patient portal conversations: ability for patients to send messages in an online portal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | At-home testing services: providers order tests and send to patient's home to complete | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sending and receiving patient reported outcomes questionnaires (e.g., quality of life, health behaviors), via an online system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Online prescription refill requests | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Online portal for patients to access medical documents, such as visit summaries and test results | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Text messaging with patients about care | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Email reminders to patients about upcoming visits | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Text reminders | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Automated phone call reminder | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Staff phone call reminder | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sending motivational reminders to help patients persist on APRETUDE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sending cabotegravir oral lead in to patient's home | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Insurance/benefits verification | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 20 | patients?" | o use the following telehealth syst | ·<br>- | T | |
| | Video consultation | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Telephone consultation | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Remote monitoring of | | | | |
| | patients | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | ŭ . | Very easy Somewhat Easy | XX (XX.X%) XX (XX.X%) | XX (XX.X%) XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| | ŭ . | , , | | | |
| | ŭ . | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | ŭ . | Somewhat Easy Neither easy nor difficult | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| | ŭ . | Somewhat Easy Neither easy nor difficult Somewhat Difficult | XX (XX.X%) XX (XX.X%) XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| | ŭ . | Somewhat Easy Neither easy nor difficult Somewhat Difficult Very Difficult | XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) | XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) | XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Patient portal conversations:<br>ability for patients to send<br>messages to providers | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | At-home testing services | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Send and receiving patient reported outcomes questionnaires (e.g., quality of life, health behaviors), via an online system | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Online prescription refills | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Online portal for patients to access medical documents, such as visit summaries and test results | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Text messaging with patients about care | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Email reminders to patient about upcoming visits | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Text reminders | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Automated phone call reminders | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Staff phone call reminder | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | Sending motivational reminders to help patients persist on APRETUDE | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Sending cabotegravir oral lead in to patient's home | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Insurance/benefits verification | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't use this system | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 21 | In the last 6 months, what proconsults, video)? | pportion of your APRETUDE visit | s would you est | imate were via teleł | nealth (e.g., tele- |
| | | None (0%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Few (1-30%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Some (31-65%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Most (66%-99%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All (100%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 23 | Why is telehealth not used by | your clinic/practice? | | | |
| | | Do not know how to use telehealth | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Telehealth is too expensive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Telehealth is too<br>impersonal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Telehealth does not allow<br>staff to do the necessary<br>physical exams | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Concerns about telehealth privacy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Lack of patient access to computers and/or the internet | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.310 Summary of Telehealth Services/Systems Used (Month 12/13), N=XX

| • | | | | ** | |
|---|---|---|---|---|---|
| 24. Which of the following telehealth services/systems is your clinic/practice using to deliver APRETUDE during the PILLAR study? | Total<br>Sample<br>n (%) | Yes, my clinic's<br>service/system<br>n (%) | Yes,<br>services/systems<br>offered through<br>PILLAR study<br>n (%) | No<br>n (%) | l don't<br>know<br>n (%) |
| A. Online system for<br>scheduling/rescheduling consultations<br>and injection appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | |
| University/Academia/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| B. Video/virtual consultations for initial and follow-up visits | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | |
| University/Academia/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| 24. Which of the following telehealth services/systems is your clinic/practice using to deliver APRETUDE during the PILLAR study? | Total<br>Sample<br>n (%) | Yes, my clinic's<br>service/system<br>n (%) | Yes,<br>services/systems<br>offered through<br>PILLAR study<br>n (%) | No<br>n (%) | l don't<br>know<br>n (%) |
|---|---|---|---|---|---|
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| C. Injection Administration: home health nurse to administer injection | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Study Arm | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | |
| University/Academia/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Social worker/case manager/PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| 24. Which of the following telehealth services/systems is your clinic/practice using to deliver APRETUDE during the PILLAR study? | Total<br>Sample<br>n (%) | Yes, my clinic's<br>service/system<br>n (%) | Yes,<br>services/systems<br>offered through<br>PILLAR study<br>n (%) | No<br>n (%) | l don't<br>know<br>n (%) |
|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D. Injection appointment reminders: text, digital, email | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | |
| University/Academia/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| E. HIV testing services: at home nurse testing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 24. Which of the following telehealth services/systems is your clinic/practice using to deliver APRETUDE during the PILLAR study? | Total<br>Sample<br>n (%) | Yes, my clinic's<br>service/system<br>n (%) | Yes,<br>services/systems<br>offered through<br>PILLAR study<br>n (%) | No<br>n (%) | I don't<br>know<br>n (%) |
|---|---|---|---|---|---|
| Clinic Type | | | | | |
| University/Academia/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.311 Summary of Ease of Use of Telehealth Services/Systems Used (Month 12/13), N=XX

| N-AA | | | | | | | |
|---|---|---|---|---|---|---|---|
| 25. How easy or difficult has each of the telehealth services/systems been for your clinic/practice to implement for the delivery of APRETUDE? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
| A. Online system for scheduling/rescheduling consultations and injection appointments | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X% |
| Site Volume | | | | | | | |
| High | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X% |
| Low | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X% |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X% |
| FQHC/Department of Health | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X% |
| Nonprofit | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X% |
| Private | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X% |
| Provider Type | | | | | | | |
| Physician | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X% |
| Mid-level providers[1] | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X% |
| Nurse | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X% |
| Medical Assistant | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X% |
| Pharmacist | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X% |
| Social worker/case<br>manager/PrEP educator/PrEP<br>navigator | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X% |



| 25. How easy or difficult has each of the telehealth services/systems been for your clinic/practice to implement for the delivery of APRETUDE? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/ot<br>her | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| B. Video/virtual consultations for initial and follow-up visits | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |



| 25. How easy or difficult has each of the telehealth services/systems been for your clinic/practice to implement for the delivery of APRETUDE? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Social worker/case<br>manager/PrEP educator/PrEP<br>navigator | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/ot<br>her | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| C. Injection Administration: home health nurse to administer injection | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |



| 25. How easy or difficult has each of the telehealth services/systems been for your clinic/practice to implement for the delivery of APRETUDE? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Pharmacist | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Social worker/case<br>manager/PrEP educator/PrEP<br>navigator | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/ot<br>her | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| D. Injection appointment reminders: text, digital, email | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |



| 25. How easy or difficult has each of the telehealth services/systems been for your clinic/practice to implement for the delivery of APRETUDE? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Medical Assistant | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Social worker/case<br>manager/PrEP educator/PrEP<br>navigator | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/ot<br>her | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| E. HIV testing services: at home nurse testing | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |



| 25. How easy or difficult has each of the telehealth services/systems been for your clinic/practice to implement for the delivery of APRETUDE? | Total<br>Sample<br>n (%) | Very<br>easy<br>n (%) | Somewhat<br>easy<br>n (%) | Neutral<br>n (%) | Somewhat<br>Difficult<br>n (%) | Very<br>difficult<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Nurse | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Social worker/case<br>manager/PrEP educator/PrEP<br>navigator | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/ot<br>her | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) |



Table 3.312 Summary of Helpfulness of Services/Systems Used (Month 12/13), N=XX

| 26. How helpful or unhelpful has each of the telehealth services/systems been to the delivery of APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>helpful<br>n (%) | Helpful<br>n (%) | Somewha<br>t helpful<br>n (%) | A little<br>Helpful<br>n (%) | Not at all<br>helpful<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| A. Online system for scheduling/rescheduling consultations and injection appointments | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Resear | XX | XX | XX | XX | XX | XX | XX |
| ch | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| FQHC/Department of Health | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Nonprofit | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Private | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Mid-level providers[1] | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Nurse | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Medical Assistant | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Pharmacist | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Social worker/case<br>manager/PrEP<br>educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| 26. How helpful or unhelpful has each of the telehealth services/systems been to the delivery of APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>helpful<br>n (%) | Helpful<br>n (%) | Somewha<br>t helpful<br>n (%) | A little<br>Helpful<br>n (%) | Not at all<br>helpful<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Laboratory<br>staff/technician/phlebotomis<br>t/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| B. Video/virtual consultations for initial and follow-up visits | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Resear | XX | XX | XX | XX | XX | XX | XX |
| ch | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| FQHC/Department of Health | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Nonprofit | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Private | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Mid-level providers[1] | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Nurse | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Medical Assistant | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Pharmacist | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Social worker/case<br>manager/PrEP<br>educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| 26. How helpful or unhelpful has each of the telehealth services/systems been to the delivery of APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>helpful<br>n (%) | Helpful<br>n (%) | Somewha<br>t helpful<br>n (%) | A little<br>Helpful<br>n (%) | Not at all<br>helpful<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Laboratory<br>staff/technician/phlebotomis<br>t/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| C. Injection Administration:<br>home health nurse to<br>administer injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Resear | XX | XX | XX | XX | XX | XX | XX |
| ch | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| FQHC/Department of Health | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Nonprofit | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Private | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Mid-level providers[1] | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Nurse | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Medical Assistant | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Pharmacist | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Social worker/case<br>manager/PrEP<br>educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| 26. How helpful or unhelpful has each of the telehealth services/systems been to the delivery of APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>helpful<br>n (%) | Helpful<br>n (%) | Somewha<br>t helpful<br>n (%) | A little<br>Helpful<br>n (%) | Not at all<br>helpful<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Laboratory<br>staff/technician/phlebotomis<br>t/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| D. Injection appointment reminders: text, digital, email | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Resear | XX | XX | XX | XX | XX | XX | XX |
| ch | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| FQHC/Department of Health | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Nonprofit | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Private | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Mid-level providers[1] | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Nurse | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Medical Assistant | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Pharmacist | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Social worker/case<br>manager/PrEP<br>educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| 26. How helpful or unhelpful has each of the telehealth services/systems been to the delivery of APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>helpful<br>n (%) | Helpful<br>n (%) | Somewha<br>t helpful<br>n (%) | A little<br>Helpful<br>n (%) | Not at all<br>helpful<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Laboratory<br>staff/technician/phlebotomis<br>t/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| E. HIV testing services: at home nurse testing | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Resear | XX | XX | XX | XX | XX | XX | XX |
| ch | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| FQHC/Department of Health | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Nonprofit | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Private | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Mid-level providers[1] | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Nurse | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Medical Assistant | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Pharmacist | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Social worker/case<br>manager/PrEP<br>educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



| 26. How helpful or unhelpful has each of the telehealth services/systems been to the delivery of APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>helpful<br>n (%) | Helpful<br>n (%) | Somewha<br>t helpful<br>n (%) | A little<br>Helpful<br>n (%) | Not at all<br>helpful<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Laboratory<br>staff/technician/phlebotomis<br>t/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 3.313 Summary of Satisfaction of Services/Systems Used (Month 12/13), N=XX

| 27. How satisfied or dissatisfied have you been with each of the telehealth services/systems for delivering APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>satisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Neither<br>satisfied<br>nor<br>dissatisfied<br>n (%) | Somewhat<br>dissatisfied<br>n (%) | Very<br>dissatisfied<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| A. Online system for scheduling/rescheduling consultations and injection appointments | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



| 27. How satisfied or dissatisfied have you been with each of the telehealth services/systems for delivering APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>satisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Neither<br>satisfied<br>nor<br>dissatisfied<br>n (%) | Somewhat<br>dissatisfied<br>n (%) | Very<br>dissatisfied<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| B. Video/virtual consultations for initial and follow-up visits | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| C. Injection Administration: home health nurse to administer injection | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



| 27. How satisfied or dissatisfied have you been with each of the telehealth services/systems for delivering APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>satisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Neither<br>satisfied<br>nor<br>dissatisfied<br>n (%) | Somewhat<br>dissatisfied<br>n (%) | Very<br>dissatisfied<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| D. Injection appointment reminders: text, digital, email | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |



| 27. How satisfied or dissatisfied have you been with each of the telehealth services/systems for delivering APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>satisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Neither<br>satisfied<br>nor<br>dissatisfied<br>n (%) | Somewhat<br>dissatisfied<br>n (%) | Very<br>dissatisfied<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| E. HIV testing services: at home nurse testing | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



| 27. How satisfied or dissatisfied have you been with each of the telehealth services/systems for delivering APRETUDE in your clinic/practice? | Total<br>Sample<br>n (%) | Very<br>satisfied<br>n (%) | Somewhat<br>satisfied<br>n (%) | Neither<br>satisfied<br>nor<br>dissatisfied<br>n (%) | Somewhat<br>dissatisfied<br>n (%) | Very<br>dissatisfied<br>n (%) | I have not<br>personally<br>used this<br>n (%) |
|---|---|---|---|---|---|---|---|
| Routine Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



Table 3.401 Summary of Utility of Proposed Implementation Strategies (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 28 | Have you used the following in the impl | ementation of AF | | | |
| 28A | Frequently Asked Questions Brochure | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 28B | Readiness Consideration | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 28C | Get Started Overview-Init/Adm Guide | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 28D | Injection Education Video | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 28E | Provider Website – location where all<br>materials and videos on APRETUDE for<br>the study is located | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 28F | Patient Materials | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 28G | Implementation Guidance Video | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 28H | Appointment Scheduler | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 281 | Pre-scheduled Appointment Guidance | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 28J | Designated Injection Days Guidance | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 28K | Drop-in Injection Visits Guidance | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 28L | Transport Support to Patient Appt | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 28M | Monthly Implement Facilitation Call | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 28N | Group Implement Facilitation Calls | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 280 | Document on How Discuss Sex Health | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 28P | PILLAR Spot | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Don't Know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29 | How often have you used the following | in the implement | ation of APRETUDE | into your practice/c | linic? |
| 29A | Frequent Ask Question Brochure | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29B | Readiness Consideration | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29C | Getting Started Overview | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29D | Injection Education Video | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29F | Patient Materials | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29G | Implementation Guidance Video | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29H | Appointment Scheduler | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 291 | Pre-scheduled Appt Guidance | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29J | Designated Inj Days Guidance | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29K | Drop-in Inj Visits Guidance | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29L | Transport Support to Pt Appt | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29M | Monthly Implement Facilit Call | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29N | Group Implement Facilit Calls | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 290 | Doc on How Discuss Sex Health | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 29P | PILLAR Spot | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |


| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 30 | How useful are the following in the impl | | | | 701 (701.7170) |
| 30A | Frequently Asked Questions Brochure | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 30B | Readiness Consideration | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 30C | OC Getting Started Overview-Init/Adm<br>Guide | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 30D | Injection Education Video | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 30E | Provider Website | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 30F | Patient Materials | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 30G | 0G Implementation Guidance Video | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 30H | Appointment Scheduler | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 301 | Pre-scheduled Appointment Guidance | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 30J | Designated Injection Days Guidance | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 30K | Drop-in Injection Visits Guidance | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 30L | Provid Transport Support to Patient<br>Appt | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 30M | OM Monthly Implementation Facilitation Call | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 30N | N Group Implementation Facilitation Calls | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 300 | Document on How to Discuss Sexual<br>Health | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 30P | PILLAR Spot | Not at all<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat<br>useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very Useful | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.501 Summary of Perceived Barriers to Delivering APRETUDE to Patients (Month 12/13), N=XX

| 55. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| A. Patients' ability to keep appointments | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



| 55. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| B. Patients' injection-related pain/soreness | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



| 55. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| C. Risk of drug resistance for patients not adherent to injections | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| D. Cost of APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



| 55. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| E. Keeping a patient engaged and motivated to continue APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | |



| 55. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP<br>educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| F. Identifying eligible individuals for<br>APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



| 55. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| G. Worried that a patient will feel stigmatized if offered APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



| 55. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| H. Patients' willingness to travel every<br>2 months for an injection<br>appointment | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | |



| 55. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| I. Patient lack of belief in the efficacy of APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



| 55. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) |



Table 3.502 Summary of Perceptions of Administering APRETUDE (Month 12/13), N=XX

| 56. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| A. Difficulty of giving the gluteal medial injection | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia<br>/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level<br>providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case<br>manager/PrEP<br>educator/PrEP<br>navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator<br>/clinic<br>administrator/front<br>desk staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phl<br>ebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 56. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| B. Understanding how<br>to manage patients<br>who miss an injection<br>dose | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia<br>/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level<br>providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case<br>manager/PrEP<br>educator/PrEP<br>navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator<br>/clinic<br>administrator/front<br>desk staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phl<br>ebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 56. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| C. How to transition patients off of APRETUDE who want to stop taking it (e.g., should other PrEP be offered) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia<br>/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level<br>providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case<br>manager/PrEP<br>educator/PrEP<br>navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator<br>/clinic<br>administrator/front<br>desk staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 56. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Laboratory<br>staff/technician/phl<br>ebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D. Understanding how<br>to use oral PrEP<br>medication for a<br><u>planned</u> missed<br>injection visit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia<br>/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level<br>providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case<br>manager/PrEP<br>educator/PrEP<br>navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator<br>/clinic | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 56. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| administrator/front<br>desk staff/scheduler | | | | | | |
| Laboratory<br>staff/technician/phl<br>ebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| E. Understanding how<br>to restart APRETUDE<br>after a missed<br>injection | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia<br>/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level<br>providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case<br>manager/PrEP<br>educator/PrEP<br>navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator<br>/clinic | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 56. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| administrator/front<br>desk staff/scheduler | | | | | | |
| Laboratory<br>staff/technician/phl<br>ebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. Managing the oral<br>lead-in phase of<br>APRETUDE before<br>starting injections if<br>needed | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia<br>/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level<br>providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case<br>manager/PrEP<br>educator/PrEP<br>navigator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 56. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat Slightly concerned concerned n (%) n (%) | | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Office administrator<br>/clinic<br>administrator/front<br>desk staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phl<br>ebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| G. Ability to provide<br>adherence counseling<br>and support when<br>injection dosing visits<br>are missed | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia<br>/Research | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level<br>providers[1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case<br>manager/PrEP | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 56. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE administration based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | Extremely<br>concerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| educator/PrEP<br>navigator | | | | | | |
| Office administrator<br>/clinic<br>administrator/front<br>desk staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phl<br>ebotomist/other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.503 Summary of Perceived Barriers to Managing Delivery of APRETUDE (Month 12/13), N=XX

| 57. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | ple con | | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| A. Management of scheduling injection appointments every 2 months during correct injection (I.e., dosing) windows | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| concerned you would be S | Total<br>ample | conc | erned | Moderately concerned | Somewhat concerned | Slightly<br>concerned | Not at all concerned |
|---|---|---|---|---|---|---|---|
| about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | n (%) | n | (%) | n (%) | n (%) | n (%) | n (%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Laboratory<br>staff/technician/phlebotomist/otl | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| B. Management of rescheduling appointments during correct injecti (I.e., dosing) windows | on I | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Study Arm | | | | | | | |
| Dynamic Implementation | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Routine Implementation | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | | | |
| High | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | | | |
| University/Academia/Research | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | | | |
| Physician | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Social worker/case manager/PrEP educator/PrEP navigator | | XX<br>X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| concerned you would be Sa | otal<br>imple<br>i (%) | cond | emely<br>cerned<br>(%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | | XX<br>(XX.X%) | XX (XX.X% | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/oth | er | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. Ability to schedule/reschedule patients who missed APRETUDE visit within correct injection (I.e., dosing) windows | | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | | XX<br>(XX.X%) | XX (XX.X% | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | | |
| Physician | | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| concerned you would be | Total<br>Sample<br>n (%) | cond | remely<br>cerned<br>(%) | CO | derately<br>ncerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| on your current expectations and knowledge. | | | | | | | | |
| Social worker/case manager/PrEl<br>educator/PrEP navigator | D | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Laboratory<br>staff/technician/phlebotomist/ot | :her | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| D. Ability to identify and flag misser injection visits to providers (in a timely manner) | d | XX<br>(XX.X%) | XX (XX.X9 | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Study Arm | | | | | | | | |
| Dynamic Implementation | | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Routine Implementation | | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | | | | |
| High | | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | | | | |
| University/Academia/Research | | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | | | | |
| Physician | | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | | XX<br>(XX.X%) | XX (XX.X% | %) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| concerned you would be about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations | otal<br>imple<br>i (%) | con | remely<br>cerned<br>(%) | Moderatel<br>concerned<br>n (%) | | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| and knowledge. Social worker/case manager/PrEP educator/PrEP navigator | // | XX<br>X.X%) | XX (XX.X% | S) XX (X | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic administrator/front desk staff/scheduler | | XX<br>XXX.X%) | XX (XX.X% | 5) XX (X) | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/oth | er (X | XX<br>X.X%) | XX (XX.X% | S) XX (X | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| E. Ability to manage patients presenting to APRETUDE injection appointments with other care needs that need to be addressed | s (X | XX<br>X.X%) | XX (XX.X% | S) XX (X) | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic Implementation | (X | XX<br>X.X%) | XX (XX.X% | S) XX (X) | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | (X | XX<br>X.X%) | XX (XX.X% | S) XX (X) | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | (X | XX<br>X.X%) | XX (XX.X% | S) XX (X) | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | (X | XX<br>X.X%) | XX (XX.X% | S) XX (X) | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | | | |
| University/Academia/Research | (X | XX<br>X.X%) | XX (XX.X% | S) XX (X) | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | (X | XX<br>X.X%) | XX (XX.X% | S) XX (X) | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | (X | XX<br>X.X%) | XX (XX.X% | S) XX (X) | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | (X | XX<br>X.X%) | XX (XX.X% | S) XX (X | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | | | |
| Physician | (X | XX<br>X.X%) | XX (XX.X% | S) XX (X) | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | (X | XX<br>X.X%) | XX (XX.X% | S) XX (X) | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | (X | XX<br>X.X%) | XX (XX.X% | S) XX (X) | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | (X | XX<br>X.X%) | XX (XX.X% | S) XX (X) | X.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| concerned you would be Sa | otal<br>mple<br>(%) | cond | remely<br>cerned<br>(%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|---|
| Pharmacist | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/oth | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. Persistence to follow up with patient on missed appointments | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Study Arm | | | | | | | |
| Dynamic Implementation | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Routine Implementation | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | | | |
| High | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | | | |
| University/Academia/Research | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | | | |
| Physician | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| 57. Please indicate how To concerned you would be Sam about each of the following n ( | ple con | remely<br>cerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat concerned n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| being a barrier or challenge<br>to APRETUDE delivery based<br>on your current expectations<br>and knowledge. | | | | | | |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| G. Provider time to discuss HIV prevention with all eligible patients | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| 57. Please indicate how concerned you would be about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations | Total<br>Sample<br>n (%) | cond | emely<br>cerned<br>(%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|---|
| and knowledge. | | | | | | | |
| Pharmacist | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrE educator/PrEP navigator | [P | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/o | ther | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| H. Ability to provide HIV screening indicated at each injection visit and provide rapid intervention/followbased on results status | d | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | | |
| Physician | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| concerned you would be Sa | otal<br>mple<br>(%) | le concerned | | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|---|
| Medical Assistant | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/oth | er (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| I. HIV monitoring requirements associated with APRETUDE | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | | |
| Physician | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| concerned you would be Sa | Fotal<br>ample<br>n (%) | le concerned | | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|---|
| Medical Assistant | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Social worker/case manager/PrEP educator/PrEP navigator | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Laboratory<br>staff/technician/phlebotomist/oth | ner (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| J. Cost/coverage of ancillary services to provide APRETUDE | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Study Arm | | | | | | | |
| Dynamic Implementation | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Routine Implementation | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | | | |
| High | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | | | |
| University/Academia/Research | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | (X | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | | | |
| Physician | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | | XX<br>X.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| 57. Please indicate how Concerned you would be San about each of the following being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | iple con | | foderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/othe | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.504 Summary of Perceived Resourcing Barriers to Support Delivery of APRETUDE (Month 12/13), N=XX

| 58. Please indicate how | | | | | | | |
|---|---|---|---|---|---|---|---|
| concerned you would be about each of the following potentially being a barrier or challenge to APRETI IDE | Fotal<br>ample<br>n (%) | con | remely<br>cerned<br>(%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
| A. Staff resourcing to ensure appropriate clinic flow | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | | | |
| High | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | | | |
| University/Academia/Research | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | | | |
| Physician | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Social worker/case manager/PrEP educator/PrEP navigator | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| 58. Please indicate how concerned you would be about each of the following potentially being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | ole con | remely<br>cerned<br>ı (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| B. Number of exam rooms for injections | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| 58. Please indicate how concerned you would be about each of the following potentially being a barrier or challenge to APRETUDE delivery based on your current expectations and | ple co | tremely<br>ncerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| knowledge. Laboratory | XX | VV (VV V0) | ) | VV (VV VV) | VV (VV V0/) | VOV (VOV VOV) |
| staff/technician/phlebotomist/other | (XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. Clinic staff to administer injections | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| potentially being a barrier or Sar | rtal<br>nple<br>(%) | Extremely concerned n (%) | | loderately<br>oncerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|---|
| knowledge. | | | | | | | |
| Laboratory<br>staff/technician/phlebotomist/othe | XX<br>(XX.X | XX (XX ) | <b>(%</b> ) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| D. Staff preparation (i.e., education, training, in-services) to implement APRETUDE | XX<br>(XX.X | XX (XX ) | <b>(%</b> ) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX<br>(XX.X | XX (XX ) | <b>(%</b> ) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Routine Implementation | XX<br>(XX.X | XX (XX ) | <b>(%</b> ) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X | XX (XX ) | <b>(%</b> ) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | XX<br>(XX.X | XXIXXX | <b>(%</b> ) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | | | |
| University/Academia/Research | XX<br>(XX.X | XXIXXX | <b>(%</b> ) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | XX<br>(XX.X | XX (XX ) | <b>(%</b> ) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | XX<br>(XX.X | XXIXXX | <b>(%</b> ) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | XX<br>(XX.X | XX (XX ) | <b>(%</b> ) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | | | |
| Physician | XX<br>(XX.X | XX (XX ) | <b>(%</b> ) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | XX<br>(XX.X | YY / YY Y | <b>(%</b> ) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | XX<br>(XX.X | XXIXXX | (%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | XX<br>(XX.X | X X ( X X ) | (%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | XX<br>(XX.X | YY / YY Y | <b>(%</b> ) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X | X X ( X X ) | (%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| potentially being a barrier or S | Total<br>ample<br>n (%) | e concerned | | Moderately<br>concerned<br>n (%) | Somewhat concerned n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|---|
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | (: | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/oth | ner ( | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| E. Staff time to provide counseling<br>and support to patients, such as<br>answering questing between visit,<br>keeping patients motivated | (: | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | (: | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | () | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | (: | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | () | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clinic Type | | | | | | | |
| University/Academia/Research | (: | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| FQHC/Department of Health | () | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nonprofit | () | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Private | () | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Provider Type | | | | | | | |
| Physician | () | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mid-level providers[1] | ( | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | () | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | (: | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | () | XX<br>XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |


| about each of the following potentially being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | ole cor | remely<br>ocerned<br>n (%) | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|
| Social worker/case manager/PrEP educator/PrEP navigator | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Laboratory<br>staff/technician/phlebotomist/other | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| F. Staff belief in the efficacy of<br>APRETUDE | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Study Arm | | | | | | |
| Dynamic Implementation | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Routine Implementation | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Site Volume | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Low | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Clinic Type | | | | | | |
| University/Academia/Research | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| FQHC/Department of Health | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nonprofit | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Private | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Provider Type | | | | | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Mid-level providers[1] | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | ) XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |



| 58. Please indicate how concerned you would be about each of the following potentially being a barrier or challenge to APRETUDE delivery based on your current expectations and knowledge. | Total<br>Sample<br>n (%) | e con | | Moderately<br>concerned<br>n (%) | Somewhat<br>concerned<br>n (%) | Slightly<br>concerned<br>n (%) | Not at all<br>concerned<br>n (%) |
|---|---|---|---|---|---|---|---|
| Social worker/case manager/PrE educator/PrEP navigator | Р | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Office administrator /clinic<br>administrator/front desk<br>staff/scheduler | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Laboratory<br>staff/technician/phlebotomist/o | ther | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.505 Summary of Perceptions of Clinic/Practice Culture and Environment (Month 12/13), N=XX

| 59. How much do you agree or disagree with the following statements about your clinic/practice? | Total<br>Sample<br>n (%) | Completely<br>Disagree<br>n (%) | Disagree<br>n (%) | Neither<br>agree nor<br>disagree<br>n (%) | Agree<br>n (%) | Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|
| A. People at all levels openly talk about what is and isn't working | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| B. Most people in this clinic<br>are willing to change how<br>they do things in response to<br>feedback from others | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. It is hard to get things to change in our clinic | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D. People in this clinic operate as a real team | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | | | | | | |
| Site Volume | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | | | | | | |
| E. Staff members often show signs of stress and strain | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 59. How much do you agree or disagree with the following statements about your clinic/practice? | Total<br>Sample<br>n (%) | Completely<br>Disagree<br>n (%) | Disagree<br>n (%) | Neither<br>agree nor<br>disagree<br>n (%) | Agree<br>n (%) | Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. We regularly take time to consider ways to improve how we do things | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| G. Leadership strongly supports clinic change efforts | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.506 Summary of Barriers to PrEP Provisioning (Month 12/13), N=XX

| <u> </u> | | | | * ** | | |
|---|---|---|---|---|---|---|
| 96. Indicate your level of agreement with the following statements: | Total<br>Sample<br>n (%) | Completely<br>Disagree<br>n (%) | Disagree<br>n (%) | Neither<br>agree nor<br>disagree<br>n (%) | Agree<br>n (%) | Completely<br>Agree<br>n (%) |
| A. The use of PrEP will cause patients to engage in riskier behaviors | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| B. Providing PrEP endorses the risk behaviors of users | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| C. Only people who engage in risky behavior need PrEP | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D. Only people with many sexual partners need PrEP | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | | | | | | |
| Site Volume | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | | | | | | |
| E. All sexually active people can benefit from PrEP | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| 96. Indicate your level of agreement with the following statements: | Total<br>Sample<br>n (%) | Completely<br>Disagree<br>n (%) | Disagree<br>n (%) | Neither<br>agree nor<br>disagree<br>n (%) | Agree<br>n (%) | Completely<br>Agree<br>n (%) |
|---|---|---|---|---|---|---|
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| F. Providing PrEP will result<br>in an increase in sexually<br>transmitted diseases among<br>patients | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| G. People do not need PrEP if they act responsibly | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.507 Distributional Characteristics of Barriers to PrEP Provisioning (Month 12/13), N=XX

| 96. Indicate your level of agreement with the following statements: | Study Arm | n | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum,<br>Maximum) | Missing | 95% CI<br>for the<br>Mean |
|---|---|---|---|---|---|---|---|---|
| | Dynamic<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| A. The use of PrEP will cause patients to engage in | Routine<br>Implementation | XX | X.XXX | x.xxxx | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| riskier behaviors | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | X.XXX | | | | | |
| | Dynamic<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| B. Providing PrEP<br>endorses the risk<br>behaviors of users | Routine<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | X.XXX | | | | | |
| | Dynamic<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| C. Only people<br>who engage in<br>risky behavior | Routine<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| need PrEP | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | X.XXX | | | | | |
| | Dynamic<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| D. Only people<br>with many sexual<br>partners need | Routine<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| PrEP | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | X.XXX | | | | | |
| E. All sexually<br>active people can<br>benefit from PrEP | Dynamic<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |



| 96. Indicate your<br>level of<br>agreement with | Study Arm | n | Mean | SD | Median | Observed<br>Range | Missing | 95% CI |
|---|---|---|---|---|---|---|---|---|
| the following statements: | | | | | (Q1, Q3) | (Minimum,<br>Maximum) | n (%) | for the<br>Mean |
| | Routine<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | X.XXX | | | | | |
| F. Providing PrEP | Dynamic<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| will result in an<br>increase in<br>sexually<br>transmitted | Routine<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| diseases among | T-test | | X.XXX | | | | | |
| patients | DF | | XX | | | | | |
| | P-Value | | X.XXX | | | | | |
| | Dynamic<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| G. People do not<br>need PrEP if they<br>act responsibly | Routine<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| act responding. | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | X.XXX | | | | | |
| | Dynamic<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| Total Score | Routine<br>Implementation | XX | X.XXX | X.XXXX | X.XX<br>(X.XX,<br>X.XX) | X.XX (X.XX,<br>X.XX) | XX (XX.X) | (X.XXX,<br>X.XXX) |
| | T-test | | X.XXX | | | | | |
| | DF | | XX | | | | | |
| | P-Value | | X.XXX | | | | | |



Table 3.508 Shift from Month 4/5 to Month 12/13 in Summary of Perceived Barriers to Delivering APRETUDE to Patients (Month 12/13), N=XX

55. Please indicate how concerned you would be about each of the following being a barrier or challenge to delivering APRETUDE to patients based on your current expectations and knowledge.

#### A. Patients' ability to keep appointments

| | | | | | | M12/13 | | | |
|---|---|---|---|---|---|---|---|---|---|
| Study Arm | N | M4/5 | Extremely<br>Concerned | Moderately<br>Concerned | Somewhat<br>Concerned | Slightly<br>Concerned | Not at all<br>Concerned | Missing | Total |
| | | Extremely<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| | | Moderately<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| | | Somewhat<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| DI | XX | Slightly Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| | | Not at all<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| | | Missing | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| | | Total | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| RI | XX | Extremely<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |



| Moderately<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
|-------------------------|------|------|------|------|------|------|------|
| Somewhat<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| Slightly Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| Not at all<br>Concerned | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| Missing | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |
| Total | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) | n(%) |

Note 1: Shift tables will be created as above for items 55b through 55i.

Note 2: Only includes respondents who completed surveys at respective months.

Missing: M4/5 = missing item at M4/5 but not M12/13. M12/13 = missing item at M12/13 but not M4/5.

Percentage calculations:

Column total %: numerator= number selecting respective response at M12/13, denominator = number responding at M12/13

Row total %: numerator= number selecting respective response at M4/5, denominator = number responding at M4/5

Cell %: numerator = number selecting respective combination of M4/5 and M12/13 responses, denominator=number of participants responding at M4/5.

Total: N = number of participants that completed the question at either M4/5 or M12/13

### Table 3.509 Shift from Month 4/5 to Month 12/13 in Summary of Perceptions of Administering APRETUDE (Month 12/13), N=XX

Note 1: Shift tables will be created as shown for Table 3.508 for items 56a through 56g.

Note 2: Only includes respondents who completed surveys at respective months.

Missing: M4/5 = missing item at M4/5 but not M12/13. M12/13 = missing item at M12/13 but not M4/5.

Percentage calculations:

Column total %: numerator= number selecting respective response at M12/13, denominator = number responding at M12/13

Row total %: numerator= number selecting respective response at M4/5, denominator = number responding at M4/5

Cell %: numerator = number selecting respective combination of M4/5 and M12/13 responses, denominator=number of participants responding at M4/5.

Total: N = number of participants that completed the question at either M4/5 or M12/13



# Table 3.510 Shift from Month 4/5 to Month 12/13 in Summary of Perceived Barriers to Managing Delivery of APRETUDE (Month 12/13), N=XX

Note 1: Shift tables will be created as shown for Table 3.508 for items 57a through 57i.

Note 2: Only includes respondents who completed surveys at respective months.

Missing: M4/5 = missing item at M4/5 but not M12/13. M12/13 = missing item at M12/13 but not M4/5.

Percentage calculations:

Column total %: numerator = number selecting respective response at M12/13, denominator = number responding at M12/13

Row total %: numerator= number selecting respective response at M4/5, denominator = number responding at M4/5

Cell %: numerator = number selecting respective combination of M4/5 and M12/13 responses, denominator=number of participants responding at M4/5.

Total: N = number of participants that completed the question at either M4/5 or M12/13

## Table 3.511 Shift from Month 4/5 to Month 12/13 in Summary of Perceived Resourcing Barriers to Support Delivery of APRETUDE (Month 12/13), N=XX

Note 1: Shift tables will be created as shown for Table 3.508 for items 58a through 58f.

Note 2: Only includes respondents who completed surveys at respective months.

Missing: M4/5 = missing item at M4/5 but not M12/13. M12/13 = missing item at M12/13 but not M4/5.

Percentage calculations:

Column total %: numerator= number selecting respective response at M12/13, denominator = number responding at M12/13

Row total %: numerator= number selecting respective response at M4/5, denominator = number responding at M4/5

Cell %: numerator = number selecting respective combination of M4/5 and M12/13 responses, denominator=number of participants responding at M4/5.

Total: N = number of participants that completed the question at either M4/5 or M12/13

# Table 3.512 Shift from Month 4/5 to Month 12/13 in Summary of Perceptions of Clinic/Practice Culture and Environment (Month 12/13), N=XX

Note 1: Shift tables will be created as shown for Table 3.508 for items 59a through 59g.

Note 2: Only includes respondents who completed surveys at respective months.

Missing: M4/5 = missing item at M4/5 but not M12/13. M12/13 = missing item at M12/13 but not M4/5.

Percentage calculations:

Column total %: numerator= number selecting respective response at M12/13, denominator = number responding at M12/13

Row total %: numerator= number selecting respective response at M4/5, denominator = number responding at M4/5



Cell %: numerator = number selecting respective combination of M4/5 and M12/13 responses, denominator=number of participants responding at M4/5.

Total: N = number of participants that completed the question at either M4/5 or M12/13

### Table 3.513 Shift from Month 4/5 to Month 12/13 in Summary of Barriers to PrEP Provisioning (Month 12/13), N=XX

Note 1: Shift tables will be created as shown for Table 3.508 for items 96a through 96g.

Note 2: Only includes respondents who completed surveys at respective months.

Missing: M4/5 = missing item at M4/5 but not M12/13. M12/13 = missing item at M12/13 but not M4/5.

Percentage calculations:

Column total %: numerator= number selecting respective response at M12/13, denominator = number responding at M12/13

Row total %: numerator= number selecting respective response at M4/5, denominator = number responding at M4/5

Cell %: numerator = number selecting respective combination of M4/5 and M12/13 responses, denominator=number of participants responding at M4/5.

Total: N = number of participants that completed the question at either M4/5 or M12/13



Table 3.601 Summary of the Sexual Health Assessment Tool (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 31 | Has your clinic/practice started | to use the Sexual Health Assessm | nent? | | |
| | | No And Not Planning To Use<br>The Sexual Health Assessment | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No But Planning To Use The<br>Sexual Health Assessment | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | l Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 32 | Who in your clinic/practice is o | r will be responsible for distributir | ng the Sexual | Health Assessment | to patients? |
| | | Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse practitioner/physician assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Medical assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Social worker/case manager | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Front desk staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Peer educator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 33 | Who in your clinic/practice is o<br>Assessment with patients? | r will be responsible for reviewing | and discussi | ng the results of th | e Sexual Health |
| | | Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse practitioner/physician assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Medical assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Social worker/case manager | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Front desk staff/scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Peer educator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The results are or will not be discussed with patients | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 34 | How often have you used the S | Sexual Health Assessment in your | clinic/practic | e? | |
| | | Rarely | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 35 | "Please indicate your level of agreement with the following statements about the Sexual Health Assessment." | | | | |
| | The Sexual Health Assessment is/will be easy to implement in my clinic/practice | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | The Sexual Health<br>Assessment is/will be an easy<br>way to identify individuals<br>interested in PrEP | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | The Sexual Health Assessment helps/will help to facilitate conversations about PrEP with patients | Completely disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 36 | Why is the Sexual Health Assessment not used by your clinic/practice? | | | | |
| | | Already have a similar assessment | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Does not integrate with the EMR | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The assessment is difficult to administer | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Concerns about patient privacy | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The assessment does not ask the right questions | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The assessment takes too much time | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The assessment is not needed | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.602 Summary of the PrEP Communication Tool (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 37 | Has your clinic/practice started to use PrEP Options Communication Tool? | | | | |
| | | No and not planning to use the PrEP<br>Options Communication Tool | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No but planning to use the PrEP<br>Options Communication Tool | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 38 | Who in your clinic/<br>patients? | practice is or will be responsible for using | the PrEP Option | ons Communication | Tool with |
| | | Physician | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse practitioner/physician assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Medical assistant | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Social worker/case manager | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Front desk staff/scheduler | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Peer educator | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 39 | How often have you used the PrEP Options Communication Tool in your clinic/practice? | | | | |
| | | Rarely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Sometimes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Often | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | All the time | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 40 | Please indicate you<br>Tool | r level of agreement with the following st | atements abo | ut the PrEP Options | Communication |
| | The PrEP Options<br>Communication<br>Tool is/will be<br>easy to<br>implement in my<br>clinic/practice | Completely disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | The PrEP Options Communication Tool helps/will help to facilitate conversations about PrEP with patients | Completely disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither agree nor disagree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 41 | Why is the PrEP Options Communication Tool not used by your clinic/practice? | | | | |
| | | Already have a similar tool | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Do not have time in a clinical visit to use the tool | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Do not understand the information in the tool | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Tool does not provide the right information | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Tool is not needed | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.701 Summaries of the Optional Oral Lead-in Phase of APRETUDE (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 79 | How do you start your patie | ents with APRETUDE? | | | |
| | | directly with injection | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | With optional oral lead-in using oral cabotegravir | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | With oral PrEP (TDF/FTC or TAF/FTC) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 80 | "Of all your patients who h | ave been prescribed APRETUDE, ple | ease estimate t | he percentage that | started:" |
| | Directly with injection<br>who switched from oral<br>PrEP | N | XX | XX | XX |
| | | Mean (SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | | Range (Min, Max) | XX (XX, XX) | XX (XX, XX) | XX (XX, XX) |
| | Directly with injection who are new to PrEP | N | XX | XX | XX |
| | | Mean (SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | | Range (Min, Max) | XX (XX, XX) | XX (XX, XX) | XX (XX, XX) |
| | With optional oral lead-in (oral Cabotegravir) | N | XX | XX | XX |
| | | Mean (SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | | Range (Min, Max) | XX (XX, XX) | XX (XX, XX) | XX (XX, XX) |
| | With oral PrEP (TDF/FTC or TAF/FTC) | N | XX | XX | XX |
| | | Mean (SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | | Range (Min, Max) | XX (XX, XX) | XX (XX, XX) | XX (XX, XX) |
| | Other | N | XX | XX | XX |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Mean (SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | | Median | XX.X | XX.X | XX.X |
| | | Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | | Range (Min, Max) | XX (XX, XX) | XX (XX, XX) | XX (XX, XX) |
| 81 | What sources of info | rmation have you drawn upon in assessin | g whether oral | lead-in is needed o | r not? |
| | | Scientific literature | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Independent Medical<br>Education | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Data from ViiV/GSK | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Scientific conferences | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Clinic rounds | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | CDC guidelines | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other medical colleagues | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other sources | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 82 | What are the main fa | actors that drive your decision to use oral | lead-in or not? | | |
| | | The ability to assess the safety/tolerability of APRETUDE in all patients | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The ability to assess the safety/tolerability of APRETUDE in patients with a history of allergy/drug intolerance | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The availability of more data from clinical trials using an oral lead-in phase | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | The ability to increase drug concentration before starting the injections | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Being cautious with a new medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Providing patient with protection against HIV until the injection arrives | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Patient request | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Enough data exists from clinical trials to start patients with injection without oral lead in | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Provide patients with immediate protection with a long acting method by not using oral lead in | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 83 | How influential are patient preferences in the decision of whether or not to use an oral lead-in phase? | | | | |
| | | Very influential | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Influential | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat influential | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not very influential | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all influential | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 84 | Have any of your pa | tients missed injection visit(s)? | | | |
| | | No, none of my patients have missed their injection visits | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Yes, some of my patients have had planned missed visits | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Yes, some of my patients have had unplanned missed visits | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 85 | For patients who have missed an injection visit, what protection were they given/offered until they received their next injection? | | | | |
| | | Cabotegravir oral tablets | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | TDF/FTC | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | TAF/FTC | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Provision of condoms | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Risk reduction education | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | None | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Do not know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 86 | For patients who pla<br>next injection? | an to miss an injection, what protection do | o you plan on of | fering them until th | ey receive their |
| | | Cabotegravir oral tablets | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | TDF/FTC | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | TAF/FTC | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Provision of condoms | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Risk reduction education | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | None | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Do not know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 87 | How easy or difficul | t was it to start patients on oral PrEP for a | | | , |
| | , | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 88 | How acceptable was it t | o start patients on oral PrEP after a mi | issed injection v | visit? | |
| | | Very acceptable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Acceptable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Acceptable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Acceptable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Acceptable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 89 | Before initiating a patier | nt on PrEP, what type of HIV test do yo | ou primarily use | ? | |
| | Oral PrEP | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4th gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/ antibody test<br>(rapid test) 4th gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test)<br>3rd gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | APRETUDE | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4th gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/ antibody test (rapid test) 4th gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test)<br>3rd gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 90 | Before initiating a patier | nt on PrEP, what type of HIV test have | you ever used? | ) | |
| | Oral PrEP | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4th gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/ antibody test<br>(rapid test) 4th gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test)<br>3rd gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | APRETUDE | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4th gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/ antibody test (rapid test) 4th gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test)<br>3rd gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 91 | For follow-up visits f | for patients who are on PrEP, what type o | f HIV test do yo | u primarily use? | |
| | Oral PrEP | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4th gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/ antibody test (rapid test) 4th gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test)<br>3rd gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | APRETUDE | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4th gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/ antibody test (rapid test) 4th gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test)<br>3rd gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 92 | For follow-up visits f | for patients who are on PrEP, what type o | f HIV test have y | ou ever used? | |
| | Oral PrEP | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4th gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/ antibody test (rapid test) 4th gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test)<br>3rd gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | APRETUDE | HIV-1 RNA, qualitative test | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV-1 RNA, quantitative test (e.g. viral load) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antigen/antibody test<br>(laboratory) 4th gen lab | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | HIV antigen/ antibody test<br>(rapid test) 4th gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | HIV antibody test (rapid test)<br>3rd gen rapid | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.702 Assessment of Alternate Sites of Administration of APRETUDE (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 93 | Have any of your APRETUDE | patients received their injections at | a location ot | her than your clinic | ? |
| | | Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 94 | At which locations have you | r APRETUDE patients received injection | ons? | | |
| | | Another clinic | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | At home | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | An infusion center | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Retail pharmacy (e.g., CVS,<br>Walgreens) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Community based organization | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Department of health | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 95 | "Please rate how appropriat | te you believe each setting would be t | for administ | ering APRETUDE." | |
| 95A | HIV-specialty clinic | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 95B | Primary care clinic/private practice | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 95C | Women's health practice/center | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 95D | Community health center | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 95E | Hospital outpatient | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 95F | Retail pharmacy (e.g.,<br>CVS, Walgreens) | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 95G | Other pharmacy | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 95H | At home/home-based caring | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 951 | Community based organization | Very Appropriate | | | |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 95J | Infusion center | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 95K | STD/STI clinic | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 95L | PrEP clinic | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 95M | Department of Health<br>Clinic | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 95N | Mobile clinic | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 950 | Other(s), (please specify) | Very Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all Appropriate | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 96 | Indicate your level of agreer | ment with the following statements: | | | |
| 96A | The use of PrEP will cause patients to engage in riskier behaviors | Completely Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither disagree nor agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 96B | Providing PrEP endorses the risk behaviors of users | Completely Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither disagree nor agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 96C | Only people who engage<br>in risky behavior need<br>PrEP | Completely Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither disagree nor agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 96D | Only people with many sexual partners need PrEP | Completely Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither disagree nor agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 96E | All sexually active people<br>can benefit from PrEP<br>(RC) | Completely Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither disagree nor agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 96F | Providing PrEP will result<br>in an increase in sexually<br>transmitted diseases<br>among patients | Completely Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither disagree nor agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 96G | People do not need PrEP if they act responsibly | Completely Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither disagree nor agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Completely agree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.801 Summary of Perceived Number of APRETUDE Patients Clinic/Practice Can Manage Per Week on an Ongoing Basis (Month 12/13), N=XX

| 60. How many APRETUDE patients do you think your clinic/practice can manage per week on an ongoing basis? | Total<br>Sample<br>n (%) | 0-10<br>Patients<br>n (%) | 11-25<br>Patients<br>n (%) | 26-50<br>Patients<br>n (%) | 51-100<br>Patients<br>n (%) | 101-200<br>Patients<br>n (%) | >200<br>Patients<br>n (%) | Unsure<br>n=xx (%) |
|---|---|---|---|---|---|---|---|---|
| Total Sample | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



Table 3.802 Distributional Characteristics of Reported Number of People in Clinic Trained and Prepared to Give APRETUDE Injections (Month 12/13), N=XX

| 61. Approximately how many people in your clinic are trained and prepared to give APRETUDE injections? | Total<br>Sample<br>n (%) | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum<br>and<br>Maximum) | Missing<br>n (%) | 95% CI for the<br>Mean | l don't know<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| Total Sample | XX<br>(XX%) | X.X | X.XX | X.X<br>(X.X,X.X) | XX<br>(XX, XX) | XX.X% | (X.XX, X.XX) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX<br>(XX%) | X.X | X.XX | X.X<br>(X.X,X.X) | XX<br>(XX, XX) | XX.X% | (X.XX, X.XX) | XX (XX.X%) |
| Routine<br>Implementation | XX<br>(XX%) | X.X | X.XX | X.X<br>(X.X,X.X) | XX<br>(XX, XX) | XX.X% | (X.XX, X.XX) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX<br>(XX%) | X.X | X.XX | X.X<br>(X.X,X.X) | XX<br>(XX, XX) | XX.X% | (X.XX, X.XX) | XX (XX.X%) |
| Low | XX<br>(XX%) | X.X | X.XX | X.X<br>(X.X,X.X) | XX<br>(XX, XX) | XX.X% | (X.XX, X.XX) | XX (XX.X%) |



Table 3.803 Distributional Characteristics of Estimated Number of Staff Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25 People (Month 12/13), N=XX

| 62. How much staff in total do you estimate is/will be needed per week to incorporate APRETUDE into your clinic/practice for approximately 25 people? | Total<br>Sample<br>n (%) | Mean | SD | Median<br>(Q1, Q3) | Observed<br>Range<br>(Minimum<br>and<br>Maximum) | Missing<br>n (%) | 95% CI for the<br>Mean | l don't know<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| Total Sample | XX<br>(XX%) | X.X | X.XX | X.X<br>(X.X,X.X) | XX<br>(XX, XX) | XX.X% | (X.XX, X.XX) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX<br>(XX%) | X.X | X.XX | X.X<br>(X.X,X.X) | XX<br>(XX, XX) | XX.X% | (X.XX, X.XX) | XX (XX.X%) |
| Routine<br>Implementation | XX<br>(XX%) | X.X | X.XX | X.X<br>(X.X,X.X) | XX<br>(XX, XX) | XX.X% | (X.XX, X.XX) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX<br>(XX%) | X.X | X.XX | X.X<br>(X.X,X.X) | XX<br>(XX, XX) | XX.X% | (X.XX, X.XX) | XX (XX.X%) |
| Low | XX<br>(XX%) | X.X | X.XX | X.X<br>(X.X,X.X) | XX<br>(XX, XX) | XX.X% | (X.XX, X.XX) | XX (XX.X%) |



Table 3.804 Summary of Estimated Percentage of Staff Time/Full-Time Equivalent Hours

Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25

People (Month 12/13), N=XX

| 63. How much staff time/full-time equivalent hours (FTE) do you estimate is/will be needed per week to incorporate APRETUDE into your clinic/practice for approximately 25 people? | Total<br>Sample<br>n (%) | 1-20% FTE<br>or 0.4 -<br>8hrs of<br>staff time<br>n (%) | 21-40% FTE<br>or 8.4 - 16hrs<br>of staff time<br>n (%) | 41-60% FTE<br>or 16.4 - 24<br>hrs of staff<br>time<br>n (%) | 61-80% FTE<br>or 24.4 –<br>32hrs of<br>staff time<br>n (%) | 81-100%<br>FTE or<br>32.4 -<br>40hrs of<br>staff<br>time<br>n (%) | l don't<br>know<br>n (%) |
|---|---|---|---|---|---|---|---|
| Total Sample | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | |
| Dynamic<br>Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Routine<br>Implementation | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | |
| High | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |



Table 3.805 Summary of Plans to Create New Roles/Positions in Clinic to Coordinate the APRETUDE Program (Month 12/13), N=XX

| 64. Have you created or do you plan to create new role(s)/new position(s) in your clinic to coordinate the APRETUDE program? | Total Sample<br>n (%) | Yes<br>n (%) | No<br>n (%) | Maybe<br>n (%) | I don't know<br>n (%) |
|---|---|---|---|---|---|
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | |
| Dynamic<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.806 Summary of Number of New Roles/Positions in Clinic to Coordinate the APRETUDE Program (Month 12/13), N=XX

| 65. How many new role(s)/new position(s) have been or will be created in your clinic to coordinate the APRETUDE program? [1] | Total<br>Sample<br>n (%) | 1<br>n (%) | 2<br>n (%) | 3<br>n (%) | 4<br>n (%) | 5<br>n (%) | More<br>than 5 n<br>(%) | l don't<br>know<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| Total Sample | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic<br>Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Routine<br>Implementation | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Site Volume | | | | | | | | |
| High | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |

<sup>[1]</sup> Only includes SSPs who responded 'yes' or 'maybe' to 'Do you plan to create new role(s)/new position(s) in your clinic to coordinate the APRETUDE program?'



Table 3.807 Summary of How Clinic/Practice Plans to Track Patients on APRETUDE (Month 12/13), N=XX

| 66. How is the clinic/practice tracking patients on APRETUDE? | Total<br>Sample<br>n (%) | Use a<br>spreadsheet<br>such as MS<br>Excel<br>n (%) | Assign<br>specific<br>staff to<br>track<br>patients<br>n (%) | Have providers track their own patients n (%) | Create<br>alerts in<br>electronic<br>medical<br>records<br>(EMRs)<br>n (%) | Other<br>[1]<br>n (%) | l don't<br>know<br>n (%) |
|---|---|---|---|---|---|---|---|
| Total Sample | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine Implementation | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |

<sup>[1]</sup> Other responses include: xxxxx


Table 3.808 Summary of How Clinic/Practice Responds to Patients who Do Not Show for a Regularly Scheduled Appointment (Month 12/13), N=XX

| 67. What does your clinic/practice do if a patient does not show for a APRETUDE visit? | Total<br>Sample<br>n (%) | Phone the<br>patient to<br>reschedule<br>n (%) | Text the patient to reschedule n (%) | Email the<br>patient to<br>reschedule<br>n (%) | Send the<br>patient a<br>postal<br>letter to<br>reschedule<br>n (%) | Wait until the patient contacts the clinic/practice to reschedule n (%) | Charge<br>the<br>patient<br>a fee<br>for not<br>showing<br>up n (%) | l don't<br>know/not<br>applicable<br>to role<br>n (%) | Other<br>[1]<br>n (%) |
|---|---|---|---|---|---|---|---|---|---|
| Total Sample | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| rotar sumple | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | | | |
| Dynamic | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| High | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| LUW | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |

<sup>[1]</sup> Other responses include: xxxxx



Table 3.809 Summary of Whether Clinic/Practice has Specific Person in Charge of Following Up on No-Shows (Month 12/13), N=XX

| 68. Is there a specific person in charge of following up on no-shows for APRETUDE appointments? | Total Sample<br>n (%) | Yes<br>n (%) | No<br>n (%) | l don't know<br>n (%) |
|---|---|---|---|---|
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.810 Summary of Type of Systems Clinic has in Place to Remind Patients of Upcoming Appointments (Month 12/13), N=XX

| 72. How do you remind patients of an upcoming APRETUDE appointment?[1] | Total<br>Sample<br>n (%) | Phone<br>Call<br>from<br>Staff n<br>(%) | Automated<br>Phone call<br>n (%) | Text<br>Message<br>n (%) | Email<br>n (%) | Postal<br>Mail n<br>(%) | Phone App<br>Notification<br>n (%) | l don't<br>know<br>n (%) | Other<br>[2]<br>n (%) |
|---|---|---|---|---|---|---|---|---|---|
| Total Sample | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | | | |
| Dynamic | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |

<sup>[1]</sup> Responses are not mutually exclusive; participants can select all that apply

<sup>[2]</sup> Other responses included: xxxxx



Table 3.811 Summary of Type of Systems Clinic has in Place to Offer Upcoming Appointments (Month 12/13), N=XX

| | Total Sample | Stud | y Arm | Site V | olume |
|---|---|---|---|---|---|
| 73. How does your practice/clinic currently offer appointments for APRETUDE injections? | | Dynamic<br>Implementation | Routine<br>Implementation | High | Low |
| | n (%) | n (%) | n (%) | n (%) | n (%) |
| Appointments each day of the week | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Appointments only on certain days of the week | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Appointments spread out over the month | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Injection only appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Allow patients to drop-in for injections on any day without an appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Allow patients to drop-in with little advanced notice (e.g., 24 hour notice) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Allow patients to drop-in on a specific injection day without an appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| After hours appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Before hours appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Weekend appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Home nursing appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mobile clinic option | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Alternate site appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Depends on the schedule of the injection nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Depends on the schedule of the APRETUDE provider | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Unsure | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

<sup>[1]</sup> Responses are not mutually exclusive; participants can select all that apply

<sup>[2]</sup> Other responses include: xxxxx



Table 3.812 Summary of Implementing APRETUDE in Practice (Month 12/13), N=XX

| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| 70 | APRETUDE must be administe | red within a two-week injectior | n window every t | wo months after th | ne loading doses. |
| | | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have not rescheduled any injections thus far | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 71 | How easy or difficult has it be | en to reschedule appointments | for APRETUDE i | njections? | |
| | | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have not rescheduled any injections thus far | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 72 | How do you remind patients o | of an upcoming APRETUDE appo | ointment? | | |
| | | Phone call from Staff | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Automated phone call | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Text message | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Email | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Postal Mail | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Phone app notification | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 73 | How does your practice/clinic | currently offer appointments for | or APRETUDE inj | ections? | |
| | | Appointments each day of the week | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appointments only on certain days of the week | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Appointments spread out over the month | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Injection-only appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Allow patients to drop-in for injections on any day without an appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | Allow patients to drop-in with little advance notice (e.g., 24 hr notice) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Allow patients to drop-in on<br>a specific injection day<br>without an appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | After hours appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Before hours appointment | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Weekend appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Home nursing appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Mobile clinic option | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Alternate site appointments | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Depends on the schedule of the injection nurse | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Depends on the schedule of the APRETUDE provider | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Unsure | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 74 | How easy or difficult has it be | en to implement APRETUDE into | o your current v | vorkflow? | |
| | | Very easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat easy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Neither easy nor difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Very difficult | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Have not rescheduled any injections thus far | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 75 | On average, how long does<br>an APRETUDE patient spend<br>in the waiting room prior to<br>an injection visit? | Up to 20 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 21-40 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 41-60 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 61-90 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | More than 90 minutes<br>(more than 1.5 hrs) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 76 | On average, how long does ar | APRETUDE patient spend in th | e exam room dı | uring an injection vis | sit? |
| | | Up to 20 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| Question<br>Number | Question | Response | Total<br>(N = XX)<br>n (%) | Dynamic<br>Implementation<br>(N = XX)<br>n (%) | Routine<br>Implementation<br>(N = XX)<br>n (%) |
|---|---|---|---|---|---|
| | | 21-40 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 41-60 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 61-90 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | More than 90 minutes<br>(more than 1.5 hrs) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 77 | What is the observation period for a patient after an APRETUDE injection? | | | | |
| | | No observation period | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Up to 10 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 11-20 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | 21-30 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | More than 30 minutes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | I don't know | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 78 | How do you feel about imple | menting APRETUDE at your clin | ic/practice? | | |
| | | Extremely positive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Positive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Somewhat positive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | A little positive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Not at all positive | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Table 3.813. Test for Differences of Implementation Arm by Site Volume on Feasibility of Intervention Measure, APRETUDE (Month 12/13), N=XX

| Source | DF | MS | F | p |
|----------------------------|------|-------|----|--------|
| Study Arm (DI vs. RI) | X.XX | X.XXX | XX | 0.XXXX |
| Volume (High vs. Low) | X.XX | X.XXX | XX | 0.XXXX |
| Interaction, Arm by Volume | X.XX | X.XXX | XX | 0.XXXX |
| Error | X.XX | X.XXX | - | - |

Table 3.814. Test for Differences of Implementation Arm by Site Volume on Feasibility of Intervention Measure, Implementation Support (Month 12/13), N=XX

| Source | DF | MS | F | p |
|----------------------------|------|-------|----|--------|
| Study Arm (DI vs. RI) | X.XX | X.XXX | XX | 0.XXXX |
| Volume (High vs. Low) | X.XX | X.XXX | XX | 0.XXXX |
| Interaction, Arm by Volume | X.XX | X.XXX | XX | 0.XXXX |
| Error | X.XX | X.XXX | - | - |

Table 3.815. Test for Differences of Implementation Arm by Site Volume on Feasibility of Intervention Measure, Telehealth (Month 12/13), N=XX

| Source | DF | MS | F | p |
|----------------------------|------|-------|----|--------|
| Study Arm (DI vs. RI) | X.XX | X.XXX | XX | 0.XXXX |
| Volume (High vs. Low) | X.XX | X.XXX | XX | 0.XXXX |
| Interaction, Arm by Volume | X.XX | X.XXX | XX | 0.XXXX |
| Error | X.XX | X.XXX | - | - |

Table 3.816. Test for Differences of Implementation Arm by Site Volume on Acceptability of Intervention Measure, APRETUDE (Month 12/13), N=XX

| Source | DF | MS | F | p |
|----------------------------|------|-------|----|--------|
| Study Arm (DI vs. RI) | X.XX | X.XXX | XX | 0.XXXX |
| Volume (High vs. Low) | X.XX | X.XXX | XX | 0.XXXX |
| Interaction, Arm by Volume | X.XX | X.XXX | XX | 0.XXXX |
| Error | X.XX | X.XXX | - | - |

Table 3.817. Test for Differences of Implementation Arm by Site Volume on Acceptability of Intervention Measure, Implementation Support (Month 12/13), N=XX

| Source | DF | MS | F | p |
|-----------------------|------|-------|----|--------|
| Study Arm (DI vs. RI) | X.XX | X.XXX | XX | 0.XXXX |
| Volume (High vs. Low) | X.XX | X.XXX | XX | 0.XXXX |



| Interaction, Arm by Volume | X.XX | X.XXX | XX | 0.XXXX |
|----------------------------|------|-------|----|--------|
| Error | X.XX | X.XXX | - | - |

Table 3.818. Test for Differences of Implementation Arm by Site Volume on Acceptability of Intervention Measure, Telehealth (Month 12/13), N=XX

| Source | DF | MS | F | p |
|----------------------------|------|-------|----|--------|
| Study Arm (DI vs. RI) | X.XX | X.XXX | XX | 0.XXXX |
| Volume (High vs. Low) | X.XX | X.XXX | XX | 0.XXXX |
| Interaction, Arm by Volume | X.XX | X.XXX | XX | 0.XXXX |
| Error | X.XX | X.XXX | - | - |



Table 3.901 Quarterly Site Reporting

| Question | | Total | Dynamic<br>Implementation | Routine<br>Implementation |
|---|---|---|---|---|
| 14. How many HIV PrEP seeking persons did the clinic/practice see in the last 3 months? | | | | |
| Baseline | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |
| Quarter X* | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |
| 15. How many patients would you estimate initiated any type of PrEP – oral or injectable – at the clinic/practice in the last 3 months? | N | VOV | VOV | VO |
| Baseline | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |
| Quarter X* | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |
| 16. How many patients would you estimate initiated APRETUDE in the last 3 months at the clinic/practice? | | | | |
| Baseline | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |



| Question | | Total | Dynamic<br>Implementation | Routine<br>Implementation |
|---|---|---|---|---|
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |
| Quarter X* | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |
| 17. Of all patients who have been prescribed PrEP at your clinic/practice, how many would you estimate have completed the Sexual Health Assessment provided by the PILLAR study? | | | | |
| Baseline | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |
| Quarter X* | N | XX | XX | XX |
| | Mean<br>(SD) | XX.X<br>(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X,<br>XX.X | XX.X, XX.X | XX.X, XX.X |
| | Min-Max | X, X | X, X | X, X |

NOTE: reporting is not compiled on schedule with Month 4/5 or Month 12/13 collections, but is instead collected quarterly \*To be populated for each quarter separately depending on available of quarterly data.



## 8 Multiple Timepoint Tables

The following tables combine reporting from Month 1, Month 4/5, and Month 12/13. Only items that were administered across all three timepoints are included in tables below. Stem wording is from Month 1 questionnaire; wording for the stem of some items differed between Month 1 and subsequent time points by verb tense.

| Table 4.01 | Summary of Staff Study Participants' Perceptions Regarding APRETUDE | 440 |
|---|---|---|
| Table 4.02 | Summary of Experiences with the Acquisition Process | 444 |
| Table 4.03 | Summary of Perceived Number of APRETUDE Patients Clinic/Practice Can Manage Per Week on an Ongoing Basis | 451 |
| Table 4.04 | Distributional Characteristics of People in Clinic Trained and Prepared to Give APRETUDE Injections | 453 |
| Table 4.05 | Distributional Characteristics of Estimated Number of Staff Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25 People | 455 |
| Table 4.06 | Summary of Estimated Percentage of Staff Time/Full-Time Equivalent Hours Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25 People | 457 |
| Table 4.07 | Summary of Plans to Create New Roles/Positions in Clinic to Coordinate the APRETUDE Program | 459 |
| Table 4.08 | Summary of Number of New Roles/Positions in Clinic to Coordinate the APRETUDE Program | 460 |
| Table 4.09 | Summary of How Clinic/Practice Plans to Track Patients on APRETUDE | 462 |
| Table 4.10 | Summary of How Clinic/Practice Responds to Patients who Do Not Show for a Regularly Scheduled Appointment | 463 |
| Table 4.11 | Summary of Whether Clinic/Practice has Specific Person in Charge of Following Up on No-Shows | 465 |
| Table 4.12 | Summary of Type of Systems Clinic has in Place to Remind Patients of Upcoming Appointments | 466 |
| Table 4.13 | Summary of Type of Systems Clinic has in Place to Offer Upcoming Appointments – Study Arm | 468 |
| Table 4.14 | Summary of Type of Systems Clinic has in Place to Offer Upcoming Appointments – Site Volume | 470 |



Table 4.01 Summary of Staff Study Participants' Perceptions Regarding APRETUDE

| | | Month 1 | | | Month 4/5 | ; | | Month 12/13 | |
|---|---|---|---|---|---|---|---|---|---|
| Outside / Bassacra | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation |
| Question / Response | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| In your opinion, APRETUDE is appropriate for which individuals? | | | | | | | | | |
| Are Sexually Active | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Have Been Sexually Active<br>With 1 Or More Partners In<br>The Last 6 Months | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Are Currently Adherent On<br>Daily Oral Prep | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Are Non-Adherent On Daily<br>Oral Prep | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Use Prep On Demand (I.E.,<br>Event-Based Prep, Prep 2-1-<br>1) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Could Benefit From Prep But<br>Do Not Want To Use Daily<br>Prep | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Have Previously Used And<br>Discontinued Daily Prep | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Feel Stigmatized About<br>Taking Oral Prep | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Request Apretude<br>Spontaneously | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Have Sex Without A Condom | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Engage In Anal Sex | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| | | Month 1 | | | Month 4/5 | 5 | | Month 12/1 | .3 |
|---|---|---|---|---|---|---|---|---|---|
| Question / Response | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation |
| Question / Response | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Have A Sexual Partner Living<br>With HIV | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Live In Areas With High HIV<br>Prevalence | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Currently Have Or Recently<br>(Within The Past 6 Months)<br>Have Had An STI Other Than<br>HIV | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Are In Monogamous<br>Relationships | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Inject Drugs | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Have Sex With A<br>Person/People Who Inject<br>Drugs | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Experience Stigma Around<br>Using HIV Prevention | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Are Concerned About Taking<br>Pills Every Day | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Experience Stress Or Anxiety<br>Over Adherence Of A Daily<br>Pill Regimen | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Have More Chaotic Lifestyles<br>(E.G., Variable Work<br>Schedules, Frequent Travel,<br>Balancing Work And School) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Have More Structured<br>Lifestyles (E.G., Regular Work | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| ne Total<br>ntation | | Month 12/13 |
|---|---|---|
| | Dynamic Routine<br>Implementation Implementati | Total Im |
| (N = XX) | (N = XX) (N = XX) | (N =<br>XX) |
| n (%) | n (%) n (%) | n (%) |
| XX (XX.X%) | XX (XX.X%) XX (XX.X%) | XX<br>(XX.X%) |
| XX<br>(XX.X%) | XX (XX.X%) XX (XX.X%) | XX<br>(XX.X%) |
| UDE? | | |
| XX<br>(XX.X%) | XX (XX.X%) XX (XX.X%) | XX<br>(XX.X%) |
| XX<br>(XX.X%) | XX (XX.X%) XX (XX.X%) | XX<br>(XX.X%) |
| XX<br>(XX.X%) | XX (XX.X%) XX (XX.X%) | XX<br>(XX.X%) |
| .) | (XX.X%) | X%) (XX.X%) XX (XX.X%) X%) XX (XX.X%) XX (XX.X%) X%) XX (XX.X%) XX (XX.X%) |



| | | Month 1 | | | Month 4/5 | 5 | | Month 12/13 | |
|---|---|---|---|---|---|---|---|---|---|
| Overtical / Bernand | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation |
| Question / Response | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| I Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| How are you or this clinic/prac | tice inform | ing patients about | APRETUDE? | | | | | | |
| Provision Of Educational<br>Materials | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| During Consultation With<br>Patient | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Through Peer Educators | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Referring Patients To Prep<br>Providers | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Posters In The Clinic/Practice | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Flyers In The Clinic/Practice | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mentions On The<br>Clinic/Practice's Website | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mentions On Social Media | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |

Results from tables 1.004, 2.004, and 3.004.



Table 4.02 Summary of Experiences with the Acquisition Process

| | | Month 1 | | | Month 4/5 | ; | | Month 12/13 | |
|---|---|---|---|---|---|---|---|---|---|
| Question / Response | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation |
| | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Are you or will you be involved in any part of acquisition process for APRETUDE, such as completing enrollment forms, prior authorization, claims, sending documents to insurance companies, and purchasing APRETUDE? | | | | | | | | | |
| Yes | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| l Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| How will your providers or clin | ic/practice | acquire APRETUDE | ? | | | | | | |
| Buy-And-Bill - Purchases<br>Apretude From A Wholesaler<br>Or Specialty Distributor And<br>Bills The Primary Third-Party<br>Payer | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| White Bagging - Submits Prescription To A Specialty Pharmacy Within ViiV's Specialty Pharmacy Network And The Specialty Pharmacy Processes The Claim And Ships Apretude For Administration | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clear Bagging - Internal<br>Pharmacy Maintains<br>Inventory Of The Medication,<br>Processes The Claim, And<br>Delivers The Medication | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| | | Month 1 | | | Month 4/5 | 5 | Month 12/13 | | |
|---|---|---|---|---|---|---|---|---|---|
| Question / Response | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation |
| | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) |
| Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| l Don't Know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Who in your clinic/practice is r | esponsible | for completing the | insurance benefits | verification | n process for specia | lty medications for | patients? | | |
| Physician | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse Practitioner/<br>Physician Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Pharmacist | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Specialty Pharmacy | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Assistant | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Social Worker/Case Manager | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Front Desk Staff/Scheduler | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Dedicated Administrator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Apretude Coordinator | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| | | | Month 1 | | | Month 4/5 | | Month 12/13 | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Question / F | Response | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation |
| | | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) |
| I Don't Know | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| For each item, p | lease indicate | how conce | rned you would be | about each of the f | ollowing b | ased on your curre | nt expectations, un | derstandin | g and knowledge of | ViiV Connect. |
| Authorization<br>Wait Times | Extremely<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Moderately<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Slightly<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Somewhat<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Not At All<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Extremely<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Moderately<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Understanding Status of Authorization | Slightly<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Adthonization | Somewhat<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Not At All<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Understanding | Extremely<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| how to seek<br>assistance | Moderately<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| | | | Month 1 | | | Month 4/5 | 5 | Month 12/13 | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Question / | Response | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation |
| | | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) |
| | Slightly<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Somewhat<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Not At All<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Extremely<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Moderately<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Amount of paperwork | Slightly<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Somewhat<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Not At All<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Extremely<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Moderately<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Clarity on<br>Coverage<br>Approval | Slightly<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Somewhat<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Not At All<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Ensuring<br>medication | Extremely<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| | | | Month 1 | | | Month 4/5 | 5 | | Month 12/13 | |
|---|---|---|---|---|---|---|---|---|---|---|
| Question / F | Response | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation |
| | | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) |
| comes to the<br>right place | Moderately<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| (e.g.,<br>clinic/practice,<br>pharmacy) | Slightly<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| <i>p</i> | Somewhat<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Not At All<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Extremely<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Potential loss | Moderately<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| of enthusiasm<br>for APRETUDE | Slightly<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| by patients | Somewhat<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Not At All<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Extremely<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Potential | Moderately<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| patient<br>dissatisfaction<br>with clinic | Slightly<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| staff | Somewhat<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Not At All<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| | | | Month 1 | | | Month 4/5 | 5 | Month 12/13 | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Question / I | Response | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation |
| | | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) |
| | Extremely<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Staff | Moderately<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| dissatisfaction<br>with the<br>acquisition | Slightly<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| process | Somewhat<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Not At All<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Extremely<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Moderately<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Potential<br>Disruption of<br>Clinic Flow | Slightly<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Cillic How | Somewhat<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Not At All<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Extremely<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Time-<br>consuming<br>Process | Moderately<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Slightly<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Somewhat<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| | | | Month 1 | | | Month 4/5 | ; | | Month 12/13 | |
|---|---|---|---|---|---|---|---|---|---|---|
| Question / I | Response | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation | Total | Dynamic<br>Implementation | Routine<br>Implementation |
| | | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) | (N =<br>XX) | (N = XX) | (N = XX) |
| | Not At All<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Extremely<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Inequitable | Moderately<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Access for<br>Eligible | Slightly<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Patients | Somewhat<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Not At All<br>Concerned | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| I would recomm | end ViiV Conn | ect to othe | r providers and clin | ics/practices to aid | in the acqu | he acquisition of ViiV medications | | | | |
| Agree | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Disagree | | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Neither Agree C | r Disagree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Completely Disa | gree | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Completely Agre | ee | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |

Results from tables 1.005, 2.005, and 3.005.



Table 4.03 Summary of Perceived Number of APRETUDE Patients Clinic/Practice Can Manage Per Week on an Ongoing Basis

| How many APRETUDE patients do you think your | Total Sample | 0-10 Patients | 11-25 Patients | 26-50 Patients | 51-100<br>Patients | 101-200<br>Patients | >200 Patients | I don't know |
|---|---|---|---|---|---|---|---|---|
| clinic/practice can manage per week on an ongoing basis? | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n=xx (%) |
| | | | Мо | nth 1 | | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | | Mon | th 4/5 | | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | | Montl | h 12/13 | | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



Results from tables 1.801, 2.801, and 3.801.



Table 4.04 Distributional Characteristics of People in Clinic Trained and Prepared to Give APRETUDE Injections

| Approximately how many people in your clinic are trained and prepared to give APRETUDE injections? | Total<br>Sample<br>n (%) | Mean | SD | Median<br>(Q1, Q3) | Observed Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% Confidence<br>Interval | l don't know<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| | | | | Month 1 | | | | |
| Total Sample | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Low | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| | | | | Month 4/5 | | | | |
| Total Sample | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Low | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| | | | | Month 12/13 | | | | |
| Total Sample | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Low | XX (XX.X%) | X.X | X.XX | X.X (X.X, X.X) | XX (XX, XX) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |



Results from tables 1.802, 2.802, and 3.802.



Table 4.05 Distributional Characteristics of Estimated Number of Staff Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25 People

| How much staff in total do you estimate will be needed per week to incorporate APRETUDE into your clinic/practice for approximately 25 people? | Total<br>Sample<br>n (%) | Mean | SD | Median<br>(Q1, Q3) | Observed Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI for the<br>Mean | I don't know<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| | | | | Month 1 | | | | |
| Total Sample | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Low | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| | | | | Month 4/5 | | | | |
| Total Sample | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Low | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| | | | | Month 12/13 | | | | |
| Total Sample | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Site Volume | | | | | | | | |



| How much staff in total do you estimate will be needed per week to incorporate APRETUDE into your clinic/practice for approximately 25 people? | Total<br>Sample<br>n (%) | Mean | SD | Median<br>(Q1, Q3) | Observed Range<br>(Minimum,<br>Maximum) | Missing<br>n (%) | 95% CI for the<br>Mean | l don't know<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| High | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |
| Low | XX (XX.X%) | X.XX | X.XXX | X.XX (X.XX,X.XX) | XX.X (XX.X, XX.X) | XX (XX.X%) | (X.XX, X.XX) | XX (XX.X%) |

Results from tables 1.803, 2.803, and 3.803.



Table 4.06 Summary of Estimated Percentage of Staff Time/Full-Time Equivalent Hours Needed Per Week to Incorporate APRETUDE into Clinic/Practice for Approximately 25 People

| How much staff time/full-time equivalent hours (FTE) do you estimate will be needed per week to incorporate APRETUDE into your clinic/practice for approximately 25 people? | Total<br>Sample<br>n (%) | 1-20% FTE or 0.4<br>- 8hrs of staff<br>time<br>n (%) | 21-40% FTE or<br>8.4 - 16hrs of<br>staff time<br>n (%) | 41-60% FTE or<br>16.4 - 24 hrs of<br>staff time<br>n (%) | 61-80% FTE or<br>24.4 – 32hrs of<br>staff time<br>n (%) | 81-100% FTE or<br>32.4 - 40hrs of<br>staff time<br>n (%) | l don't know<br>n (%) |
|---|---|---|---|---|---|---|---|
| | | | Month 1 | | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | | Month 4/5 | | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | | Month 12/13 | | | | |



| How much staff time/full-time equivalent hours (FTE) do you estimate will be needed per week to incorporate APRETUDE into your clinic/practice for approximately 25 people? | Total<br>Sample<br>n (%) | 1-20% FTE or 0.4<br>- 8hrs of staff<br>time<br>n (%) | 21-40% FTE or<br>8.4 - 16hrs of<br>staff time<br>n (%) | 41-60% FTE or<br>16.4 - 24 hrs of<br>staff time<br>n (%) | 61-80% FTE or<br>24.4 – 32hrs of<br>staff time<br>n (%) | 81-100% FTE or<br>32.4 - 40hrs of<br>staff time<br>n (%) | I don't know<br>n (%) |
|---|---|---|---|---|---|---|---|
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Results from tables 1.804, 2.804, and 3.804.



Table 4.07 Summary of Plans to Create New Roles/Positions in Clinic to Coordinate the APRETUDE Program

| Do you plan to create new role(s)/new position(s) in your clinic | Total<br>Sample | Yes | No | Maybe | l don't<br>know |
|---|---|---|---|---|---|
| to coordinate the APRETUDE program? | n (%) | n (%) | n (%) | n (%) | n (%) |
| | | Month 1 | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Month 4/5 | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | Month 12/13 | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Results from tables 1.805, 2.805, and 3.805.



Table 4.08 Summary of Number of New Roles/Positions in Clinic to Coordinate the APRETUDE Program

| How many new role(s)/new position(s) are you planning to create in | Total<br>Sample | 1 | 2 | 3 | 4 | 5 | More<br>than 5 | l don't<br>know |
|---|---|---|---|---|---|---|---|---|
| your clinic to coordinate the APRETUDE program? | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | | | Mont | h 1 | | | | |
| Total Sample | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | Month | 4/5 | | | | |
| Total Sample | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Low | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| | | | Month 1 | 12/13 | | | | |
| Total Sample | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Routine | XX | XX | XX | XX | XX | XX | XX | XX |
| Implementation | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX | XX | XX | XX | XX | XX | XX | XX |
| | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) | (XX.X%) |



| How many new role(s)/new position(s) are you planning to create in your clinic to coordinate | Total<br>Sample<br>n (%) | <b>1</b><br>n (%) | <b>2</b><br>n (%) | <b>3</b><br>n (%) | <b>4</b><br>n (%) | <b>5</b><br>n (%) | More<br>than 5 | l don't<br>know<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| the APRETUDE program? | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) |
| Low | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) |

Results from tables 1.806, 2.806, and 3.806.



Table 4.09 Summary of How Clinic/Practice Plans to Track Patients on APRETUDE

| How does your clinic/practice plan to track patients on APRETUDE? | Total<br>Sample<br>n (%) | Use a<br>spreadsheet<br>such as MS<br>Excel<br>n (%) | Assign<br>specific<br>staff to<br>track<br>patients<br>n (%) | Have<br>providers<br>track their<br>own<br>patients<br>n (%) | Create<br>alerts in<br>electronic<br>medical<br>records<br>(EMRs)<br>n (%) | Other [1]<br>n (%) | I don't<br>know<br>n (%) |
|---|---|---|---|---|---|---|---|
| Month 1 | | | | | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Month 4/5 | | | ı | ı | ı | ı | 1 |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Month 12/13 | | | | | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | |
| Dynamic<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine<br>Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Results from tables 1.807, 2.807, and 3.807.



Table 4.10 Summary of How Clinic/Practice Responds to Patients who Do Not Show for a Regularly Scheduled Appointment

| What does your clinic/practice do if a patient does not show for a regularly scheduled appointment? | Total<br>Sample<br>n (%) | Phone the<br>patient to<br>reschedule<br>n (%) | Text the patient to reschedule n (%) | Email the<br>patient to<br>reschedule<br>n (%) | Send the<br>patient a<br>postal letter<br>to<br>reschedule<br>n (%) | Wait until the patient contacts the clinic/practice to reschedule n (%) | Charge the<br>patient a<br>fee for not<br>showing up<br>n (%) | I don't<br>know/not<br>applicable<br>to role<br>n (%) | Other<br>n (%) |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Month 1 | | | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | | | Month 4/5 | | | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | | | Month 12/13 | | | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | | | |



| What does your clinic/practice do if a patient does not show for a regularly scheduled appointment? | Total<br>Sample<br>n (%) | Phone the<br>patient to<br>reschedule<br>n (%) | Text the<br>patient to<br>reschedule<br>n (%) | Email the<br>patient to<br>reschedule<br>n (%) | Send the<br>patient a<br>postal letter<br>to<br>reschedule<br>n (%) | Wait until the patient contacts the clinic/practice to reschedule n (%) | Charge the<br>patient a<br>fee for not<br>showing up<br>n (%) | I don't<br>know/not<br>applicable<br>to role<br>n (%) | Other<br>n (%) |
|---|---|---|---|---|---|---|---|---|---|
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Results from tables 1.808, 2.808, and 3.808.



Table 4.11 Summary of Whether Clinic/Practice has Specific Person in Charge of Following Up on No-Shows

| Is there a specific person in charge of | Total Sample | Yes | No | I don't know |
|---|---|---|---|---|
| following up on no-shows? | n (%) | n (%) | n (%) | n (%) |
| | Mont | h 1 | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Month | 4/5 | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Month 1 | 12/13 | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Results from tables 1.809, 2.809, and 3.809.



Table 4.12 Summary of Type of Systems Clinic has in Place to Remind Patients of Upcoming Appointments

| What type of systems does your clinic have in place to remind patients of an upcoming appointment? | Total Sample<br>n (%) | Phone<br>Call<br>from<br>Staff<br>n (%) | Automated<br>Phone<br>call<br>n (%) | Text<br>Message<br>n (%) | Email<br>n (%) | Postal<br>Mail<br>n (%) | Phone<br>App Notification<br>n (%) | Other<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| | | | Month: | 1 | | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | | Month 4 | /5 | | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | | | Month 12 | /13 | | | | |
| Total Sample | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Arm | | | | | | | | |
| Dynamic Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Routine Implementation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Site Volume | | | | | | | | |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |



| What type of systems does your clinic have in place to remind patients of an upcoming appointment? | Total Sample<br>n (%) | Phone<br>Call<br>from<br>Staff<br>n (%) | Automated<br>Phone<br>call<br>n (%) | Text<br>Message<br>n (%) | Email<br>n (%) | Postal<br>Mail<br>n (%) | Phone<br>App Notification<br>n (%) | Other<br>n (%) |
|---|---|---|---|---|---|---|---|---|
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Results from tables 1.810, 2.810, and 3.810.



Table 4.13 Summary of Type of Systems Clinic has in Place to Offer Upcoming Appointments – Study Arm

| | | | | | | | | - | |
|---|---|---|---|---|---|---|---|---|---|
| How do you | | Month 1 | | | Mon | th 4/5 | Month 12 | 2/13 | |
| plan to offer | Total | Study | y Arm | Total | Study Arm | | | Study A | rm |
| appointments<br>for APRETUDE<br>injections? | Total<br>Sample | Dynamic<br>Implementation | Routine<br>Implementation | Total<br>Sample | Dynamic<br>Implementation | Routine<br>Implementation | Total<br>Sample | Dynamic<br>Implementation | Routine<br>Implementation |
| injections: | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Appointments<br>each day of the<br>week | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Appointments<br>only on certain<br>days of the<br>week | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Appointments spread out over the month | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Injection-only appointments | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Allow patients<br>to drop-in for<br>injections on<br>any day<br>without an<br>appointment | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Allow patients<br>to drop-in with<br>little advanced<br>notice (e.g., 24<br>hour notice) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Allow patients<br>to drop-in on a<br>specific<br>injection day<br>without an<br>appointment | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| After hours appointments | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| How do you<br>plan to offer | | Month 1 | y Arm | | | th 4/5<br>y Arm | | Month 1<br>Study A | |
|---|---|---|---|---|---|---|---|---|---|
| appointments<br>for APRETUDE<br>injections? | Total<br>Sample | Dynamic<br>Implementation | Routine<br>Implementation | Total<br>Sample | Dynamic<br>Implementation | Routine<br>Implementation | Total<br>Sample | Dynamic<br>Implementation | Routine<br>Implementation |
| injections | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Before hours appointment | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Weekend<br>appointments | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Home nursing appointments | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mobile clinic option | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Alternate site appointments | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Depends on the schedule of the injection nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Depends on the<br>schedule of the<br>APRETUDE<br>provider | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |

Results from tables 1.811, 2.811, and 3.811.



Table 4.14 Summary of Type of Systems Clinic has in Place to Offer Upcoming Appointments – Site Volume

| How do you | | Month 1 | | | Mon | Month 12/13 | | | |
|---|---|---|---|---|---|---|---|---|---|
| plan to offer appointments | Total | Site V | olume | Total | Site V | olume | Site | Site Volu | ime |
| for APRETUDE | Sample | High Volume | Low Volume | Sample | High Volume | Low Volume | Volume | High Volume | Low Volume |
| injections? | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Appointments<br>each day of the<br>week | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Appointments<br>only on certain<br>days of the<br>week | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Appointments<br>spread out over<br>the month | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Injection-only appointments | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Allow patients<br>to drop-in for<br>injections on<br>any day<br>without an<br>appointment | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Allow patients<br>to drop-in with<br>little advanced<br>notice (e.g., 24<br>hour notice) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Allow patients to drop-in on a specific injection day without an appointment | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| After hours<br>appointments | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Before hours<br>appointment | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |



| How do you | | Month 1 | | | Mon | th 4/5 | | Month 12/13 | |
|---|---|---|---|---|---|---|---|---|---|
| plan to offer appointments | Total | Site V | olume olume | Total | Site V | olume on the second | Site | Site Volu | ıme |
| for APRETUDE | Sample | High Volume | Low Volume | Sample | High Volume | Low Volume | Volume | High Volume | Low Volume |
| injections? | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Weekend appointments | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Home nursing appointments | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mobile clinic option | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Alternate site appointments | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Depends on the schedule of the injection nurse | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Depends on the<br>schedule of the<br>APRETUDE<br>provider | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |
| I don't know | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) | XX<br>(XX.X%) | XX (XX.X%) | XX (XX.X%) |

Results from tables 1.811, 2.811, and 3.81